# S1: Study protocol

# Specification for Herd immunity April, 2019

## Overview:

This study is a PhD project conducted by Ms. Hina Hakim, supervised by Dr. Holly O. Witteman, PhD, and co-supervised by Dr. Daniel Reinharz, professors, and researchers at the Faculty of Medicine at Laval University. The purpose of this study is to evaluate the effects of visualization conveying the concept of community immunity or herd immunity on risk perception (towards individual, family, community and vulnerable people in communities) (primary outcome) and on emotions, attitudes, knowledge, and behavioural intentions (secondary outcomes).

# People Involved:

Hakim, H (PhD candidate)
Witteman, H (Research supervisor)
Parent, E (Designer and adviser on designing)
Aziaka, D (Developer/Programmer)
Noubi, M (Developer/Programmer)
Toudjeu, NT (Developer/Programmer)

## Collaborating with:

- The members of the National Institute of Public Health of Quebec (INSPQ) whose comments
  we have received as we planned this project are: Eve Dubé, Marc Dionne, Rodica Gilca,
  Manale Ouakki and Dominique Gagnon.
- The members of Public Health Ontario whose comments we have received as we planned this
  project are: Beate Sander and Bryna Warshawsky.

## Co-investigators:

Hina Hakim, Christine T. Chambers, Eve Dubé, S. Michelle Driedger, Teresa Gavaruzzi, Anik M. C. Giguere, Noah M. Ivers, Éric Kavanagh, Shannon MacDonald, Rita Orji, Elizabeth Parent, Jean-Sébastien Paquette, Jacynthe Roberge, Beate Sander, Aaron Scherer, Bryna Warshawsky, Kumanan Wilson, Daniel Reinharz, Holly O. Witteman

# INTRODUCTION

## Background and rationale

Herd immunity or community immunity exists when enough people in a given population are vaccinated. This provides an indirect protection to those who cannot get vaccinated due to a weak immune system as either they are too young, too old or immunocompromised (vulnerable people). Recent drop in vaccine uptake results in an outbreak of vaccine-preventable diseases which increases the risk of everyone to be in at high risk of being infected, especially vulnerable people. Research suggested that effective communication about herd immunity may increase vaccination intention (Betsch et al. 2017).

Visualization is a powerful communication mechanism that uses pre-attentive processing to communicate large amounts of information rapidly in understandable and compelling ways (Healey and Enns 2012). A systematic review demonstrates that there are some interventions available for conveying the concept of community immunity, and very few evaluate interventions for their effects

on vaccine intentions and uptake as well as their precursors, such as knowledge, attitudes, and none on emotions (Hakim et al. 2018).

The purpose of this study is to evaluate the effects of visualization conveying the concept of community immunity on risk perception (to individual, family, community and vulnerable people in communities) (primary outcome) and on emotions, attitudes, knowledge, and behavioural intentions (secondary outcomes).

## INTRODUCTION

## Contexte et justification

L'immunité collective existe quand suffisamment de personnes dans une population donnée sont vaccinées. Cela fournit une protection indirecte aux personnes qui ne peuvent pas se faire vacciner en raison de la faiblesse de leur système immunitaire, du fait qu'elles soient trop jeunes, trop âgées ou immunodéprimées (personnes vulnérables). La récente baisse des taux de vaccination a entraîné une épidémie des maladies pouvant être prévenues par la vaccination, ce qui augmente le risque pour chacun d'être infecté, en particulier les personnes vulnérables. Les recherches ont suggéré qu'une communication efficace sur l'immunité collective pourrait augmenter l'intention de vaccination (Betsch et al. 2017).

La visualisation est un mécanisme de communication puissant qui utilise un traitement préattentif pour communiquer rapidement de grandes quantités d'informations de manière compréhensible et convaincante (Healey et Enns 2012). Une revue systématique a montré que certaines interventions permettent de véhiculer le concept d'immunité collective et que très peu évaluent leurs effets sur les intentions liées à la vaccination ainsi que sur leurs précurseurs, telles que les connaissances, les attitudes, mais aucune ne portant sur les émotions (Hakim et al 2018).

Le but de cette étude est d'évaluer les effets de la visualisation transmettant le concept d'immunité collective sur la perception du risque (pour l'individu, la famille, la communauté et les personnes vulnérables dans les communautés) (résultat principal) et sur les émotions, les attitudes, les connaissances et les intentions comportementales (résultats secondaires).

# Objectives

To evaluate the effects of visualization conveying the concept of community immunity on risk perception (to individual, family, community and vulnerable people in communities) (primary outcome) and on emotions, attitudes, knowledge, and behavioural intentions (secondary outcomes). We hypothesize that the new visualization "Herdimm" (A visualization developed iteratively in our previous study) will help people understand the concept of community immunity better than the control condition or comparator:

- Control: No information about community immunity or herd immunity
- Intervention: Herdimm visualization

We will also conduct secondary analyses comparing the effects of visualization (Herdimm) versus five comparators:

- Measles: Guardian visualization (<a href="https://www.theguardian.com/society/ng-interactive/2015/feb/05/-sp-watch-how-measles-outbreak-spreads-when-kids-get-vaccinated">https://www.theguardian.com/society/ng-interactive/2015/feb/05/-sp-watch-how-measles-outbreak-spreads-when-kids-get-vaccinated</a>)
- Measles: Visualization by theotheredmund: (https://imgur.com/gallery/8M7q8#J7LANQ4)
- Generic: Robert Koch Institut visualization (http://rocs.hu-berlin.de/D3/herd/)
- Generic: SBS News visualization: (<a href="https://www.sbs.com.au/news/two-sydney-babies-too-young-to-be-vaccinated-infected-with-measles?fbclid=IwAR1Rns\_ycauiZeTeY1HC22eJe8JE6dwcQG0A9fgq305WCskIHBT\_AGZExLE">https://www.sbs.com.au/news/two-sydney-babies-too-young-to-be-vaccinated-infected-with-measles?fbclid=IwAR1Rns\_ycauiZeTeY1HC22eJe8JE6dwcQG0A9fgq305WCskIHBT\_AGZExLE</a>)
- Influenza: Public Health Agency of Canada Flu: Don't Pass It On! (https://www.canada.ca/en/public-health/services/video/the-flu-don-t-pass-it-on.html)

## **Objectifs**

Évaluer les effets de la visualisation traduisant le concept d'immunité communautaire sur la perception du risque (pour l'individu, la famille, la communauté et les personnes vulnérables dans la communauté) (résultat principal) et sur les émotions, les attitudes, les Connaissances et les intentions comportementales (résultats secondaires).

Nous émettons l'hypothèse que la nouvelle visualisation « Herdimm » (visualisation développée de manière itérative dans notre précédente étude) aidera les gens à mieux comprendre le concept d'immunité collective que la condition de contrôle ou le comparateur :

- Contrôle : aucune éducation sur l'immunité de la communauté ou l'immunité collective
- Intervention: visualisation « Herdimm »

Nous effectuerons également des analyses secondaires comparant les effets de la visualisation (Herdimm) à ceux de six comparateurs :

- Rougeole: Visualisation de The Guardian (<a href="https://www.theguardian.com/society/ng-interactive/2015/feb/05/-sp-watch-how-measles-outbreak-spreads-when-kids-get-vaccinated">https://www.theguardian.com/society/ng-interactive/2015/feb/05/-sp-watch-how-measles-outbreak-spreads-when-kids-get-vaccinated</a>)
- Rougeole: Visualisation par theotheredmund: (https://imgur.com/gallery/8M7q8#J7LANQ4)
- Générique : Visualisation de l'Institut Robert Koch (http://rocs.hu-berlin.de/D3/herd/)
- Générique: Visualisation de SBS (The Special Broadcasting Service):
   (https://www.sbs.com.au/news/two-sydney-babies-too-young-to-be-vaccinated-infected-with-measles?fbclid=IwAR1Rns\_ycauiZeTeY1HC22eJe8JE6dwcQG0A9fgq305WCskIHBT\_AGZExLE)
- Influenza : Agence de la santé publique du Canada Grippe: ne le transmettez pas! (<a href="https://www.canada.ca/fr/sante-publique/services/video/la-grippe-n-en-passez-pas-les-maux.html">https://www.canada.ca/fr/sante-publique/services/video/la-grippe-n-en-passez-pas-les-maux.html</a>)

# METHODS: Study design, participants, interventions, and outcomes Study/Trial Design

A factor is a variable that is controlled and varied during the course of an experiment. In the clinical trial, treatment can be a factor i.e., treatment vs. control. Factorial clinical trials are experiments that test the effect of more than one treatment using a type of design that permits an assessment of potential interactions among the treatments. The randomized controlled trial is the robust research method for determining whether a cause and effect relation exists between an intervention and an outcome. By using randomized controlled trial one can generate high-quality evidence when evaluating the effectiveness of an intervention.

This study will be a multi-armed factorial randomized controlled trial. Factorial experiments allow for the estimation of main effects of multiple factors in a single experiment by combining experimental conditions (Gallis et al. 2019). Thus, such designs are useful options in health behaviour research to efficiently compare more than one intervention. In this study, our primary analysis will be no education about community immunity or herd immunity (control) versus our developed visualization (herdimm).

Each participant will be randomly allocated to focus on one of four possible vaccine-preventable diseases that is: measles, pertussis, flu (influenza), or a generic vaccine-preventable disease (hereby referred to as "generic"). All aspects of the study (visualization, questionnaire) will be focused on that one disease for that participant.

For secondary analyses, we will compare effects of disease-specific interventions (e.g., the measles version of the visualization) to the effects of disease-matched interventions (comparators)

drawn from existing visualizations available online. Specifically, we will compare our measles visualization to other measles visualizations, and so on. The comparators are:

- Measles: Guardian visualization (<a href="https://www.theguardian.com/society/ng-interactive/2015/feb/05/-sp-watch-how-measles-outbreak-spreads-when-kids-get-vaccinated">https://www.theguardian.com/society/ng-interactive/2015/feb/05/-sp-watch-how-measles-outbreak-spreads-when-kids-get-vaccinated</a>)
- Measles: Gif by theotheredmund: (https://imgur.com/gallery/8M7q8#J7LANQ4)
- Generic: Robert Koch Institut visualization (http://rocs.hu-berlin.de/D3/herd/)
- Generic: SBS News visualization: (<a href="https://www.sbs.com.au/news/two-sydney-babies-too-young-to-be-vaccinated-infected-with-measles?fbclid=IwAR1Rns\_ycauiZeTeY1HC22eJe8JE6dwcQG0A9fgq305WCskIHBT\_AGZExLE">https://www.sbs.com.au/news/two-sydney-babies-too-young-to-be-vaccinated-infected-with-measles?fbclid=IwAR1Rns\_ycauiZeTeY1HC22eJe8JE6dwcQG0A9fgq305WCskIHBT\_AGZExLE</a>)
- Generic: NHS visualization (https://www.nhs.uk/Video/Pages/Vaccinationanimation2.aspx)
- Influenza: Public Health Agency of Canada Flu: Don't Pass It On! (https://www.canada.ca/en/public-health/services/video/the-flu-don-t-pass-it-on.html)

The primary and secondary outcomes of the study which are risk perception, emotion, knowledge,trust (in information provided), attitudes and a validated scale about vaccination (Betsch et al. 2018) will be assessed in an online questionnaire.

Because three online visualizations are available only in English whereas our study will be conducted in both English and French, we will use slightly different randomization patterns for English- and French-speaking participants.

# MÉTHODES: Conception de l'étude, participants, interventions et résultats Conception de l'étude

Un facteur est une variable contrôlée et variée au cours d'une expérience. Dans l'essai clinique, le traitement peut être un facteur, par exemple traitement versus contrôle. Les essais cliniques factoriels sont des expériences qui testent l'effet de plus d'un traitement en utilisant un type de conception permettant d'évaluer les interactions potentielles entre les traitements. L'essai contrôlé randomisé est la méthode de recherche robuste pour déterminer s'il existe une relation de cause à effet entre une intervention et un résultat. En utilisant des essais contrôlés randomisés, on peut générer des preuves de haute qualité lors de l'évaluation de l'efficacité d'une intervention.

Cette étude sera un essai contrôlé randomisé factoriel multi-bras. Les expériences factorielles permettent d'estimer les effets principaux de plusieurs facteurs dans une seule expérience en combinant des conditions expérimentales. Ainsi, de tels modèles sont des options utiles dans la recherche sur les comportements en matière de santé pour comparer efficacement plus d'une intervention. Dans cette étude, notre analyse principale portera sur l'absence d'éducation concernant l'immunité de la communauté ou l'immunité collective (contrôle) par rapport à notre visualisation développée (herdimm).

Chaque participant se verra attribuer au hasard une des quatre maladies pouvant être prévenues par un vaccin aux fins de l'étude : rougeole, coqueluche, grippe ou une maladie générique évitable par un vaccin (ci-après dénommée « générique »). Tous les aspects de l'étude (visualisation, questionnaire) seront centrés sur cette maladie pour ce participant.

Pour les analyses secondaires, nous comparerons les effets des interventions spécifiques à une maladie (par exemple, la version de la visualisation portant sur la rougeole) avec les effets des interventions appariées à la maladie (comparateurs) tirés des visualisations existantes disponibles en ligne. Plus précisément, nous comparerons notre visualisation de la rougeole à d'autres visualisations de la rougeole, et ainsi de suite. Les comparateurs sont :

- Rougeole: visualisation de The Guardian (https://www.theguardian.com/society/ng-interactive/2015/feb/05/-sp-watch-how-measles-outbreak-spreads-when-kids-get-vaccinated)
- Rougeole: Visualisation par theotheredmund: (https://imgur.com/gallery/8M7q8#J7LANQ4)
- Générique : Visualisation de l'Institut Robert Koch (http://rocs.hu-berlin.de/D3/herd/)
- Générique : Visualisation de SBS (The Special Broadcasting Service) : (https://www.sbs.com.au/news/two-sydney-babies-too-young-to-be-vaccinated-infected-with-

- measles?fbclid=IwAR1Rns\_ycauiZeTeY1HC22eJe8JE6dwcQG0A9fgq305WCskIHBT\_AGz ExLE)
- Générique: visualisation NHS (National Health Service) (https://www.nhs.uk/Video/Pages/Vaccinationanimation2.aspx)
- Influenza: Agence de la santé publique du Canada Grippe: ne le transmettez pas! (<a href="https://www.canada.ca/fr/sante-publique/services/video/la-grippe-n-en-passez-pas-les-maux.html">https://www.canada.ca/fr/sante-publique/services/video/la-grippe-n-en-passez-pas-les-maux.html</a>)

Les résultats primaires et secondaires de l'étude (perception du risque, émotion, connaissances et une échelle validée concernant la vaccination (Betsch et al. 2018) seront évalués à l'aide d'un questionnaire en ligne.

Puisque trois visualisations en ligne sont disponibles uniquement en anglais alors que notre étude sera menée en anglais et en français, nous utiliserons des schémas de randomisation légèrement différents pour les participants anglophones et francophones.

## Flow chart: Overall randomization



<sup>\*</sup> Sample size doubled for an embedded study of male versus female voice narration

## Study setting

 The online randomized controlled trial will be running in Qualtrics, an online survey software. • Eligible participants will be adult members (18 years and over) of the general public in Canada (with a minimum of 25% of the sample with French as their preferred language compared to English).

#### Cadre de l'étude

- L'essai contrôlé randomisé en ligne sera exécuté dans Qualtrics, un logiciel de sondage en ligne.
- Les participants admissibles seront des membres adultes (de 18 ans et plus) du grand public au Canada (au moins 25% de l'échantillon ayant le français comme langue préférée par rapport à l'anglais).

# Eligibility criteria

#### Inclusion Criteria:

- Members of the general population
- Be at least 18 years old
- To be able to provide free and informed consent and to be able to read and understand
   French or English
- Do not have vision problems not corrected
- To be able to use computer

## Exclusion Criteria:

- Be under 18 years old
- Not being able to provide free and informed consent
- Have difficulty understanding and answering questions in French or English
- Have uncorrected vision problems

# Critères d'éligibilité

### Critères d'inclusion:

- Membres de la population générale
- Avoir au moins 18 ans
- Être capable de donner son consentement libre et éclairé et savoir lire et comprendre le français ou l'anglais
- Ne pas avoir des problèmes de vision non corrigés
- Être en mesure d'utiliser un ordinateur

## Critères d'exclusion:

- Avoir moins de 18 ans
- Être dans l'incapacité de donner un consentement libre et éclairé
- Avoir de la difficulté à comprendre et à répondre aux questions en français ou en anglais
- Avoir des problèmes de vision non corrigés

## **Interventions/Interventions**

- Explained above (in section study design)
- Expliqué ci-dessus (dans la section conception de l'étude)

## **Incentive / Incitatif**

We will use paid panels that offer a small incentive (typically \$1-1.50) to members of panels to complete surveys.

Nous aurons recours à des panels rémunérés offrant un petit incitatif (généralement de 1 à 50 USD) aux membres des panels pour leur permettre de répondre aux sondages.

## Outcomes / Résultats

In this study we are evaluating the effects of visualization on risk perception (for the individual, family, community, and vulnerable people in communities) (1st outcome) and on emotions, attitudes, knowledge, and behavioural intentions (2nd outcome) with trust as a covariate.

Dans cette étude, nous évaluons les effets de la visualisation sur la perception du risque (pour l'individu, la famille, la communauté et les personnes vulnérables dans les communautés) (1<sup>er</sup> résultat) et sur les émotions, les attitudes, les Connaissances et les intentions comportementales (2<sup>e</sup> résultat) en utilisant la confiance comme covariable.

# Participant timeline / Calendrier

Following ethics approval from Laval University, we will collect data online from **December 2020 to February 2021**.

Suite à l'approbation éthique de l'Université Laval, nous collecterons les données en ligne du décembre 2020 au février 2021.

# Sample size / Taille de l'échantillon

To determine the sample size for this between-subjects design, we assumed a small effect size (Cohen's f=0.10) and a statistical test power of 80% and 5% type 1 error, resulting in a required N of 320 participants for each arm with 75% of English and 25% of French speaking respondents which were sufficient to run our two-way analysis of variance. We estimated the sample size by using g power (Universität Düsseldorf: gpower) for continuous outcome.

Pour déterminer la taille de l'échantillon pour ce plan inter-sujets, nous avons supposé une petite taille d'effet (f=0,10 de Cohen) et une puissance de test statistique de 80% et 5% d'erreur de type 1, ce qui a donné un N requis de 320 participants pour chaque bras avec 75% de répondants anglophones et 25% de répondants francophones qui étaient suffisants pour effectuer notre analyse de variance à deux voies. Nous avons estimé la taille de l'échantillon en utilisant la puissance (Universität Düsseldorf: gpower ) pour un résultat continu.

# Recruitment / Recrutement

- The online randomized controlled trial will be run in Qualtrics, an online survey software.
- Eligible participants will be adult members of the general public in Canada (with a minimum of 25% of the sample with French as their preferred language compared to English).
- Participants will be recruited using established survey panels (subcontracted in Qualtrics).
- L'essai contrôlé randomisé en ligne sera exécuté dans Qualtrics, un logiciel de sondage en ligne.
- Les participants admissibles seront des membres adultes du grand public au Canada (au moins 25% de l'échantillon ayant le français comme langue préférée par rapport à l'anglais).
- Les participants seront recrutés sur des panels d'enquêtes établis (sous-traités dans Qualtrics)

# METHODS: Assignment of interventions (for controlled trials)/MÉTHODES: Attribution des interventions (pour les essais contrôlés)

## Allocation/Allocation:

# Sequence generation/Génération de séquences

This study will be simple randomized (computer generated randomization) to eliminate selection bias, balancing both known and unknown prognostic factors, in the assignment of interventions.

Cette étude utilisera une randomisation simple(randomisation générée par ordinateur) pour éliminer le biais de sélection, en équilibrant les facteurs pronostiques connus et inconnus, dans l'attribution des interventions.

## Allocation concealment mechanism/Mécanisme de dissimulation des attributions

This will be a single-blinded study because we cannot mask participants to the fact that they have been randomized to a visualization e.g., about measles. However, participants will not necessarily know the purpose of the study arm to which they are assigned, and investigators will be blinded to study arm during data analysis (investigators are not aware of whether the next eligible participant will be receiving treatment or control intervention).

Les participants et les investigateurs seront aveugles (à double insu) quant au processus d'attribution (les investigateurs ou les participants ne savent pas si le prochain participant éligible se verra attribué un traitement ou une intervention de contrôle).

# Implementation/ Implémentation

Qualtrics (computerized survey software) will use computerized randomization to automatically assign participants to interventions.

Qualtrics (logiciel d'enquête informatisé) utilisera la randomisation informatisée pour affecter automatiquement les participants aux interventions.

## Blinding (masking)/ Aveuglement (masquage)

This will be a single-blinded study because we cannot mask participants to the fact that they have been randomized to a visualization e.g., about measles. However, participants will not necessarily know the purpose of the study arm to which they are assigned, and investigators will be blinded to study arm during data analysis.

Ce sera une étude à simple insu car nous ne pouvons pas masquer aux participants le fait qu'ils ont été randomisés pour obtenir une visualisation p. ex., de la rougeole. Cependant, les participants ne connaîtront pas nécessairement le but du groupe d'étude auquel ils sont affectés et les investigateurs seront aveuglés pour étudier le groupe lors de l'analyse des données.

# METHODS: Data collection, management, and analysis/MÉTHODES: collecte, traitement et analyse des données

## Data collection methods/Méthodes de collecte des données

After seeking eligible participants' consent, participants will be randomized into different arms of the study and the effects of visualization on risk perception (for the individual, family, community, and vulnerable people in communities) (primary outcome) and on emotions, attitudes, knowledge, and behavioural intentions (secondary outcome) will be measured by questionnaire.

Après avoir recherché le consentement des participants éligibles, les participants seront randomisés dans différentes parties de l'étude et sur les effets de la visualisation sur la perception du risque (pour l'individu, la famille, la communauté et les personnes vulnérables dans les communautés) (résultat principal) et sur les émotions, les attitudes, les Connaissances et les intentions comportementales (résultat secondaire) seront mesurées par questionnaire.

# Data management/Traitement des données

All the information we collect will be confidential and used for research purposes only. In other words:

- Participant credentials will not be associated with the results of the study and no individual information will be presented in reports, publications or presentations.
- All data will be presented in aggregate form without individual identifiers.
- Data will be stored on Qualtrics servers located in Canada. When we work with data, the only
  people who will have access to our Qualtrics account will be the investigators and our team
  members who have complete and relevant ethics training. When the data is stored on our
  computers, each of our computers will be protected by a password. The data will be stored on
  a secure server, to which access is maintained and reserved for the members of the team
  (members of the team affiliated with Université Laval).

# After the end of the study:

- Anonymized data (answers to questions in the survey including socio-demographic
  information) will be deposited in a public repository (Dataverse de l'Université Laval (Laval
  University)) which will allow data sharing with the scientific community. No information that
  would allow anyone to identify a person will be deposited in this public repository.
- Any other electronic data will be destroyed in June 2027.

Toutes les informations que nous recueillons seront confidentielles et utilisées uniquement à des fins de recherche. En d'autres termes:

- Les informations d'identification des participants ne seront pas associées aux résultats de l'étude et aucune information individuelle ne sera présentée dans des rapports, des publications ou des présentations.
- Toutes les données seront présentées sous forme agrégée, sans identificateurs individuels.
- Les données seront enregistrées sur les serveurs de Qualtrics situés au Canada. Lorsque nous travaillons avec des données, les seules personnes qui auront accès à notre compte Qualtrics seront les enquêteurs et les membres de notre équipe qui ont toute la formation éthique complète et pertinente. Lorsque les données seront stockées sur nos ordinateurs, chacun de nos ordinateurs sera protégé par un mot de passe. Les données seront stockées sur un serveur sécurisé, auquel l'accès est maintenu et réservé aux membres de l'équipe (membres de l'équipe affiliés à l'Université Laval).

# Après la fin de l'étude :

- Les données anonymisées (réponses aux questions de l'enquête y inclus les informations sociodémographiques) seront déposées dans un dépôt public (Dataverse de l'Université Laval) qui permettra le partage des données avec la communauté scientifique. Aucune information qui permettrait d'identifier une personne ne sera déposée dans ce dépôt public.
- Toute autre donnée électronique sera détruite en juin 2027.

# Statistical methods/Méthodes statistiques

The type of comparison between intervention and control groups will be analyzed and reported as a superiority trial. The comparison will be done by using a linear regression for statistical analysis of continuous data.

Le type de comparaison entre le groupe d'intervention et le groupe de contrôle sera analysé et présenté comme un essai de supériorité. La comparaison sera effectuée en utilisant une régression linéaire pour l'analyse statistique des données continues.

| Variables/ outcomes | Visualization (Herdimm) | Control 1(no visualization/ no education about community immunity) |
|---|---|---|
| Risk perception | | |
| Emotions | | |
| Attitudes | | |
| Knowledge | | |
| Behavioural intentions | | |
| Trust | | |

| Variables/<br>outcomes | Visualization<br>(Herdimm) | Measles:<br>Guardian<br>visualization | Measles:<br>theotheredmun<br>d visualization | Influenza: Public<br>Health Agency of<br>Canada Flu:<br>Don't Pass It On! |
|---|---|---|---|---|
| Risk<br>perception | | | | |
| Emotions | | | | |
| Attitudes | | | | |
| knowledge | | | | |
| Behavioural intentions | | | | |
| Trust | | | | |

| Variables/<br>outcomes | Visualization<br>(Herdimm) | Generic: Robert<br>Koch Institut<br>visualization | Generic: SBS<br>News<br>visualization | Generic: NHS<br>visualization |
|---|---|---|---|---|
| Risk<br>perception | | | | |
| Emotions | | | | |
| Attitudes | | | | |
| Knowledge | | | | |
| Behavioural intentions | | | | |
| Trust | | | | |

# ETHICS AND DISSEMINATION/ÉTHIQUE ET DIFFUSION

# Research ethics approval/Approbation de l'éthique de la recherche

This study is approved from the Laval University ethics committee (Approval No. 2017-137 Phase II A-6/10-09-2020).

Approbation de l'éthique de la recherche Cette étude est approuvée par le comité d'éthique de l'Université Laval (Approbation  $n^{\circ}$  2017-137 Phase II A-6/10-09-2020).

## Consent/Consentement

The free and informed consent will be seeked before the start of the study. Participants will be able to withdraw from the study at anytime if they don't want to take part in the study. Participants who withdrew from the study in the middle and has not completed the study their data won't be analysed.

Le consentement libre et éclairé sera recherché avant le début de l'étude. Les participants pourront se retirer de l'étude à tout moment s'ils ne veulent pas participer à l'étude. Les participants qui se sont retirés de l'étude au milieu et qui n'ont pas terminé l'étude ne seront pas analysés.

# Confidentiality/Confidentialité

- Explained in the data management section above.
- Expliqué dans la section sur le **traitement des données** ci-dessus.

## Declaration of interests/Déclaration d'intérêts

- No competing interests.
- Pas de conflits d'intérêts.

## Access to data/Accès aux données

The data will be kept in the principal investigator's laboratory located on the campus of Laval University and only members of the research team will have access to data.

The data will be stored on Qualtrics Canadian servers, located in Canada and subject to Canadian data protection laws. When we work with data the only people who will have access to our Qualtrics account will be investigators and our team members who have all complete and relevant ethics training. When the data will be held on our computers each of our computers will be protected by the password. The data will be stored on a secure server, to which access is maintained and restricted to team members (team members affiliated at Laval university).

Les données seront conservées dans le laboratoire du chercheur principal situé sur le campus de l'Université Laval et seuls les membres de l'équipe de recherche auront accès aux données.

Les données seront stockées sur des serveurs canadiens de Qualtrics, situés au Canada. Lorsque nous travaillons avec des données, les seules personnes qui auront accès à notre compte Qualtrics seront les enquêteurs et les membres de notre équipe qui ont toute la formation éthique complète et pertinente. Lorsque les données seront stockées sur nos ordinateurs, chacun de nos ordinateurs sera protégé par un mot de passe. Les données seront stockées sur un serveur sécurisé, auquel l'accès est maintenu et réservé aux membres de l'équipe (membres de l'équipe affiliés à l'université Laval).

# Dissemination policy/Politique de diffusion

We intend to publish our results in a peer reviewed journal for healthcare professionals, the public, and other relevant groups to access.

Nous avons l'intention de publier nos résultats dans une revue évaluée par des pairs, à laquelle les professionnels de la santé, le public et d'autres groupes concernés pourront accéder.

## Factors:

| Factors: | <u>Facteurs</u> : |
|---|---|
| Visualization (Herdimm) | Visualization (Herdimm) |
| Control 1(no visualization/ no education about community immunity) | Contrôle 1 (pas de visualisation / pas d'éducation sur l'immunité de la communauté) |
| Control 2 (Guardian visualization) | Contrôle 2 (visualization Guardian) |
| Control 3(Robert Koch Institut visualization) | Contrôle 3 (visualization Robert Koch Institut ) |
| Control 4(theotheredmund visualization) | Contrôle 4 (visualization theotheredmund) |
| Control 5 (SBS news visualization) | Contrôle 5 (SBS news visualization) |
| Control 6 (NHS visualization) | Contrôle 6 (NHS visualization) |
| Control 7 (Flu: Public Health Agency of Canada<br>Flu: Don't Pass It On!) | Contrôle 7 (Flu: Public Health Agency of<br>Canada Flu: Don't Pass It On!) |

## Measures

| Measures: | Mesures : |
|---|---|
| Risk perception (primary outcome) | Perception du risque (résultat principal) |
| Emotions (secondary outcome) | Émotions (résultat secondaire) |
| Attitudes (secondary outcome) | Attitudes (résultat secondaire) |
| Knowledge (secondary outcome) | Connaissances (résultat secondaire) |
| Behavioural intentions (secondary outcome) | Intentions comportementales (résultat secondaire) |
| Trust (Covariates) | Confiance (covariables) |

## Randomized variables:

| Randomized variables: | | Valeurs randomisées : |
|---|---|---|
| visualization | 0= No education 1 = Herdimm 2 = Guardian visualization 3 = Robert Koch Institut visualization 4= theotheredmund visualization 5=SBS news visualization 6= NHS visualization 7= Flu: Public Health Agency of Canada | 0= No education 1 = Herdimm 2 = visualization Guardian 3 = visualization Robert Koch Institut 4= visualization theotheredmund 5= SBS news visualization 6= NHS visualization 7= Flu: Public Health Agency of Canada |

## References:

- Betsch, Cornelia, Robert Böhm, Lars Korn, and Cindy Holtmann. 2017. "On the Benefits of Explaining Herd Immunity in Vaccine Advocacy." *Nature Human Behaviour* 1 (3): s41562–017 0056.
- Betsch, Cornelia, Philipp Schmid, Dorothee Heinemeier, Lars Korn, Cindy Holtmann, and Robert Böhm. 2018. "Beyond Confidence: Development of a Measure Assessing the 5C Psychological Antecedents of Vaccination." *PloS One* 13 (12): e0208601.
- Gallis, John A., Gary G. Bennett, Dori M. Steinberg, Sandy Askew, and Elizabeth L. Turner. 2019. "Randomization Procedures for Multicomponent Behavioral Intervention Factorial

- Trials in the Multiphase Optimization Strategy Framework: Challenges and Recommendations." *Translational Behavioral Medicine*. https://doi.org/10.1093/tbm/iby131.
- Hakim, Hina, Thierry Provencher, Christine T. Chambers, S. Michelle Driedger, Eve Dube, Teresa Gavaruzzi, Anik M. C. Giguere, et al. 2018. "Interventions to Help People Understand Community Immunity: A Systematic Review." *Vaccine*, December. https://doi.org/10.1016/j.vaccine.2018.11.016.
- Healey, Christopher G., and James T. Enns. 2012. "Attention and Visual Memory in Visualization and Computer Graphics." *IEEE Transactions on Visualization and Computer Graphics* 18 (7): 1170–88.
- "Universität Düsseldorf: Gpower." n.d. Accessed July 28, 2020. https://www.psychologie.hhu.de/arbeitsgruppen/allgemeine-psychologie-und-arbeitspsychologie/gpower.html.

# S2: Study questionnaire

# contag\_phase3b

Start of Block: Introduction

Intro Project Description

# **Project Description**

## Introduction

Thank you for participating in this study. This project is a collaboration with University Laval, Public Health Ontario (PHO) and The National Institute of Public Health of Quebec (INSPQ).

In this study, we will first give you some information to do with contagious diseases and then ask you to answer some questions.

The survey will take about 15 to 20 minutes. Your name will not be recorded anywhere in this survey. Researchers will not be able to associate your name with your answers. If you choose to leave the study, you can stop at any time. You may choose not to answer any questions you don't want to answer. If, for some reason, you cannot complete the survey, you may **restart** the survey at a later time by clicking on the survey link in your email invitation. You will have to **restart** the survey from the beginning.

If you become worried about your health while taking this survey, please talk to a healthcare provider.

### About the researchers

This study is a PhD project conducted by Ms. Hina Hakim, PhD student, supervised by Holly O. Witteman, PhD, professor and researcher in the Faculty of Medicine at Laval University. Ms. Hakim is co-supervised by Dr. Daniel Reinharz, professor and researcher in the Faculty of Medicine at Laval University.

## Purpose of the study

The purpose of this study is to evaluate the effects of information to do with contagious diseases on risk perception, knowledge, emotions, attitudes, beliefs, and behavioural intentions.

# What your participation entails

Participating in this study will involve following:

- Answering survey questions.
- You may be asked to view or listen to information, which will require either the ability to read or hear.

You may be asked to briefly visit another website in the middle the survey.

## Risks and benefits

The risks associated with participating in the study, specifically:

- Information and questions, we ask may make you feel uncomfortable or anxious. We suggest you to consult your healthcare professional, as the case may be;
- You may feel some discomfort having to focus on a computer screen.
- You may feel some fatigue from concentrating throughout the survey.

There is no personal benefit to participate in this study, however, the information we gather will help us to evaluate the effects of the information, which may help in improving the way health information is shared, and population health.

Your help means a lot to us. We thank you again for taking the time to complete this survey.

## Confidentiality and data protection

All information we collect will be confidential and used only for research purposes. In other words:

- Participant credentials will not be associated with the results of the study and no individual information will be presented in reports, publications or presentations.
- All data will be presented in aggregate form without individual identifiers.
- Data will be stored on Qualtrics servers located in Canada. When we work with data, the
  only people who will have access to our Qualtrics account will be the investigators and
  our team members who have complete and relevant ethics training. When the data is
  stored on our computers, each of our computers will be protected by a password. The
  data will be stored on a secure server, to which access is maintained and reserved for the
  members of the team (members of the team affiliated with Université Laval).

# After the end of the study:

- Anonymized data (answers to questions in the survey including socio-demographic
  information) will be deposited in a public repository (Dataverse de l'Université Laval
  (Laval University)) which will allow data sharing with the scientific community. No
  information that would allow anyone to identify a person will be deposited in this public
  repository.
- Any other electronic data will be destroyed in June 2027.

# Contact people

If you have any questions about the research study, or if you experience a problem as a result of participating in the study, please contact:

Holly Witteman Laval University

Tel: (418) 656-2131 ext: 403981 Email: holly.witteman@fmed.ulaval.ca

If you have concerns about your rights as a participant in this study or any complaints, you can communicate with the University Laval Ombudsman at:

Pavillon Alphonse-Desjardins 2325, rue de l'Université, Local 3320 Québec, QC G1V 0A6 Tel: 418-656-3081

Toll free: 1-866-323-2271

Email: info@ombudsman.ulaval.ca

This project has been approved by Laval University Research Ethics Board: Approval No. 2017-137 Phase II A-6/10-09-2020

## Description du projet

## Introduction

Merci de participer à cette étude. Ce projet est réalisé en collaboration avec l'Université Laval, Santé publique Ontario (SPO) et l'Institut national de la santé publique du Québec (INSPQ).

Dans cette étude, nous vous donnerons d'abord quelques informations sur les maladies contagieuses et nous vous demanderons ensuite de répondre à quelques questions.

L'enquête durera environ 15 à 20 minutes. Votre nom ne sera enregistré nulle part dans cette enquête. Les chercheurs et les chercheuses ne pourront pas associer votre nom à vos réponses. Si vous choisissez de quitter l'étude, vous pouvez y mettre fin à tout moment. Vous pouvez choisir d'ignorer les questions auxquelles vous ne voulez pas répondre. Si, pour une raison quelconque, vous ne pouvez pas compléter le sondage, vous pourrez le recommencer ultérieurement en cliquant sur le lien du sondage dans votre invitation par courrier électronique. Vous devrez alors **recommencer** le sondage depuis le début.

Si vous ressentez de l'inquiétude pour votre santé en répondant à cette enquête, parlez-en à un.e professionnel.le de la santé.

## À propos des chercheurs

Cette étude est un projet de doctorat conduit par Mme Hina Hakim, candidate au doctorat en santé communautaire, supervisée par Mme Holly Witteman, Ph.D., professeure et chercheuse à la Faculté de médecine de l'Université Laval. Mme Hakim est co-dirigée par le Dr Daniel Reinharz, professeur et chercheur à la Faculté de médecine de l'Université Laval.

# Aperçu de l'étude

Le but de cette étude est d'évaluer l'effet de certaines informations relatives aux maladies contagieuses sur la perception du risque, la connaissance, les émotions, les attitudes, les croyances et les intentions comportementales.

# Ce que votre participation implique

Participer à cette étude impliquera de :

- Répondre aux questions du sondage
- Il se peut qu'on vous demande de lire ou d'écouter des informations, ce qui nécessiterait la capacité de voir ou d'entendre
- Il se peut que l'on vous demande de visiter brièvement un autre site web au milieu de l'enquête.

# Risques et avantages

Il existe certains risques associés à la participation à l'étude, notamment :

- Les informations et questions posées pourraient vous rendre mal à l'aise ou anxieux. Nous vous suggérons de consulter votre professionnel.le de la santé;
- Vous pouvez ressentir un certain inconfort à fixer un écran d'ordinateur.
- Vous pourriez ressentir de la fatigue due à la concentration demandée tout au long du sondage.

Il n'y a aucun avantage personnel à participer à cette étude. Toutefois, les données recueillies nous aideront à évaluer les effets des informations transmises, ce qui pourrait aider à améliorer le partage des informations sur la santé ainsi que la santé de la population.

Votre aide compte beaucoup pour nous. Nous vous remercions encore de prendre le temps de répondre à ce sondage.

## Confidentialité et protection des données

Toutes les informations que nous recueillons seront confidentielles et utilisées uniquement à des fins de recherche.

En d'autres termes:

- Les informations d'identification des participant.e.s ne seront pas associées aux résultats de l'étude et aucune information individuelle ne sera présentée dans des rapports, des publications ou des présentations.
- Toutes les données seront présentées sous forme agrégée, sans identificateurs individuels.
- Les données seront enregistrées sur les serveurs de Qualtrics situés au Canada. Lorsque nous travaillons avec des données, les seules personnes qui auront accès à notre compte Qualtrics seront les enquêteurs et les membres de notre équipe qui ont toute la formation éthique complète et pertinente. Lorsque les données seront stockées sur nos ordinateurs, chacun de nos ordinateurs sera protégé par un mot de passe. Les données seront stockées sur un serveur sécurisé, auquel l'accès est maintenu et réservé aux membres de l'équipe (membres de l'équipe affiliés à l'Université Laval).

# Après la fin de l'étude :

- Les données anonymisées (réponses aux questions de l'enquête y inclus les informations sociodémographiques) seront déposées dans un dépôt public (Dataverse de l'Université Laval) qui permettra le partage des données avec la communauté scientifique. Aucune information qui permettrait d'identifier une personne ne sera déposée dans ce dépôt public.
- Toute autre donnée électronique sera détruite en juin 2027.

## Contact

Si vous avez des questions sur le projet de recherche, ou si vous rencontrez un problème en participant à l'étude, veuillez contacter:

Prof. Holly Witteman Université Laval

Téléphone: (418) 656-2131 ext: 403981 Courriel: holly.witteman@fmed.ulaval.ca

Si vous avez des plaintes ou des préoccupations au sujet de vos droits en tant que participant à cette étude, vous pouvez communiquer avec l'Ombudsman de l'Université Laval à:

Pavillon Alphonse-Desigrdins 2325, rue de l'Université, Local 3320

Québec, QC G1V 0A6 Téléphone: 418-656-3081 Sans frais: 1-866-323-2271

Courriel: info@ombudsman.ulaval.ca

« Ce projet a été approuvé par le Comité d'éthique de la recherche de l'Université Laval : No d'approbation 2017-137 Phase II A-6/10-09-2020 »

t\_intro Timing

First Click (1)

Last Click (2)

Page Submit (3)

Click Count (4)

t intro Durée

First Click (1)

Last Click (2)

Page Submit (3)

Click Count (4)

End of Block: Introduction

Start of Block: Consent for participation:



### Consent

- 1. I have been informed about the nature and purpose of this study and the research procedures.
- 2. I was informed in English which is a language I understand fluently.
- 3. I understand that my participation in this study is voluntary and that I can withdraw at any time without penalty or consequences of any kind.
- 4. I understand that the information collected is confidential and will only be used for research purposes.
- 5. I have read the project description and informed consent form and I voluntarily agree to participate in this study.

| $\bigcirc$ | Yes | I Consent | (1) |
|---------------|------|-----------|------|
| $\overline{}$ | 1 00 | CONSCIIL | ('') |

No I do not Consent (0)

#### Consent

- 1. J'ai été informé.e de la nature et du but de cette étude et des procédures de recherche.
- 2. J'ai été informé.e en français, une langue que je comprends et parle couramment.
- 3. Je comprends que ma participation à cette étude est volontaire et que je peux me retirer à tout moment sans pénalité ni conséquence d'aucune sorte.

| 5. | Je comprends que les informations recueillies sont confidentielles et ne seront utilisées qu'à des fins de recherche. J'ai lu la description du projet et le formulaire de consentement éclairé et j'accepte volontairement de participer à cette étude. |
|---|---|
| $\circ$ | Oui, je consens (1) |
| $\circ$ | Non, je n'y consens pas (0) |
| Skip To<br>researc | : End of Survey If I have been informed about the nature and purpose of this study and the<br>h procedures. I wa = No I do not Consent |
| First Cl<br>Last Cl<br>Page S | |
| First Cl<br>Last Cl<br>Page S | |
| Page E | Break ———————————————————————————————————— |

| End of Block: Consent for participation: |
|--------------------------------------------------------------------|
| Start of Block: Standard Sociodemo Canada |
| yearofbirth In what year were you born? |
| ▼ Prefer not to answer (888) 2010 (2010) |
| yearofbirth Quelle est votre année de naissance? |
| ▼ Je préfère ne pas répondre (888) 2010 (2010) |
| $\chi_{\rightarrow}$ |
| bornincanada Were you born in Canada? (Check one only.) |
| O Prefer not to answer (888) |
| O Yes (1) |
| O No - What year did you arrive in Canada? (0) |
| bornincanada Êtes-vous né(e) au Canada? (Cochez une seule réponse) |
| O Je préfère ne pas répondre (888) |
| Oui (1) |
| O Non - en quelle année êtes-vous arrivé(e) au Canada? (0) |
| Display This Question: If If False |

*^* 

| ΠP | hp Were you born outside North America? (Check one only.) |
|---|---|
| | O Prefer not to answer (888) |
| | ○ Yes (1) |
| | No - What year did you arrive in North America? (0) |
| hp l | ites-vous né(e) hors de l'Amérique du Nord? (Cochez une seule réponse) |
| | O Je préfère ne pas répondre (888) |
| | Oui (1) |
| | Non - en quelle année êtes-vous arrivé(e) au Canada? (0) |
| X→ | |
| | uage What language would you feel most comfortable speaking in with your healthcare ider? (doctor, nurse, dentist, pharmacist)? (Check all that apply.) |
| | Prefer not to answer (888) |
| | ☐ English (1) |
| | English (1) |
| | ☐ French (2) |

| a santé (méd | decin, infirmière, dentiste, pharmacien)? (Cochez tout ce qui s'applique) |
|---|---|
| | Je préfère ne pas répondre (888) |
| | Anglais (1) |
| | Français (2) |
| | Autre, précisez : (3) |

language Dans quelle(s) langue(s) êtes-vous à l'aise pour parler avec un.e professionnel.le de

| ethnicity Which apply.) | h of the following best describes your racial or ethnic group(s)? (Check all that |
|---|---|
| | Prefer not to answer (888) |
| | Asian - East (e.g., Chinese, Japanese, Korean) (1) |
| | Asian - Central (e.g., Kazakhstani, Uzbekistani) (2) |
| | Asian - South (e.g., Indian, Pakistani, Sri Lankan) (3) |
| | Asian - South-East (e.g., Malaysian, Filipino, Vietnamese) (4) |
| | Black - African (e.g., Ghanaian, Kenyan, Somali) (13) |
| | Black - Caribbean (e.g., Barbadian, Jamaican) (14) |
| | Black - North American (e.g., Canadian, American) (15) |
| | First Nations (16) |
| Quechua) | Indigenous or aboriginal person from outside of North America (e.g., Maori, (5) |
| | Inuit (8) |
| | Latin American (e.g., Chilean, Mexican, Salvadorian) (9) |
| | Metis (Metis Nation in Canada) (10) |
| | Middle Eastern (e.g., Egyptian, Iranian, Lebanese) (12) |
| | North African (e.g., Moroccan, Tunisian) (11) |
| | White - European (e.g., English, Italian, Portuguese, Russian) (6) |
| | White - North American (e.g., Canadian, American) (7) |

| Other, please specify: (17) |
|-----------------------------|
|-----------------------------|

| | Je préfère ne pas répondre (888) |
|---|---|
| | Asiatique de l'est (p.ex. : Chinois, Japonais, Coréen) (1) |
| | Asiatique du centre (p.ex. : Kazakh, Ouzbek) (2) |
| | Asiatique du sud (p.ex.: Indien, Pakistanais, Sri Lankais) (3) |
| | Asiatique du sud-est (p.ex.: Malaisien, Philippin, Vietnamien) (4) |
| | Noir Africain (p.ex. : Ghanéen, Kenyan, Somalien) (13) |
| | Noir Caribéen (p.ex. : Barbadien, Jamaïcain) (14) |
| | Noir Nord-américain (p.ex.: Canadien, États-Unien) (15) |
| | Premières Nations (16) |
| (5) | Autochtone ou aborigène de hors de l'Amérique du Nord (p.ex.: Maori, Quechua) |
| | Inuit (8) |
| | Latino-américain (p.ex. : Chilien, Mexicain, Salvadorien) (9) |
| | Métis (Nation métisse du Canada) (10) |
| | Moyen-oriental (p.ex. : Égyptien, Iranien, Libanais) (12) |
| | Maghrébin (p.ex. : Marocain, Tunisien) (11) |
| | Blanc Européen (p.ex.: Français, Anglais, Italien, Portugais, Russe) (6) |

ethnicity Laquelle ou lesquelles des catégories suivantes représente(nt) vos groupes raciaux ou

ethniques? (Cochez tout ce qui s'applique.)

| Blanc Nord-Américain (p.ex.: Canadien, États-Unien) (7) |
|---|
| Autre, précisez : (17) |
| X+ |
| disability Do you consider yourself to have a disability (e.g, physical disability, sensory disability (e.g., hearing or vision loss), chronic illness, learning disability, mental illness, developmental disability or other)? (Check one only.) |
| ☐ Prefer not to answer (888) |
| ○ □ No disability (0) |
| ☐ Yes, at least one disability (1) |
| disability Considérez-vous avoir une limitation ou un handicap (p.ex. : limitation ou déficience physique, limitation ou déficience sensorielle (p.ex. perte de vision ou d'audition), maladie chronique, trouble d'apprentissage, trouble de santé mentale, trouble du développement ou autre)? (Cochez une seule réponse.) |
| O Je préfère ne pas répondre (888) |
| O Non, aucune limitation ou handicap (0) |
| Oui, au moins une limitation ou handicap (1) |
| $X^{\Rightarrow}$ |
| techdisability Do you have a disability that limits your access to technology and computer based tools (p.ex. : computer, tablet, interactive terminal)? (Check one only.) |
| ☐ Prefer not to answer (888) |
| O No (0) |
| ○ Yes (1) |

| techdisability Selon vous, avez-vous une limitation ou un handicap qui vous limite l'accès à certains outils technologiques ou informatiques (p.ex. : ordinateur, tablette, borne interactive)? (Cochez une seule réponse.) |
|---|
| O Je préfère ne pas répondre (888) |
| O Non (0) |
| Oui (1) |
| $\chi_{\to}$ |
| sexatbirth What sex were you assigned at birth, meaning on your original birth certificate? (Check one only.) |
| O Prefer not to answer (888) |
| O Female (1) |
| O Male (2) |
| sexatbirth Quel sexe vous a-t-on assigné à la naissance, sur votre certificat de naissance original? (Cochez une seule réponse.) |
| O Je préfère ne pas répondre (888) |
| O Féminin (1) |
| O Masculin (2) |
| X+ |

| genderidentity Do you consider yourself: (Check one only.) |
|---|
| O Female (1) |
| O Male (2) |
| O Indigenous or other cultural gender minority identity (e.g., two-spirit) (3) |
| O Something else (e.g. non-binary, gender fluid) (4) |
| O Prefer not to answer (888) |
| genderidentity Vous considérez-vous comme : (Cochez une seule réponse.) |
| O Une femme (1) |
| O Un homme (2) |
| <ul> <li>Un(e) minorité de genre culturelle, autochtone ou autre (p.ex. : bispiritualité, « two-spirit</li> <li>») (3)</li> </ul> |
| O Autre (p.ex. : non-binaire, « gender fluid ») (4) |
| O Je préfère ne pas répondre (888) |
| X |
| income What was your total family income before taxes last year? (Check one only.) |
| ☐ Prefer not to answer (888) |
| ◯ □ 24 999 or less (1) |
| ○ □ 25 000 to 49 999 (2) |
| ○ □ 50 000 to 99 999 (3) |
| ☐ 100 000 or more (4) |
| ◯ □ Do not know (5) |

| seule réponse.) |
|-----------------------------------------------------------------|
| O Je préfère ne pas répondre (888) |
| O 24 999 et moins (1) |
| O 25 000 à 49 999 (2) |
| O 50 000 à 99 999 (3) |
| O 100 000 ou plus (4) |
| O Je ne sais pas (5) |
| supportedbyincome How many people does this income support? |
| O Number of people: (1) |
| O Prefer not to answer (888) |
| supportedbyincome Combien de personnes ce revenu supporte-t-il? |
| O Nombre de personnes : (1) |
| O Je préfère ne pas répondre (888) |

| educatio | onlevel What is the highest level of education you have completed? (Check one only.) |
|---|---|
| 0 | Prefer not to answer (888) |
| 0 | Elementary School (completed or not) (1) |
| 0 | High School Diploma (2) |
| 0 | Apprenticeship or trade certificate or diploma (3) |
| 0 | College or polytechnical school certificate or diploma (4) |
| 0 | University degree, bachelor level or below (5) |
| 0 | University graduate degree (Master's level) (6) |
| 0 | University graduate degree (Doctorate level) (7) |
| 0 | Do not know (8) |
| education<br>réponse | onlevel Quel est votre plus haut niveau de scolarité complété? (Cochez une seule s.) |
| 0. | Je préfère ne pas répondre (888) |
| O E | ○ Études primaires (complétées ou non) (1) |
| $\circ$ | O Diplôme d'études secondaires (2) |
| $\bigcirc$ ( | Certificat ou diplôme d'apprentissage ou de métier (3) |
| $\bigcirc$ A | Attestation ou diplôme d'études professionnelles (DES, ASP, DEP) (4) |
| O E | Études universitaires de premier cycle (Certificat, Baccalauréat) ou moins (5) |
| O E | Études universitaires de deuxième cycle (DESS, Maîtrise) (6) |
| ○ Études universitaires de troisième cycle (Doctorat) (7) | |
| 0. | Je ne sais pas (8) |

| t_sociodemographic Timing First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
|---|
| t_sociodemographic Durée First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
| End of Block: Standard Sociodemo Canada |
| Start of Block: Individualism and Collectivism Scale - Triandis1998 - EN/FR |
| ih1 Evaluate how well each of the following statements applies to you: |
| I'd rather depend on myself rather than others. |
| O Never or definitely not =1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| Always or definitely yes = 9 (9) |

ih1
Évaluez à quel point chacun des énoncés suivants s'applique à vous :

Je préfère dépendre de moi-même que des autres

Jamais ou définitivement non = 1 (1)

2 (2)

3 (3)

4 (4)

5 (5)

6 (6)

7 (7)

8 (8)

O Toujours ou définitivement oui = 9 (9)

| ih2 I rely on myself most of the time, I rarely rely on others. |
|--------------------------------------------------------------------|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Always or definitely yes = 9 (9) |
| ih2 Je me fie à moi-même la plupart du temps, rarement aux autres. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |
| ih3 | I often do "my own thing." |
|-----|------------------------------------------|
| | O Never or definitely not = 1 (1) |
| | O 2 (2) |
| | O 3 (3) |
| | O 4 (4) |
| | O 5 (5) |
| | O 6 (6) |
| | O 7 (7) |
| | O 8 (8) |
| | Always or definitely yes = 9 (9) |
| ih3 | Je fais souvent « ma propre affaire. » |
| | O Jamais ou définitivement non = 1 (1) |
| | O 2 (2) |
| | O 3 (3) |
| | O 4 (4) |
| | O 5 (5) |
| | O 6 (6) |
| | O 7 (7) |
| | O 8 (8) |
| | O Toujours ou définitivement oui = 9 (9) |

| ih4 My personal identity, independent of others, is very important to me. |
|---|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Always or definitely yes = 9 (9) |
| ih4 Mon identité personnelle, indépendante des autres, est très importante pour moi. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |

| iv1 It is important that I do my job better than others. |
|--------------------------------------------------------------------------|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Always or definitely yes = 9 (9) |
| iv1 II est important pour moi de faire mon travail mieux que les autres. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |

| iv2 Winning is everything. |
|------------------------------------------|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Always or definitely yes = 9 (9) |
| iv2 Gagner, c'est tout ce qui compte. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |

| iv3 Competition is the law of nature. |
|---------------------------------------------|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| ○ 8 (8) |
| O Always or definitely yes = 9 (9) |
| iv3 La compétition est la loi de la nature. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |

| 174 When another person does better than 1 do, 1 get tense and aroused. |
|-----------------------------------------------------------------------------|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Always or definitely yes = 9 (9) |
| iv4 Quand une autre personne fait mieux que moi, je deviens tendu et agité. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |

| ch'i if a coworker gets a prize, i would feel proud. |
|--------------------------------------------------------------|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| ○ 8 (8) |
| O Always or definitely yes = 9 (9) |
| ch1 Si un collègue remportait un prix, je me sentirais fier. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |

| ch2 The well-being of my coworkers is important to me. |
|-----------------------------------------------------------|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| ○ 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| ○ 8 (8) |
| O Always or definitely yes = 9 (9) |
| ch2 Le bien-être de mes collègues est important pour moi. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| ○ 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |

| ch3 To me, pleasure is spending time with others. |
|--------------------------------------------------------------------|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| ○ 8 (8) |
| O Always or definitely yes = 9 (9) |
| ch3 Pour moi, le plaisir c'est de passer du temps avec les autres. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |

| ch4 I feel good when I cooperate with others. |
|---------------------------------------------------------|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Always or definitely yes = 9 (9) |
| ch4 Je me sens bien lorsque je coopère avec les autres. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |

| cvi Falents and children must stay together as much as possible. |
|-----------------------------------------------------------------------------|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Always or definitely yes = 9 (9) |
| cv1 Les parents et les enfants doivent rester ensemble autant que possible. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |

| cv2 It is my duty to take care of my family, even when I have to sacrifice what I want. |
|---|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Always or definitely yes = 9 (9) |
| cv2 C'est mon devoir de prendre soin de ma famille, même si je dois sacrifier mes propres |
| désirs. |
| O Jamais ou définitivement non = 1 (1) |
| O Jamais ou définitivement non = 1 (1) |
| <ul><li>Jamais ou définitivement non = 1 (1)</li><li>2 (2)</li></ul> |
| <ul><li>Jamais ou définitivement non = 1 (1)</li><li>2 (2)</li><li>3 (3)</li></ul> |
| <ul> <li>Jamais ou définitivement non = 1 (1)</li> <li>2 (2)</li> <li>3 (3)</li> <li>4 (4)</li> </ul> |
| <ul> <li>Jamais ou définitivement non = 1 (1)</li> <li>2 (2)</li> <li>3 (3)</li> <li>4 (4)</li> <li>5 (5)</li> </ul> |
| <ul> <li>Jamais ou définitivement non = 1 (1)</li> <li>2 (2)</li> <li>3 (3)</li> <li>4 (4)</li> <li>5 (5)</li> <li>6 (6)</li> </ul> |
| <ul> <li>Jamais ou définitivement non = 1 (1)</li> <li>2 (2)</li> <li>3 (3)</li> <li>4 (4)</li> <li>5 (5)</li> <li>6 (6)</li> <li>7 (7)</li> </ul> |

| cv3 Family members should stick together, no matter what sacrifices are required. |
|---|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| ○ 8 (8) |
| O Always or definitely yes = 9 (9) |
| cv3 Les membres d'une même famille devraient être solidaires peu importe les sacrifices requis. |
| O Jamais ou définitivement non = 1 (1) |
| O Jamais ou définitivement non = 1 (1) O 2 (2) |
| O 2 (2) |
| O 2 (2) O 3 (3) |
| <ul><li>2 (2)</li><li>3 (3)</li><li>4 (4)</li></ul> |
| <ul><li>2 (2)</li><li>3 (3)</li><li>4 (4)</li><li>5 (5)</li></ul> |
| <ul> <li>2 (2)</li> <li>3 (3)</li> <li>4 (4)</li> <li>5 (5)</li> <li>6 (6)</li> </ul> |
| <ul> <li>2 (2)</li> <li>3 (3)</li> <li>4 (4)</li> <li>5 (5)</li> <li>6 (6)</li> <li>7 (7)</li> </ul> |

| cv4 It is important to me that I respect the decisions made by my groups. |
|---|
| O Never or definitely not = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Always or definitely yes = 9 (9) |
| cv4 II est important pour moi de respecter les décisions prises par mes groupes. |
| O Jamais ou définitivement non = 1 (1) |
| O 2 (2) |
| O 3 (3) |
| O 4 (4) |
| O 5 (5) |
| O 6 (6) |
| O 7 (7) |
| O 8 (8) |
| O Toujours ou définitivement oui = 9 (9) |

t\_ic Timing
First Click (1)

Last Click (2)

Page Submit (3)

Click Count (4)

t ic Durée

First Click (1)

Last Click (2)

Page Submit (3)

Click Count (4)

End of Block: Individualism and Collectivism Scale - Triandis1998 - EN/FR

Start of Block: media

## Display This Question:

If viz = 0

control Now we need your answers to some questions about contagious diseases.

control Nous avons maintenant également besoin de votre avis sur certaines questions concernant les maladies contagieuses.

\_\_\_\_\_

## Display This Question:

If viz = 1

Or viz = 2

robertkochgeneric Now you will visit another website with some information about contagious diseases.

When you are done, please come back here to finish the survey.

robertkochgeneric Vous allez maintenant visiter un autre site web contenant des informations sur les maladies contagieuses.

Lorsque vous aurez terminé, revenez ici pour terminer ce sondage, s'il vous plaît.

\_\_\_\_\_

```
Display This Question:

If viz = 1

And disease = 0

And voice = 1
```

herdimmgenericmale Please click here to go to the other website

herdimmgenericmale Veuillez cliquer ici pour accéder à l'autre site web

\_\_\_\_\_

```
Display This Question:

If viz = 1

And disease = 0

And voice = 2
```

herdimmgenericfemale Please click here to go to the other website

herdimmgenericfemale Veuillez cliquer ici pour accéder à l'autre site web

\_\_\_\_\_

```
Display This Question:

If viz = 1

And disease = 1

And voice = 1
```

herdimmmeaslesmale Please click here to go to the other website

herdimmmeaslesmale Veuillez cliquer ici pour accéder à l'autre site web

\_\_\_\_\_

```
Display This Question:

If viz = 1

And disease = 1

And voice = 2
```

herdimmmeaslesfemale Please click here to go to the other website

herdimmmeaslesfemale Veuillez cliquer ici pour accéder à l'autre site web

\_\_\_\_\_

```
Display This Question:

If viz = 1

And disease = 2

And voice = 1

herdimmpertussismale Please click here to go to the other website
```

herdimmpertussismale <u>Veuillez cliquer ici pour accéder à l'autre site web</u>

```
Display This Question:

If viz = 1

And disease = 2

And voice = 2
```

herdimmpertussisfema Please click here to go to the other website

herdimmpertussisfema Veuillez cliquer ici pour accéder à l'autre site web

```
Display This Question:

If viz = 1

And disease = 3

And voice = 1
```

herdimmflumale Please click here to go to the other website

herdimmflumale Veuillez cliquer ici pour accéder à l'autre site web

.....

```
Display This Question:

If viz = 1

And disease = 3

And voice = 2
```

herdimmflufemale Please click here to go to the other website

herdimmflufemale Veuillez cliquer ici pour accéder à l'autre site web

\_\_\_\_\_\_

```
Display This Question:

If Q_Language = EN

And viz = 2
```

robertkoch Please click here to go to the other website

robertkoch NA

\_\_\_\_\_\_

```
Display This Question:

If Q_Language = EN
```

And viz = 3

sbsnewsgeneric Now we ask you to please watch the video below with some information to do with contagious diseases and then continue the survey.

sbsnewsgeneric NA

```
Display This Question:
```

If Q\_Language = EN And viz = 5

guardianmeasles

Now we ask you to please watch the video below with some information to do with contagious diseases and then continue the survey.

guardianmeasles NA

\_\_\_\_\_\_

```
Display This Question:

If Q_Language = EN

And viz = 6
```

theotheredmundmeasle Now we ask you to please watch the video below with some information to do with contagious diseases and then continue the survey.

## theotheredmundmeasle NA

\_\_\_\_\_

## Display This Question:

If viz = 7

publichealthagencyca Now we ask you to please watch the video below with some information to do with contagious diseases and then continue the survey.

publichealthagencyca Nous vous demandons maintenant de visionner la vidéo ci-dessous, qui contient des informations sur les maladies contagieuses, puis de poursuivre le sondage.

\_\_\_\_\_

t\_media Timing

First Click (1)

Last Click (2)

Page Submit (3)

Click Count (4)

t media Durée

First Click (1)

Last Click (2)

Page Submit (3)

Click Count (4)

End of Block: media

Start of Block: Risk Perception

riskpercep1 Imagine there are two groups of 100 people each. In one group, there is 1 UNvaccinated person surrounded by 99 vaccinated people. In the other group, there is 1 vaccinated person surrounded by 99 UNvaccinated people. Who is at higher risk of getting infected with \${e://Field/diseasedescEN}?



riskpercep1 Imaginez deux groupes composés de 100 personnes dans chacun d'eux. Dans un des groupes, il y a 99 individus vaccinés et une personne NON vaccinée. Dans l'autre groupe, il y a 1 personne vaccinée et 99 NON vaccinées. Qui serait le plus à risque de contracter \${e://Field/diseasedescFR-CA}?



| \${e://Field/diseasedescEN} affects only them, individually. |
|---|
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| Slightly agree (5) |
| O moderately agree (6) |
| ostrongly agree (7) |
| riskpercep2 La décision d'une personne de se faire vacciner ou non contre \${e://Field/diseasedescFR-CA} ne touche que cette personne individuellement. |
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |

riskpercep2 A person's decision to be vaccinated or not against

| | ep3 People who are vaccinated it on to others. | against \${e://Field/diseasedescEN} are | less likely |
|---|---|---|---|
| 0 | strongly disagree (1) | | |
| 0 | moderately disagree (2) | | |
| 0 | slightly disagree (3) | | |
| 0 | neutral (4) | | |
| $\bigcirc$ | slightly agree (5) | | |
| 0 | moderately agree (6) | | |
| 0 | strongly agree (7) | | |
| - | ep3 Les personnes qui sont vaccir<br>usceptibles de la transmettre. | ées contre \${e://Field/diseasedescFR-CA} | sont |
| O 1 | ortement en désaccord (1) | | |
| 0 | modérément en désaccord (2) | | |
| $\circ$ | égèrement en désaccord (3) | | |
| 0 | neutre (4) | | |
| $\circ$ | égèrement en accord (5) | | |
| 0 | modérément en accord (6) | | |
| O 1 | ortement en accord (7) | | |

| anyone else's chances of catching \${e://Field/diseasedescEN}. |
|---|
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| Slightly agree (5) |
| O moderately agree (6) |
| O strongly agree (7) |
| riskpercep4 Ma décision de me faire vacciner ou non contre $ext{ge://Field/diseasedescFR-CA} $ <b>n'a aucune incidence</b> sur les chances des autres de contracter $ext{ge://Field/diseasedescFR-CA}.$ |
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |
| X+ |

riskpercep4 My decision to be vaccinated against \${e://Field/diseasedescEN} has **no impact** on

| impact on anyone else's chances of catching \${e://Field/diseasedescEN}. |
|---|
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| O slightly agree (5) |
| O moderately agree (6) |
| O strongly agree (7) |
| riskpercep5 Ma décision de ne PAS me faire vacciner contre \${e://Field/diseasedescFR-CA} <b>n'a aucune incidence</b> sur les chances des autres de contracter \${e://Field/diseasedescFR-CA}. |
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |
| $\chi_{\rightarrow}$ |

riskpercep5 My decision NOT to be vaccinated against \${e://Field/diseasedescEN} has no

| riskpercep6 If I get vaccinated against \${e://Field/diseasedescEN}, it lowers the risk of vulnerable people in my community (babies, young children, older people, cancer patients) getting sick. |
|---|
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| O slightly agree (5) |
| O moderately agree (6) |
| O strongly agree (7) |
| riskpercep6 Si je me fais vacciner contre \${e://Field/diseasedescFR-CA}, cela réduit le risque que des personnes vulnérables de ma communauté (bébés, jeunes enfants, personnes âgées, patients atteints de cancer) tombent malades. |
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |

| t-riskpercp Timing First Click (1) Last Click (2) Page Submit (3) Click Count (4) t-riskpercp Durée First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
|---|
| End of Block: Risk Perception |
| Start of Block: 5CScale X→ |
| confidence1 I am completely confident that vaccines are safe. |
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| O slightly agree (5) |
| O moderately agree (6) |
| O strongly agree (7) |

| COI | nfidence1 Je suis complètement confiant que les vaccins sont sans danger. |
|---|---|
| | O fortement en désaccord (1) |
| | O modérément en désaccord (2) |
| | O légèrement en désaccord (3) |
| | O neutre (4) |
| | O légèrement en accord (5) |
| | O modérément en accord (6) |
| | O fortement en accord (7) |
| X- | nfidence2 Vaccinations are effective. |
| | O strongly disagree (1) |
| | O moderately disagree (2) |
| | O slightly disagree (3) |
| | O neutral (4) |
| | O slightly agree (5) |
| | O moderately agree (6) |
| | O strongly agree (7) |

| CO | nfidence2 Les vaccins sont efficaces. |
|---|---|
| | O fortement en désaccord (1) |
| | O modérément en désaccord (2) |
| | O légèrement en désaccord (3) |
| | O neutre (4) |
| | O légèrement en accord (5) |
| | O modérément en accord (6) |
| | O fortement en accord (7) |
| | nfidence3 Regarding vaccines, I am confident that public authorities decide in the best erest of the community. |
| | erest of the community. |
| | O strongly disagree (1) |
| | o strongly disagree (1) o moderately disagree (2) |
| | erest of the community. O strongly disagree (1) O moderately disagree (2) O slightly disagree (3) |
| | erest of the community. O strongly disagree (1) O moderately disagree (2) O slightly disagree (3) O neutral (4) |

| dé | dent dans le meilleur intérêt de la communauté. |
|---|---|
| | Offortement en désaccord (1) |
| | modérément en désaccord (2) |
| | Olégèrement en désaccord (3) |
| | neutre (4) |
| | Olégèrement en accord (5) |
| | modérément en accord (6) |
| | Offortement en accord (7) |
| | placency1 Vaccination is unnecessary because vaccine-preventable diseases are not mon anymore. Strongly disagree (1) moderately disagree (2) slightly disagree (3) |
| | mon anymore. Strongly disagree (1) moderately disagree (2) |
| | mon anymore. strongly disagree (1) moderately disagree (2) slightly disagree (3) |
| | mon anymore. strongly disagree (1) moderately disagree (2) slightly disagree (3) neutral (4) |
| | mon anymore. strongly disagree (1) moderately disagree (2) slightly disagree (3) neutral (4) slightly agree (5) |

confidence3 En ce qui concerne les vaccins, je suis convaincu que les autorités publiques

| complacency1 La vaccination est inutile car les maladies évitables par la vaccination ne sont plus courantes. |
|---|
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |
| X |
| complacency2 My immune system is so strong, it also protects me against diseases. |
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| O slightly agree (5) |
| O moderately agree (6) |
| O strongly agree (7) |

| CO | mplacency2 Mon système immunitaire est suffisamment fort pour me protéger des maladies. |
|---|---|
| | O fortement en désaccord (1) |
| | O modérément en désaccord (2) |
| | O légèrement en désaccord (3) |
| | O neutre (4) |
| | O légèrement en accord (5) |
| | O modérément en accord (6) |
| | O fortement en accord (7) |
| X- | mplacency3 Vaccine-preventable diseases are not so severe that I should get vaccinated. |
| | O strongly disagree (1) |
| | O moderately disagree (2) |
| | O slightly disagree (3) |
| | O neutral (4) |
| | O slightly agree (5) |
| | O moderately agree (6) |
| | ostrongly agree (7) |

| complacency3 Les maladies évitables par la vaccination ne sont pas graves au point de devoir me faire vacciner. |
|---|
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |
| $X \rightarrow$ |
| constraints1 Everyday stress prevents me from getting vaccinated. |
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| O slightly agree (5) |
| O moderately agree (6) |
| O strongly agree (7) |

| constraints1 Le stress quotidien m'empêche de me faire vacciner. |
|------------------------------------------------------------------|
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |
| X |
| constraints2 For me, it is inconvenient to receive vaccinations. |
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| O slightly agree (5) |
| O moderately agree (6) |
| O strongly agree (7) |

| СО | constraints2 Pour moi, il est peu pratique de recevoir des vaccins. |
|---|---|
| | O fortement en désaccord (1) |
| | O modérément en désaccord (2) |
| | O légèrement en désaccord (3) |
| | O neutre (4) |
| | O légèrement en accord (5) |
| | O modérément en accord (6) |
| | O fortement en accord (7) |
| | nstraints3 Visiting the doctor's makes me feel uncomfortable; this keeps me from getting ccinated. |
| | ccinated. |
| | O strongly disagree (1) |
| | O strongly disagree (1) O moderately disagree (2) |
| | coinated. Strongly disagree (1) moderately disagree (2) slightly disagree (3) |
| | coinated. Strongly disagree (1) moderately disagree (2) slightly disagree (3) neutral (4) |
| | coinated. Strongly disagree (1) moderately disagree (2) slightly disagree (3) neutral (4) slightly agree (5) |

| constraints3 Visiter le médecin me met mal à l'aise; cela m'empêche de me faire vacciner. | |
|---|---|
| O fortement en désaccord (1) | |
| O modérément en désaccord (2) | |
| O légèrement en désaccord (3) | |
| O neutre (4) | |
| O légèrement en accord (5) | |
| O modérément en accord (6) | |
| O fortement en accord (7) | |
| V-3 | - |
| calculation1 When I think about getting vaccinated, I weigh benefits and risks to make the best decision possible. | |
| best decision possible. | |
| best decision possible. O strongly disagree (1) | |
| best decision possible. O strongly disagree (1) O moderately disagree (2) | |
| <ul> <li>best decision possible.</li> <li>strongly disagree (1)</li> <li>moderately disagree (2)</li> <li>slightly disagree (3)</li> </ul> | |
| best decision possible. O strongly disagree (1) O moderately disagree (2) O slightly disagree (3) O neutral (4) | |
| best decision possible. Strongly disagree (1) moderately disagree (2) slightly disagree (3) neutral (4) slightly agree (5) | |

| calculation1 Quand je pense à me faire vacciner, je mesure les avantages et les risques pour prendre la meilleure décision possible. | |
|---|--|
| O fortement en désaccord (1) | |
| O modérément en désaccord (2) | |
| O légèrement en désaccord (3) | |
| O neutre (4) | |
| O légèrement en accord (5) | |
| O modérément en accord (6) | |
| O fortement en accord (7) | |
| $\chi_{\Rightarrow}$ | |
| calculation2 For each and every vaccination, I closely consider whether it is useful for me. | |
| O strongly disagree (1) | |
| O moderately disagree (2) | |
| O slightly disagree (3) | |
| O neutral (4) | |
| O slightly agree (5) | |
| O moderately agree (6) | |
| O strongly agree (7) | |
| calculat | tion2 Pour chaque vaccin, j'évalue de près si cela m'est utile. |
|---|---|
| 0 | fortement en désaccord (1) |
| $\circ$ | modérément en désaccord (2) |
| $\circ$ | légèrement en désaccord (3) |
| 0 | neutre (4) |
| $\circ$ | légèrement en accord (5) |
| 0 | modérément en accord (6) |
| 0 | fortement en accord (7) |
| X→ | |
| calculat<br>vaccina | tion3 It is important for me to fully understand the topic of vaccination, before I get ited. |
| vaccina | |
| vaccina | ited. |
| vaccina | strongly disagree (1) |
| vaccina | strongly disagree (1) moderately disagree (2) |
| vaccina | strongly disagree (1) moderately disagree (2) slightly disagree (3) |
| vaccina | strongly disagree (1) moderately disagree (2) slightly disagree (3) neutral (4) |
| vaccina | strongly disagree (1) moderately disagree (2) slightly disagree (3) neutral (4) slightly agree (5) |

| calculation3 II est important pour moi de bien comprendre tout ce qu'englobe la vaccination avant de me faire vacciner. |
|---|
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |
| X- |
| collectiverespon1 When everyone else is vaccinated, I don't have to get vaccinated, too. |
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| O neutral (4) O slightly agree (5) |
| O slightly agree (5) |

| collectiverespon1 Quand tous les autres sont vaccinés, je n'ai pas à me | faire vacciner aussi. |
|---|---|
| O fortement en désaccord (1) | |
| O modérément en désaccord (2) | |
| O légèrement en désaccord (3) | |
| O neutre (4) | |
| O légèrement en accord (5) | |
| O modérément en accord (6) | |
| O fortement en accord (7) | |
| collectiverespon2 I get vaccinated because I can also protect people wit system. | h a weaker immune |
| | h a weaker immune |
| system. | h a weaker immune |
| System. O strongly disagree (1) | h a weaker immune |
| system. O strongly disagree (1) O moderately disagree (2) | h a weaker immune |
| system. O strongly disagree (1) O moderately disagree (2) O slightly disagree (3) | h a weaker immune |
| system. Strongly disagree (1) moderately disagree (2) slightly disagree (3) neutral (4) | h a weaker immune |
| system. Strongly disagree (1) moderately disagree (2) slightly disagree (3) neutral (4) slightly agree (5) | h a weaker immune |

| système immunitaire est plus faible. | |
|---|---|
| O fortement en désaccord (1) | |
| O modérément en désaccord (2) | |
| O légèrement en désaccord (3) | |
| O neutre (4) | |
| O légèrement en accord (5) | |
| O modérément en accord (6) | |
| O fortement en accord (7) | |
| $X \rightarrow$ | - |
| collectiverespon3 Vaccination is a collective action to prevent the spread of diseases. | |
| collectiverespon3 Vaccination is a collective action to prevent the spread of diseases. O strongly disagree (1) | |
| O strongly disagree (1) | |
| <ul><li>strongly disagree (1)</li><li>moderately disagree (2)</li></ul> | |
| <ul><li>strongly disagree (1)</li><li>moderately disagree (2)</li><li>slightly disagree (3)</li></ul> | |
| <ul> <li>strongly disagree (1)</li> <li>moderately disagree (2)</li> <li>slightly disagree (3)</li> <li>neutral (4)</li> </ul> | |
| <ul> <li>strongly disagree (1)</li> <li>moderately disagree (2)</li> <li>slightly disagree (3)</li> <li>neutral (4)</li> <li>slightly agree (5)</li> </ul> | |

collectiverespon2 Je me fais vacciner parce que je peux aussi protéger les personnes dont le

| maladies |
|---|
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |
| _5Cscale Timing First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
| _5Cscale Durée First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
| End of Block: 5CScale |
| Start of Block: Emotion X→ |

collectiverespon3 La vaccination est une action collective visant à prévenir la propagation des

| emotion1 I am worried about getting \${e://Field/diseasedescEN}. | |
|------------------------------------------------------------------------|---|
| O strongly disagree (1) | |
| O moderately disagree (2) | |
| O slightly disagree (3) | |
| O neutral (4) | |
| O slightly agree (5) | |
| O moderately agree (6) | |
| O strongly agree (7) | |
| emotion1 Je suis inquiet de contracter \${e://Field/diseasedescFR-CA}. | |
| O fortement en désaccord (1) | |
| O modérément en désaccord (2) | |
| O légèrement en désaccord (3) | |
| O neutre (4) | |
| O légèrement en accord (5) | |
| O modérément en accord (6) | |
| O fortement en accord (7) | |
| | _ |

Page 63 of 80

| emotion2 I am worried about people in my life (family, friends) getting \${e://Field/diseasedescEN}. |
|---|
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| O slightly agree (5) |
| O moderately agree (6) |
| O strongly agree (7) |
| emotion2 Je suis inquiet que mon entourage (famille, amis) contracte \${e://Field/diseasedescFR-CA}. |
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |

| emotion3 I am worried about vulnerable people in my community (babies, young older people, cancer patients) getting \${e://Field/diseasedescEN}. | , |
|---|---|
| O strongly disagree (1) | |
| O moderately disagree (2) | |
| O slightly disagree (3) | |
| O neutral (4) | |
| O slightly agree (5) | |
| O moderately agree (6) | |
| O strongly agree (7) | |
| emotion3 Je suis inquiet que des gens vulnérables de ma communauté (bébés, jeunes enfait personnes âgées, patients atteints du cancer) contractent \${e://Field/diseasedescFR-CA}. | nts, |
| O fortement en désaccord (1) | |
| O modérément en désaccord (2) | |
| O légèrement en désaccord (3) | |
| O neutre (4) | |
| O légèrement en accord (5) | |
| O modérément en accord (6) | |
| O fortement en accord (7) | |

| \${e://Field/diseasedescEN} from me. |
|---|
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| O slightly agree (5) |
| O moderately agree (6) |
| O strongly agree (7) |
| emotion4 Je me sentirais coupable si je transmettais à quelqu'un de mon entourage (famille, amis) \${e://Field/diseasedescFR-CA}. |
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |

| emotion5 I would feel guilty if a vulnerable person (a baby, a young child, an older person, a cancer patient) got \${e://Field/diseasedescEN} from me. |
|---|
| O strongly disagree (1) |
| O moderately disagree (2) |
| O slightly disagree (3) |
| O neutral (4) |
| O slightly agree (5) |
| O moderately agree (6) |
| O strongly agree (7) |
| emotion5 Je me sentirais coupable si je transmettais à une personne vulnérable (un bébé, un jeune enfant, une personne âgée, un patient atteint du cancer) \${e://Field/diseasedescFR-CA}. |
| O fortement en désaccord (1) |
| O modérément en désaccord (2) |
| O légèrement en désaccord (3) |
| O neutre (4) |
| O légèrement en accord (5) |
| O modérément en accord (6) |
| O fortement en accord (7) |
| t_emotion Timing First Click (1) |
| Last Click (2) |
| Page Submit (3) Click Count (4) |

| t_emotion Durée First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
|---|
| End of Block: Emotion |
| Start of Block: Knowledge X+ |
| know01 When a person gets vaccinated, it can help protect: (check one) |
| ○ The person (1) |
| O The people around them (2) |
| O Vulnerable people in their community (3) |
| O All of the above (4) |
| know01 Quand une personne est vaccinée, cela peut aider à protéger : (cochez une réponse) |
| O La personne elle-même (1) |
| O Les gens autour d'elle (2) |
| O Les personnes vulnérables dans sa communauté (3) |
| O Toutes ces réponses (4) |

| | people are considered more vulnerable to contagious diseases, either because them more easily, or the diseases can make them sicker? (check all that apply) |
|---|---|
| | People who are very old (1) |
| | People who are very young (babies, etc.) (2) |
| | People who are athletes (3) |
| | People who have cancer (4) |
| | People who are healthy adults (5) |
| maladies conta | es personnes peuvent être considérées comme étant plus vulnérables aux agieuses, soit parce qu'ils peuvent attraper les maladies plus facilement, et les vent les rendre plus malades? (Cochez toutes les réponses qui s'appliquent) |
| | Les personnes très âgées (1) |
| | Les personnes très jeunes (bébés, etc.) (2) |
| | Les personnes qui sont des athlètes (3) |
| | Les personnes atteintes du cancer (4) |
| | Les adultes en bonne santé (5) |
| X→ | |

statement For the following statements, please indicate whether they are true, false, or you don't know:

| | True (1) | False (0) | I don't know (77) |
|---|---|---|---|
| \${e://Field/diseasedescEN_CAP} can spread from one person to another person. (know03) | 0 | 0 | 0 |
| When you come into contact with someone who is infected with \${e://Field/diseasedescEN}, there is a chance you could get the disease. (know04) | 0 | 0 | 0 |
| The only way to get<br>\${e://Field/diseasedescEN} is to<br>touch someone who has the<br>disease. (know05) | 0 | 0 | 0 |
| \${e://Field/diseasedescEN_CAP} always spread through groups of people at the same speed. (know07) | 0 | 0 | 0 |
| Some vaccines provide less protection than others. (know08) | 0 | 0 | 0 |
| Every vaccine provides full protection from a single dose (one needle/shot, one dose of drops in the mouth, or a one spray up the nose). (know10) | 0 | 0 | 0 |
| Some vaccines only provide partial protection after one dose and require multiple doses to get protected. (know11) | 0 | 0 | 0 |
| Some vaccines become less effective over time and need booster doses. (know12) | 0 | 0 | 0 |
| Community protection (or herd immunity) means everyone in the community has been vaccinated. (know13) | 0 | 0 | 0 |
| Unvaccinated people in a population can be protected from infections when enough people in their community are vaccinated. (know14) | 0 | 0 | 0 |

| Every person in a community (100%) must be vaccinated to achieve community protection. (know15) | 0 | 0 | 0 |
|---|---|---|---|
| The percentage of people (that is, how many members of a community) who must be vaccinated for the community to achieve community protection depends on the disease and the vaccine. (know16) | 0 | 0 | 0 |
| An individual's decision to get vaccinated or not affects only that individual. (know17) | 0 | 0 | 0 |

statement Pour les énoncés suivants, veuillez indiquer s'ils sont vrais, faux ou si vous ne savez pas :

| | Vrai (1) | Faux (0) | Je ne sais pas (77) |
|---|---|---|---|
| \${e://Field/diseasedescFR-<br>CA_CAP} peut se<br>propager d'une personne<br>à l'autre (know03) | 0 | 0 | 0 |
| Lorsque vous entrez en contact avec une personne infectée par \${e://Field/diseasedescFR-CA}, vous risquez de contracter cette maladie. (know04) | 0 | 0 | 0 |
| La seule façon de contracter \${e://Field/diseasedescFR-CA} est d'être en contact direct avec une personne infectée. (know05) | 0 | 0 | 0 |
| \${e://Field/diseasedescFR-<br>CA_CAP} se propage à<br>travers une communauté à<br>la même vitesse. (know07) | 0 | 0 | 0 |
| Certains vaccins offrent<br>moins de protection que<br>d'autres. (know08) | 0 | 0 | 0 |
| Chaque vaccin offre une protection complète avec une seule dose (une injection par aiguille, une dose de gouttes dans la bouche ou une seule pulvérisation dans le nez). (know10) | 0 | 0 | 0 |
| Certains vaccins ne<br>procurent qu'une<br>protection partielle après<br>une dose et nécessitent<br>plusieurs doses pour être<br>protégé. (know11) | 0 | 0 | 0 |
| Certains vaccins<br>deviennent moins<br>efficaces avec le temps et<br>nécessitent des doses de | 0 | 0 | 0 |

| rappel. (know12) | | | |
|---|---|---|---|
| La protection<br>communautaire (ou<br>l'immunité collective)<br>signifie que tout le monde<br>dans la communauté a été<br>vacciné. (know13) | 0 | 0 | 0 |
| Les gens non-vaccinés<br>d'une population peuvent<br>être protégés des<br>infections quand assez de<br>gens de leur communauté<br>sont vaccinés. (know14) | 0 | 0 | 0 |
| 100% des membres d'une<br>communauté doivent être<br>vaccinés pour assurer la<br>protection communautaire.<br>(know15) | 0 | 0 | 0 |
| Le pourcentage de personnes (c'est-à-dire combien de membres d'une communauté) qui doivent être vaccinées pour que la communauté puisse assurer la protection communautaire dépend de la maladie et du vaccin. (know16) | 0 | 0 | 0 |
| La décision d'un individu<br>de se faire vacciner ou<br>non affecte seulement cet<br>individu. (know17) | 0 | 0 | 0 |

t\_know Timing First Click (1)

Last Click (2)

Page Submit (3)

Click Count (4)

| :_know Duree First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
|-----------------------------------------------------------------------------|
| End of Block: Knowledge |
| Start of Block: Trust |
| $X \rightarrow$ |
| trustinfo \${e://Field/trustq_EN} |
| O not at all trustworthy (1) |
| O moderately untrustworthy (2) |
| Slightly untrustworthy (3) |
| O neutral (4) |
| O slightly trustworthy (5) |
| O moderately trustworthy (6) |
| ostrongly trustworthy (7) |
| trustinfo \${e://Field/trustq_FR-CA} |
| O pas du tout digne de confiance (1) |
| O modérément NON digne de confiance (2) |
| O légèrement NON digne de confiance (3) |
| O neutre (4) |
| O légèrement digne de confiance (5) |
| O moyennement digne de confiance (6) |
| O fortement digne de confiance (7) |

| t_trustinfo Timing First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
|---|
| t_trustinfo Durée First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
| End of Block: Trust |
| Start of Block: Behavioural intentions |
| Display This Question: |
| If disease = 1 Or disease = 2 |
| Or disease = 3 |
| $\chi_{\Rightarrow}$ |
| immune To the best of your knowledge, are you already immune to \${e://Field/diseasedescEN}? |
| O Yes (1) |
| O No (0) |
| O I don't know (77) |
| immune A votre connaissance, êtes-vous déjà immunisé contre \${e://Field/diseasedescFR-CA}? |
| Oui (1) |
| O Non (0) |
| O Je ne sais pas (77) |

| t_immune Timing First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
|---|
| t_immune Durée<br>First Click (1)<br>Last Click (2)<br>Page Submit (3)<br>Click Count (4) |
| Page Break ————— |

Display This Question: If To the best of your knowledge, are you already immune to \$\{e://Field/diseasedescEN}\? = Yes Or If disease = 0 Q For the next question, imagine you were **not** already immune to \${e://Field/diseasedescEN}. Q Imaginez que vous **n'étiez pas** déjà immunisé contre \${e://Field/diseasedescFR-CA}. vaxintention If you were eligible to receive a free vaccine against \${e://Field/diseasedescEN}, how likely would you be to get vaccinated? Extremely unlikely, I Extremely likely, I would would definitely NOT bedefinitely BE vaccinated vaccinated 1 () vaxintention Si vous étiez admissible à recevoir gratuitement un vaccin contre \$\{e://Field/diseasedescFR-CA\}, quelle serait votre probabilité de recevoir le vaccin ? Extrêmement Extrêmement probable, improbable, je ne serais ie SERAIS certainement PAS certainement vacciné vacciné t vaxintention Timing First Click (1) Last Click (2) Page Submit (3)

Click Count (4)

| t_vaxintention Durée |
|----------------------|
| First Click (1) |
| Last Click (2) |
| Page Submit (3) |
| Click Count (4) |
| Page Break ———— |



| c19vax Have you already received a COVID-19 vaccine (between Dec 2020 and now)? |
|---|
| ○ Yes (1) |
| O No (0) |
| O I don't know (77) |
| c19vax Avez-vous déjà reçu un vaccin contre la COVID-19 (entre décembre 2020 et maintenant) ? |
| Oui (1) |
| O Non (0) |
| O Je ne sais pas (77) |
| t_c19vax Timing First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
| t_c19vax Durée First Click (1) Last Click (2) Page Submit (3) Click Count (4) |
| Page Break ———————————————————————————————————— |

Display This Question:

If Have you already received a COVID-19 vaccine (between Dec 2020 and now)? = No Or Have you already received a COVID-19 vaccine (between Dec 2020 and now)? = I don't know

c19vaxintention Assuming you will be eligible to get a COVID-19 vaccine this year, how likely are you to get the vaccine?

COVID-19 vaccine

Extremely unlikely, I will Extremely likely, I will definitely NOT get a definitely get a COVID-19 vaccine

1 ()

c19vaxintention En supposant que vous soyez éligible pour recevoir un vaccin COVID-19 cette année, quelle est la probabilité que vous receviez le vaccin?

> Extrêmement improbable (c.-à-d. je ne me ferai certainement PAS vacciner contre la COVID-19)

Extrêmement probable, (c.-à-d. je me ferai certainement vacciner contre la COVID-19)

1 ()

t c19vaxintention Timing

First Click (1)

Last Click (2)

Page Submit (3)

Click Count (4)

t c19vaxintention Durée

First Click (1)

Last Click (2)

Page Submit (3)

Click Count (4)

**End of Block: Behavioural intentions** 

```
$3: Study statistal analysis plan
# Project: herdimm
 1
 2
     # Description: code for analysing the results of Hina Hakim's final PhD study
 3
     # Script developed by: Hina Hakim Jul 2019 - Dec 2020 with the collaboration of
 4
     Anne-Sophie Julien
 5
     # (statistician) and Holly Witteman (PhD advisor). Reviewed externally by a statistician
 6
     # unaffiliated with the project in October 2020; report received 2020-10-30.
 7
8
     # Last run: 2021-09-20 with real data from 2021-07-05
9
10
     #### RESEARCH QUESTIONS ####
11
12
     # This project uses the herdimm intervention to convey the concept of community
     immunity or herd
13
     # immunity. The herdimm intervention is described in detail here: DOI: 10.2196/20113
14
     # Research question 1 (primary): Across 4 vaccine-preventable diseases, does the herdimm
15
16
     # intervention influence risk perception compared to a control?
17
18
     # Research question 2 (secondary): Across 4 vaccine-preventable diseases, does the
     herdimm
19
     # intervention influence other outcomes (5C scale, emotions, trust, knowledge,
     behavioural
20
     # intentions) compared to a control?
21
22
     # Research question 3 (secondary): For any of the 4 diseases, do existing interventions
     already
23
     # available online outperform the herdimm intervention?
24
25
     # Research question 4 (add-on, may be reported separately from Hina Hakim's thesis):
     Are the effects
26
     # of the herdimm intervention different when the narration uses a female or male voice?
27
28
29
     #### LOAD LIBRARIES ####
30
31
     # Libraries are required to run different packages for running the code below.
32
     library(psych) # describeBy
33
    library(emmeans) # emmeans
34
    library(moments) # kurtosis, skewness
35
    library(car) # Anova
36 library (MASS) # Box-Cox
37
    library(olsrr) # testing collinearity
38 library(readr) # read files
39 library(tidyverse)
40
    library(dplyr)
     library(ggplot2) # for plots
41
     library(BlandAltmanLeh) # for Bland Altman test
42
43
     library(ltm) # to determine Cronbach alpha
44
    library(mice) # for multiple imputations
45
    library(naniar)
46
     library (R2HTML) #CHANGELOG ASJ: to output results 2021-08-06.
47
     library (mitml) #CHANGELOG ASJ: add global test after multiple imputation 21-09-20.
48
49
     sessionInfo() # for citing packages in paper
50
51
     #### IMPORT DATA ####
52
53
     # Import CSV file of raw data, removing Qualtrics artifacts in rows 1-2 (unneeded
54
     # and columns 1-16 (unneeded data automatically collected by default by Qualtrics.)
55
56
    datRaw = (
57
58
         "./contag phase3b July 5, 2021 08.19.csv",
59
        header = T,
         sep = ","
60
       ) [-c(1, 2)]
61
62
     ) #CHANGELOG Changed to new file name 2021-07-05
```

```
63
      # View(datRaw)
 64
 65
      # Subset the data we need: people who started (Consent == 1) and finished (Finished == 1)
 66
      #CHANGELOG ASJ: Replace subset by qc = 1 equivalent to Consent + Finished + Quality,
      21-08-06
      dat<-subset (datRaw, gc==1)</pre>
 67
      # View(dat)
 68
 69
 70
      #CHANGELOG ASJ: save and print results 2021-09-03.
 71
      HTMLStart(outdir=".\\",
                 file = "Herdimm Descriptive210903", extension = "html", echo=TRUE, HTMLframe =
 72
                 TRUE)
 73
 74
      #### CLEAN DATA ####
 75
 76
 77
      #### + Risk Perception ####
 78
 79
      # First change the columns (variables) from character to numeric form so that we can
      work with them.
 80
 81
      dat$riskpercep1 1 <- as.numeric(as.character(dat$riskpercep1 1))</pre>
 82
      dat$riskpercep2 <- as.numeric(as.character(dat$riskpercep2))</pre>
 83
      dat$riskpercep3 <- as.numeric(as.character(dat$riskpercep3))</pre>
 84
      dat$riskpercep4 <- as.numeric(as.character(dat$riskpercep4))</pre>
 85
      dat$riskpercep5 <- as.numeric(as.character(dat$riskpercep5))</pre>
      dat$riskpercep6 <- as.numeric(as.character(dat$riskpercep6))</pre>
 86
 87
 88
      # Then recode reverse-coded items riskpercep2, riskpercep4, riskpercep5.
 89
 90
      dat$riskpercep2rev <- 8-dat$riskpercep2</pre>
 91
      dat$riskpercep4rev <- 8-dat$riskpercep4
 92
      dat$riskpercep5rev <- 8-dat$riskpercep5</pre>
 93
      # To check if risk percep_1 measures the same construct as riskpercep 2-6, we rescale
 94
      riskpercep 1
 95
      # so that it is measured on the same scale as the other items.
 96
 97
      dat$score riskpercep1 1 <- dat$riskpercep1 1*6/100+1
 98
      summary(dat$score riskpercep1 1)
 99
100
      # To calculate the mean of the six other risk perception items (that is: riskpercep 2,
      riskpercep 3,
101
      # riskpercep 4, riskpercep 5, riskpercep 6), first, we create a subset of the items we
      need.
102
103
      dat riskpercep2 6 <-
104
       subset (
105
          dat,
106
          select = c(
107
           riskpercep2rev,
108
            riskpercep3,
109
            riskpercep4rev,
110
            riskpercep5rev,
111
            riskpercep6
112
          )
113
        )
114
115
      # Sum all items (riskpercept 2 to riskpercep 6) for each participant.
116
117
      risk sumrows <-rowSums(dat riskpercep2 6, na.rm=T)</pre>
118
119
      # Count the number of missing items (no response in items riskpercept 2 to
      riskpercep 6) for each
120
      # participant.
121
122
      risk summissing <-
123
        is.na(dat riskpercep2 6$riskpercep2rev) +
```

```
124
        is.na(dat riskpercep2 6$riskpercep3) +
125
        is.na(dat riskpercep2 6$riskpercep4rev) +
        is.na(dat riskpercep2 6$riskpercep5rev) +
126
127
        is.na(dat riskpercep2 6$riskpercep6)
128
129
      table(risk summissing)
130
      prop.table(table(risk summissing))*100
131
132
      # Calculate the mean value (mean risk perception) from riskpercept 2 to riskpercep 6 of
      all answered
133
      # items.
134
135
      dat$mean riskperception2 6<-risk sumrows/(5-risk summissing)
136
      summary(dat$mean riskperception2 6)
137
138
      # To see if the item risk percep 1 and risk percept 2 to 6 are all measuring the same
      thing, we need
139
      # a Bland Altman plot. To create a Bland Altman plot, we need the difference between 1
      and the mean
140
      # of 2 to 6. So, for that purpose, we will create 2 new variables then create the plot.
141
142
      dat$diff riskp1 6 <-dat$score riskpercep1 1-dat$mean riskperception2 6
143
      summary(dat$diff riskp1 6)
144
145
      dat$mean riskp1 6<- (dat$score riskpercep1 1+dat$mean riskperception2 6)/2
146
      summary(dat$mean riskp1 6)
147
148
      plot(dat$score riskpercep1 1,dat$mean riskperception2 6)
149
150
      # We are using two = 1.96 (two standard deviations) rather than two = 2.0. If there are
      data points
151
      # outside these limits, this raises concerns that these two measures may not, in fact,
     measure the
      # same construct.
152
153
154
      bland.altman.plot(
155
        dat$mean riskperception2 6,
156
        dat$score riskpercep1 1,
157
        two = 1.96,
158
        mode = 1,
        graph.sys = "base",
159
160
        conf.int = 0,
161
        silent = TRUE,
162
        sunflower = FALSE,
163
        geom count = FALSE
164
165
      # Then we formally test the hypothesis. If this test is statistically significant, it
166
      means the
167
      # difference between the two new variables is not zero, which implies a lack of
      similarity between
168
      # the two original measurement methods (i.e., riskpercep 1 and riskpercep 2 to 6.)
169
170
      summary(lm(dat$mean riskp1 6 ~ dat$diff riskp1 6))
171
172
      # If riskpercep_1 and riskpercep_2 to _6 are similar, we will combine them into a
      single measure if
173
      # their combined Cronbach alpha is >=0.8 and will consider doing so if their combined
      Cronbach alpha
174
      # can be raised to >=0.8 by removing inconsistent items. We will explore removing items
      because this
175
      # measure is an ad hoc measure created specifically for this study.
176
177
      # Create a subset for riskpercep 2 to 6 to determine Cronbach alpha more easily
178
179
      dat riskpercep2 6 alpha <-
180
        subset (
181
          dat,
182
          select = c(
```

```
183
            riskpercep2rev,
184
            riskpercep3,
185
            riskpercep4rev,
186
            riskpercep5rev,
187
            riskpercep6
188
          )
189
        )
190
191
      # Cronbach alpha value for riskpercep 2-6
192
193
     cronbach.alpha(
194
        dat riskpercep2 6 alpha,
195
        standardized = FALSE,
196
        CI = FALSE,
197
        probs = c(0.025, 0.975),
198
        B = 1000,
199
        na.rm = TRUE
      ) \# CHANGELOG Change na.rm = FALSE to TRUE 2021-07-14
200
201
202
      # Create a subset for riskpercep 1 to 6 to determine Cronbach alpha more easily
203
204
      dat riskpercep1 6 alpha <-
205
        subset (
206
          dat,
207
          select = c(
208
            score riskpercep1 1,
209
            riskpercep2rev,
210
            riskpercep3,
211
            riskpercep4rev,
212
            riskpercep5rev,
213
            riskpercep6
214
          )
215
        )
216
217
      # Cronbach alpha value for riskpercep 1-6
218
219
      cronbach.alpha(
220
        dat riskpercep1 6 alpha,
221
        standardized = FALSE,
222
        CI = FALSE,
223
        probs = c(0.025, 0.975),
224
        B = 1000,
225
        na.rm = TRUE
226
      ) # CHANGELOG Change na.rm = FALSE to TRUE 2021-07-14
227
228
      # 1. If we can combine the measures (based on Bland Altman & Cronbach alpha) then we
      create a single
229
      # measure using the same series of steps as above (subset, sum of all items, number of
      missing
230
      # items, calculate mean). This is our preferred approach, so we are prioritizing this
      option in the
231
      # pre-registered code.
232
233
      # subset
234
     dat riskpercep <-
235
        subset (
236
          dat,
237
          select = c(
238
            score riskpercep1 1,
239
            riskpercep2rev,
240
            riskpercep3,
241
            riskpercep4rev,
242
            riskpercep5rev,
243
            riskpercep6
244
          )
245
        )
246
247
      # sum of all items for each person
248
      risk sumrows <-rowSums(dat riskpercep, na.rm=T)</pre>
```

```
249
250
      # count of missing values
251
      risk summissing <-
252
        is.na(dat riskpercep$score riskpercep1 1) +
        is.na(dat_riskpercep$riskpercep2rev) +
253
254
        is.na(dat_riskpercep$riskpercep3) +
255
        is.na(dat riskpercep$riskpercep4rev) +
256
        is.na(dat riskpercep$riskpercep5rev) +
257
        is.na(dat riskpercep$riskpercep6)
258
259
      # mean
260
      dat$mean riskperception<-risk sumrows/(6-risk summissing)
261
262
      # 2. If we cannot combine the measures, we will run the rest of the script once with
      risk perception
263
      # being the first item only, and then re-run the rest of the script with risk
      perception being items
264
      # 2 to 6. In that case, we will add a comment for which condition we are running the
      ANOVA each
265
      # time. For now, we have commented these out, as we hope not to have to use them.
266
267
      # dat$mean riskperception<-(dat$score riskpercep1 1)</pre>
268
269
      dat$mean riskperception<- (dat$mean riskperception2 6)
270
      # CHANGELOG: As mentioned above that if risk perception item 1 and 2 to 6 are measuring
271
      differently, we will use in our analysis ANOVA model separately
272
      # CHANGELOG ASJ: Since riskperception 1 is asymetric, no ANOVA will be run on it, so
      the mean can be directly equal to 2-6, 2021-08-03
273
274
      #### + Betsch et al 5C measure ####
275
276
      # Variables are coming in as data type character. Force them to be numeric so we can
      work with them.
277
278
      cols.num <- c(
279
        "confidence1"
280
        "confidence2",
281
        "confidence3".
282
        "complacency1",
283
        "complacency2",
284
        "complacency3",
        "constraints1",
285
286
        "constraints2",
287
        "constraints3",
        "calculation1",
288
289
        "calculation2",
        "calculation3",
290
        "collectiverespon1",
291
292
        "collectiverespon2"
293
        "collectiverespon3"
294
295
296
      dat[cols.num] <- sapply(dat[cols.num],as.numeric)</pre>
297
298
      # Recode reverse-coded item collectiverespon1
299
300
      dat$collectiverespon1rev <- 8-dat$collectiverespon1</pre>
301
302
      # Calculate mean (subset, sum of all items, number of missing items, calculate mean).
303
304
      dat 5c <-
305
        subset (
306
          dat,
307
          select = c(
308
            confidence1,
309
            confidence2,
310
            confidence3,
311
            complacency1,
```

```
complacency2,
313
            complacency3,
314
            constraints1,
315
            constraints2,
316
            constraints3,
317
            calculation1,
318
            calculation2,
319
            calculation3,
320
            collectiverespon1rev,
321
            collectiverespon2,
322
            collectiverespon3
323
          )
324
        )
325
326
      C5 sumrows <- rowSums(dat 5c, na.rm = T)
327
328
      C5 summissing <-
329
        is.na(dat 5c$confidence1) +
330
        is.na(dat 5c$confidence2) +
331
        is.na(dat 5c$confidence3) +
332
        is.na(dat 5c$complacency1) +
333
        is.na(dat 5c$complacency2) +
334
        is.na(dat 5c$complacency3) +
335
        is.na(dat 5c$constraints1) +
        is.na(dat_5c$constraints2) +
is.na(dat_5c$constraints3) +
336
337
338
        is.na(dat_5c$calculation1) +
        is.na(dat_5c$calculation2) +
339
        is.na(dat_5c$calculation3) +
340
        is.na(dat 5c$collectiverespon1rev) +
341
342
        is.na(dat 5c$collectiverespon2) +
343
        is.na(dat 5c$collectiverespon3)
344
345
      dat$mean C5 <- C5 sumrows / (15 - C5 summissing)
346
347
      # Determine Cronbach alpha of overall 5C scale.
348
      #CHANGELOG ASJ: Overall consistency is low, while it's high for subscales. Analysis of
      subscales instead of total score, 2021-08-06
349
      cronbach.alpha(dat_5c, standardized = FALSE, CI = FALSE,
350
                      probs = c(0.025, 0.975), B = 1000, na.rm = TRUE) # CHANGELOG Change na.rm
                      = FALSE to TRUE 2021-07-14
351
352
353
      # Create subsets for each subscale .
354
355
      dat 5c confidence <-subset(dat,select=c(confidence1,confidence2,confidence3))</pre>
356
      dat 5c complacency<-subset(dat, select=c(complacency1, complacency2, complacency3))</pre>
357
          5c constraints<-subset(dat,select=c(constraints1,constraints2,constraints3))</pre>
          _5c_calculation<-subset(dat, select=c(calculation1, calculation2, calculation3))
358
359
      dat_5c_collectiverespon<-subset (dat, select=c (collectiverespon1rev, collectiverespon2, colle</pre>
      ctiverespon3))
360
361
      # Determine Cronbach alpha values for each of 5C subscales.
362
363
      # Confidence
364
      cronbach.alpha(
365
        dat 5c confidence,
366
        standardized = FALSE,
367
        CI = FALSE,
368
        probs = c(0.025, 0.975),
        B = 1000,
369
370
        na.rm = TRUE
371
      ) # CHANGELOG Change na.rm = FALSE to TRUE 2021-07-14
372
373
      # Complacency
374
      cronbach.alpha(
375
        dat 5c complacency,
376
        standardized = FALSE,
377
        CI = FALSE,
```

```
378
        probs = c(0.025, 0.975),
379
        B = 1000,
380
       na.rm = TRUE
381
      ) # CHANGELOG Change na.rm = FALSE to TRUE 2021-07-14
382
383
      # Constraints
384
     cronbach.alpha(
385
       dat 5c constraints,
386
        standardized = FALSE,
387
        CI = FALSE,
388
        probs = c(0.025, 0.975),
389
       B = 1000,
390
       na.rm = TRUE
391
      ) # CHANGELOG Change na.rm = FALSE to TRUE 2021-07-14
392
393
      # Calculation
394
     cronbach.alpha(
395
        dat 5c calculation,
396
        standardized = FALSE,
397
        CI = FALSE,
398
        probs = c(0.025, 0.975),
399
        B = 1000,
400
       na.rm = TRUE
      ) \# CHANGELOG Change na.rm = FALSE to TRUE 2021-07-14
401
402
403
     # Collective responsibility
404
     cronbach.alpha(
405
        dat_5c_collectiverespon,
406
        standardized = FALSE,
407
        CI = FALSE,
       probs = c(0.025, 0.975),
408
409
       B = 1000,
410
       na.rm = TRUE
      ) \# CHANGELOG Change na.rm = FALSE to TRUE 2021-07-14
411
412
413
      #CHANGELOG ASJ: Calculate mean for each subscale because of low overall consistency,
      2021-08-06.
414
      C5conf_sumrows <- rowSums(dat_5c_confidence, na.rm = T)</pre>
415
      C5comp_sumrows <- rowSums(dat_5c_complacency, na.rm = T)</pre>
416
      C5cons_sumrows <- rowSums(dat_5c_constraints, na.rm = T)
417
      C5calc sumrows <- rowSums(dat 5c calculation, na.rm = T)
418
      C5coll sumrows <- rowSums(dat 5c collectiverespon, na.rm = T)
419
420
421
      C5conf summissing <-
                               is.na(dat 5c$confidence1) + is.na(dat 5c$confidence2) +
      is.na(dat 5c$confidence3)
422
                               is.na(dat 5c$complacency1) + is.na(dat 5c$complacency2) +
      C5comp summissing <-
      is.na(dat 5c$complacency3)
423
                              is.na(dat 5c$constraints1) + is.na(dat 5c$constraints2) +
      C5cons summissing <-
      is.na(dat_5c$constraints3)
424
                              is.na(dat 5c$calculation1) + is.na(dat 5c$calculation2) +
      C5calc summissing <-
      is.na(dat 5c$calculation3)
425
                               is.na(dat 5c$collectiverespon1rev) +
      C5coll summissing <-
      is.na(dat 5c$collectiverespon2) + is.na(dat 5c$collectiverespon3)
426
427
      dat$mean_C5_conf <- C5conf_sumrows / (3 - C5conf_summissing)</pre>
428
      dat$mean C5 comp <- C5comp sumrows / (3 - C5comp summissing)
      dat$mean C5 cons <- C5cons sumrows / (3 - C5cons summissing)
429
      dat$mean C5 calc <- C5calc sumrows / (3 - C5calc summissing)
430
      dat$mean C5 coll <- C5coll sumrows / (3 - C5coll summissing)
431
432
433
      #CHANGELOG ASJ: Dichotomize the five subscales because they are highly asymetric,
      21-09-03
434
      hist(dat$mean C5 conf)
435
      hist(dat$mean C5 comp)
436
      hist(dat$mean C5 cons)
437
      hist(dat$mean C5 calc)
438
      hist(dat$mean C5 coll)
439
```

```
440
      summary(dat$mean C5 conf) #6
441
      summary(dat$mean C5 comp) #2.33
442
      summary(dat$mean C5 cons) #2
443
      summary(dat$mean C5 calc) #5.33
444
      summary(dat$mean C5 coll) #6.33
445
      dat$mean C5 conf2<-ifelse(dat$mean C5 conf>=6,1,0)
446
447
      dat$mean C5 comp2<-ifelse(dat$mean C5 comp<=2.34,1,0)
448
      dat$mean C5 cons2<-ifelse(dat$mean C5 cons<=2,1,0)
449
      dat$mean C5 calc2<-ifelse(dat$mean C5 calc>=5.33,1,0)
450
      dat$mean C5 coll2<-ifelse(dat$mean C5 coll>=6.33,1,0)
451
452
      table (dat$mean C5 conf2, dat$mean C5 conf)
      table(dat$mean C5 comp2, dat$mean_C5_comp)
453
      table(dat$mean_C5_cons2,dat$mean_C5_cons)
454
455
      table(dat$mean C5 calc2, dat$mean C5 calc)
      table(dat$mean_C5_coll2, dat$mean_C5_coll)
456
457
458
      table(dat$mean C5 conf2)
459
      table(dat$mean C5 comp2)
460
      table (dat$mean C5 cons2)
461
      table (dat$mean C5 calc2)
462
      table (dat$mean C5 coll2)
463
464
465
      #### + Emotions ####
466
467
      # Variables are coming in as data type character. Force them to be numeric so we can
      work with them.
468
469
      cols.num <- c("emotion1", "emotion2", "emotion3", "emotion4", "emotion5")</pre>
470
      dat[cols.num] <- sapply(dat[cols.num],as.numeric)</pre>
471
472
      # Calculate mean (subset, sum of all items, number of missing items, calculate mean).
473
474
      dat emotion <-
475
        subset(dat, select = c(emotion1, emotion2, emotion3, emotion4, emotion5))
476
477
      emotion sumrows <- rowSums(dat emotion, na.rm = T)</pre>
478
479
      emotion summissing <-
480
        is.na(dat_emotion$emotion1) +
481
        is.na(dat emotion$emotion2) +
482
        is.na(dat emotion$emotion3) +
483
        is.na(dat emotion$emotion4) +
484
        is.na(dat emotion$emotion5)
485
486
      dat$mean emotion <- emotion summows / (5 - emotion summissing)
487
488
      # Calculate Cronbach alpha for emotions questions.
489
490
     cronbach.alpha(
491
        dat emotion,
492
        standardized = FALSE,
493
        CI = FALSE,
494
        probs = c(0.025, 0.975),
495
        B = 1000,
496
        na.rm = TRUE
497
      ) # CHANGELOG Change na.rm = FALSE to TRUE 2021-07-14
498
      #### + Knowledge ####
499
500
501
      # Variables are coming in as data type character. Force them to be numeric so we can
      work with them.
      # The original knowledge scale included slightly repetitive items know06 and know09
502
503
      # removed to shorten the overall survey.
504
505
      cols.num <-
```

```
507
           "know01",
508
           "know02 1",
           "know02
509
510
           "know02
                   3",
511
          "know02_4",
512
           "know02 5",
           "know03",
513
          "know04",
514
          "know05",
515
          "know07",
516
          "know08",
517
          "know10",
518
           "know11",
519
           "know12",
520
           "know13",
521
           "know14",
522
           "know15",
523
           "know16",
524
           "know17"
525
526
527
528
      dat[cols.num] <- lapply(dat[cols.num],as.numeric)</pre>
529
530
      # Calculate the knowledge score. If the participant selected the correct response, they
      get 1 point
531
      # for that item. Otherwise they get 0 for that item. know01 and know02 are multiple
      choice.
532
      # know03-17 are true/false. For know01, we required a single correct choice. For
      know02, we require
      # all correct options selected. For know03-17, we require the correct choice (true or
533
      false.)
534
535
      dat$know01 score <- ifelse(dat$know01 == 4, 1, 0)</pre>
536
      dat$know02 score <- ifelse(dat$know02 1 == 1 &</pre>
537
                                    dat$know02 2 == 1 &
                                    dat$know02 3 == 0 &
538
539
                                    dat$know02 4 == 1 &
540
                                    dat$know02_5 == 0,1,0)
541
      dat$know03 score <- ifelse(dat$know03 == 1, 1, 0)</pre>
542
      dat$know04 score <- ifelse(dat$know04 == 1, 1, 0)</pre>
543
      dat$know05 score <- ifelse(dat$know05 == 1, 1, 0)
544
      dat$know07 score <- ifelse(dat$know07 == 0, 1, 0)</pre>
545
      dat$know08 score <- ifelse(dat$know08 == 1, 1, 0)</pre>
546
      dat$know10 score <- ifelse(dat$know10 == 0, 1, 0)</pre>
547
      dat$know11 score <- ifelse(dat$know11 == 1, 1, 0)</pre>
      dat$know12 score <- ifelse(dat$know12 == 1, 1, 0)</pre>
548
549
      dat$know13 score <- ifelse(dat$know13 == 0, 1, 0)</pre>
      dat$know14_score <- ifelse(dat$know14 == 1, 1, 0)</pre>
550
551
      dat$know15_score <- ifelse(dat$know15 == 0, 1, 0)</pre>
552
      dat$know16 score <- ifelse(dat$know16 == 1, 1, 0)</pre>
553
      dat$know17 score <- ifelse(dat$know17 == 0, 1, 0)</pre>
554
555
      # Subset the items so we can easily calculate total score.
556
557
      dat know <-
558
        subset (
559
           dat,
560
           select = c(
561
             know01_score,
             know02_score,
562
563
             know03 score,
564
             know04_score,
565
             know05 score,
566
             know07 score,
567
             know08 score,
568
             know10 score,
             know11 score,
569
             know12 score,
570
```

506

```
571
            know13 score,
572
            know14 score,
573
            know15 score,
574
            know16 score,
575
            know17 score
576
          )
577
        )
578
579
      # Calculate sum of correct answers out of 15 total.
580
581
      dat$sum knowledge <- rowSums(dat know,na.rm=T)</pre>
582
583
     # If we want to know the number of NA's in the data we can run the line below. This
      would allow us
     # to distinguish between people who selected the wrong answer and people who indicated
584
      they didn't
585
     # know. We will do this if knowledge scores are very low across all conditions (e.g.,
      mean scores
586
     # less than about 5.) It is commented out for the preregistered code because we hope
      not to need it.
587
588
      #CHANGELOG ASJ: the mean of sum knowledge is 8.9, so no need for it, 2021-08-03
589
     # dat$sum knowledge <-rowSums(dat know,na.rm=F)</pre>
590
      #### + Trust ####
591
592
593
      # Variable is coming in as data type character. Force it to be numeric so we can work
      with it.
594
595
     dat$trustinfo <- as.numeric(dat$trustinfo)</pre>
596
597
      #### + Behavourial Intentions ####
598
599
     # Variables are coming in as data type character. Force them to be numeric so we can
      work with them.
600
601
      cols.num <-
602
        C (
          "immune",
603
604
         "vaxintention 1",
          "c19vax",
605
          "c19vaxintention 1"
606
607
608
609
      dat[cols.num] <- sapply(dat[cols.num], as.numeric)</pre>
610
611
      #### + Individualism and Collectivism Scale ####
612
613
      # Variables are coming in as data type character. Force them to be numeric so we can
      work with them.
614
615
     cols.num <-
616
617
          "ih1",
          "ih2",
618
          "ih3",
619
          "ih4",
620
621
          "iv1",
          "iv2",
622
623
          "iv3",
624
          "iv4",
625
          "ch1",
          "ch2",
626
627
          "ch3",
          "ch4",
628
         "cv1",
629
630
         "cv2",
         "cv3",
631
          "cv4"
632
```

```
633
        )
634
635
      dat[cols.num] <- sapply(dat[cols.num], as.numeric)</pre>
636
637
      # This scale may have up to 4 dimensions, so we need to check for collinearity. To do
      this, we
638
      # calculate mean scores for each participant for each of the 4 subscales, using the
      same method as
      # above (subset, sum, count missing, calculate mean scores.) Then we enter these in a
639
      linear model
      # on our primary outcome and check VIF for indications of multicollinearity. If all the
640
      # below 10, it means there is no multicollinearity. If some of the VIF values are more
641
      than 10, it
      # means that variables are correlated. If there is collinearity then we can not use the 4
642
643
      # dimensions in the model. In that case, we can use either 2 dimensions or just one or
      3 dimensions.
644
      # If there is no collinearity then we can use the 4 dimensions.
645
646
      dat indivhorz <-subset(dat, select=c(ih1, ih2, ih3, ih4))</pre>
647
      dat indivvertical <-subset(dat, select=c(iv1, iv2, iv3, iv4))</pre>
648
      dat collhorz <-subset(dat, select=c(ch1, ch2, ch3, ch4))</pre>
649
      dat collvertical <-subset(dat, select=c(cv1, cv2, cv3, cv4))</pre>
650
      dat indiv coll <-
      subset (dat, select=c(ih1, ih2, ih3, ih4, iv1, iv2, iv3, iv4, ch1, ch2, ch3, ch4, cv1, cv2, cv3, cv4))
651
652
      # Cronbach alpha for subscales (each dimension) of the scale.
653
      # CHANGELOG Change below na.rm = FALSE to TRUE 2021-07-14
654
655
      cronbach.alpha(dat indivhorz, standardized = FALSE, CI = FALSE,
656
                      probs = c(0.025, 0.975), B = 1000, na.rm = TRUE)
657
      cronbach.alpha (dat indivvertical, standardized = FALSE, CI = FALSE,
658
                      probs = c(0.025, 0.975), B = 1000, na.rm = TRUE)
659
      cronbach.alpha(dat collhorz, standardized = FALSE, CI = FALSE,
660
                      probs = c(0.025, 0.975), B = 1000, na.rm = TRUE)
661
      cronbach.alpha(dat collvertical, standardized = FALSE, CI = FALSE,
                      probs = c(0.025, 0.975), B = 1000, na.rm = TRUE)
662
663
      cronbach.alpha(dat_indiv_coll, standardized = FALSE, CI = FALSE,
664
                      probs = c(0.025, 0.975), B = 1000, na.rm = TRUE)
665
666
      # Sum all items
667
668
      indivhorz sumrows <- rowSums(dat indivhorz, na.rm=T)</pre>
669
      indivvertical sumrows <- rowSums(dat indivvertical,na.rm=T)</pre>
670
      collhorz sumrows <- rowSums(dat collhorz,na.rm=T)</pre>
671
      collvertical sumrows <- rowSums(dat collvertical,na.rm=T)</pre>
672
673
      # Count missing items
674
675
      indivhorz summissing <-</pre>
676
        is.na(dat indivhorz$ih1) + is.na(dat indivhorz$ih2) + is.na(dat indivhorz$ih3) +
        is.na(dat_indivhorz$ih4)
677
678
679
      indivvertical summissing <-</pre>
        is.na(dat indivvertical$iv1) + is.na(dat indivvertical$iv2) +
680
        is.na(dat indivvertical$iv3) +
681
        is.na(dat indivvertical$iv4)
682
683
      collhorz summissing <-</pre>
684
        is.na(dat collhorz$ch1) + is.na(dat collhorz$ch2) + is.na(dat collhorz$ch3) +
        is.na(dat collhorz$ch4)
685
686
687
      collvertical summissing <-
688
        is.na(dat collvertical$cv1) + is.na(dat collvertical$cv2) +
        is.na(dat collvertical$cv3) +
        is.na(dat_collvertical$cv4)
689
690
691
      # Calculate mean scores
692
```

```
dat$mean indivhorz <- indivhorz sumrows/(4- indivhorz summissing)
693
694
      dat$mean indivvertical <- indivvertical sumrows/(4 -indivvertical summissing)
695
      dat$mean collhorz <- collhorz sumrows/(4 - collhorz summissing)
696
      dat$mean collvertical <- collvertical sumrows/(4 - collvertical summissing)
697
698
      # Test for collinearity
699
      #CHANGELOG ASJ: no collineary, the 4 variables will be kept for analysis as covariates,
      2021-08-03
700
701
     model <-
702
        lm(
          mean riskperception ~ mean indivhorz + mean indivvertical + mean collhorz +
703
          mean collvertical,
704
          data = dat
705
        )
706
      vif(model)
707
      ols coll diag(model)
708
709
      #### + Other data cleaning for demographics ####
710
711
      # Force year of birth as numeric and calculate age accordingly.
712
713
      dat$yearofbirth <- as.numeric(dat$yearofbirth)</pre>
714
      dat$yearofbirth[dat$yearofbirth==888] <- NA
715
      #CHANGELOG ASJ: year of the survey was postponed to 2021 instead of 2020, 2021-08-03
716
      dat$age <- 2021 - dat$yearofbirth</pre>
717
718
719
      dat$agecat <- as.numeric(dat$agecat)</pre>
720
721
      # Recode multiple answers for language and ethnicity so that people are appropriately
      counted in
722
      # each group. These questions are set up so that people "check all that apply." Each of
723
      # questions also includes a single option to indicate "I prefer not to answer." For
      each language
724
      # and ethnicity, we want to count the number of participants who affirmatively checked it
      # (indicating 'yes' for that option), those who did not check it but did check other
725
      options in the
726
      # list (indicating 'no' for that option), and those who checked that they prefer not to
727
      # (indicating 'prefer not to answer' for each option in the list). To do this, we use a
728
      # process in which we first recode the true 'no' values for each option as 0, meaning
      that all 'yes'
729
      # answers are 1 and all 'no' answers are 0. Then we assign any 'prefer not to answer'
      to be 'NA'.
730
731
      # Force variables to be numeric.
732
733
     cols.num <-
734
735
          "bornincanada",
736
          "language 1",
737
          "language 2",
738
          "language 3",
739
          "language 888",
740
          "ethnicity 1",
741
          "ethnicity 2",
742
          "ethnicity_3",
743
          "ethnicity_4",
744
          "ethnicity 5",
745
          "ethnicity 6",
          "ethnicity 7",
746
747
          "ethnicity 8",
748
          "ethnicity 9",
          "ethnicity 10",
749
750
          "ethnicity 11",
751
          "ethnicity 12",
```
```
752
          "ethnicity 13",
753
          "ethnicity 14",
754
          "ethnicity 15",
755
          "ethnicity 16",
          "ethnicity_17",
"ethnicity_888",
756
757
758
          "disability",
759
          "techdisability",
760
          "sexatbirth",
761
          "genderidentity",
762
          "supportedbyincome",
          "educationlevel",
763
764
          "studyarm",
765
          "viz",
766
          "disease",
767
          "immune",
768
          "c19vax"
769
770
771
      dat[cols.num] <- lapply(dat[cols.num],as.numeric)</pre>
772
773
      # NB. language 1=English, language 2=French, language 3=Other
774
775
      dat$language 1[is.na(dat$language 1)] <- 0</pre>
776
      dat$language 2[is.na(dat$language 2)] <- 0</pre>
      dat$language 3[is.na(dat$language 3)] <- 0</pre>
777
778
779
      dat$language 1[dat$language 888==1&dat$language 1==0&dat$language 2==0&dat$language 3==0]
780
      dat$language 2[dat$language 888==1&dat$language 1==0&dat$language 2==0&dat$language 3==0]
       <- NA
781
      dat$language 3[dat$language 888==1&dat$language 1==0&dat$language 2==0&dat$language 3==0]
782
783
      # ethnicity 1=Asian - East (e.g., Chinese, Japanese, Korean)
784
      dat$ethnicity 1[is.na(dat$ethnicity 1)] <- 0</pre>
785
      # ethnicity_2=Asian - Central (e.g., Kazakhstani, Uzbekistani)
786
      dat$ethnicity_2[is.na(dat$ethnicity_2)] <- 0</pre>
787
      # ethnicity_3=Asian - South (e.g., Indian, Pakistani, Sri Lankan)
788
      dat$ethnicity 3[is.na(dat$ethnicity 3)] <- 0</pre>
789
      # ethnicity 4=Asian - South-East (e.g., Malaysian, Filipino, Vietnamese)
790
      dat$ethnicity 4[is.na(dat$ethnicity 4)] <- 0</pre>
791
      # ethnicity 5=Indigenous or aboriginal person from outside of North America (e.g.,
      Maori, Quechua)
792
      dat$ethnicity 5[is.na(dat$ethnicity 5)] <- 0</pre>
      # ethnicity_6=White / European (e.g., English, Italian, Portuguese, Russian)
793
794
      dat$ethnicity 6[is.na(dat$ethnicity 6)] <- 0</pre>
795
      # ethnicity 7=White / North American (e.g., Canadian, American)
796
      dat$ethnicity_7[is.na(dat$ethnicity_7)] <- 0</pre>
797
      # ethnicity_8=Inuit
798
      dat$ethnicity 8[is.na(dat$ethnicity 8)] <- 0</pre>
799
      # ethnicity 9=Latin American (e.g., Chilean, Mexican, Salvadorian)
800
      dat$ethnicity 9[is.na(dat$ethnicity 9)] <- 0</pre>
801
      # ethnicity 10=Metis (Metis Nation in Canada)
802
      dat$ethnicity 10[is.na(dat$ethnicity 10)] <- 0</pre>
803
      # ethnicity_11=North African (e.g., Moroccan, Tunisian)
804
      dat$ethnicity 11[is.na(dat$ethnicity 11)] <- 0</pre>
805
      # ethnicity_12=Middle Eastern (e.g., Egyptian, Iranian, Lebanese)
806
      dat$ethnicity 12[is.na(dat$ethnicity 12)] <- 0</pre>
807
      # ethnicity_13=Black - African (e.g., Ghanaian, Kenyan, Somali)
808
      dat$ethnicity_13[is.na(dat$ethnicity_13)] <- 0</pre>
809
      # ethnicity 14=Black - Caribbean (e.g., Barbadian, Jamaican)
810
      dat$ethnicity 14[is.na(dat$ethnicity 14)] <- 0</pre>
811
      # ethnicity 15=Black - North American (e.g., Canadian, American)
812
      dat$ethnicity 15[is.na(dat$ethnicity 15)] <- 0</pre>
813
      # ethnicity 16=First Nations
814
      dat$ethnicity_16[is.na(dat$ethnicity_16)] <- 0</pre>
815
      # ethnicity 17 = 0ther
816
      dat$ethnicity 17[is.na(dat$ethnicity 17)] <- 0</pre>
```

```
818
      # Subset ethnicity values
819
820
      dat ethnicity <-
821
        subset (
822
          dat,
823
          select = c(
824
            ethnicity 1,
825
            ethnicity 2,
826
            ethnicity 3,
827
            ethnicity 4,
            ethnicity 5,
828
829
            ethnicity 6,
830
            ethnicity
831
            ethnicity 8,
            ethnicity 9,
833
            ethnicity_10,
            ethnicity_11,
834
835
            ethnicity 12,
836
            ethnicity 13,
837
            ethnicity 14,
838
            ethnicity 15,
839
            ethnicity 16,
840
            ethnicity 17
841
          )
842
        )
843
844
      # Sum of the 17 ethnicity catogories checked
845
846
      dat$sum ethnicity <-rowSums(dat ethnicity, na.rm=T)</pre>
847
848
      # Assign NA when the participant selected prefer not to answer ( 888) and no other
      option.
849
850
      dat$ethnicity 1[dat$ethnicity 888==1&dat$sum ethnicity==0] <- NA
      dat$ethnicity 2[dat$ethnicity 888==1&dat$sum ethnicity==0] <- NA
851
      dat$ethnicity_3[dat$ethnicity_888==1&dat$sum_ethnicity==0] <- NA
852
853
      dat$ethnicity_4[dat$ethnicity_888==1&dat$sum_ethnicity==0] <- NA</pre>
854
      dat$ethnicity_5[dat$ethnicity_888==1&dat$sum_ethnicity==0] <- NA
855
      dat$ethnicity_6[dat$ethnicity_888==1&dat$sum_ethnicity==0] <- NA
856
      dat$ethnicity 7[dat$ethnicity 888==1&dat$sum ethnicity==0] <- NA
857
      dat$ethnicity 8[dat$ethnicity 888==1&dat$sum ethnicity==0] <- NA
858
      dat$ethnicity 9[dat$ethnicity 888==1&dat$sum ethnicity==0] <- NA
859
      dat$ethnicity 10[dat$ethnicity 888==1&dat$sum ethnicity==0] <- NA
860
      dat$ethnicity 11[dat$ethnicity 888==1&dat$sum ethnicity==0] <- NA
861
      dat$ethnicity 12[dat$ethnicity 888==1&dat$sum ethnicity==0] <- NA
      dat$ethnicity 13[dat$ethnicity 888==1&dat$sum ethnicity==0] <- NA
862
      dat$ethnicity 14[dat$ethnicity 888==1&dat$sum ethnicity==0] <- NA
863
864
      dat$ethnicity_15[dat$ethnicity_888==1&dat$sum_ethnicity==0] <- NA
865
      dat$ethnicity_16[dat$ethnicity_888==1&dat$sum_ethnicity==0] <- NA
866
      dat$ethnicity 17 [dat$ethnicity 888==1&dat$sum ethnicity==0] <- NA
867
868
      # Regrouping ethnicities for later covariate analyses. E.g., if participant checked one
      or more of
      # Asian options, they get a 1 for Asian group. If they checked no Asian options, they
      get a 0 for
870
      # Asian group.
871
872
      dat$Asian group <-
873
        ifelse(
874
          dat$ethnicity_1 == 1 |
875
            dat$ethnicity 2 == 1 |
876
            dat$ethnicity_3 == 1 |
877
            dat$ethnicity 4 == 1,
878
          1,
879
880
        )
881
882
      dat$Black group <-
```

```
883
        ifelse(
884
          dat$ethnicity 13 == 1 |
885
            dat$ethnicity 14 == 1 |
886
            dat$ethnicity 15 == 1,
887
          1,
888
889
        )
890
891
      dat$Indigenous group <-
892
        ifelse(
893
          dat$ethnicity 16 == 1 |
894
            dat$ethnicity 5 == 1 |
895
            dat$ethnicity 8 == 1 |
896
            dat$ethnicity 10 == 1,
897
          1,
898
899
        )
900
901
      dat$MaghrebMiddleEast group <-
902
        ifelse(
903
          dat$ethnicity 11 == 1 |
904
            dat$ethnicity 12 == 1,
905
906
907
        )
908
909
     dat$White group <-
910
        ifelse(
911
          dat$ethnicity 6 == 1 |
912
            dat$ethnicity 7 == 1,
913
914
          0
915
        )
916
917
      # CHANGELOG: We are creating a new variable for high and low edcation to be later used
      in 2 way and one way ANOVA analysis 2021-07-28
918
      #CHANGELOG ASJ: We need to exclude the do not know and prefer not to answer from the
      falses, 2021-08-03
919
      dat$edhi <- ifelse(dat$educationlevel == 4 |</pre>
920
                            dat$educationlevel == 5|
921
                            dat$educationlevel == 6|
922
                            dat$educationlevel == 7, TRUE,
923
                          ifelse (dat$educationlevel == 8 | dat$educationlevel == 888, NA, FALSE))
924
      table(dat$educationlevel,dat$edhi)
925
926
      # Now we assign NA for 'prefer not to answer' responses for the rest of the
      socidemographic items.
927
      # We will report the count of 'prefer not to answer' responses in the paper, but for
      our statistical
928
      # analyses, we group these with the other responses indicating a lack of affirmative
      response.
929
930
      dat$bornincanada[dat$bornincanada==888] <- NA
931
      dat$disability[dat$disability==888] <- NA
932
      dat$techdisability[dat$techdisability==888] <- NA
933
      dat$sexatbirth[dat$sexatbirth==888] <- NA
934
      dat$genderidentity[dat$genderidentity==888] <- NA
935
      dat$income[dat$income==888] <- NA
936
      dat$income[dat$income==5] <- NA</pre>
937
      dat$supportedbyincome[dat$supportedbyincome==888] <- NA
938
      dat$educationlevel[dat$educationlevel==888] <- NA
939
      dat$educationlevel[dat$educationlevel==8] <- NA</pre>
940
941
      #CHANGELOG ASJ: i prefer not to answer also put to NA, 2021-08-03
942
      dat$agecat[dat$agecat==888 | dat$agecat==1] <- NA</pre>
943
944
      # Now we force all categorical variables as factors and add labels for ease of
      interpretation later.
945
```

```
946
       dat$bornincanada <-
 947
         factor(dat$bornincanada,
 948
                 levels = c(1, 0),
 949
                 labels = c("Yes", "No"))
 950
      dat$language_1 <-
 951
 952
         factor(dat$language_1,
 953
                levels = c(1, 0),
                labels = c("Yes", "No"))
 954
 955
 956
       dat$language 2 <-
 957
         factor(dat$language 2,
 958
                 levels = c(1, 0),
                labels = c("Yes", "No"))
 959
 960
 961
       dat$language 3 <-
         factor(dat$language_3,
 962
                levels = c(1, 0),
 963
 964
                labels = c("Yes", "No"))
 965
 966
      dat$ethnicity 1 <-
         factor(dat$\int ethnicity 1,
 967
 968
                 levels = c(1, 0),
                labels = c("Yes", "No"))
 969
 970
 971
      dat$ethnicity 2 <-
         factor(dat$ethnicity 2,
 972
 973
                 levels = c(1, 0),
 974
                labels = c("Yes", "No"))
 975
 976
       dat$ethnicity 3 <-
         factor(dat$ethnicity_3,
 977
 978
                 levels = c(1, 0),
 979
                labels = c("Yes", "No"))
 980
 981
       dat$ethnicity 4 <-
 982
         factor(dat$ethnicity 4,
 983
                 levels = c(1, 0),
                labels = c("Yes", "No"))
 984
 985
 986
       dat$ethnicity 5 <-
         factor(dat$ethnicity_5,
 987
                 levels = c(1, 0),
 988
                labels = c("Yes", "No"))
 989
 990
 991
       dat$ethnicity 6 <-
 992
         factor(dat$ethnicity 6,
 993
                 levels = c(1, 0),
                 labels = c("Yes", "No"))
 994
 995
 996
      dat$ethnicity 7 <-
 997
         factor(dat$ethnicity 7,
 998
                 levels = c(1, 0),
 999
                labels = c("Yes", "No"))
1000
1001
       dat$ethnicity 8 <-
1002
         factor(dat$ethnicity_8,
1003
                 levels = c(1, 0),
                 labels = c("Yes", "No"))
1004
1005
1006
       dat$ethnicity 9 <-
1007
         factor(dat$ethnicity 9,
1008
                 levels = c(1, 0),
                labels = c("Yes", "No"))
1009
1010
1011
       dat$ethnicity 10 <-
1012
         factor(dat$ethnicity_10,
1013
                 levels = c(1, 0),
1014
                 labels = c("Yes", "No"))
```

```
1015
1016
       dat$ethnicity 11 <-
1017
         factor(dat$ethnicity_11,
1018
                levels = c(1, 0),
                labels = c("Yes", "No"))
1019
1020
1021
      dat$ethnicity 12 <-
1022
         factor(dat$ethnicity 12,
1023
                levels = c(1, 0),
                labels = c("Yes", "No"))
1024
1025
1026
      dat$ethnicity 13 <-
1027
         factor(dat$ethnicity 13,
1028
                levels = c(1, 0),
                labels = c("Yes", "No"))
1029
1030
1031
       dat$ethnicity 14 <-
1032
         factor(dat$ethnicity 14,
1033
                levels = c(1, 0),
1034
                labels = c("Yes", "No"))
1035
1036
      dat$ethnicity 15 <-
1037
         factor(dat$ethnicity 15,
1038
                levels = c(1, 0),
1039
                labels = c("Yes", "No"))
1040
1041
      dat$ethnicity 16 <-
1042
        factor(dat$ethnicity_16,
1043
                levels = c(1, 0),
                labels = c("Yes", "No"))
1044
1045
1046
      dat$ethnicity 17 <-
1047
         factor(dat$ethnicity 17,
1048
                levels = c(1, 0),
                labels = c("Yes", "No"))
1049
1050
1051
       dat$Asian group <-
1052
         factor(dat$Asian_group,
1053
                levels = c(1, 0),
1054
                labels = c("Yes", "No"))
1055
1056
       dat$MaghrebMiddleEast group <-</pre>
1057
         factor(dat$MaghrebMiddleEast group,
1058
                levels = c(1, 0),
                labels = c("Yes", "No"))
1059
1060
1061
       dat$Black group <-
1062
         factor(dat$Black_group,
1063
                levels = c(1, 0),
1064
                labels = c("Yes", "No"))
1065
1066
      dat$White group <-
1067
         factor(dat$White group,
1068
                levels = c(1, 0),
1069
                labels = c("Yes", "No"))
1070
1071
       dat$Indigenous group <-
1072
         factor(dat$Indigenous group,
1073
                levels = c(1, 0),
                labels = c("Yes", "No"))
1074
1075
1076
      dat$disability <-
1077
         factor(
1078
           dat$disability,
1079
           levels = c(0, 1),
1080
           labels = c("No disability", "yes, at least one")
1081
1082
1083
       dat$techdisability <-
```

```
1084
         factor (dat$techdisability,
1085
                 levels = c(0, 1),
1086
                 labels = c("No", "Yes"))
1087
1088
      dat$sexatbirth <-
1089
         factor(dat$sexatbirth,
1090
                 levels = c(1, 2),
1091
                labels = c("Female", "Male"))
1092
1093
      dat$genderidentity <- factor(</pre>
1094
         dat$genderidentity,
1095
         levels = c(1, 2, 3, 4),
         labels = c(
1096
           "Female",
1097
1098
           "Male",
1099
           "Indigenous or other cultural gender minority identity",
1100
           "Something else"
1101
1102
       )
1103
1104
      dat$income <-
1105
         factor (
1106
           dat$income,
1107
           levels = c(1, 2, 3, 4),
           labels = c("24 999 \text{ or less"}, "25 000 to 49 999",
1108
                       "50 000 to 99 999", "100 000 or more")
1109
1110
1111
      dat$educationlevel <- factor(
1112
1113
         dat$educationlevel,
1114
         levels = c(1, 2, 3, 4, 5, 6, 7),
1115
         labels = c(
1116
           "Some Elementary School",
1117
           "High School Diploma",
1118
           "Apprenticeship or trade certificate or diploma",
1119
           "College or polytechnical school certificate or diploma",
1120
           "University degree bachelor level or below",
1121
           "University graduate degree Master level",
1122
            "University graduate degree Doctorate level"
1123
         )
1124
       )
1125
1126
      dat$agecat<-
1127
         factor(
1128
           dat$agecat,
1129
           levels = c(2, 3, 4),
1130
           labels = c("18-34 \text{ years}", "35-49 \text{ years}", "50 \text{ years and more}")
1131
1132
1133
       dat$UserLanguage <- as.factor(dat$UserLanguage)</pre>
1134
1135
      dat$studyarm <-
1136
        factor (
1137
           dat$studyarm,
1138
           levels = c(0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 11, 12, 13),
1139
           labels = c(
1140
             "controlgeneric",
             "controlmeasles",
1141
             "controlpertussis",
1142
             "controlflu",
1143
             "herdimmgeneric",
1144
1145
             "herdimmmeasles",
1146
             "herdimmpertussis",
             "herdimmflu",
1147
             "robertkochgeneric",
1148
1149
             "sbsnewsgeneric",
             "guardianmeasles",
1150
1151
             "theotheredmundmeasles",
             "publichealthagencycanadaflu"
1152
```

```
1153
           )
1154
         )
1155
1156
      dat$viz <- factor (
1157
         dat$viz,
         levels = c(0, 1, 2, 3, 5, 6, 7),
1158
1159
         labels = c(
1160
           "no visualization",
           "herdimm",
1161
           "robertkoch",
1162
           "sbsnews",
1163
           "quardian",
1164
1165
           "theotheredmund",
1166
           "publichealthagencycanada"
1167
1168
1169
1170
      dat$disease <-
1171
       factor (
1172
           dat$disease,
1173
           levels = c(0, 1, 2, 3),
1174
           labels = c("Generic", "Measles", "Pertussis", "Flu")
1175
         )
1176
1177
       #Keep I don't know categories as is, not as NA, to distinguish them, for these special
1178
       variables (COVID-19)
1179
      dat$immune <-
1180
         factor(
1181
           dat$immune,
1182
           levels = c(1, 0, 77),
1183
           labels = c("Yes", "No", "I don't know")
1184
1185
1186
       dat$c19vax <-
1187
         factor(
1188
           dat$c19vax,
1189
           levels = c(1, 0, 77),
1190
           labels = c("Yes", "No", "I don't know")
1191
         )
1192
1193
       #CHANGELOG ASJ: All variables related to children were removed from the final survey
       and are deleted in the rest of the code (children, childimmune, childfluvax), 2021-08-06.
1194
1195
1196
       #Make restrictions on the dataset for analysis of patients kept for analysis vs not
       kept for analysis
1197
       #CHANGELOG ASJ: Variables were different than planned, subset done differently because
       of gc, 2021-08-06.
1198
       datConsent<- subset (datRaw, Consent==1)</pre>
1199
       datConsent$used<-ifelse(datConsent$gc==1 & datConsent$Finished ==1, 1,0) #used in our
       analysis (n = 5516 vs others with consent (not finished, no quality))
1200
       table(datConsent$used)
1201
1202
1203
       # Note re: possibly recoding low-frequency data after collecting data
1204
1205
       # If we observe low frequencies (below 5%) among socio demographic variables, we will
       recode these
1206
       # groups. This is because small subgroups are unlikely to work well in our planned
       statistical
1207
       # models.
1208
       # Descriptive statistics of all original variables will be examined. The following
1209
       steps will be
1210
       # used if a category has frequency smaller than 5% of the total sample. We anticipate
       this may be
1211
       # necessary for gender identity and education level.
1212
```

```
# For gender identity, we will remove smaller categories from inclusion in analytical
1213
       models since
1214
       # they cannot be combined with other category. We still still report these statistics
       in the
1215
       # sociodemographic statistics of the same and will otherwise use these participants'
       data as usual.
1216
       # This means that if categories 3 and 4 have frequencies smaller than 5 % than we will
       use this
1217
       # code:
1218
1219
       #CHANGELOG ASJ: the variable is a factor, need to exclude with text instead of numbers,
1220
       #CHANGELOG ASJ: this is removed from comments since <5% answered the two last categories
1221
       dat$genderidentity[dat$genderidentity == "Something else" |
1222
                             dat$genderidentity == "Indigenous or other cultural gender
                             minority identity"] <- NA
1223
       dat$genderidentity <- droplevels(dat$genderidentity)</pre>
1224
1225
       # For education level, we will regroup smaller categories with the closest bigger
       categories with
       # which it makes sense to group them. If, for example, there are small frequencies for
1226
1227
       # elementary school' we will regroup it with high school diploma. Potential code would
       be:
1228
       # dat$educationlevel[dat$educationlevel== 1] <- 2; dat$educationlevel <-</pre>
1229
       \# factor(dat$educationlevel,levels = c(2,3,4,5,6,7), labels = c("Some Elementary School")
1230
       or High
1231
       # School Diploma", "Apprenticeship or trade certificate or diploma College or
       polytechnical school
       # certificate or diploma", "University degree bachelor level or below", "University
1232
       graduate degree
1233
       # Master level", "University graduate degree Doctorate level", "Do not know"))
1234
1235
       #CHANGELOG ASJ: Education was recoded as high vs low in edhi variable above, instead of
       using this code, 2021-08-03.
1236
1237
       # The rest won't change unless we need to. If we observe another category with
       frequency below 5%,
1238
       # we will follow similar procedures.
1239
1240
       #CHANGELOG ASJ: Several covariates have categories with <5% (language 3,
       MaghrebMiddleEast group, Black group, Indigenous group, ethnicity 9, techdisability).
       However, they are dichotomous variable, so it is not possible to combine categories.
       They will simply be dropped from the models.
1241
       #CHANGELOG ASJ: However, for techdisability, it will be combined with disability, we
       don't want to loose that information. 2021-08-03.
1242
       dat$disability any <-ifelse(dat$disability =="yes,at least one" | dat$techdisability ==</pre>
       "Yes", 1, 0)
1243
       dat$disability any <-
1244
         factor(
1245
           dat$disability any,
1246
           levels = c(1, 0),
           labels = c("Yes", "No")
1247
1248
         )
1249
1250
       #CHANGELOG ASJ: As mentioned later on in the preregistered code, we are recoding here
       trust info because it is asymetric, 2021-08-03
1251
       dat$Htrustinfo <- ifelse(dat$trustinfo >= 5, 1, 0)
1252
       dat$Htrustinfo <-
1253
         factor(
1254
           dat$Htrustinfo,
           levels = c(1, 0),
1255
           labels = c("Yes", "No")
1256
1257
1258
1259
       #CHANGELOG ASJ: Because 1st variable of risk perception does not have enough variance
       and is asymetric, recode as dichotomic variable, 2021-08-03
1260
       #CHANGELOG ASJ: Cutpoint = 80, keep people who correctly identified a high risk,
```

```
2021-08-06.
1261
       hist(dat$riskpercep1 1)
1262
       dat$RP1_dicho <- ifelse(dat$riskpercep1_1 >= 80, 1, 0)
1263
      dat$RP1 dicho <-
1264
         factor(
           dat$RP1 dicho,
1265
1266
           levels = c(1, 0),
1267
           labels = c("High", "Low")
1268
1269
      table(dat$RP1 dicho)
1270
1271
       #CHANGELOG ASJ: Because vaxintention does not have enough variance and is asymetric,
       recode as dichotomic variable, 2021-08-06.
1272
       #CHANGELOG ASJ: Cutpoint = 91, at or above median.
1273
       hist(dat$vaxintention 1)
1274
       summary(dat$vaxintention 1)
1275
       dat$vaxintent<-ifelse(dat$vaxintention 1>=91,1,0)
1276
1277
       dat$vaxintent <-
1278
        factor(
1279
           dat$vaxintent,
1280
           levels = c(1, 0),
1281
           labels = c("High", "Low")
1282
1283
1284
       table(dat$vaxintent)
1285
1286
       #CHANGELOG ASJ: Because c19vaxintention does not have enough variance and is asymetric,
       recode as dichotomic variable, 2021-08-06.
1287
       #CHANGELOG ASJ: Cutpoint = 90, at or above median.
      hist(dat$c19vaxintention_1)
1288
1289
       summary(dat$c19vaxintention 1)
1290
       dat$c19vaxintent<-ifelse(dat$c19vaxintention 1>=90,1,0)
1291
1292
       dat$c19vaxintent <-
1293
        factor(
1294
           dat$c19vaxintent,
1295
           levels = c(1, 0),
           labels = c("High", "Low")
1296
1297
1298
1299
       table (dat$c19vaxintent)
1300
1301
       #### + Subsets for primary and secondary analyses ####
1302
1303
       # We create new subsets for primary and secondary analyses. The first subset (datMain)
       is for our
1304
       # primary research question. The other subsets are for the secondary question.
1305
1306
      datMain <-
1307
       subset (
1308
           dat,
1309
           dat$studyarm == "controlgeneric" |
1310
             dat$studyarm == "controlmeasles" |
1311
             dat$studyarm == "controlpertussis" |
             dat$studyarm == "controlflu" |
1312
1313
             dat$studyarm == "herdimmgeneric" |
1314
             dat$studyarm == "herdimmmeasles" |
             dat$studyarm == "herdimmpertussis" |
1315
             dat$studyarm == "herdimmflu"
1316
1317
         )
1318
1319
       don<-subset(datMain, select=c(studyarm, mean riskperception, viz, disease, mean indivhorz,</pre>
1320
                                    mean indivvertical,
1321
                                     mean collhorz ,
1322
                                     mean collvertical,
1323
                                     bornincanada ,
1324
                                     language 1 ,
1325
                                     language 2 ,
```

```
Asian group ,
1326
1327
                                    White group,
1328
                                     disability any ,
1329
                                      genderidentity ,
1330
                                      income ,
1331
                                     edhi,
1332
                                     age,
1333
                                    mean riskperception2 6,RP1 dicho, vaxintent, mean emotion, sum k
                                    nowledge, Htrustinfo,
1334
                                    mean C5 conf2, mean C5 comp2, mean C5 cons2, mean C5 calc2, mean
                                    C5 coll2)) # CHANGELOG ASJ updated restrictions
1335
                                             #Added the code to determine the missing data
1336
                                           # for variables later used in ANOVA analysis, only
                                           those with >5\%, 2021-08-03
1337
                                           #remove c19vaxintent, too many missing values
1338
1339
1340
1341
      datGeneric <-
1342
         subset (
1343
           dat.
1344
1345
             dat$studyarm == "controlgeneric" |
1346
                dat$studyarm == "herdimmgeneric" |
                dat$studyarm == "robertkochgeneric" |
1347
1348
               dat$studyarm == "sbsnewsgeneric"
1349
           . &
1350
             UserLanguage == "EN"
1351
1352
1353
      datMeasles <-
        subset (
1354
1355
           dat,
           dat$studyarm == "controlmeasles" |
1356
1357
             dat$studyarm == "herdimmmeasles" |
1358
             dat$studyarm == "guardianmeasles" |
1359
             dat$studyarm == "theotheredmundmeasles"
1360
         )
1361
1362
      datFlu <-
1363
        subset (
1364
           dat,
1365
           dat$studyarm == "controlflu" |
1366
             dat$studyarm == "herdimmflu" |
1367
             dat$studyarm == "publichealthagencycanadaflu"
1368
1369
1370
       datMain$studyarm <- droplevels(datMain$studyarm)</pre>
1371
       datGeneric$studyarm <- droplevels(datGeneric$studyarm)</pre>
1372
       datMeasles$studyarm <- droplevels(datMeasles$studyarm)</pre>
1373
       datFlu$studyarm <- droplevels(datFlu$studyarm)</pre>
1374
1375
      #CHANGELOG ASJ, save r dataset for analysis, 2021-09-03
1376
      write.csv(dat, file="./datMain.csv", row.names=T)
1377
       write.csv(dat, file="./datGeneric.csv", row.names=T)
       write.csv(dat, file="./datMeasles.csv", row.names=T)
1378
1379
       write.csv(dat, file="./datFlu.csv", row.names=T)
1380
1381
       save (dat, file="dat.RData")
1382
       save (datMain, file="datMain.RData")
1383 save (datGeneric, file="datGeneric.RData")
1384 save (datMeasles, file="datMeasles.RData")
1385
       save (datFlu, file="datFlu.RData")
1386
       save (datConsent, file="datConsent.RData")
1387
1388
       #### DESCRIPTIVE STATISTICS ####
1389
```

```
1390
      # For each variable separately
1391
1392
      ### Nominal variables - independent variables to which people were randomized
1393
1394
      # frequencies - study arm
1395
      table (dat$studyarm)
1396
     # proportion of each study arm that is
1397
      # 0 = controlgeneric
1398
     # 1 = controlmeasles
1399
     # 2 = controlpertussis
1400
     # 3 = controlflu
      # 4 = herdimmgeneric
1401
      #5 = herdimmmeasles
1402
1403
      # 6 = herdimmpertussis
      #7 = herdimmflu
1404
1405
      # 8 = robertkochgeneric
      # 9 = sbsnewsgeneric
1406
1407
     # 10 = nhsgeneric (no longer included because has been taken down)
1408 # 11 = guardianmeasles
1409 # 12 = theotheredmundmeasles
1410 # 13 = publichealthagencycanadaflu
1411 prop.table(table(dat$studyarm)) * 100
1412
1413
     # frequencies - Visualization
      table(dat$viz, exclude = NULL)
1414
1415
      # proportion of each visualization that is
1416
      # 0 = no visualization
1417
      #1 = herdimm
1418
      #2 = robertkoch
1419
     # 3 = sbsnews
1420 # 4 = nhs (no longer included because has been taken down)
1421 # 5 = quardian
1422
     # 6 = theotheredmund
1423
     # 7 = publichealthagencycanada
1424
      prop.table(table(dat$viz, exclude = NULL)) * 100
1425
      # frequencies - Disease
1426
1427
      table (dat$disease, exclude = NULL)
1428
      # proportion of each disease that is
1429
      # 0 = Generic
1430 # 1 = Measles
1431
      #2 = Pertussis
1432
      #3 = Flu
1433
     prop.table(table(dat$disease, exclude = NULL)) * 100
1434
1435
      ### Nominal variables - in what language did the person complete the survey
1436
1437
      # frequencies - User-language for survey
1438
      table(dat$UserLanguage, exclude = NULL)
1439
      # proportion of language that is
1440
     # English (EN)
1441
      # French (FR-CA)
1442
      prop.table(table(dat$UserLanguage, exclude = NULL)) * 100
1443
1444
      ### Nominal variables - Demographics # proportion of each demographic variable
1445
      # CHANGELOG exclude = NULL added in code below to detemine NA's in the variable
      2021-05-10
1446
1447
       # frequencies - place of birth (Canada or outside Canada)
1448
       table (dat$bornincanada, exclude = NULL)
1449
      prop.table(table(dat$bornincanada, exclude = NULL)) * 100
1450
1451
       # frequencies - Language English
1452
      table(dat$language 1, exclude = NULL)
1453
      prop.table(table(dat$language 1, exclude = NULL)) * 100
1454
1455
      # frequencies - Language_French
1456
      table(dat$language 2,exclude = NULL)
1457
       prop.table(table(dat$language 2,exclude = NULL)) * 100
```

```
1458
1459
       # frequencies - Language Other
1460
       table(dat$language 3,exclude = NULL)
1461
       prop.table(table(dat$language 3,exclude = NULL)) * 100
1462
       # frequencies - Ethnicity_Asian - East (e.g., Chinese, Japanese, Korean)
1463
1464
       table(dat$ethnicity 1, exclude = NULL)
1465
       prop.table(table(dat$ethnicity 1, exclude = NULL)) * 100
1466
1467
       # frequencies - Ethnicity Asian - Central (e.g., Kazakhstani, Uzbekistani)
       table(dat$ethnicity 2, exclude = NULL)
1468
1469
       prop.table(table(dat$ethnicity 2,exclude = NULL)) * 100
1470
1471
       # frequencies - Ethnicity Asian - South (e.g., Indian, Pakistani, Sri Lankan)
1472
       table(dat$ethnicity 3, exclude = NULL)
1473
       prop.table(table(dat$ethnicity 3, exclude = NULL)) * 100
1474
1475
       # frequencies - Ethnicity Asian - South-East (e.g., Malaysian, Filipino, Vietnamese)
1476
       table(dat$ethnicity 4, exclude = NULL)
1477
       prop.table(table(dat$ethnicity 4, exclude = NULL)) * 100
1478
1479
       # frequencies - Ethnicity Indigenous or aboriginal person from outside of North America
       (e.g.,
1480
       # Maori, Quechua)
1481
       table(dat$ethnicity 5, exclude = NULL)
       prop.table(table(dat$ethnicity 5, exclude = NULL)) * 100
1482
1483
       # frequencies - Ethnicity_White / European (e.g., English, Italian, Portuguese, Russian)
1484
1485
      table(dat$ethnicity 6, exclude = NULL)
1486
       prop.table(table(dat$ethnicity 6, exclude = NULL)) * 100
1487
1488
       # frequencies - Ethnicity White / North American (e.g., Canadian, American)
1489
       table(dat$ethnicity 7, exclude = NULL)
1490
       prop.table(table(dat$ethnicity 7, exclude = NULL)) * 100
1491
1492
       # frequencies - Ethnicity Inuit
1493
       table(dat$ethnicity 8, exclude = NULL)
1494
       prop.table(table(dat$ethnicity 8,exclude = NULL)) * 100
1495
1496
       # frequencies - Ethnicity Latin American (e.g., Chilean, Mexican, Salvadorian)
1497
       table(dat$ethnicity 9,exclude = NULL)
1498
       prop.table(table(dat$ethnicity 9, exclude = NULL)) * 100
1499
1500
       # frequencies - Ethnicity Metis (Metis Nation in Canada)
1501
       table (dat$ethnicity 10, exclude = NULL)
1502
       prop.table(table(dat$ethnicity_10,exclude = NULL)) * 100
1503
1504
       # frequencies - Ethnicity North African (e.g., Moroccan, Tunisian)
1505
       table(dat$ethnicity 11,exclude = NULL)
1506
       prop.table(table(dat$ethnicity 11,exclude = NULL)) * 100
1507
1508
       # frequencies - Ethnicity Middle Eastern (e.g., Egyptian, Iranian, Lebanese)
1509
       table (dat$ethnicity 12, exclude = NULL)
1510
       prop.table(table(dat$ethnicity 12,exclude = NULL)) * 100
1511
1512
       # frequencies - Ethnicity_Black - African (e.g., Ghanaian, Kenyan, Somali)
1513
       table(dat$ethnicity 13,exclude = NULL)
1514
       prop.table(table(dat$ethnicity 13,exclude = NULL)) * 100
1515
1516
       # frequencies - Ethnicity Black - Caribbean (e.g., Barbadian, Jamaican)
1517
       table(dat$ethnicity_14,exclude = NULL)
1518
       prop.table(table(dat$ethnicity 14,exclude = NULL)) * 100
1519
1520
       # frequencies - Ethnicity Black - North American (e.g., Canadian, American)
1521
       table (dat$ethnicity 15, exclude = NULL)
1522
       prop.table(table(dat$ethnicity 15,exclude = NULL)) * 100
1523
1524
       # frequencies - Ethnicity First Nations
1525
       table(dat$ethnicity 16,exclude = NULL)
```

```
1526
       prop.table(table(dat$ethnicity 16,exclude = NULL)) * 100
1527
1528
       # frequencies - Ethnicity Other
1529
       table(dat$ethnicity 17, exclude = NULL)
1530
      prop.table(table(dat$ethnicity 17,exclude = NULL)) * 100
1531
1532
       # frequencies - Asian group
1533
      table(dat$Asian group, exclude = NULL)
1534
      prop.table(table(dat$Asian group, exclude = NULL)) * 100
1535
       # frequencies - Black group
1536
1537
      table(dat$Black group, exclude = NULL)
1538
       prop.table(table(dat$Black group, exclude = NULL)) * 100
1539
1540
       # frequencies - Indigenous group
1541
       table (dat$Indigenous group, exclude = NULL)
       prop.table(table(dat$Indigenous group, exclude = NULL)) * 100
1542
1543
1544
       # frequencies - MaghrebMiddleEast group
1545
      table(dat$MaghrebMiddleEast group, exclude = NULL)
1546
       prop.table(table(dat$MaghrebMiddleEast group, exclude = NULL)) * 100
1547
1548
      # frequencies - White group
1549
      table (dat$White group, exclude = NULL)
1550
       prop.table(table(dat$White group, exclude = NULL)) * 100
1551
1552
       # frequencies - disability
1553
      table (dat$disability, exclude = NULL)
1554
      prop.table(table(dat$disability,exclude = NULL)) * 100
1555
1556
       # frequencies - tech disability
1557
      table (dat$techdisability, exclude = NULL)
1558
      prop.table(table(dat$techdisability, exclude = NULL)) * 100
1559
1560
      #CHANGELOG ASJ: frequencies - any disability, 2021-08-03
1561
       table (dat$disability any, exclude = NULL)
1562
      prop.table(table(dat$disability any, exclude = NULL)) * 100
1563
1564
       # frequencies - sex at birth
1565
      table(dat$sexatbirth, exclude = NULL)
1566
      prop.table(table(dat$sexatbirth, exclude = NULL)) * 100
1567
1568
       # frequencies - gender identity
1569
      table(dat$genderidentity, exclude = NULL)
1570
      prop.table(table(dat$genderidentity, exclude = NULL)) * 100
1571
1572
      # frequencies - income
1573
      table(dat$income, exclude = NULL)
1574
      prop.table(table(dat$income, exclude = NULL)) * 100
1575
1576
       # frequencies - supportedbyincome
1577
      table(dat$supportedbyincome, exclude = NULL)
1578
      prop.table(table(dat$supportedbyincome, exclude = NULL)) * 100
1579
1580
       # frequencies - education level
1581
      table (dat$educationlevel, exclude = NULL)
1582
       prop.table(table(dat$educationlevel, exclude = NULL)) * 100
1583
1584
       #CHANGELOG ASJ: frequencies - education level high vs low, 2021-08-03
1585
       table(dat$edhi, exclude = NULL)
1586
      prop.table(table(dat$edhi, exclude = NULL)) * 100
1587
1588
       # frequencies - age category
1589
       table(dat$agecat,exclude = NULL)
1590
      prop.table(table(dat$agecat, exclude = NULL)) * 100
1591
1592
       # frequencies - already immune
1593
      table(dat$immune, exclude = NULL)
1594
       prop.table(table(dat$immune, exclude = NULL)) * 100
```

```
1595
1596
       # frequencies - COVID-19 vax
1597
       table (dat$c19vax, exclude = NULL)
1598
       prop.table(table(dat$c19vax, exclude = NULL)) * 100
1599
1600
1601
       ### Nominal variables - Other variables
1602
      #CHANGELOG ASJ: Section added for new variables created, 2021-08-03
1603
      table(dat$Htrustinfo)
1604
      prop.table(table(dat$Htrustinfo)) * 100
1605
1606
      table (dat$RP1 dicho)
1607
       prop.table(table(dat$RP1 dicho)) * 100
1608
1609
       table(dat$c19vaxintent)
1610
      prop.table(table(dat$c19vaxintent)) * 100
1611
1612
       table (dat$vaxintent)
1613
       prop.table(table(dat$vaxintent)) * 100
1614
1615
       #CHANGELOG ASJ: Add new variables 21-09-03
1616
       table (dat$mean C5 conf2)
1617
       prop.table(table(dat$mean C5 conf2)) * 100
1618
1619
       table(dat$mean C5 comp2)
1620
       prop.table(table(dat$mean C5 comp2)) * 100
1621
1622
      table(dat$mean C5 cons2)
1623
      prop.table(table(dat$mean C5 cons2)) * 100
1624
1625
      table(dat$mean C5 calc2)
1626
      prop.table(table(dat$mean C5 calc2)) * 100
1627
      table (dat$mean C5 coll2)
1628
1629
       prop.table(table(dat$mean C5 coll2)) * 100
1630
       ### Continuous variables - Demographics, scales, etc.
1631
1632
1633
       # Summary statistics for each continuous variable for all participants
1634
       summary (dat$mean riskperception) #CHANGELOG ASJ: this is equivalent to
       riskperception2 6 2021-08-03
1635
       summary(dat$score riskpercep1 1) # CHANGELOG Added separate analysis for risk
       perception item 1 2021-07-08
1636
       summary (dat$mean riskperception2 6) # CHANGELOG Added separate analysis for risk
       perception item 2 to 6 2021-07-08
1637
       summary (dat$mean C5) #CHANGELOG Added separate analysis for 5 subscales, 2021-08-06
1638
       summary(dat$mean C5 conf)
1639
       summary(dat$mean C5 comp)
      summary(dat$mean_C5_cons)
1640
1641
      summary(dat$mean_C5_calc)
1642
     summary(dat$mean C5 coll)
1643 summary (dat$mean emotion)
1644 summary(dat$sum_knowledge)
1645
      summary(dat$trustinfo)
1646
       summary(dat$vaxintention 1)
1647
       summary(dat$age)
1648
       summary(dat$c19vaxintention 1)
1649
       summary(dat$mean indivhorz)
1650
       summary(dat$mean indivvertical)
       summary(dat$mean_collhorz)
1651
1652
       summary(dat$mean collvertical)
1653
1654
       #### + Descriptive statistics per study arm ####
1655
       ### Continuous variables
1656
1657
1658
       # The describeBy function in the psych package returns the number of observations,
       mean, median,
1659
       # trimmed means, minimum, maximum, range, skew, kurtosis, and standard error of the
```

```
mean for grouped
1660
       # data.
1661
1662
       describeBy (dat$mean riskperception, dat$studyarm) #CHANGELOG ASJ: this is equivalent to
       riskperception2 6 2021-08-03
1663
       describeBy(dat$riskpercep1 1,dat$studyarm) # CHANGELOG Added separate analysis for risk
       perception item 1 2021-07-08
1664
       describeBy(dat$mean riskperception2 6,dat$studyarm) # CHANGELOG Added separate analysis
       for risk perception item 2 to 6 202\overline{1}-07-08
       describeBy(dat$mean C5,dat$studyarm) #CHANGELOG Added separate analysis for 5
1665
       subscales, 2021-08-06
       describeBy(dat$mean C5 conf,dat$studyarm)
1666
       describeBy (dat$mean C5 comp, dat$studyarm)
1667
       describeBy(dat$mean C5 cons, dat$studyarm)
1668
       describeBy (dat$mean C5 calc, dat$studyarm)
1669
       describeBy(dat$mean_C5_coll,dat$studyarm)
1670
1671
       describeBy(dat$mean_emotion, dat$studyarm)
1672
       describeBy(dat$sum knowledge,dat$studyarm)
1673
       describeBy (dat$age, dat$studyarm)
1674
       describeBy (dat$trustinfo, dat$studyarm)
1675
       describeBy(dat$vaxintention 1, dat$studyarm)
1676
       describeBy(dat$c19vaxintention 1, dat$studyarm)
1677
       describeBy(dat$mean indivhorz, dat$studyarm)
1678
       describeBy(dat$mean indivvertical, dat$studyarm)
1679
       describeBy(dat$mean collhorz, dat$studyarm)
1680
       describeBy(dat$mean collvertical, dat$studyarm)
1681
1682
       ### Nominal variables - frequencies and proportion per arm
1683
1684
      t1<-data.frame(dat$bornincanada,dat$studyarm)
1685
      table(t1)
1686
      prop.table(table(t1), 2) * 100
1687
      # Language English
1688
1689
      t1<-data.frame(dat$language 1,dat$studyarm)</pre>
1690
       table(t1)
1691
       prop.table(table(t1), 2) * 100
1692
1693
       # Language French
       t1<-data.frame(dat$language 2,dat$studyarm)</pre>
1694
1695
       table(t1)
1696
       prop.table(table(t1), 2) * 100
1697
1698
       # Language Other
1699
       t1<-data.frame(dat$language 3,dat$studyarm)</pre>
1700
       table (t1)
1701
       prop.table(table(t1), 2) * 100
1702
1703
       # Asian - East (e.g., Chinese, Japanese, Korean)
1704
       t1<-data.frame(dat$ethnicity 1,dat$studyarm)
1705
       table(t1)
1706
       prop.table(table(t1), 2) * 100
1707
1708
       # Asian - Central (e.g., Kazakhstani, Uzbekistani)
1709
       t1<-data.frame(dat$ethnicity 2,dat$studyarm)
1710
       table(t1)
1711
       prop.table(table(t1), 2) * 100
1712
1713
       # Asian - South (e.g., Indian, Pakistani, Sri Lankan)
1714
       t1<-data.frame(dat$ethnicity 3,dat$studyarm)
1715
       table (t1)
1716
       prop.table(table(t1), 2) * 100
1717
1718
       # Asian - South-East (e.g., Malaysian, Filipino, Vietnamese)
1719
       t1<-data.frame(dat$ethnicity 4,dat$studyarm)
1720
       table (t1)
1721
       prop.table(table(t1), 2) * 100
1722
1723
       # Indigenous or aboriginal person from outside of North America (e.g., Maori, Quechua)
```

```
1724
       t1<-data.frame(dat$ethnicity 5, dat$studyarm)
1725
      table(t1)
1726
      prop.table(table(t1), 2) * 100
1727
       # White / European (e.g., English, Italian, Portuguese, Russian)
1728
1729
      t1<-data.frame(dat$ethnicity 6,dat$studyarm)
1730
     table(t1)
1731
      prop.table(table(t1), 2) * 100
1732
1733
      # White / North American (e.g., Canadian, American)
1734 t1<-data.frame(dat$ethnicity 7, dat$studyarm)
1735 table(t1)
1736
      prop.table(table(t1), 2) * 100
1737
1738
      # Inuit
1739
      t1<-data.frame(dat$ethnicity 8, dat$studyarm)
1740 table(t1)
1741 prop.table(table(t1), 2) * 100
1742
1743
     # Latin American (e.g., Chilean, Mexican, Salvadorian)
1744 t1<-data.frame(dat$ethnicity 9,dat$studyarm)
1745
     table(t1)
1746
      prop.table(table(t1), 2) * 100
1747
1748
      # Metis (Metis Nation in Canada)
1749
      t1<-data.frame(dat$ethnicity 10,dat$studyarm)
1750
      table(t1)
1751
      prop.table(table(t1), 2) * 100
1752
1753
      # North African (e.g., Moroccan, Tunisian)
1754 t1<-data.frame(dat$ethnicity_11,dat$studyarm)
1755
     table(t1)
1756
      prop.table(table(t1), 2) * 100
1757
1758
      # Middle Eastern (e.g., Egyptian, Iranian, Lebanese)
1759
     t1<-data.frame(dat$ethnicity 12,dat$studyarm)
1760
      table(t1)
1761
      prop.table(table(t1), 2) * 100
1762
1763
      # Black - African (e.g., Ghanaian, Kenyan, Somali)
1764 t1<-data.frame(dat$ethnicity 13,dat$studyarm)
1765 table(t1)
1766
      prop.table(table(t1), 2) * 100
1767
1768
      # Black - Caribbean (e.g., Barbadian, Jamaican)
1769 t1<-data.frame(dat$ethnicity 14,dat$studyarm)
1770
      table(t1)
1771
      prop.table(table(t1), 2) * 100
1772
1773
       # Black - North American (e.g., Canadian, American)
1774
     t1<-data.frame(dat$ethnicity 15,dat$studyarm)
1775
      table(t1)
1776
      prop.table(table(t1), 2) * 100
1777
1778
     # First Nations
1779 t1<-data.frame(dat$ethnicity 16,dat$studyarm)
1780
     table(t1)
1781
      prop.table(table(t1), 2) * 100
1782
1783
       # Other
1784
      t1<-data.frame(dat$ethnicity 17, dat$studyarm)
1785
      table(t1)
1786
      prop.table(table(t1), 2) * 100
1787
1788
       # Asian group
1789 t1<-data.frame(dat$Asian group,dat$studyarm)
1790
      table(t1)
1791
       prop.table(table(t1), 2) * 100
1792
```

```
1793
     # MaghrebMiddleEast group
1794 t1<-data.frame(dat$MaghrebMiddleEast group,dat$studyarm)
1795
      table(t1)
1796
     prop.table(table(t1), 2) * 100
1797
1798
     # Black_group
1799
     t1<-data.frame(dat$Black group,dat$studyarm)
1800 table(t1)
1801 prop.table(table(t1), 2) * 100
1802
1803 # White group
1804 t1<-data.frame(dat$White group,dat$studyarm)
1805 table(t1)
      prop.table(table(t1), 2) * 100
1806
1807
1808
     # Indigenous group
1809
     t1<-data.frame(dat$Indigenous group,dat$studyarm)
1810 table(t1)
1811 prop.table(table(t1), 2) * 100
1812
1813
     # disability
1814 t1<-data.frame(dat$disability,dat$studyarm)
1815 table(t1)
1816 prop.table(table(t1), 2) * 100
1817
1818
     # tech disability
     t1<-data.frame(dat$techdisability,dat$studyarm)
1819
1820 table(t1)
1821
     prop.table(table(t1), 2) * 100
1822
1823
     #CHANGELOG ASJ: add any disability, 2021-08-03
1824 t1<-data.frame(dat$disability any,dat$studyarm)
1825 table(t1)
1826
     prop.table(table(t1), 2) * 100
1827
1828
     # sex at birth
1829
     t1<-data.frame(dat$sexatbirth,dat$studyarm)
1830
     table(t1)
1831
     prop.table(table(t1), 2) * 100
1832
1833 # gender identity
1834 t1<-data.frame(dat$genderidentity,dat$studyarm)
1835 table(t1)
1836 prop.table(table(t1), 2) * 100
1837
1838
     # income
1839 t1<-data.frame(dat$income,dat$studyarm)
1840
      table(t1)
     prop.table(table(t1), 2) * 100
1841
1842
     # education level
1843
1844 t1<-data.frame(dat$educationlevel,dat$studyarm)
1845 table(t1)
1846 prop.table(table(t1), 2) * 100
1847
1848
     #CHANGELOG ASJ: add education level high/low, 2021-08-03
1849 t1<-data.frame(dat$edhi,dat$studyarm)
1850 table(t1)
1851
     prop.table(table(t1), 2) * 100
1852
1853
     # immune
1854
     t1<-data.frame(dat$immune,dat$studyarm)
1855 table(t1)
1856 prop.table(table(t1), 2) * 100
1857
1858 # COVID-19 vax
1859 t1<-data.frame(dat$c19vax,dat$studyarm)
1860 table(t1)
1861
      prop.table(table(t1), 2) * 100
```

```
1862
1863
1864
       #CHANGELOG ASJ: add 4 new variables, 2021-08-06
1865
      #Trust Info
1866
      t1<-data.frame(dat$Htrustinfo,dat$studyarm)
1867
      table(t1)
     prop.table(table(t1), 2) * 100
1868
1869
1870 #Risk Perception 1
1871 t1<-data.frame(dat$RP1 dicho, dat$studyarm)
1872 table(t1)
     prop.table(table(t1), 2) * 100
1873
1874
1875
      #VaxIntention
1876
      t1<-data.frame(dat$vaxintent,dat$studyarm)
1877
      table(t1)
      prop.table(table(t1), 2) * 100
1878
1879
1880 #Covid19 VaxIntention
1881 t1<-data.frame(dat$c19vaxintent,dat$studyarm)
1882 table(t1)
1883 prop.table(table(t1), 2) * 100
1884
1885
      #### + Graphics per arm ####
1886
1887
      # Boxplots (NB. find nicer colours for publication/thesis)
1888
     par (mar=c(12,5,1,1)) #CHANGELOG ASJ: change margins to see the labels properly,
1889
      2021-08-03
1890
1891
      # Risk perception
1892
     # RECALL: Risk perception item 1 and item 2 to 6 are not measuring the same thing (item
      1 will be analysed as dichotomous variable)
1893
      # Box plot of risk perception item 2 to 6 for overall data
1894
      boxplot(
1895
        dat$mean riskperception2 6 ~ dat$studyarm, las=2,
         xlab = "",
1896
1897
        ylab = "Risk Perception2 6",
1898
       main = "Boxplot",
1899
       col = c(
           "white",
1900
          "darksalmon",
1901
          "darkolivegreen1",
1902
1903
          "lightcyan",
          "bisque3",
1904
1905
          "indianred4",
          "green4",
1906
1907
          "darkslateblue",
1908
          "khaki",
1909
          "gray75",
1910
           "gray85",
           "firebrick3",
1911
1912
           "dodgerblue"
1913
1914
       ) # CHANGELOG Added seperate analysis for risk perception item 2 to 6 2021-07-08
1915
1916
1917
1918
       # Box plot of risk perception item 2 to 6 for subset Main data
1919
       boxplot(
1920
         datMain$mean riskperception2 6 ~ datMain$studyarm, las=2,
         xlab = "",
1921
        ylab = "Risk Perception2 6",
1922
       main = "Boxplot",
1923
1924
       col = c(
1925
          "white",
          "darksalmon",
1926
1927
          "darkolivegreen1",
          "lightcyan",
1928
```

```
1929
           "bisque3",
1930
           "indianred4",
1931
           "green4",
1932
           "darkslateblue"
1933
1934
      )
1935
1936
       # Box plot of risk perception item 2 to 6 for subset Generic data
1937
      boxplot (
1938
         datGeneric$mean riskperception2 6 ~ datGeneric$studyarm,las=2,
1939
         xlab = "",
         ylab = "Risk Perception2 6",
1940
1941
         main = "Boxplot"
        col = c("white", "bisque3", "khaki", "gray75", "gray85")
1942
1943
       ) # CHANGELOG Added seperate analysis for risk perception item 2 to 6 2021-07-08
1944
1945
1946
       par(mar=c(12,5,1,1)) #CHANGELOG ASJ: change margins to see the labels properly,
       2021-08-03
1947
1948
1949
       # Box plot of risk perceptiom item 2 to 6 for subset Measles data
1950
      boxplot(
1951
         datMeasles$mean riskperception2 6 ~ datMeasles$studyarm, las=2,
1952
         xlab = "",
1953
         ylab = "Risk Perception2 6",
1954
        main = "Boxplot",
1955
        col = c("darksalmon", "indianred4", "firebrick3", "firebrick1")
1956
       ) # CHANGELOG Added seperate analysis for risk perception item 2 to 6 2021-07-08
1957
1958
1959
       # Box plot of risk perception item 2 to 6 for subset Flu data
1960
      boxplot(
1961
         datFlu$mean riskperception2 6 ~ datFlu$studyarm, las=2,
1962
         xlab = "",
         ylab = "Risk Perception2_6",
1963
1964
         main = "Boxplot",
1965
         col = c("lightcyan", "darkslateblue", "dodgerblue")
1966
       ) # CHANGELOG Added seperate analysis for risk perception item 2 to 6 2021-07-08
1967
1968
       # Betsch et al C5
1969
       #CHANGELOG ASJ: add boxplot for each subscales, 2021-08-06.
1970
1971
1972
      boxplot(
1973
         datMain$mean C5 conf ~ datMain$studyarm, las=2,
1974
         xlab = "",
         ylab = "C5 Confidence",
1975
1976
         main = "Boxplot",
1977
         col = c(
1978
           "white",
1979
           "darksalmon",
1980
           "darkolivegreen1",
1981
           "lightcyan",
1982
           "bisque3",
1983
           "indianred4",
1984
           "green4",
1985
           "darkslateblue"
1986
1987
1988
1989
      boxplot(
1990
         datMain$mean C5 comp ~ datMain$studyarm, las=2,
1991
         xlab = "",
         ylab = "C5 complacency",
1992
1993
         main = "Boxplot",
         col = c(
1994
1995
           "white",
1996
           "darksalmon",
```

```
1997
           "darkolivegreen1",
1998
           "lightcyan",
1999
           "bisque3",
2000
          "indianred4",
2001
          "green4",
2002
          "darkslateblue"
2003
         )
2004
     )
2005
2006
     boxplot(
2007
        datMain$mean C5 cons ~ datMain$studyarm, las=2,
        xlab = "",
2008
        ylab = "C5 constraints",
2009
        main = "Boxplot",
2010
2011
        col = c(
          "white",
2012
          "darksalmon",
2013
2014
           "darkolivegreen1",
           "lightcyan",
2015
2016
          "bisque3",
          "indianred4",
2017
2018
          "green4",
2019
          "darkslateblue"
2020
        )
2021
      )
2022
      boxplot(
2023
2024
        datMain$mean C5 calc ~ datMain$studyarm, las=2,
2025
        xlab = "",
2026
        ylab = "C5 calculation",
       main = "Boxplot",
2027
2028
       col = c(
2029
          "white",
          "darksalmon",
2030
2031
          "darkolivegreen1",
          "lightcyan",
2032
          "bisque3",
2033
2034
          "indianred4",
2035
          "green4",
2036
           "darkslateblue"
2037
        )
2038
      )
2039
2040
      boxplot(
2041
        datMain$mean C5 coll ~ datMain$studyarm, las=2,
        xlab = "",
2042
2043
        ylab = "C5 Collective Respons.",
2044
        main = "Boxplot",
2045
        col = c(
2046
          "white",
2047
          "darksalmon",
2048
           "darkolivegreen1",
2049
           "lightcyan",
          "bisque3",
2050
2051
          "indianred4",
2052
           "green4",
2053
           "darkslateblue"
2054
2055
2056
2057
2058
      boxplot(
2059
       datGeneric$mean C5 conf ~ datGeneric$studyarm,las=2,
        xlab = "",
2060
        ylab = "C5 confidence",
2061
        main = "Boxplot",
2062
2063
        col = c("white", "bisque3", "khaki", "gray75", "gray85")
2064
2065
```

```
2066
      boxplot (
2067
         datGeneric$mean C5 comp ~ datGeneric$studyarm, las=2,
         xlab = "",
2068
2069
         ylab = "C5 complacency",
        main = "Boxplot",
2070
        col = c("white", "bisque3", "khaki", "gray75", "gray85")
2071
2072
2073
2074
      boxplot(
2075
        datGeneric$mean C5 cons ~ datGeneric$studyarm,las=2,
2076
        xlab = "",
2077
         ylab = "C5 constraints",
2078
        main = "Boxplot",
        col = c("white", "bisque3", "khaki", "gray75", "gray85")
2079
2080
2081
2082
      boxplot (
2083
        datGeneric$mean C5 calc ~ datGeneric$studyarm, las=2,
         xlab = "",
2084
        ylab = "C5 calculation",
2085
        main = "Boxplot",
2086
2087
        col = c("white", "bisque3", "khaki", "gray75", "gray85")
2088
      )
2089
2090
      boxplot(
2091
        datGeneric$mean C5 coll ~ datGeneric$studyarm, las=2,
2092
         xlab = "",
        ylab = "C5 collective respons.",
2093
2094
        main = "Boxplot",
2095
        col = c("white", "bisque3", "khaki", "gray75", "gray85")
2096
       )
2097
2098
2099
2100
      boxplot(
2101
         datMeasles$mean C5 conf ~ datMeasles$studyarm, las=2,
         xlab = "",
2102
2103
        ylab = "C5 confidence",
2104
        main = "Boxplot",
2105
        col = c("darksalmon", "indianred4", "firebrick3", "firebrick1")
2106
       )
2107
2108
      boxplot(
2109
        datMeasles$mean C5 comp ~ datMeasles$studyarm, las=2,
2110
        xlab = "",
         ylab = "C5 complacency",
2111
2112
        main = "Boxplot",
2113
        col = c("darksalmon", "indianred4", "firebrick3", "firebrick1")
2114
      )
2115
2116
      boxplot(
2117
        datMeasles$mean C5 cons ~ datMeasles$studyarm,las=2,
2118
        xlab = "",
2119
        ylab = "C5 contraints",
2120
        main = "Boxplot",
2121
         col = c("darksalmon", "indianred4", "firebrick3", "firebrick1")
2122
       )
2123
2124
      boxplot(
2125
         datMeasles$mean C5 calc ~ datMeasles$studyarm, las=2,
2126
         xlab = "",
        ylab = "C5 calculation",
2127
        main = "Boxplot",
2128
        col = c("darksalmon", "indianred4", "firebrick3", "firebrick1")
2129
2130
2131
2132
       boxplot(
2133
         datMeasles$mean C5 coll ~ datMeasles$studyarm, las=2,
2134
         xlab = "",
```

```
ylab = "C5 collective respons.",
2135
2136
       main = "Boxplot",
2137
        col = c("darksalmon", "indianred4", "firebrick3", "firebrick1")
2138
2139
2140
2141
      boxplot(
2142
       datFlu$mean C5 conf ~ datFlu$studyarm, las=2,
2143
        xlab = "",
2144
        ylab = "C5 confidence",
       main = "Boxplot",
2145
        col = c("lightcyan", "darkslateblue", "dodgerblue")
2146
2147
2148
2149
      boxplot(
2150
        datFlu$mean C5 comp ~ datFlu$studyarm, las=2,
2151
         xlab = "",
        ylab = "C5 complacency",
2152
        main = "Boxplot",
2153
2154
        col = c("lightcyan", "darkslateblue", "dodgerblue")
2155
2156
2157
      boxplot(
2158
        datFlu$mean C5 cons ~ datFlu$studyarm, las=2,
         xlab = "",
2159
2160
         ylab = "C5 constraints",
2161
        main = "Boxplot",
        col = c("lightcyan", "darkslateblue", "dodgerblue")
2162
2163
      )
2164
2165
      boxplot(
2166
       datFlu$mean C5 calc ~ datFlu$studyarm, las=2,
2167
        xlab = "",
2168
        ylab = "C5 calculation",
        main = "Boxplot",
2169
        col = c("lightcyan", "darkslateblue", "dodgerblue")
2170
2171
2172
2173
      boxplot(
2174
       datFlu$mean C5 coll ~ datFlu$studyarm, las=2,
        xlab = "",
2175
        ylab = "C5 collective respons.",
2176
        main = "Boxplot",
2177
2178
        col = c("lightcyan", "darkslateblue", "dodgerblue")
2179
      )
2180
2181
      # Emotion
2182
2183
      boxplot(
2184
        dat$mean_emotion ~ dat$studyarm,las=2,
2185
        xlab = "",
2186
       ylab = "emotion",
2187
       main = "Boxplot",
2188
        col = c(
2189
           "white",
2190
          "darksalmon",
2191
          "darkolivegreen1",
           "lightcyan",
2192
           "bisque3",
2193
           "indianred4",
2194
2195
           "green4",
2196
           "darkslateblue",
2197
           "khaki",
2198
           "gray75",
          "gray85",
2199
2200
          "firebrick3",
          "firebrick1",
2201
2202
           "dodgerblue"
2203
        )
```

```
2204
     )
2205
2206 boxplot(
2207
        datMain$mean emotion ~ datMain$studyarm,las=2,
       xlab = "",
2208
       ylab = "emotion",
2209
       main = "Boxplot",
2210
       col = c(
2211
          "white",
2212
         "darksalmon",
2213
2214
         "darkolivegreen1",
         "lightcyan",
2215
2216
         "bisque3",
2217
         "indianred4",
2218
         "green4",
2219
          "darkslateblue"
2220
        )
2221 )
2222
2223 boxplot(
2224
       datGeneric$mean emotion ~ datGeneric$studyarm,las=2,
2225
       xlab = "",
2226
       ylab = "emotion",
       main = "Boxplot",
2227
2228
        col = c("white", "bisque3", "khaki", "gray75", "gray85")
2229
2230
2231 boxplot(
2232
       datMeasles$mean emotion ~ datMeasles$studyarm,las=2,
2233
       xlab = "",
       ylab = "emotion",
2234
2235
       main = "Boxplot",
2236
       col = c("darksalmon", "indianred4", "firebrick3", "firebrick1")
2237
2238
2239
     boxplot(
2240
       datFlu$mean emotion ~ datFlu$studyarm, las=2,
2241
        xlab = "",
       ylab = "emotion",
2242
2243
       main = "Boxplot",
2244
       col = c("lightcyan", "darkslateblue", "dodgerblue")
2245
     )
2246
2247
      # Knowledge
2248
2249
     boxplot(
2250
       dat$sum knowledge ~ dat$studyarm, las=2,
2251
        xlab = "",
       ylab = "knowledge",
2252
       main = "Boxplot",
2253
2254
       col = c(
          "white",
2255
2256
          "darksalmon",
2257
         "darkolivegreen1",
2258
         "lightcyan",
2259
         "bisque3",
          "indianred4",
2260
2261
          "green4",
          "darkslateblue",
2262
          "khaki",
2263
          "gray75",
2264
         "gray85",
2265
2266
          "firebrick3",
2267
          "firebrick1",
2268
          "dodgerblue"
2269
        )
2270
2271
2272
     boxplot(
```

```
2273
         datMain$sum knowledge ~ datMain$studyarm, las=2,
2274
        xlab = "",
2275
        ylab = "knowledge",
2276
        main = "Boxplot",
2277
       col = c(
          "white",
2278
          "darksalmon",
2279
2280
           "darkolivegreen1",
           "lightcyan",
2281
          "bisque3",
2282
2283
          "indianred4",
          "green4",
2284
2285
           "darkslateblue"
2286
2287
       )
2288
2289
      boxplot(
2290
         datGeneric$sum knowledge ~ datGeneric$studyarm, las=2,
         xlab = "",
2291
        ylab = "knowledge",
2292
       main = "Boxplot",
2293
2294
        col = c("white", "bisque3", "khaki", "gray75", "gray85")
2295
2296
2297
      boxplot(
2298
        datMeasles$sum knowledge ~ datMeasles$studyarm, las=2,
2299
        xlab = "",
2300
        ylab = "knowledge",
2301
       main = "Boxplot",
2302
        col = c("darksalmon", "indianred4", "firebrick3", "firebrick1")
2303
      )
2304
2305
      boxplot(
        datFlu$sum knowledge ~ datFlu$studyarm, las=2,
2306
2307
        xlab = "",
2308
        ylab = "knowledge",
        main = "Boxplot",
2309
2310
        col = c("lightcyan", "darkslateblue", "dodgerblue")
2311
       )
2312
2313
2314
       #CHANGELOG ASJ: Boxplot removed for variables that will be analysed as dichotomous
       variables (trust info & vax intention), 2021-08-06
2315
2316
       #### MISSING DATA EXPLORATION ####
2317
2318
       # CHANGELOG The code added to determine percentage of the missing data 2021-07-08
2319
2320
      don %>%
2321
        naniar::vis_miss(.,
2322
                          sort miss = TRUE,
2323
                          cluster = TRUE)
2324
2325
      don %>%
2326
         naniar::gg miss upset(., nsets = 6) # CHANGELOG Descriptive data of missing 2021-07-08
2327
2328
       don %>%
2329
         summarise(n complete = sum(stats::complete.cases(.)),
2330
                   pct complete = 100 * naniar::prop complete case(.),
2331
                   n missing = sum(!stats::complete.cases(.)),
2332
                   pct_missing = 100 * naniar::prop_miss_case(.))
2333
       don %>%
2334
       naniar::miss case table() # CHANGELOG Missing numbers
2335
2336
      don %>%
2337
         naniar::miss var summary() %>%
2338
         dplyr::filter(n_miss > 0) # CHANGELOG nvar missing
2339
2340
       don %>%
```

```
naniar::miss prop summary() # CHANGELOG percentage of missing overall, % de var avec
         missing, % obs avec missingdon %>% #résumé des missing stat + plot avec VIM
2342
2343
2344
       HTMLStop() #CHANGELOG ASJ: Stop output html 2021-08-06.
2345
2346
2347
       #CHANGELOG ASJ Add descriptive statistic per visualization, 21-09-20.
2348
      HTMLStart(outdir=".\\",
2349
                 file = "Herdimm Descriptive+ 210921", extension = "html", echo=TRUE, HTMLframe
                 = TRUE)
2350
2351
2352
       describeBy(dat$mean riskperception2 6,dat$viz)
2353
       describeBy (dat$mean emotion, dat$viz)
2354
       describeBy(dat$sum knowledge,dat$viz)
2355
       describeBy(dat$mean_C5_calc,dat$viz)
2356
       describeBy(dat$mean_C5_conf,dat$viz)
2357
       describeBy(dat$mean C5 cons,dat$viz)
2358
       describeBy(dat$mean C5 comp,dat$viz)
2359
       describeBy(dat$mean C5 coll,dat$viz)
2360
       describeBy(dat$trustinfo,dat$viz)
2361
       describeBy(dat$vaxintention 1, dat$viz)
2362
       describeBy(dat$c19vaxintention 1,dat$viz)
2363
       describeBy(dat$riskpercep1 1,dat$viz)
2364
2365
2366
      t1<-data.frame(dat$RP1 dicho, dat$viz)
2367
      table(t1)
2368
      prop.table(table(t1), 2) * 100
2369
2370
      t1<-data.frame(dat$Htrustinfo,dat$viz)
2371
      table(t1)
       prop.table(table(t1), 2) * 100
2372
2373
2374
       t1<-data.frame(dat$vaxintent,dat$viz)</pre>
2375
       table (t1)
2376
       prop.table(table(t1), 2) * 100
2377
2378
       t1<-data.frame(dat$c19vaxintent,dat$viz)
2379
       table(t1)
2380
      prop.table(table(t1), 2) * 100
2381
2382
       t1<-data.frame(dat$mean C5 calc2, dat$viz)
2383
       table(t1)
2384
       prop.table(table(t1), 2) * 100
2385
2386
       t1<-data.frame(dat$mean C5 conf2,dat$viz)
2387
       table(t1)
2388
      prop.table(table(t1), 2) * 100
2389
2390
      t1<-data.frame(dat$mean C5 comp2,dat$viz)
2391
      table(t1)
2392
      prop.table(table(t1), 2) * 100
2393
2394
       t1<-data.frame(dat$mean C5 cons2,dat$viz)
2395
       table(t1)
       prop.table(table(t1), 2) * 100
2396
2397
2398
       t1<-data.frame(dat$mean C5 coll2,dat$viz)
2399
       table (t1)
2400
       prop.table(table(t1), 2) * 100
2401
       HTMLStop()
2402
2403
       #### MULTIPLE IMPUTATION ####
2404
2405
       # Create new data sets for imputed values to make analyses easier
2406
2407
       #CHANGELOG ASJ: change list of variables for imputation according to above recoding,
```

```
2408
     datMain4Imputation <-
2409
        subset (
2410
           dat,
2411
           dat$studyarm == "controlgeneric" |
2412
             dat$studyarm == "controlmeasles"
             dat$studyarm == "controlpertussis" |
2413
2414
             dat$studyarm == "controlflu"|
             dat$studyarm == "herdimmgeneric" |
2415
2416
             dat$studyarm == "herdimmmeasles" |
2417
            dat$studyarm == "herdimmpertussis" |
            dat$studyarm == "herdimmflu",
2418
2419
          select = c(
2420
            viz,
2421
            disease,
2422
           mean riskperception2 6,
2423
           mean_C5_conf,
2424
            mean C5 comp,
2425
            mean C5 cons,
2426
            mean C5 calc,
2427
           mean C5 coll,
2428
           mean emotion,
2429
            sum knowledge,
2430
           mean indivhorz,
            mean indivvertical,
2431
2432
            mean collhorz,
2433
            mean collvertical,
2434
            bornincanada,
2435
             language 1,
2436
             language 2,
2437
            Asian group,
2438
            White group,
2439
           disability any,
2440
             genderidentity,
2441
            income,
2442
             edhi,
2443
             age,
2444
            Htrustinfo,
2445
            RP1 dicho,
2446
           vaxintent
2447
           )
2448
         )
2449
2450
2451
      datGeneric4Imputation <-
2452
        subset (
2453
           dat,
2454
           dat$studyarm == "controlgeneric" |
2455
             dat$studyarm == "herdimmgeneric" |
2456
             dat$studyarm == "robertkochgeneric" |
2457
             dat$studyarm == "sbsnewsgeneric" & UserLanguage == "EN",
2458
          select = c(
2459
            studyarm,
2460
             UserLanguage,
2461
            mean riskperception2 6,
2462
            mean C5 conf,
2463
            mean C5 comp,
2464
            mean C5 cons,
2465
            mean C5 calc,
2466
            mean_C5_coll,
2467
            mean emotion,
2468
            sum knowledge,
2469
            mean indivhorz,
2470
             mean indivvertical,
2471
             mean collhorz,
2472
             mean collvertical,
2473
             bornincanada,
2474
             language 1,
2475
             language 2,
```

2021-08-06

```
2476
             Asian group,
2477
             White group,
2478
             disability any,
2479
             genderidentity,
2480
             income,
2481
             edhi,
2482
             age,
2483
             Htrustinfo,
2484
             RP1 dicho,
2485
             vaxintent
2486
           )
2487
         )
2488
2489
       datMeasles4Imputation <-</pre>
2490
         subset (
2491
           dat,
2492
           dat$studyarm == "controlmeasles" |
             dat$studyarm == "herdimmmeasles" |
2493
2494
             dat$studyarm == "guardianmeasles" |
2495
             dat$studyarm == "theotheredmundmeasles",
2496
           select = c(
2497
             studyarm,
2498
             UserLanguage,
2499
             mean riskperception2 6,
2500
             mean C5 conf,
2501
             mean C5 comp,
2502
             mean C5 cons,
2503
             mean_C5_calc,
2504
             mean C5 coll,
2505
             mean emotion,
2506
             sum knowledge,
2507
             mean indivhorz,
2508
             mean indivvertical,
2509
             mean collhorz,
2510
             mean collvertical,
2511
             bornincanada,
2512
             language 1,
2513
             language 2,
2514
             Asian_group,
2515
             White_group,
2516
             disability any,
2517
             genderidentity,
2518
             income,
2519
             edhi,
2520
             age,
2521
             Htrustinfo,
2522
             RP1 dicho,
2523
             vaxintent
2524
           )
2525
         )
2526
2527
      datFlu4Imputation <-
2528
       subset (
2529
2530
           dat$studyarm == "controlflu" |
2531
             dat$studyarm == "herdimmflu" |
2532
             dat$studyarm == "publichealthagencycanadaflu",
2533
           select = c(
2534
             studyarm,
2535
              UserLanguage,
2536
             mean riskperception2 6,
2537
             mean C5 conf,
2538
             mean C5 comp,
2539
             mean C5 cons,
2540
             mean C5 calc,
2541
             mean C5 coll,
2542
             mean emotion,
2543
             sum knowledge,
2544
             mean indivhorz,
```

```
2545
             mean indivvertical,
2546
             mean collhorz,
2547
             mean collvertical,
2548
             bornincanada,
2549
             language 1,
2550
             language 2,
2551
             Asian group,
2552
             White_group,
2553
             disability any,
2554
             genderidentity,
2555
             income,
2556
             edhi,
2557
             age,
2558
             Htrustinfo,
2559
             RP1 dicho,
2560
             vaxintent
2561
           )
2562
         )
2563
2564
       # Drop any unused levels to clean up the dataset
2565
2566
       datMain4Imputation$viz <- droplevels(datMain4Imputation$viz)</pre>
2567
2568
       datGeneric4Imputation$studyarm <- droplevels(datGeneric4Imputation$studyarm)</pre>
2569
2570
       datMeasles4Imputation$studyarm <- droplevels(datMeasles4Imputation$studyarm)</pre>
2571
2572
       datFlu4Imputation$studyarm <- droplevels(datFlu4Imputation$studyarm)
2573
2574
       # Impute the missing values, using parameters:
2575
       # m: Refers to 15 imputed data sets
2576
       # maxit: Refers to number of iterations taken to impute missing values: 15
2577
       #CHANGELOG ASJ: method removed from mice, use pmm, logreg or polyreg according to
       datatype, 21-09-20.
2578
2579
       #CHANGELOG ASJ: Set the seed for reproducibility 2021-08-03
2580
       seed for imp <- 20210920
2581
2582
       datMainImputed <-
2583
         mice(
2584
           datMain4Imputation,
2585
           m = 15,
2586
           maxit = 15,
2587
2588
           seed = seed for imp,
2589
         )
2590
       summary(datMainImputed)
2591
2592
       #CHANGELOG ASJ: added to validate imputation. 2021-09-20.
2593
       plot (datMainImputed, c ("bornincanada", "language 1", "Asian group", "White group", "disability
       _any",
2594
                                "genderidentity", "income", "edhi", "age", "Htrustinfo", "RP1 dicho", "
2595
       stripplot(datMainImputed,age)
2596
       bwplot (datMainImputed, age)
2597
       densityplot(datMainImputed, ~age)
2598
       densityplot(datMainImputed, ~bornincanada)
2599
       densityplot(datMainImputed, ~language 1)
       densityplot(datMainImputed, ~Asian group)
2600
2601
       densityplot(datMainImputed, ~White group)
2602
       densityplot(datMainImputed, ~disability any)
2603
       densityplot(datMainImputed, ~genderidentity)
2604
       densityplot(datMainImputed, ~income)
2605
       densityplot(datMainImputed, ~edhi)
2606
       densityplot(datMainImputed, ~Htrustinfo) #only one missing obs
2607
       densityplot(datMainImputed, ~RP1 dicho)
2608
       densityplot(datMainImputed, ~vaxintent)
2609
       save (datMainImputed, file="datMainImputed.RData")
```

```
2610
2611
2612
       datGenericImputed <-
2613
        mice(
2614
           datGeneric4Imputation,
2615
           m = 15,
2616
           maxit = 15,
2617
           seed = seed for imp
2618
2619
       summary(datGenericImputed)
2620
2621
       #CHANGELOG ASJ: added to validate imputation. 2021-09-20.
2622
       plot (datGenericImputed, c ("bornincanada", "language 1", "Asian group", "White group", "disabil
       ity any",
2623
                              "genderidentity", "income", "edhi", "age", "Htrustinfo", "RP1 dicho", "va
                              xintent"))
2624
       stripplot(datGenericImputed,age)
2625
       bwplot (datGenericImputed, age)
2626
       densityplot(datGenericImputed, ~age)
2627
       densityplot(datGenericImputed, ~bornincanada)
2628
       densityplot(datGenericImputed, ~language 1)
2629
       densityplot(datGenericImputed, ~Asian group)
2630
       densityplot(datGenericImputed, ~White group)
2631
       densityplot(datGenericImputed, ~disability any)
2632
       densityplot(datGenericImputed, ~genderidentity)
2633
       densityplot(datGenericImputed, ~income)
       densityplot(datGenericImputed, ~edhi)
2634
2635
       densityplot(datGenericImputed,~Htrustinfo) #only one missing obs
2636
       densityplot(datGenericImputed, ~RP1 dicho)
2637
       densityplot(datGenericImputed, ~vaxintent)
2638
       save (datGenericImputed, file="datGenericImputed.RData")
2639
2640
2641
2642
       datMeaslesImputed <-
2643
         mice(
2644
           datMeasles4Imputation,
2645
           m = 15,
2646
           maxit = 15,
2647
           seed = seed for imp
2648
         )
2649
       summary(datMeaslesImputed)
2650
       #CHANGELOG ASJ: added to validate imputation. 2021-09-20.
2651
2652
       plot (datMeaslesImputed, c ("bornincanada", "language 1", "Asian group", "White group", "disabil
       ity any",
2653
                                 "genderidentity", "income", "edhi", "age", "RP1 dicho", "vaxintent"))
2654
       stripplot(datMeaslesImputed,age)
2655
       bwplot (datMeaslesImputed, age)
2656
       densityplot(datMeaslesImputed, ~age)
2657
       densityplot(datMeaslesImputed, ~bornincanada)
2658
       densityplot(datMeaslesImputed,~language 1) #only 1 missing
2659
       densityplot(datMeaslesImputed, ~Asian group)
2660
       densityplot(datMeaslesImputed, ~White group)
2661
       densityplot(datMeaslesImputed, ~disability any)
2662
       densityplot(datMeaslesImputed, ~genderidentity)
2663
       densityplot(datMeaslesImputed, ~income)
2664
       densityplot(datMeaslesImputed, ~edhi)
2665
       densityplot(datMeaslesImputed, ~RP1 dicho)
2666
       densityplot(datMeaslesImputed, ~vaxintent)
2667
       save (datMeaslesImputed, file="datMeaslesImputed.RData")
2668
2669
       datFluImputed <-
2670
         mice(
2671
           datFlu4Imputation,
           m = 15,
2672
2673
           maxit = 15,
2674
          seed = seed for imp
```

```
2675
2676
       summary(datFluImputed)
2677
2678
       #CHANGELOG ASJ: added to validate imputation. 2021-09-20.
       plot (datFluImputed, c ("bornincanada", "language 1", "Asian group", "White group", "disability
2679
       any",
                                 "qenderidentity", "income", "edhi", "age", "RP1 dicho", "vaxintent"))
2680
2681
       stripplot(datFluImputed, age)
2682
       bwplot (datFluImputed, age)
2683
       densityplot(datFluImputed, ~age)
2684
       densityplot(datFluImputed, ~bornincanada)
2685
       densityplot(datFluImputed, ~language 1) #only 1 missing
2686
       densityplot(datFluImputed, ~Asian group)
2687
       densityplot(datFluImputed, ~White group)
2688
       densityplot(datFluImputed, ~disability any)
2689
       densityplot(datFluImputed, ~genderidentity)
2690
       densityplot(datFluImputed, ~income)
2691
       densityplot(datFluImputed, ~edhi)
2692
       densityplot(datFluImputed, ~RP1 dicho)
2693
       densityplot(datFluImputed, ~vaxintent)
2694
       save (datFluImputed, file="datFluImputed.RData")
2695
2696
       #### ANALYSES ####
2697
2698
2699
       #### RESEARCH QUESTION 1 (PRIMARY): EFFECT OF HERDIMM ON RISK PERCEPTION ####
2700
2701
       # + 2-way ANOVA (adjusted for covariates and with moderators) ####
2702
2703
       # Recall: Research question 1 (primary): Across 4 vaccine-preventable diseases, does
       the herdimm
2704
       # intervention influence risk perception compared to a control?
2705
       #### + Model 1: Check for direct effects of factors without any covariates (Risk
2706
       perception1 1) ####
2707
       # We have made a new variable with transformation. We want to know that when we look at
       model 1 to model 3
2708
       # what we get the significant results e.g., do we get significant results from
       interaction for all, or between which diseases, or viz,
       # if it doesn't change then we use risk perception 2-6 without any transformation, and
2709
       we will be good with that
2710
       # because yes, transformation makes residual better but it doesnt change the conclusion.
2711
       # Note: if we do not see changes in the model 1-3 for datMain, we do not use transform
       in imputation data,
2712
       # if there is change then we use transformation variable in the imputation data.
2713
2714
       #CHANGELOG. Analysis of RiskPerception2-6 only in anova model, 2021-08-04
2715
       #CHANGELOG ASJ: After analysis of residuals, model also run with transformed variable
       #CHANGELOG ASJ: results are similar and residuals not that improved, keep original
2716
       variable
2717
       hist(datMain$mean riskperception2 6)
2718
       datMain$mean riskperception2 6trans<-datMain$mean riskperception2 6 ** 2
2719
       hist(datMain$mean riskperception2 6trans)
2720
       datMain$mean riskperception2 6transinv<-log(8-datMain$mean riskperception2 6)
2721
       hist(datMain$mean riskperception2 6transinv)
2722
2723
       #### + Model 1: Check for direct effects of factors without any covariates (for risk
       perception 2 to 6) ####
2724
       options(contrasts=c("contr.sum", "contr.poly")) # CHANGELOG: The statement below is
2725
       added to calculate properly the type III sum of squares with lm 2021-07-27
2726
2727
       mRP1 2 6 <- lm(mean riskperception2 6 ~ viz * disease, data = datMain)
2728
       Anova(mRP1 2 6, type="III")
2729
       summary(mRP1 2 6)
2730
2731
       # Model 2: Check for direct effects of factors with adjustment for other covariates
2732
       #CHANGELOG ASJ: change list of covariates after recoding and deletion for <5%
       categories, 2021-08-04
```

```
2733
2734
      mRP2 2 6 <-
2735
         lm (
2736
           mean riskperception2 6 ~ viz * disease +
2737
             mean indivhorz +
2738
             mean_indivvertical +
             mean_collhorz +
2739
2740
             mean collvertical +
2741
             bornincanada +
2742
             language 1 +
2743
             language 2 +
2744
             Asian group +
2745
             White group +
2746
             disability any +
2747
             genderidentity +
2748
             income +
2749
             edhi +
2750
             age,
2751
           data = datMain
2752
         )
2753
       Anova (mRP2 2 6, type = "III")
2754
       summary (mRP2 2 6)
2755
2756
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other
2757
       # covariates
2758
2759
      mRP3 2 6 <-
2760
       lm (
2761
           mean riskperception2 6 ~
2762
             viz * disease * mean indivhorz +
2763
             viz * disease * mean indivvertical +
             viz * disease * mean collhorz +
2764
             viz * disease * mean collvertical +
2765
2766
             bornincanada +
2767
             language 1 +
2768
             language 2 +
2769
             Asian group +
2770
             White_group +
2771
             disability any +
2772
             genderidentity +
2773
             income +
2774
             edhi +
2775
             age,
2776
           data = datMain
2777
         )
2778
       Anova (mRP3 2 6, type = "III")
2779
       summary(mRP3 2 6)
2780
2781
       #### + Adding interaction for high and low education with herdimm vizsualization ####
2782
       # CHANGELOG We have added 2 new models to check the interaction between
2783
       # high and low education with herdimm vizualization 2021-07-22
2784
2785
       #### + Model 4: Check for interaction viz*edhi without any covariates (for risk
       perception 2 to 6) ####
2786
2787
       mRP4 2 6 <- lm(mean riskperception2 6 ~ viz * disease + viz * edhi, data = datMain)
2788
       Anova (mRP4 2 6, type="III")
2789
       summary(mRP4 2 6)
2790
2791
       # Model 5: Check for interaction viz*edhi with covariates
2792
2793
      mRP5 2 6 <-
2794
2795
           mean riskperception2 6 ~ viz * disease +
2796
             viz * edhi +
2797
             mean_indivhorz +
2798
             mean indivvertical +
2799
             mean collhorz +
```

```
2800
                         mean collvertical +
2801
                         bornincanada +
2802
                         language 1 +
2803
                          language 2 +
2804
                         Asian group +
2805
                         White_group +
                         disability_any +
2806
2807
                         genderidentity +
2808
                         income +
2809
                         age,
2810
                     data = datMain
2811
                 )
2812
             Anova (mRP5 2 6, type = "III")
2813
              summary(mRP5 2 6)
2814
2815
2816
              #### + Validating assumptions ####
2817
2818
              # Check to see if the assumptions of the models are respected. If not, we will
             transform the
2819
             # outcome.
2820
2821
              # First, create an assumption-checking function that we can run on each model for
             efficiency.
2822
             checkassumptions <- function(modelname) {</pre>
2823
                boxcox (modelname, lambda = seq(-2, 2, 0.1), plotit = T)
2824
                 # Extract the residuals from the model
2825
2826
               res <- studres (modelname)
2827
               # Check their normality
2828
               print(kurtosis(res) - 3)
2829
               print(skewness(res))
2830
               hist(res)
2831
               qqnorm(res)
2832
               qqline(res)
2833
                 print(ks.test(res, "pnorm", 0, 1))
2834
                 print(shapiro.test(res))
2835
                  # Homoscedasticity (homogeneity of variance)
2836
                 fitted <- fitted (modelname)</pre>
2837
               plot(fitted, res)
2838
                 abline (h = c(-3, 0, 3))
2839
             }
2840
2841
              # Then run the function to check the assumptions for each model.
2842
2843
             checkassumptions (mRP1 2 6)
2844
             checkassumptions (mRP2 2 6)
2845
             checkassumptions (mRP3 2 6)
2846
             \hbox{checkassumptions (mRP4\_2\_6) $\#$ CHANGELOG We have added check assumptions function for the control of the c
             Model 4, 5 and 6 2021-07-22
2847
             checkassumptions (mRP5 2 6)
2848
2849
2850
              #### + Interpretation (Risk perception 2 to 6) ####
2851
2852
              #CHANGELOG ASJ: only the appropriate section (with or without interaction) is kept for
              each model, 2021-08-09
2853
2854
              # Interpretation of model 1 in the case of an interaction
2855
2856
             mRP1_2_6_vd <- emmeans(mRP1 2 6,~viz|disease)</pre>
2857
             mRP1 2 6 vd
2858
              pairs (mRP1 2 6 vd) # Only do multiple comparisons if type 3 test is significant
2859
             plot (mRP1 2 6 vd) # Explore options for less ugly plot for publication/thesis
2860
2861
            mRP1 2 6 dv <- emmeans (mRP1 2 6, ~disease|viz)
            mRP1 2 6 dv
2862
2863
             pairs (mRP1 2 6 dv) # Only do multiple comparisons if type 3 test is significant
2864
              plot(mRP1 2 6 dv)
```

```
2865
2866
2867
       # Interpretation of model 2 in the case of an interaction
2868
       mRP2 2 6 vd <- emmeans (mRP2 2 6,~viz|disease)
2869
       mRP2_2_6_vd
2870
2871
       pairs (mRP2 2 6 vd) # Only do multiple comparisons if type 3 test is significant
2872
       plot (mRP2 2 6 vd) # Explore options for less ugly plot for publication/thesis
2873
2874
      mRP2 2 6 dv <- emmeans (mRP2 2 6, ~disease | viz)
2875
       mRP2 2 6 dv
       pairs (mRP2 2 6 dv) # Only do multiple comparisons if type 3 test is significant
2876
2877
       plot (mRP2 2 6 dv)
2878
2879
       # Interpretation of model 3 moderating effects
2880
       #CHANGELOG ASJ: change the focus of the interpretation 2021-08-11.
2881
2882
       emmip (mRP3 2 6, disease ~ mean indivhorz, cov.reduce = range)
2883
       emmip(mRP3 2 6, viz ~ mean indivvertical, cov.reduce = range)
2884
       emmip (mRP3 2 6, viz ~ mean collhorz, cov.reduce = range)
2885
2886
       emmeans(mRP3 2 6, ~ viz, at=list(mean indivvertical=(2.5)))
2887
       pairs(emmeans(mRP3 2 6, ~ viz, at=list(mean indivvertical=(2.5))))
       emmeans(mRP3_2_6, ~ viz, at=list(mean_indivvertical=(5.0)))
2888
       pairs(emmeans(mRP3_2_6, ~ viz, at=list(mean_indivvertical=(5.0))))
emmeans(mRP3_2_6, ~ viz, at=list(mean_indivvertical=(7.5)))
2889
2890
2891
       pairs(emmeans(mRP3 2 6, ~ viz, at=list(mean indivvertical=(7.5))))
2892
2893
       # Interpretation of model 4 in the case of an interaction viz*edhi
2894
       # CHANGELOG We have added interpretation of model 4 2021-07-22
2895
2896
      mRP4 2 6 ve <- emmeans (mRP4 2 6, ~viz|edhi)
2897
       mRP4 2 6 ve
2898
       pairs (mRP4 2 6 ve) # Only do multiple comparisons if type 3 test is significant
2899
       plot (mRP4 2 6 ve) # Explore options for less ugly plot for publication/thesis
2900
2901
       mRP4 2 6 ev <- emmeans (mRP4 2 6, ~edhi|viz)
2902
       mRP4\_2\_6\_ev
2903
       pairs (mRP4 2 6 ev) # Only do multiple comparisons if type 3 test is significant
2904
       plot (mRP4 2 6 ev)
2905
2906
2907
       # Interpretation of model 5 in the case of an interaction viz*edhi
2908
       #No interaction
2909
2910
2911
       #### + Analyses on imputed data ####
2912
2913
       #CHANGELOG ASJ: No missing data for mean riskperception2 6, no model with imputation
       performed, 21-09-20.
2914
2915
2916
       #### RESEARCH QUESTION 2: EFFECT OF HERDIMM ON OTHER OUTCOMES ####
2917
2918
       # Recall: Research question 2 (secondary): Across 4 vaccine-preventable diseases, does
       the herdimm
2919
       # intervention influence other outcomes (5C scale, emotions, trust, knowledge,
       behavioural
2920
       # intentions) compared to a control?
2921
       # The same analysis as above will be done for the secondary outcomes: mean C5,
2922
       mean emotions,
2923
       # sum knowledge, and behavioural intentions. For trustinfo the same analysis will be
       done if the
2924
       # distribution has enough variance (2-way ANOVA). However, if it's not the case the
2925
       # dichotomised into 1 to 4 (low trust) and 5 to 7 (high trust) and we will run a
       logistic
2926 # regression.
```

```
2928
2929
       #### +++ Emotions ####
2930
2931
       options (contrasts=c("contr.sum", "contr.poly")) # CHANGELOG: The statement below is
       added to calculate properly the type III sum of squares with lm 2021-07-27
2932
       #### + Model 1: Check for direct effects of factors without any covariates (Emotions)
2933
2934
      mEmotions 1 <- lm(mean emotion ~ viz * disease, data = datMain)
2935
      Anova (mEmotions 1, type="III")
2936
       summary(mEmotions 1)
2937
2938
       # Model 2: Check for direct effects of factors with adjustment for other covariates
2939
2940
      mEmotions 2 <-
2941
         lm (
2942
           mean emotion ~ viz * disease +
2943
            mean indivhorz +
2944
             mean indivvertical +
2945
            mean collhorz +
2946
             mean collvertical +
2947
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
2948
             language 1 +
2949
             language 2 +
2950
             Asian group +
2951
             White group +
2952
             disability any +
2953
             genderidentity +
2954
             income +
2955
             edhi +
2956
             age,
2957
           data = datMain
2958
         )
2959
      Anova (mEmotions 2, type = "III")
2960
       summary(mEmotions 2)
2961
2962
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other
2963
      # covariates
2964
2965
      mEmotions 3 <-
2966
         lm (
2967
           mean emotion ~
2968
             viz * disease * mean indivhorz +
             viz * disease * mean indivvertical +
2969
2970
             viz * disease * mean collhorz +
2971
             viz * disease * mean collvertical +
2972
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
2973
             language 1 +
2974
             language 2 +
2975
             Asian group +
2976
             White group +
2977
             disability any +
2978
             genderidentity +
2979
             income +
2980
             edhi +
2981
             age,
2982
           data = datMain
2983
2984
       Anova (mEmotions_3, type = "III")
2985
       summary(mEmotions 3)
2986
2987
       # + Adding interaction for high and low education with herdimm vizsualization
2988
       # CHANGELOG We have added 2 new models to check the interaction between
2989
       # high and low education with herdimm vizualization 2021-07-26
2990
2991
       #### + Model 4: Check for interaction edhi*viz without any covariates (for Emotions) ####
2992
```

```
mEmotions 4 <- lm(mean emotion ~ viz * disease + viz * edhi, data = datMain)
2993
2994
      Anova (mEmotions 4, type="III")
2995
       summary(mEmotions 4)
2996
2997
       # Model 5: Check for interaction edhi*viz with covariates
2998
2999
      mEmotions 5 <-
3000
       lm (
3001
          mean emotion ~ viz * disease +
3002
            viz * edhi +
3003
            mean indivhorz +
3004
            mean indivvertical +
3005
            mean collhorz +
3006
             mean collvertical +
3007
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
3008
             language 1 +
3009
             language_2 +
3010
             Asian group +
3011
            White group +
3012
            disability any +
3013
            genderidentity +
3014
            income +
3015
             age,
3016
           data = datMain
3017
         )
3018
      Anova (mEmotions 5, type = "III")
3019
       summary(mEmotions 5)
3020
3021
3022
      #### + Validating assumptions ####
3023
3024 # Check to see if the assumptions of the models are respected. If not, we will
      transform the
3025
      # outcome.
3026
3027
       checkassumptions (mEmotions 1)
3028
       checkassumptions (mEmotions 2)
3029
      checkassumptions (mEmotions 3)
3030
       checkassumptions (mEmotions 4)
3031
       checkassumptions (mEmotions 5)
3032
3033
3034
       #### + Interpretation (Emotions) ####
3035
3036
      # Interpretation of model 1 in the case of no interaction
3037
3038
      memory.size(max = TRUE)
3039
3040 mEmotions_1_v <- emmeans(mEmotions_1,~viz)
3041 mEmotions_1_v
3042
      plot(mEmotions 1 v)
3043
3044 mEmotions 1 d <- emmeans (mEmotions 1, ~ disease)
3045
      mEmotions 1 d
3046
      pairs (mEmotions 1 d) # Only do multiple comparisons if type 3 test is significant
3047
      plot (mEmotions 1 d)
3048
3049
3050
       # Interpretation of model 2 in the case of no interaction
3051
3052
      mEmotions_2_v <- emmeans(mEmotions_2,~viz)</pre>
3053
      mEmotions 2 v
3054
      plot(mEmotions_2_v)
3055
3056
      mEmotions 2 d <- emmeans (mEmotions 2, ~ disease)
3057
      mEmotions 2 d
3058
      pairs (mEmotions 2 d) # Only do multiple comparisons if type 3 test is significant
3059
       plot(mEmotions 2 d)
3060
```

```
3062
3063
       # Interpretation of model 3 in the case of an interaction with moderator
3064
       emmip (mEmotions 3, viz*disease ~ mean collhorz, cov.reduce = range)
3065
3066
       # Interpretation of model 4 in the case of an interaction viz edhi
3067
      # CHANGELOG We have added interpretation of model 4 2021-07-26
3068
3069
     mEmotions 4 ve <- emmeans (mEmotions 4,~viz|edhi)
3070 mEmotions 4 ve
3071
      pairs (mEmotions 4 ve) # Only do multiple comparisons if type 3 test is significant
3072
      plot (mEmotions 4 ve)
3073
3074
      mEmotions 4 ev <- emmeans (mEmotions 4,~edhi|viz)
3075
      mEmotions 4 ev
3076
      pairs (mEmotions 4 ev) # Only do multiple comparisons if type 3 test is significant
3077
      plot(mEmotions 4 ev)
3078
3079
       # Interpretation of model 5 in the case of an interaction viz edhi
3080
      # CHANGELOG We have added interpretation of model 5 2021-07-26
3081
3082
      mEmotions 5 ve <- emmeans (mEmotions 5, ~viz|edhi)
3083 mEmotions 5 ve
3084
      pairs (mEmotions 5 ve) # Only do multiple comparisons if type 3 test is significant
3085
      plot(mEmotions 5 ve)
3086
3087
      mEmotions 5 ev <- emmeans (mEmotions 5, ~edhi|viz)
3088
     mEmotions_5_ev
3089
      pairs (mEmotions 5 ev) # Only do multiple comparisons if type 3 test is significant
3090
      plot(mEmotions 5 ev)
3091
3092
3093
       # Now we run the models on imputed data.
3094
3095
      #CHANGELOG ASJ: No missing data for mean emotion, no model with imputation performed,
       21-09-20.
3096
3097
3098
       #### +++ Knowledge ####
3099
       #### + Model 1: Check for direct effects of factors without any covariates (Knowledge)
       ####
3100
3101
       options (contrasts=c("contr.sum", "contr.poly")) # CHANGELOG: The statement below is
       added to calculate properly the type III sum of squares with lm 2021-07-27
3102
3103
      mKnowledge 1 <- lm(sum knowledge ~ viz * disease, data = datMain)</pre>
3104
       Anova (mKnowledge 1, type="III")
3105
       summary(mKnowledge 1)
3106
3107
       # Model 2: Check for direct effects of factors with adjustment for other covariates
3108
3109
      mKnowledge 2 <-
3110
       lm (
3111
           sum knowledge ~ viz * disease +
3112
             mean indivhorz +
3113
             mean indivvertical +
3114
            mean collhorz +
3115
            mean collvertical +
3116
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
3117
             language_1 +
3118
             language_2 +
3119
            Asian group +
3120
            White group +
3121
            disability any +
3122
            genderidentity +
3123
            income +
3124
            edhi +
3125
            age,
3126
          data = datMain
```
```
3127
3128
       Anova (mKnowledge 2, type = "III")
3129
       summary(mKnowledge 2)
3130
3131
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other
3132
      # covariates
3133
3134
      mKnowledge 3 <-
3135
         lm (
3136
           sum knowledge ~
3137
             viz * disease * mean indivhorz +
3138
             viz * disease * mean indivvertical +
             viz * disease * mean_collhorz +
3139
3140
             viz * disease * mean collvertical +
3141
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
3142
             language 1 +
             language_2 +
3143
3144
             Asian group +
3145
             White group +
3146
             disability any +
3147
             genderidentity +
3148
             income +
3149
             edhi +
3150
             age,
3151
           data = datMain
3152
         )
3153
      Anova(mKnowledge 3, type = "III")
3154
      summary(mKnowledge 3)
3155
3156
       # + Adding interaction for high and low education with herdimm vizsualization
3157
       # CHANGELOG We have added 2 new models to check the interaction between
3158
       # high and low education with herdimm vizualization 2021-07-26
3159
3160
       #### + Model 4: Check for interaction viz*edhi without any covariates (for Knowledge)
       ####
3161
3162
       mKnowledge 4 <- lm(sum knowledge ~ viz * disease + viz * edhi, data = datMain)
3163
       Anova (mKnowledge 4, type="III")
3164
       summary(mKnowledge 4)
3165
3166
       # Model 5: Check for interaction disease*viz with covariates
3167
3168
      mKnowledge 5 <-
3169
         1m(
3170
           sum knowledge ~ viz * disease +
3171
             viz * edhi +
             mean indivhorz +
3172
3173
             mean_indivvertical +
3174
             mean collhorz +
3175
             mean collvertical +
3176
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
3177
             language 1 +
3178
             language 2 +
3179
             Asian group +
3180
             White group +
3181
             disability any +
3182
             genderidentity +
3183
             income +
3184
             age,
3185
           data = datMain
3186
3187
       Anova (mKnowledge 5, type = "III")
3188
       summary(mKnowledge 5)
3189
3190
3191
       #### + Validating assumptions ####
3192
3193
       # Check to see if the assumptions of the models are respected. If not, we will
```

```
transform the
3194
      # outcome.
3195
3196
       checkassumptions (mKnowledge 1)
3197
       checkassumptions (mKnowledge 2)
      checkassumptions(mKnowledge_3)
3198
3199
       checkassumptions (mKnowledge 4)
3200
       checkassumptions (mKnowledge 5)
3201
3202
       #### + Interpretation (Knowledge) ####
3203
       # Interpretation of model 1 in the case of no interaction
3204
3205
3206
       memory.size (max = TRUE)
3207
3208
       mKnowledge 1 v <- emmeans (mKnowledge 1, ~viz)
       {\tt mKnowledge\_1\_v}
3209
3210
      plot (mKnowledge 1 v)
3211
3212
      mKnowledge 1 d <- emmeans (mKnowledge 1, ~ disease)
3213 mKnowledge 1 d
3214
      pairs (mKnowledge 1 d) # Only do multiple comparisons if type 3 test is significant
3215
      plot (mKnowledge 1 d)
3216
3217
3218
       # Interpretation of model 2 in the case of an interaction
3219
3220
      mKnowledge_2_vd <- emmeans (mKnowledge_2, ~viz|disease)</pre>
      mKnowledge 2 vd
3221
      pairs (mKnowledge 2 vd) # Only do multiple comparisons if type 3 test is significant
3222
3223
      plot(mKnowledge 2 vd)
3224
3225
      mKnowledge 2 dv <- emmeans (mKnowledge 2,~disease|viz)
3226
      mKnowledge 2 dv
3227
       pairs (mKnowledge 2 dv) # Only do multiple comparisons if type 3 test is significant
3228
       plot(mKnowledge 2 dv)
3229
3230
      mKnowledge 3 d
       pairs(mKnowledge_3_d) # Only do multiple comparisons if type 3 test is significant
3231
3232
      plot (mKnowledge 3 d)
3233
3234
       # Interpretation of model 3
3235
       emmip (mKnowledge 3, viz ~ mean indivvertical, cov.reduce = range)
3236
3237
3238
       # Interpretation of model 4 in the case of an interaction viz edhi
3239
       # CHANGELOG We have added interpretation of model 4 2021-07-26
3240
3241
      mKnowledge 4 ve <- emmeans (mKnowledge 4,~viz|edhi)
3242
      mKnowledge 4 ve
      pairs (mKnowledge 4 ve) # Only do multiple comparisons if type 3 test is significant
3243
3244
      plot(mKnowledge 4 ve)
3245
3246
      mKnowledge 4 ev <- emmeans (mKnowledge 4,~edhi|viz)
3247
      mKnowledge 4 ev
3248
       pairs (mKnowledge 4 ev) # Only do multiple comparisons if type 3 test is significant
3249
       plot (mKnowledge_4_ev)
3250
3251
       # Interpretation of model 5 in case of an interaction viz*edhi
3252
       # CHANGELOG We have added interpretation of model 5 2021-07-26
3253
3254
      mKnowledge 5 ve <- emmeans (mKnowledge 5, ~viz|edhi)
3255
       mKnowledge 5 ve
3256
       pairs (mKnowledge 5 ve) # Only do multiple comparisons if type 3 test is significant
3257
      plot(mKnowledge 5 ve)
3258
3259
      mKnowledge 5 ev <- emmeans (mKnowledge 5, ~edhi|viz)
3260
      mKnowledge 5 ev
3261
       pairs (mKnowledge 5 ev) # Only do multiple comparisons if type 3 test is significant
```

```
3262
       plot (mKnowledge 5 ev)
3263
3264
       # Now we run the models on imputed data.
3265
3266
3267
       #CHANGELOG ASJ: No missing data for sum knowledge, no model with imputation performed,
       21-09-20.
3268
3269
3270
       #CHANGELOG ASJ: Add logistic regression models for dichotomous outcomes, 2021-08-05.
3271
3272
3273
3274
       #### +++ Logistic regression for RP1 ####
3275
3276
       #### + Model 1: Check for direct effects of factors without any covariates ####
3277
3278
3279
3280
       options(contrasts=c("contr.sum", "contr.poly"))
       rlog RP1 1 <- glm(relevel(RP1 dicho, ref="Low") ~ viz * disease, data =</pre>
3281
       datMain, family=binomial("logit"))
       Anova(rlog RP1 1,type="III")
3282
3283
       summary(rlog RP1 1)
3284
3285
       # Interpretation of model 1
3286
      mRP1 v <- emmeans(rlog RP1 1,~viz,type = "response") #proportions
3287
      mRP1_v
3288
      plot (mRP1 v)
3289
       confint (pairs (mRP1 v, reverse = TRUE)) #Odds ratios
3290
3291
      mRP1 d <- emmeans(rlog RP1 1, ~ disease, type = "response") #proportions
3292
      mRP1 d
       plot (mRP1_d)
3293
3294
       confint(pairs(mRP1 d,reverse = TRUE)) #Odds ratios
3295
3296
3297
       # Model 2: Check for direct effects of factors with adjustment for other covariates
3298
       rlog RP1_2 <-
3299
3300
         glm(relevel(RP1 dicho, ref="Low") ~ viz * disease +
3301
               mean indivhorz +
3302
               mean indivvertical +
3303
               mean collhorz +
3304
               mean collvertical +
3305
               bornincanada +
3306
               language 1 +
3307
               language 2 +
3308
               Asian group +
3309
               White_group +
3310
               disability any +
3311
               genderidentity +
3312
               income +
3313
               edhi +
3314
               age,
3315
             data = datMain, family=binomial("logit")
3316
         )
3317
       Anova(rlog RP1 2, type = "III")
3318
       summary(rlog RP1 2)
3319
3320
3321
       # Interpretation of model 2
3322
      mRP1 2 v <- emmeans (rlog RP1 2, ~viz, type = "response")
3323
      mRP1 2 v
3324
      plot (mRP1 2 v)
3325
       confint(pairs(mRP1_2_v,reverse = TRUE))
3326
3327
       mRP1_2_d <- emmeans(rlog_RP1_2, ~ disease, type = "response")</pre>
3328
       mRP1 2 d
```

```
3329
       plot (mRP1 2 d)
3330
       confint(pairs(mRP1 2 d, reverse = TRUE))
3331
3332
3333
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
3334
      rlog RP1 3 <-
3335
         glm(relevel(RP1 dicho, ref="Low")
3336
               viz * disease * mean indivhorz +
3337
               viz * disease * mean indivvertical +
3338
              viz * disease * mean collhorz +
              viz * disease * mean collvertical +
3339
3340
               bornincanada +
3341
               language 1 +
3342
               language 2 +
3343
               Asian group +
3344
              White_group +
3345
              disability any +
3346
              genderidentity +
3347
              income +
3348
               edhi +
3349
3350
             data = datMain, family=binomial("logit")
3351
         )
3352
       Anova(rlog RP1 3, type = "III")
3353
       summary(rlog RP1 3)
3354
3355
       ## Interpretation of model 3 : no interaction with moderator to interpret
3356
3357
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
3358
3359
       rlog RP1 4 <- glm(relevel(RP1 dicho, ref="Low") ~ viz * disease + viz * edhi, data =</pre>
       datMain, family=binomial("logit"))
3360
      Anova(rlog RP1 4, type="III")
3361
       summary(rlog RP1 4)
3362
3363
       # Interpretation of model 4
3364
       mRP1 4 v <- emmeans(rlog RP1 4,~viz|edhi,type = "response")
3365
       mRP1_4_v
3366
       confint(pairs(mRP1 4 v,reverse = TRUE))
3367
       pairs (mRP1 4 v, reverse = TRUE, type = "response")
3368
      plot(mRP1 4 v)
3369
3370
      mRP1 4 e <- emmeans(rlog RP1 4, ~ edhi|viz, type = "response")
      mRP1 4 e
3371
3372
       confint(pairs(mRP1 4 e, reverse = TRUE))
3373
       pairs (mRP1 4 e, reverse = TRUE, type = "reponse")
3374
       plot(mRP1 4 e)
3375
3376
3377
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
3378
3379
      rlog RP1 5 <-
3380
         glm(relevel(RP1 dicho, ref="Low") ~ viz * disease +
3381
               viz * edhi +
3382
               mean indivhorz +
3383
               mean indivvertical +
3384
               mean collhorz +
3385
               mean collvertical +
3386
               bornincanada +
3387
               language_1 +
3388
              language 2 +
3389
              Asian group +
3390
              White group +
3391
              disability any +
3392
              genderidentity +
3393
              income +
3394
               age,
3395
            data = datMain, family=binomial("logit")
```

```
3396
3397
       Anova(rlog RP1 5, type = "III")
3398
       summary(rlog_RP1 5)
3399
3400
       # Interpretation of model 5
      mRP1_5_v <- emmeans(rlog RP1 5,~viz|edhi,type = "response")</pre>
3401
3402
      mRP1 5 v
3403
      confint(pairs(mRP1 5 v, reverse = TRUE))
3404
      pairs (mRP1 5 v, reverse = TRUE, type = "response")
3405
      plot(mRP1 5 v)
3406
3407
      mRP1 5 e <- emmeans(rlog RP1 5, ~ edhi|viz, type = "response")
3408
      mRP1 5 e
3409
       confint(pairs(mRP1 5 e, reverse = TRUE))
       pairs (mRP1_5_e, reverse = TRUE, type = "reponse")
3410
3411
       plot (mRP1 5 e)
3412
3413
3414
       # Now we run the models on imputed data.
3415
3416
       #### + Imputed Model 1: Check for direct effects of factors without any covariates ####
3417
3418
       imprlog RP1 1 <-
3419
         with(data = datMainImputed,
3420
              exp = glm(relevel(RP1 dicho, ref="Low") ~ viz * disease, family =
              binomial("logit")))
3421
       combineimprlog_RP1_1 <- pool(imprlog_RP1_1)</pre>
3422
       summary(combineimprlog RP1 1)
3423
3424
3425
       #### +++ Logistic regression for C19 vax intention ####
3426
3427
       #### + Model 1: Check for direct effects of factors without any covariates ####
3428
3429
       options(contrasts=c("contr.sum", "contr.poly"))
       rlog c19vi 1 <- glm(relevel(c19vaxintent, ref="Low") ~ viz * disease, data =</pre>
3430
       datMain, family=binomial("logit"))
3431
       Anova(rlog c19vi 1, type="III")
3432
       summary(rlog c19vi 1)
3433
3434
       # Interpretation of model 1
3435
      mc19vi 1 v <- emmeans(rlog c19vi 1,~viz,type = "response") #proportions
3436
      mc19vi 1 v
3437
       plot (mc19vi 1 v)
3438
       confint(pairs(mc19vi 1 v, reverse = TRUE)) #Odds ratios
3439
3440
      mc19vi 1 d <- emmeans(rlog c19vi 1, ~ disease, type = "response") #proportions</pre>
      mc19vi 1 d
3441
3442
      plot (mc19vi 1 d)
3443
      confint(pairs(mc19vi 1 d, reverse = TRUE)) #Odds ratios
3444
3445
       # Model 2: Check for direct effects of factors with adjustment for other covariates
3446
3447
      rlog c19vi 2 <-
3448
         glm(relevel(c19vaxintent,ref="Low") ~ viz * disease +
3449
               mean indivhorz +
3450
               mean indivvertical +
3451
               mean collhorz +
3452
               mean collvertical +
3453
               bornincanada +
3454
               language_1 +
3455
               language 2 +
3456
              Asian group +
3457
              White group +
3458
              disability any +
3459
              genderidentity +
3460
              income +
3461
               edhi +
3462
               age,
```

```
3463
             data = datMain, family=binomial("logit")
3464
        )
3465
       Anova(rlog c19vi 2, type = "III")
3466
       summary(rlog c19vi 2)
3467
3468
3469
      # Interpretation of model 2
3470 mc19vi 2 v <- emmeans(rlog c19vi 2,~viz,type = "response")
3471 mc19vi 2 v
3472
     plot (mc19vi 2 v)
3473
      confint(pairs(mc19vi 2 v,reverse = TRUE))
3474
3475
      mc19vi 2 d <- emmeans(rlog c19vi 2, ~ disease, type = "response")
      mc19vi 2 d
3476
3477
      plot (mc19vi 2 d)
3478
      confint(pairs(mc19vi 2 d, reverse = TRUE))
3479
3480
3481
      # Model 3: Check for moderating effects of individualism & collectivism with adjustment
      for other covariates
3482
      rlog c19vi 3 <-
3483
         glm(relevel(c19vaxintent, ref="Low")
3484
               viz * disease * mean indivhorz +
               viz * disease * mean indivvertical +
3485
3486
               viz * disease * mean collhorz +
               viz * disease * mean_collvertical +
3487
3488
               bornincanada +
3489
               language 1 +
3490
              language 2 +
3491
              Asian group +
3492
              White group +
3493
              disability any +
3494
              genderidentity +
              income +
3495
3496
              edhi +
3497
               age,
             data = datMain, family=binomial("logit")
3498
3499
3500
       Anova(rlog c19vi 3, type = "III")
3501
      summary(rlog c19vi 3)
3502
3503
       # Interpretation of model 3
3504
       emmip(rlog c19vi 3, viz ~ mean collvertical, cov.reduce = range, type = "response")
3505
3506
3507
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
3508
3509
       rlog c19vi 4 <- glm(relevel(c19vaxintent,ref="Low") ~ viz * disease + viz * edhi,</pre>
       data = datMain, family=binomial("logit"))
3510
       Anova(rlog_c19vi_4,type="III")
3511
      summary(rlog c19vi 4)
3512
3513
      # Interpretation of model 4 (no significant interaction viz edhi)
3514
      mc19vi 4 v <- emmeans(rlog c19vi 4,~viz|edhi,type = "response")
3515
      mc19vi 4 v
3516
      confint(pairs(mc19vi 4 v,reverse = TRUE))
3517
       plot(mc19vi 4 v)
3518
3519
      mc19vi 4 e <- emmeans(rlog c19vi 4, ~ edhi|viz, type = "response")
3520
      mc19vi 4 e
3521
      confint(pairs(mc19vi 4 e, reverse = TRUE))
3522
      plot(mc19vi 4 e)
3523
3524
3525
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
3526
3527
      rlog c19vi 5 <-
3528
         glm(relevel(c19vaxintent, ref="Low") ~ viz * disease +
3529
               viz * edhi +
```

```
3530
              mean indivhorz +
3531
              mean indivvertical +
3532
              mean collhorz +
3533
              mean collvertical +
3534
              bornincanada +
3535
              language_1 +
3536
              language 2 +
3537
              Asian group +
3538
              White group +
3539
               disability any +
3540
               genderidentity +
3541
               income +
3542
               age,
3543
             data = datMain, family=binomial("logit")
3544
         )
3545
       Anova(rlog c19vi 5, type = "III")
3546
      summary(rlog c19vi 5)
3547
3548
       # Interpretation of model 5
3549
      mc19vi 5 v <- emmeans(rlog c19vi 5,~viz|edhi,type = "response")</pre>
3550
      mc19vi 5 v
3551
      confint(pairs(mc19vi 5 v, reverse = TRUE))
3552
      plot(mc19vi 5 v)
3553
3554
      mc19vi 5 e <- emmeans(rlog c19vi 5, ~ edhi|viz, type = "response")
      mc19vi 5 e
3555
3556
      confint(pairs(mc19vi 5 e, reverse = TRUE))
3557
      plot(mc19vi 5 e)
3558
3559
3560
       # Now we run the models on imputed data.
3561
3562
       #CHANGELOG ASJ: No imputation for c19vaxintention, since 51% missing values, 21-09-20.
3563
3564
3565
3566
       #### +++ Logistic regression for vax intention ####
3567
3568
       #In order for the pairs function to work properly, relevel function must be removed
       from the model.
3569
       datMain$vaxintentRel<-relevel (datMain$vaxintent, ref="Low")</pre>
3570
3571
       #### + Model 1: Check for direct effects of factors without any covariates ####
3572
3573
       options(contrasts=c("contr.sum", "contr.poly"))
3574
       rlog vi 1 <- glm(vaxintentRel ~ viz * disease, data = datMain, family=binomial("logit"))</pre>
3575
       Anova(rlog vi 1, type="III")
3576
       summary(rlog vi 1)
3577
3578
       # Interpretation of model 1
3579
      mvi 1 v <- emmeans (rlog vi 1, ~viz, type = "response") #proportions
3580 mvi 1 v
3581
      plot(mvi 1 v)
3582
      confint(pairs(mvi 1 v, reverse = TRUE)) #Odds ratios
3583
3584
      mvi 1 d <- emmeans(rlog vi 1, ~ disease, type = "response") #proportions
3585
      mvi 1 d
3586
       plot (mvi 1 d)
       pairs (mvi 1 d, reverse = TRUE, type = "response")
3587
3588
       confint(pairs(mvi 1 d, reverse = TRUE)) #Odds ratios
3589
3590
       # Model 2: Check for direct effects of factors with adjustment for other covariates
3591
3592
      rlog vi 2 <-
3593
         glm(vaxintentRel ~ viz * disease +
3594
               mean indivhorz +
3595
               mean indivvertical +
3596
               mean collhorz +
3597
               mean collvertical +
```

```
3598
              bornincanada +
3599
              language 1 +
3600
              language 2 +
3601
              Asian group +
3602
              White group +
3603
              disability any +
3604
              genderidentity +
3605
              income +
3606
              edhi +
3607
               age,
3608
             data = datMain, family=binomial("logit")
3609
         )
3610
      Anova(rlog vi 2, type = "III")
3611
       summary(rlog vi 2)
3612
3613
      # Interpretation of model 2
3614
3615 mvi 2 v <- emmeans(rlog vi 2,~viz,type = "response")
3616 mvi_2_v
3617
     plot (mvi 2 v)
3618
      confint(pairs(mvi 2 v,reverse = TRUE))
3619
3620 mvi 2 d <- emmeans(rlog vi 2, ~ disease, type = "response")
3621
      mvi 2 d
3622
      plot (mvi 2 d)
3623
      confint(pairs(mvi 2 d, reverse = TRUE))
3624
      pairs (mvi 2 d, reverse=TRUE, type="response")
3625
     # Model 3: Check for moderating effects of individualism & collectivism with adjustment
3626
      for other covariates
     rlog vi 3 <-
3627
3628
        glm(vaxintentRel ~
3629
              viz * disease * mean indivhorz +
3630
              viz * disease * mean indivvertical +
              viz * disease * mean collhorz +
3631
3632
               viz * disease * mean_collvertical +
3633
              bornincanada +
3634
               language 1 +
3635
               language_2 +
3636
              Asian group +
3637
              White group +
3638
              disability any +
3639
              genderidentity +
3640
              income +
3641
              edhi +
3642
               age,
3643
             data = datMain, family=binomial("logit")
3644
3645
      Anova(rlog vi 3, type = "III")
3646
      summary(rlog_vi_3)
3647
3648
       # Interpretation of model 3
3649
       emmip(rlog vi 3, disease ~ mean indivvertical, cov.reduce = range, type = "response")
3650
3651
3652
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
3653
3654
       rlog vi 4 <- glm (vaxintentRel</pre>
                                      ~ viz * disease + viz * edhi, data =
       datMain, family=binomial("logit"))
3655
       Anova(rlog vi 4, type="III")
3656
      summary(rlog_vi_4)
3657
3658
       # Interpretation of model 4 (no significant interaction viz edhi)
3659
     mvi 4 v <- emmeans(rlog vi 4,~viz|edhi,type = "response")</pre>
3660 mvi 4 v
      confint (pairs (mvi_4_v, reverse = TRUE))
3661
3662
      plot(mvi 4 v)
3663
      mvi 4 e <- emmeans(rlog vi 4, ~ edhi|viz, type = "response")</pre>
3664
```

```
3665
       mvi 4 e
3666
       confint(pairs(mvi 4 e, reverse = TRUE))
3667
       plot(mvi 4 e)
3668
3669
3670
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
3671
3672
      rlog vi 5 <-
3673
        glm (vaxintentRel
                             ~ viz * disease +
3674
               viz * edhi +
3675
               mean indivhorz +
3676
               mean indivvertical +
3677
               mean collhorz +
3678
               mean collvertical +
3679
               bornincanada +
3680
               language 1 +
3681
               language_2 +
3682
               Asian group +
3683
               White group +
3684
               disability any +
3685
               genderidentity +
3686
               income +
3687
               age,
3688
             data = datMain, family=binomial("logit")
3689
         )
       Anova(rlog vi 5, type = "III")
3690
3691
       summary(rlog vi 5)
3692
3693
       # Interpretation of model 5 ( no significant interaction)
3694
      mvi 5 v <- emmeans(rlog vi 5,~viz|edhi,type = "response")</pre>
3695
      mvi 5 v
3696
      confint(pairs(mvi 5 v,reverse = TRUE))
3697
       plot(mvi 5 v)
3698
3699
      mvi 5 e <- emmeans(rlog vi 5, ~ edhi|viz, type = "response")</pre>
3700
       mvi 5 e
3701
       confint(pairs(mvi 5 e, reverse = TRUE))
3702
       plot(mvi 5 e)
3703
3704
3705
       # Now we run the models on imputed data.
3706
3707
       #### + Imputed Model 1: Check for direct effects of factors without any covariates ####
3708
       imprlog_vi 1 <-</pre>
3709
3710
         with(data = datMainImputed,
3711
              exp = glm(relevel(vaxintent, ref="Low") ~ viz * disease, family =
              binomial("logit")))
3712
       combineimprlog_vi_1 <- pool(imprlog_vi_1)</pre>
3713
       summary(combineimprlog vi 1)
3714
3715
3716
       #### +++ Logistic regression for Trust info ####
3717
3718
       datMain$Htrustinfo<-relevel(datMain$Htrustinfo,ref="No")</pre>
3719
3720
       \#\#\# + Model 1: Check for direct effects of factors without any covariates \#\#\#
3721
       options(contrasts=c("contr.sum", "contr.poly"))
3722
3723
       rlog_ti_1 <- glm(Htrustinfo ~ viz * disease, data = datMain, family=binomial("logit"))</pre>
3724
       Anova(rlog_ti_1, type="III")
3725
       summary(rlog ti 1)
3726
3727
       # Interpretation of model 1
3728
      mti 1 v <- emmeans(rlog ti 1,~viz|disease,type = "response") #proportions
      \mathtt{mti}^-1 v
3729
3730
       plot (mti_1_v)
3731
       confint(pairs(mti_1 v,reverse = TRUE)) #Odds ratios
3732
       pairs(mti 1 v,reverse=TRUE, type = "response")
```

```
3733
3734
      mti 1 d <- emmeans(rlog ti 1, ~ disease|viz, type = "response") #proportions</pre>
3735
      mti 1 d
3736
       plot (mti 1 d)
3737
       pairs (mti 1 d, reverse = TRUE, type = "response")
       confint(pairs(mti_1 d, reverse = TRUE)) #Odds ratios
3738
3739
3740
       # Model 2: Check for direct effects of factors with adjustment for other covariates
3741
3742
      rlog ti 2 <-
3743
         glm(Htrustinfo ~ viz * disease +
3744
               mean indivhorz +
3745
               mean indivvertical +
3746
               mean collhorz +
3747
               mean collvertical +
3748
               bornincanada +
3749
               language_1 +
3750
               language 2 +
3751
               Asian group +
3752
              White group +
3753
              disability any +
3754
               genderidentity +
3755
               income +
3756
               edhi +
3757
               age,
             data = datMain, family=binomial("logit")
3758
3759
         )
3760
      Anova(rlog_ti_2, type = "III")
3761
      summary(rlog ti 2)
3762
3763
3764
      # Interpretation of model 2
3765 mti 2 v <- emmeans(rlog ti 2,~viz|disease,type = "response")
3766 mti 2 v
3767
       plot (mti 2 v)
3768
       confint(pairs(mti 2 v,reverse = TRUE))
3769
      pairs (mti 2 v, reverse=TRUE, type = "response")
3770
3771 mti_2_d <- emmeans(rlog_ti_2, ~ disease|viz, type = "response")
3772
      mti 2 d
3773
      plot(mti 2 d)
3774
       confint(pairs(mti 2 d, reverse = TRUE))
3775
      pairs (mti 2 d, reverse=TRUE, type="response")
3776
3777
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
3778
       rlog ti 3 <-
3779
         glm (Htrustinfo ~
3780
               viz * disease * mean_indivhorz +
3781
               viz * disease * mean_indivvertical +
3782
               viz * disease * mean collhorz +
3783
               viz * disease * mean collvertical +
3784
               bornincanada +
3785
               language 1 +
3786
               language 2 +
3787
               Asian_group +
3788
               White group +
3789
               disability any +
3790
               genderidentity +
3791
               income +
3792
               edhi +
3793
               age,
3794
             data = datMain, family=binomial("logit")
3795
3796
       Anova(rlog ti 3, type = "III")
3797
       summary(rlog ti 3)
3798
3799
       #No interaction with moderators
3800
```

```
3801
3802
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
3803
3804
       rlog ti 4 <- glm (Htrustinfo
                                    ~ viz * disease + viz * edhi, data =
       datMain, family=binomial("logit"))
3805
       Anova(rlog_ti_4, type="III")
3806
       summary(rlog ti 4)
3807
3808
       # Interpretation of model 4 (no significant interaction viz edhi)
3809
      mti 4 v <- emmeans(rlog ti 4,~viz|edhi,type = "response")</pre>
3810
      mti 4 v
3811
       confint(pairs(mti 4 v,reverse = TRUE))
3812
       plot (mti 4 v)
3813
3814
      mti 4 e <- emmeans(rlog_ti_4, ~ edhi|viz, type = "response")</pre>
3815
       confint(pairs(mti 4 e, reverse = TRUE))
3816
       plot(mti 4 e)
3817
3818
3819
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
3820
3821
      rlog ti 5 <-
3822
         glm (Htrustinfo
                         ~ viz * disease +
3823
               viz * edhi +
               mean indivhorz +
3824
3825
               mean indivvertical +
3826
              mean collhorz +
3827
              mean_collvertical +
3828
              bornincanada +
3829
              language 1 +
3830
              language 2 +
3831
              Asian group +
3832
              White group +
3833
              disability any +
3834
               genderidentity +
3835
               income +
3836
               age,
3837
             data = datMain, family=binomial("logit")
3838
         )
3839
       Anova(rlog ti 5, type = "III")
3840
      summary(rlog ti 5)
3841
3842
       # Interpretation of model 5 ( no significant interaction)
3843 mti 5 v <- emmeans(rlog ti 5,~viz|edhi,type = "response")
3844
      mti 5 v
3845
       confint(pairs(mti_5_v,reverse = TRUE))
3846
      plot(mti 5 v)
3847
3848
      mti_5_e <- emmeans(rlog_ti_5, ~ edhi|viz, type = "response")</pre>
3849
      mti_5_e
3850
      confint (pairs (mti 5 e, reverse = TRUE))
3851
      plot(mti 5 e)
3852
3853
3854
       # Now we run the models on imputed data.
3855
3856
       #### + Imputed Model 1: Check for direct effects of factors without any covariates ####
3857
3858
3859
       imprlog_ti_1 <-</pre>
3860
         with(data = datMainImputed,
              exp = glm(relevel(Htrustinfo, ref="No") ~ viz * disease, family =
3861
              binomial("logit")))
3862
       combineimprlog ti 1 <- pool(imprlog ti 1)
3863
       summary(combineimprlog ti 1)
3864
3865
       #### +++ Logistic regression for Mean C5 Confidence ####
3866
3867
       datMain$mean C5 conf2<-relevel(as.factor(datMain$mean C5 conf2),ref="0")
```

```
3868
3869
       #### + Model 1: Check for direct effects of factors without any covariates ####
3870
3871
       options(contrasts=c("contr.sum", "contr.poly"))
3872
       rlog c5conf 1 <- glm(mean C5 conf2 ~ viz * disease, data =</pre>
       datMain, family=binomial("logit"))
3873
      Anova(rlog c5conf 1, type="III")
3874
      summary(rlog c5conf 1)
3875
3876
      # Interpretation of model 1
3877 mc5conf v <- emmeans(rlog c5conf 1,~viz,type = "response") #proportions
3878 mc5conf v
3879
      plot(mc5conf v)
3880
      confint(pairs(mc5conf v, reverse = TRUE)) #Odds ratios
3881
3882
      mc5conf d <- emmeans(rlog c5conf 1, ~ disease, type = "response") #proportions</pre>
3883
      mc5conf d
3884
     plot (mc5conf d)
3885
      confint (pairs (mc5conf d, reverse = TRUE)) #Odds ratios
3886
3887
3888
       # Model 2: Check for direct effects of factors with adjustment for other covariates
3889
      rlog_c5conf 2 <-
3890
3891
        glm(mean C5 conf2 ~ viz * disease +
3892
               mean indivhorz +
               mean indivvertical +
3893
3894
              mean collhorz +
3895
              mean collvertical +
3896
              bornincanada +
3897
              language 1 +
3898
              language 2 +
3899
              Asian group +
3900
              White group +
3901
              disability any +
3902
               genderidentity +
3903
               income +
3904
               edhi +
3905
               age,
3906
             data = datMain, family=binomial("logit")
3907
3908
       Anova(rlog c5conf 2, type = "III")
3909
       summary(rlog c5conf 2)
3910
3911
3912
      # Interpretation of model 2
3913
      mc5conf 2 v <- emmeans(rlog c5conf 2,~viz,type = "response")</pre>
      mc5conf 2 v
3914
3915
      plot (mc5conf 2 v)
3916
      confint (pairs (mc5conf_2_v, reverse = TRUE))
3917
3918
      mc5conf 2 d <- emmeans(rlog c5conf 2, ~ disease, type = "response")</pre>
3919 mc5conf_2_d
3920
      plot (mc5conf 2 d)
3921
       confint(pairs(mc5conf 2 d,reverse = TRUE))
3922
3923
3924
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
3925
       rlog_c5conf_3 <-</pre>
3926
         glm (mean_C5_conf2 ~
3927
               viz * disease * mean indivhorz +
3928
               viz * disease * mean indivvertical +
3929
              viz * disease * mean collhorz +
3930
              viz * disease * mean collvertical +
3931
              bornincanada +
3932
              language 1 +
               language 2 +
3933
3934
              Asian group +
```

```
3935
               White group +
3936
              disability any +
3937
               genderidentity +
3938
               income +
3939
               edhi +
3940
               age,
3941
             data = datMain, family=binomial("logit")
3942
         )
3943
      Anova(rlog c5conf 3, type = "III")
3944
      summary(rlog c5conf 3)
3945
3946
      ## Interpretation of model 3
3947
       emmip(rlog c5conf 3, viz ~ mean collvertical , cov.reduce = range, type = "response")
3948
3949
3950
3951
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
3952
3953
      rlog c5conf 4 <- glm(mean C5 conf2 ~ viz * disease + viz * edhi, data =</pre>
       datMain, family=binomial("logit"))
3954
       Anova(rlog c5conf 4, type="III")
3955
       summary(rlog c5conf 4)
3956
      # Interpretation of model 4
3957
3958
      mc5conf 4 v <- emmeans(rlog c5conf 4,~viz|edhi,type = "response")</pre>
      mc5conf 4 v
3959
3960
     confint(pairs(mc5conf 4 v,reverse = TRUE))
3961
     pairs (mc5conf_4_v, reverse = TRUE, type = "response")
3962
      plot(mc5conf 4 v)
3963
3964
     mc5conf 4 e <- emmeans(rlog c5conf 4, ~ edhi|viz, type = "response")</pre>
3965 mc5conf 4 e
3966 confint (pairs (mc5conf 4 e, reverse = TRUE))
3967
      pairs (mc5conf 4 e, reverse = TRUE, type = "reponse")
3968
       plot(mc5conf 4 e)
3969
3970
3971
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
3972
3973
      rlog c5conf 5 <-
3974
         glm (mean C5 conf2 ~ viz * disease +
3975
              viz * edhi +
3976
              mean indivhorz +
3977
              mean indivvertical +
3978
              mean collhorz +
3979
              mean collvertical +
3980
              bornincanada +
3981
               language 1 +
3982
              language_2 +
3983
              Asian group +
3984
              White group +
3985
              disability any +
3986
              genderidentity +
3987
              income +
3988
              age,
3989
             data = datMain, family=binomial("logit")
3990
         )
3991
       Anova(rlog c5conf 5, type = "III")
3992
       summary(rlog c5conf 5)
3993
3994
       # Interpretation of model 5
3995
      mc5conf 5 v <- emmeans(rlog c5conf 5,~viz|edhi,type = "response")</pre>
3996
      mc5conf 5 v
3997
      confint(pairs(mc5conf 5 v, reverse = TRUE))
3998
      pairs (mc5conf 5 v, reverse = TRUE, type = "response")
3999
      plot(mc5conf 5 v)
4000
4001
       mc5conf_5_e <- emmeans(rlog_c5conf_5, ~ edhi|viz, type = "response")</pre>
4002
      mc5conf 5 e
```

```
4003
       confint(pairs(mc5conf 5 e, reverse = TRUE))
4004
       pairs (mc5conf 5 e, reverse = TRUE, type = "reponse")
       plot (mc5conf \overline{5} \overline{e})
4005
4006
4007
4008
       # Now we run the models on imputed data.
4009
       #CHANGELOG ASJ: No missing data for mean C5 conf2, no model with imputation performed,
       21-09-20.
4010
4011
       #### +++ Logistic regression for Mean C5 Complacency ####
4012
       datMain$mean C5 comp2<-relevel(as.factor(datMain$mean C5 comp2), ref="0")</pre>
4013
4014
4015
       #### + Model 1: Check for direct effects of factors without any covariates ####
4016
       options(contrasts=c("contr.sum", "contr.poly"))
4017
4018
       rlog_c5comp_1 <- glm(mean_C5_comp2 ~ viz * disease, data =</pre>
       datMain, family=binomial("logit"))
4019
       Anova(rlog c5comp 1, type="III")
4020
      summary(rlog c5comp 1)
4021
4022
       # Interpretation of model 1
4023 mc5comp_v <- emmeans(rlog_c5comp_1,~viz,type = "response") #proportions
4024
      mc5comp v
4025
       plot (mc5comp v)
4026
       confint(pairs(mc5comp v, reverse = TRUE)) #Odds ratios
4027
4028
      mc5comp_d <- emmeans(rlog_c5comp_1, ~ disease, type = "response") #proportions</pre>
4029 mc5comp d
4030
     plot(mc5comp d)
4031
      confint(pairs(mc5comp d,reverse = TRUE)) #Odds ratios
4032
4033
4034
       # Model 2: Check for direct effects of factors with adjustment for other covariates
4035
4036
      rlog_c5comp 2 <-
4037
         glm (mean C5 comp2 ~ viz * disease +
4038
               mean\_indivhorz +
4039
               mean_indivvertical +
4040
              mean collhorz +
4041
              mean collvertical +
4042
              bornincanada +
4043
              language 1 +
4044
              language 2 +
4045
              Asian group +
4046
              White group +
4047
               disability any +
4048
               genderidentity +
4049
               income +
4050
               edhi +
4051
               age,
4052
             data = datMain, family=binomial("logit")
4053
4054
      Anova(rlog c5comp 2, type = "III")
4055
       summary(rlog c5comp 2)
4056
4057
4058
       # Interpretation of model 2
4059
       mc5comp 2 v <- emmeans(rlog c5comp 2,~viz,type = "response")</pre>
      mc5comp_2_v
4060
4061
      plot (mc5comp 2 v)
4062
      confint(pairs(mc5comp 2 v,reverse = TRUE))
4063
4064 mc5comp 2 d <- emmeans(rlog_c5comp_2, ~ disease, type = "response")
4065 mc5comp 2 d
4066
      plot (mc5comp 2 d)
4067
       confint(pairs(mc5comp_2_d,reverse = TRUE))
4068
4069
```

```
# Model 3: Check for moderating effects of individualism & collectivism with adjustment
4070
       for other covariates
4071
      rlog_c5comp 3 <-</pre>
4072
         glm (mean C5 comp2 ~
4073
               viz * disease * mean indivhorz +
4074
               viz * disease * mean_indivvertical +
4075
              viz * disease * mean collhorz +
4076
              viz * disease * mean collvertical +
4077
              bornincanada +
4078
              language 1 +
4079
              language 2 +
4080
              Asian group +
              White group +
4081
4082
              disability any +
4083
               genderidentity +
4084
               income +
4085
               edhi +
4086
               age,
4087
             data = datMain, family=binomial("logit")
4088
4089
       Anova(rlog c5comp 3, type = "III")
4090
       summary(rlog c5comp 3)
4091
4092
       ## Interpretation of model 3 : no moderating effect to interpret
4093
4094
4095
4096
      #### + Model 4: Check for interaction viz*edhi without any covariates ####
4097
                                           ~ viz * disease + viz * edhi, data =
4098
      rlog c5comp 4 <- glm (mean C5 comp2
       datMain, family=binomial("logit"))
4099
      Anova(rlog c5comp 4, type="III")
      summary(rlog_c5comp_4)
4100
4101
4102
      # Interpretation of model 4
4103
      mc5comp 4 v <- emmeans(rlog c5comp 4,~viz|edhi,type = "response")</pre>
4104
      mc5comp 4 v
4105
      confint(pairs(mc5comp 4 v,reverse = TRUE))
4106
     pairs (mc5comp_4_v, reverse = TRUE, type = "response")
4107
      plot(mc5comp 4 v)
4108
4109
      mc5comp 4 e <- emmeans(rlog c5comp 4, ~ edhi|viz, type = "response")</pre>
4110 mc5comp 4 e
      confint(pairs(mc5comp 4 e,reverse = TRUE))
4111
      pairs (mc5comp 4 e, reverse = TRUE, type = "reponse")
4112
4113
      plot(mc5comp 4 e)
4114
4115
4116
      # Model 5: Check for interaction viz*edhi with adjustment for other covariates
4117
4118 rlog c5comp 5 <-
4119
       glm(mean C5 comp2 ~ viz * disease +
4120
              viz * edhi +
4121
              mean indivhorz +
4122
              mean indivvertical +
4123
              mean collhorz +
4124
              mean collvertical +
4125
              bornincanada +
4126
               language 1 +
4127
               language_2 +
4128
              Asian_group +
4129
              White group +
4130
              disability any +
4131
              genderidentity +
4132
              income +
4133
4134
             data = datMain, family=binomial("logit")
4135
4136
      Anova(rlog c5comp 5, type = "III")
```

```
4137
       summary(rlog c5comp 5)
4138
4139
      # Interpretation of model 5
4140 mc5comp 5 v <- emmeans(rlog c5comp 5,~viz|edhi,type = "response")
4141
      mc5comp 5 v
4142
      confint(pairs(mc5comp_5_v,reverse = TRUE))
4143
     plot(mc5comp 5 v)
4144
4145 mc5comp 5 e <- emmeans(rlog c5comp 5, ~ edhi|viz, type = "response")
4146 mc5comp 5 e
4147
      confint(pairs(mc5comp 5 e,reverse = TRUE))
4148
      plot (mc5comp 5 e)
4149
4150
4151
      # Now we run the models on imputed data.
4152
      #CHANGELOG ASJ: No missing data for mean C5 comp2, no model with imputation performed,
       21-09-20.
4153
4154
4155
4156
4157
       #### +++ Logistic regression for Mean C5 Constraints ####
4158
       datMain$mean_C5_cons2<-relevel(as.factor(datMain$mean C5 cons2),ref="0")</pre>
4159
4160
4161
      #### + Model 1: Check for direct effects of factors without any covariates ####
4162
4163
      options(contrasts=c("contr.sum", "contr.poly"))
4164 rlog c5cons 1 <- glm(mean C5 cons2 ~ viz * disease, data =
      datMain, family=binomial("logit"))
4165
      Anova(rlog c5cons 1, type="III")
4166
      summary(rlog c5cons 1)
4167
4168
      # Interpretation of model 1
4169
     mc5cons v <- emmeans(rlog c5cons 1,~viz,type = "response") #proportions
4170
      mc5cons v
4171
      plot(mc5cons v)
4172
      confint(pairs(mc5cons v, reverse = TRUE)) #Odds ratios
4173
4174
      mc5cons d <- emmeans(rlog c5cons 1, ~ disease, type = "response") #proportions
4175
      mc5cons d
4176
      plot (mc5cons d)
4177
      confint(pairs(mc5cons d, reverse = TRUE)) #Odds ratios
4178
4179
4180
      # Model 2: Check for direct effects of factors with adjustment for other covariates
4181
4182
      rlog c5cons 2 <-
4183
       glm (mean_C5_cons2 ~ viz * disease +
4184
              mean_indivhorz +
4185
              mean indivvertical +
4186
              mean collhorz +
4187
              mean collvertical +
4188
              bornincanada +
4189
              language 1 +
4190
              language 2 +
4191
              Asian group +
4192
              White group +
4193
              disability any +
4194
              genderidentity +
4195
              income +
4196
              edhi +
4197
               age,
4198
             data = datMain, family=binomial("logit")
4199
4200
       Anova(rlog c5cons 2, type = "III")
4201
       summary(rlog_c5cons_2)
4202
4203
```

```
4204
     # Interpretation of model 2
4205 mc5cons 2 v <- emmeans(rlog c5cons 2,~viz,type = "response")
4206 mc5cons 2 v
      plot(mc5cons 2 v)
4207
4208
      confint(pairs(mc5cons 2 v,reverse = TRUE))
4209
4210 mc5cons 2 d <- emmeans(rlog c5cons 2, ~ disease, type = "response")
4211 mc5cons 2 d
4212 plot (mc5cons 2 d)
4213 confint (pairs (mc5cons 2 d, reverse = TRUE))
4214
4215
4216 # Model 3: Check for moderating effects of individualism & collectivism with adjustment
      for other covariates
4217 rlog c5cons 3 <-
4218
       glm (mean C5 cons2 ~
4219
              viz * disease * mean indivhorz +
4220
              viz * disease * mean indivvertical +
4221
              viz * disease * mean collhorz +
              viz * disease * mean collvertical +
4222
4223
             bornincanada +
4224
              language 1 +
4225
             language 2 +
4226
             Asian group +
             White group +
4227
4228
              disability any +
4229
              genderidentity +
              income +
4230
              edhi +
4231
4232
              age,
4233
            data = datMain, family=binomial("logit")
4234
4235 Anova(rlog c5cons 3, type = "III")
      summary(rlog c5cons 3)
4236
4237
4238
      ## Interpretation of model 3
4239
       emmip(rlog c5cons 3, viz ~ mean indivvertical, cov.reduce = range, type = "response")
4240
4241
4242
4243
      #### + Model 4: Check for interaction viz*edhi without any covariates ####
4244
4245 rlog c5cons 4 <- glm (mean C5 cons2
                                         ~ viz * disease + viz * edhi, data =
      datMain, family=binomial("logit"))
4246
      Anova(rlog c5cons 4, type="III")
4247
      summary(rlog_c5cons_4)
4248
4249
      # Interpretation of model 4
4250 mc5cons_4_v <- emmeans(rlog_c5cons_4,~viz|edhi,type = "response")
4251 mc5cons_4_v
4252 confint (pairs (mc5cons 4 v, reverse = TRUE))
4253 pairs (mc5cons 4_v,reverse = TRUE, type = "response")
4254 plot (mc5cons_4_v)
4255
4256 mc5cons 4 e <- emmeans(rlog c5cons 4, ~ edhi|viz, type = "response")
4257 mc5cons 4 e
4258
      confint(pairs(mc5cons_4_e, reverse = TRUE))
4259
      pairs(mc5cons 4 e,reverse = TRUE, type = "reponse")
4260
      plot (mc5cons 4 e)
4261
4262
4263
      # Model 5: Check for interaction viz*edhi with adjustment for other covariates
4264
4265 rlog c5cons_5 <-
4266
       glm(mean C5 cons2 ~ viz * disease +
4267
              viz * edhi +
4268
              mean indivhorz +
4269
              mean indivvertical +
4270
              mean collhorz +
```

```
4271
              mean collvertical +
4272
              bornincanada +
4273
              language 1 +
4274
              language 2 +
4275
              Asian group +
              White_group +
4276
              disability_any +
4277
4278
              genderidentity +
4279
              income +
4280
4281
            data = datMain, family=binomial("logit")
4282
         )
      Anova(rlog c5cons 5, type = "III")
4283
4284
      summary(rlog c5cons 5)
4285
4286
      # Interpretation of model 5
     mc5cons_5_v <- emmeans(rlog_c5cons_5,~viz|edhi,type = "response")</pre>
4287
4288 mc5cons 5 v
4289 confint (pairs (mc5cons 5 v, reverse = TRUE))
4290 pairs (mc5cons 5 v, reverse = TRUE, type = "response")
4291
     plot(mc5cons 5 v)
4292
4293 mc5cons 5 e <- emmeans(rlog c5cons 5, ~ edhi|viz, type = "response")
4294 mc5cons 5 e
4295
      confint(pairs(mc5cons 5 e, reverse = TRUE))
      pairs(mc5cons_5_e,reverse = TRUE, type = "reponse")
4296
4297
      plot(mc5cons 5 e)
4298
4299
4300
       # Now we run the models on imputed data.
4301 #CHANGELOG ASJ: No missing data for mean C5 cons2, no model with imputation performed,
       21-09-20.
4302
4303
4304
4305
       #### +++ Logistic regression for Mean C5 Calculation ####
4306
4307
       datMain$mean C5 calc2<-relevel(as.factor(datMain$mean C5 calc2),ref="0")
4308
4309
       #### + Model 1: Check for direct effects of factors without any covariates ####
4310
4311
       options(contrasts=c("contr.sum", "contr.poly"))
4312
       rlog c5calc 1 <- glm(mean C5 calc2 ~ viz * disease, data =</pre>
       datMain, family=binomial("logit"))
4313
      Anova(rlog c5calc 1, type="III")
4314
      summary(rlog_c5calc_1)
4315
4316
      # Interpretation of model 1
4317
      mc5calc v <- emmeans(rlog c5calc 1,~viz,type = "response") #proportions
4318 mc5calc_v
4319
     plot(mc5calc v)
4320
     confint(pairs(mc5calc v, reverse = TRUE)) #Odds ratios
4321
4322
     mc5calc d <- emmeans(rlog c5calc 1, ~ disease, type = "response") #proportions
4323 mc5calc d
4324
      plot (mc5calc d)
4325
       confint(pairs(mc5calc d, reverse = TRUE)) #Odds ratios
4326
4327
4328
       # Model 2: Check for direct effects of factors with adjustment for other covariates
4329
4330
      rlog c5calc 2 <-
4331
       glm(mean C5 calc2 ~ viz * disease +
4332
              mean indivhorz +
4333
              mean indivvertical +
4334
              mean collhorz +
4335
              mean collvertical +
4336
              bornincanada +
              language 1 +
4337
```

```
4338
               language 2 +
4339
              Asian group +
4340
              White group +
4341
              disability any +
4342
               genderidentity +
4343
               income +
4344
               edhi +
4345
               age,
4346
             data = datMain, family=binomial("logit")
4347
         )
      Anova(rlog c5calc 2, type = "III")
4348
4349
       summary(rlog c5calc 2)
4350
4351
4352
      # Interpretation of model 2
4353
      mc5calc 2 v <- emmeans(rlog c5calc 2,~viz,type = "response")</pre>
4354
     mc5calc_2_v
4355
     plot(mc5calc 2 v)
4356
     confint(pairs(mc5calc 2 v, reverse = TRUE))
4357
4358
      mc5calc 2 d <- emmeans(rlog c5calc 2, ~ disease, type = "response")
4359
     mc5calc 2 d
4360
      plot (mc5calc 2 d)
4361
      confint(pairs(mc5calc 2 d, reverse = TRUE))
4362
4363
4364
      # Model 3: Check for moderating effects of individualism & collectivism with adjustment
      for other covariates
4365
     rlog c5calc 3 <-
4366
        glm (mean C5 calc2 ~
4367
               viz * disease * mean indivhorz +
4368
               viz * disease * mean indivvertical +
4369
               viz * disease * mean collhorz +
               viz * disease * mean collvertical +
4370
4371
              bornincanada +
4372
               language 1 +
4373
               language 2 +
4374
               Asian group +
4375
               White_group +
4376
              disability any +
4377
              genderidentity +
4378
              income +
4379
              edhi +
4380
               age,
4381
             data = datMain, family=binomial("logit")
4382
         )
4383
      Anova(rlog c5calc 3, type = "III")
4384
      summary(rlog c5calc 3)
4385
4386
       ## Interpretation of model 3 : no moderation effect to interpret
4387
4388
4389
4390
       #### + Model 4: Check for interaction viz*edhi without any covariates
4391
4392
      rlog c5calc 4 <- glm (mean C5 calc2
                                            ~ viz * disease + viz * edhi, data =
       datMain, family=binomial("logit"))
4393
       Anova(rlog c5calc 4, type="III")
4394
       summary(rlog c5calc 4)
4395
4396
       # Interpretation of model 4
4397
      mc5calc 4 v <- emmeans(rlog c5calc 4,~viz|edhi,type = "response")</pre>
4398
      mc5calc 4 v
4399
      confint(pairs(mc5calc 4 v,reverse = TRUE))
4400
      plot(mc5calc 4 v)
4401
4402
      mc5calc_4_e <- emmeans(rlog_c5calc_4, ~ edhi|viz, type = "response")</pre>
4403
      mc5calc 4 e
4404
       confint(pairs(mc5calc 4 e,reverse = TRUE))
```

```
4405
      plot(mc5calc 4 e)
4406
4407
4408
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
4409
     rlog_c5calc 5 <-
4410
4411
       glm(mean C5 calc2 ~ viz * disease +
4412
              viz * edhi +
4413
              mean indivhorz +
4414
              mean indivvertical +
4415
              mean collhorz +
4416
              mean collvertical +
4417
              bornincanada +
4418
               language 1 +
              language 2 +
4419
4420
              Asian group +
4421
              White_group +
4422
              disability any +
4423
              genderidentity +
4424
              income +
4425
               age,
4426
            data = datMain, family=binomial("logit")
4427
        )
      Anova(rlog_c5calc_5, type = "III")
4428
4429
      summary(rlog c5calc 5)
4430
4431
      # Interpretation of model 5
4432 mc5calc_5_v <- emmeans(rlog_c5calc_5,~viz|edhi,type = "response")
4433 mc5calc 5 v
4434 confint (pairs (mc5calc 5 v, reverse = TRUE))
4435
     plot(mc5calc 5 v)
4436
4437
     mc5calc 5 e <- emmeans(rlog c5calc 5, ~ edhi|viz, type = "response")</pre>
4438 mc5calc 5 e
4439
      confint(pairs(mc5calc 5 e, reverse = TRUE))
4440
      plot(mc5calc 5 e)
4441
4442
4443
       # Now we run the models on imputed data.
4444
      #CHANGELOG ASJ: No missing data for mean C5 calc2, no model with imputation performed,
       21-09-20.
4445
4446
4447
4448
      #### +++ Logistic regression for Mean C5 Collective Response ####
4449
4450
       datMain$mean C5 coll2<-relevel(as.factor(datMain$mean C5 coll2),ref="0")
4451
4452
       #### + Model 1: Check for direct effects of factors without any covariates ####
4453
4454
     options(contrasts=c("contr.sum", "contr.poly"))
4455
     rlog c5coll 1 <- glm(mean C5 coll2 ~ viz * disease, data =</pre>
      datMain, family=binomial("logit"))
4456
      Anova(rlog c5coll 1, type="III")
4457
      summary(rlog c5coll 1)
4458
4459
      # Interpretation of model 1
4460
      mc5coll v <- emmeans(rlog c5coll 1,~viz,type = "response") #proportions
4461
      mc5coll v
4462
      plot (mc5coll v)
4463
      confint(pairs(mc5coll_v,reverse = TRUE)) #Odds ratios
4464
4465
      mc5coll d <- emmeans(rlog c5coll 1, ~ disease, type = "response") #proportions</pre>
4466 mc5coll d
4467
      plot (mc5coll d)
4468
      confint(pairs(mc5coll d, reverse = TRUE)) #Odds ratios
4469
4470
4471
       # Model 2: Check for direct effects of factors with adjustment for other covariates
```

```
4472
4473
      rlog c5coll 2 <-
4474
         glm (mean C5 coll2 ~ viz * disease +
4475
              mean indivhorz +
4476
               mean indivvertical +
4477
              mean collhorz +
4478
              mean collvertical +
4479
              bornincanada +
4480
              language 1 +
4481
              language 2 +
4482
              Asian group +
              White_group +
4483
4484
              disability any +
4485
               genderidentity +
4486
               income +
4487
               edhi +
4488
               age,
4489
             data = datMain, family=binomial("logit")
4490
         )
4491
       Anova(rlog c5coll 2, type = "III")
4492
       summary(rlog c5coll 2)
4493
4494
      # Interpretation of model 2
4495
      mc5coll_2_v <- emmeans(rlog_c5coll_2,~viz,type = "response")
mc5coll_2_v</pre>
4496
4497
     plot(mc5coll 2 v)
4498
4499
      confint(pairs(mc5coll_2_v,reverse = TRUE))
4500
4501 mc5coll 2 d <- emmeans(rlog c5coll 2, ~ disease, type = "response")
4502 mc5coll 2 d
4503 pairs (mc5coll 2 d, reverse = TRUE)
4504 plot (mc5coll 2 d)
4505
      confint(pairs(mc5coll 2 d, reverse = TRUE))
4506
4507
4508
      # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
4509
       rlog c5coll 3 <-
4510
         glm (mean C5 coll2 ~
4511
               viz * disease * mean indivhorz +
4512
               viz * disease * mean indivvertical +
4513
              viz * disease * mean collhorz +
4514
              viz * disease * mean collvertical +
4515
              bornincanada +
4516
               language 1 +
4517
               language 2 +
              Asian group +
4518
4519
              White_group +
4520
              disability any +
4521
               genderidentity +
4522
              income +
4523
               edhi +
4524
4525
             data = datMain, family=binomial("logit")
4526
         )
4527
       Anova(rlog_c5coll 3, type = "III")
4528
       summary(rlog c5coll 3)
4529
4530
       ## Interpretation of model 3
4531
       emmip(rlog_c5coll_3, viz ~ mean_indivvertical , cov.reduce = range, type = "response")
4532
       emmip(rlog c5coll 3, viz ~ mean collhorz , cov.reduce = range, type = "response")
4533
4534
4535
4536
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
4537
4538
       rlog c5coll 4 <- glm (mean C5 coll2  ~ viz * disease + viz * edhi, data =</pre>
       datMain, family=binomial("logit"))
```

```
4539
      Anova(rlog c5coll 4, type="III")
4540
      summary(rlog c5coll 4)
4541
4542
       # Interpretation of model 4
4543
      mc5coll 4 v <- emmeans(rlog c5coll 4,~viz|edhi,type = "response")</pre>
4544 mc5coll_4_v
4545
     confint(pairs(mc5coll 4 v,reverse = TRUE))
4546
     plot (mc5coll 4 v)
4547
4548
     mc5coll 4 e <- emmeans(rlog c5coll 4, ~ edhi|viz, type = "response")</pre>
4549 mc5coll 4 e
4550
      confint(pairs(mc5coll 4 e, reverse = TRUE))
4551
      plot (mc5coll 4 e)
4552
4553
4554
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
4555
      rlog c5coll 5 <-
4556
4557
         glm (mean C5 coll2 ~ viz * disease +
4558
              viz * edhi +
4559
              mean indivhorz +
4560
              mean indivvertical +
4561
              mean collhorz +
4562
              mean collvertical +
4563
              bornincanada +
4564
              language 1 +
4565
              language 2 +
4566
              Asian group +
4567
              White group +
4568
              disability any +
4569
              genderidentity +
4570
              income +
4571
              age,
            data = datMain, family=binomial("logit")
4572
4573
         )
4574
       Anova(rlog c5coll 5, type = "III")
4575
      summary(rlog c5coll 5)
4576
4577
      # Interpretation of model 5
4578 mc5coll_5_v <- emmeans(rlog_c5coll_5,~viz|edhi,type = "response")
4579 mc5coll_5_v
4580 confint (pairs (mc5coll 5 v, reverse = TRUE))
4581
      plot(mc5coll 5 v)
4582
4583 mc5coll 5 e <- emmeans(rlog_c5coll_5, ~ edhi|viz, type = "response")
4584 mc5coll 5 e
4585
      confint(pairs(mc5coll 5 e, reverse = TRUE))
4586
      plot (mc5coll 5 e)
4587
4588
4589
     # Now we run the models on imputed data.
4590
     #CHANGELOG ASJ: No missing data for mean C5 coll2, no model with imputation performed,
       21-09-20.
4591
4592
4593
4594
       #### RESEARCH QUESTION 3: EXISTING INTERVENTIONS VS HERDIMM ####
4595
4596
      # Recall: Research question 3 (secondary): For any of the 4 diseases, do existing
       interventions
4597
       # already available online outperform the herdimm intervention?
4598
4599
       # 1-way ANOVA (adjusted for covariates and with moderators)
4600
      # Here, we test to see if there is an existing intervention to convey the concept of
4601
      herd immunity
     # that outperforms our intervention. Because the existing interventions each only
4602
      represent one
4603 # disease whereas ours was built to explicitly represent to the epidemiology of
```

```
different infectious
4604
       # diseases, we do this by comparing relevant study arms for one disease at a time.
       These models are
       # therefore similar to our models for two-way analyses, but disease*viz collapses into
4605
       a single
       # variable (study arm).
4606
4607
4608
       #### +++ ONE WAY ANOVA FOR RISK PERCEPTION 2-6 ####
4609
       #### + Generic ####
4610
       #CHANGELOG ASJ: Mean risk perception replaced by MRP2 6 in the rest of the section,
4611
       2021-08-05.
4612
4613
       # Model 1: Check for direct effects of factors without any covariates
       options(contrasts=c("contr.sum", "contr.poly")) # CHANGELOG: Added to calculate
4614
       properly the type III sum of squares with lm 2021-07-27
4615
       mG RP1 <- lm(mean riskperception2 6 ~ studyarm, data=datGeneric)
4616
       Anova (mG RP1, type="III")
      summary(mG_RP1)
4617
4618
4619
       # Model 2: Check for direct effects of factors with adjustment for other covariates
4620
      mG RP2 <-
4621
         lm (
4622
           mean riskperception2 6 ~
4623
             studyarm +
4624
             mean indivhorz +
             mean_indivvertical +
4625
4626
             mean collhorz +
4627
             mean collvertical +
4628
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
4629
             language 1 +
4630
             language 2 +
4631
             Asian group +
4632
             White group +
4633
             disability any +
4634
             genderidentity +
4635
             income +
4636
             edhi +
4637
             age,
4638
           data = datGeneric
4639
         )
4640
       Anova (mG RP2, type="III")
4641
      summary(mG RP2)
4642
4643
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
4644
      mG RP3 <-
4645
        lm(
4646
           mean riskperception2 6 ~
4647
             studyarm * mean indivhorz +
4648
             studyarm * mean indivvertical +
4649
             studyarm * mean collhorz +
4650
             studyarm * mean collvertical +
4651
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
4652
             language 1 +
4653
             language_2 +
4654
             Asian group +
4655
             White group +
4656
             disability any +
4657
             genderidentity +
4658
             income +
4659
             edhi +
4660
             age,
4661
           data = datGeneric
4662
         )
4663
       Anova (mG RP3, type="III")
4664
       summary(mG_RP3)
4665
4666
       \# CHANGELOG: Model 4 + 5 : To check the interaction between the study arm and education
```

```
4667
       # Model 4: Check for interaction studyarm*edhi
4668
       mG RP4 <- lm(mean riskperception2 6 ~ studyarm*edhi, data=datGeneric)
       Anova (mG RP4, type="III")
4669
4670
       summary (mG RP4)
4671
4672
       # Model 5: Check for interaction studyarm*edhi with adjustment for other covariates
       mG_RP5 <- lm(mean_riskperception2 6 ~ studyarm*edhi +</pre>
4673
4674
                      mean indivhorz +
4675
                      mean indivvertical +
4676
                      mean collhorz +
4677
                      mean collvertical +
4678
                      bornincanada +
4679
                      language 1 +
                      language 2 +
4680
                      Asian group +
4681
4682
                      White_group +
4683
                      disability any +
4684
                      genderidentity +
4685
                      income +
4686
                      age, data=datGeneric)
4687
       Anova (mG RP5, type="III")
4688
       summary(mG RP5)
4689
4690
      #### ++ Validating assumptions ####
4691
4692
       # Check to see if the assumptions of the models are respected. If not, we will
       transform the
4693
      # outcome.
4694
4695 checkassumptions (mG RP1)
4696 checkassumptions (mG_RP2)
4697 checkassumptions (mG RP3)
      checkassumptions (mG RP4)
4698
4699
      checkassumptions (mG RP5)
4700
4701
       #### ++ Interpretation ####
4702
4703
      mG RP1 arm <- emmeans (mG RP1, ~studyarm)
4704
      mG RP1 arm
4705
      pairs (mG RP1 arm)
4706
      plot (mG RP1 arm)
4707
4708
      mG RP2 arm <- emmeans (mG RP2, ~studyarm)
4709
       mG RP2 arm
4710
       pairs (mG RP2 arm)
4711
       plot (mG_RP2_arm)
4712
4713
       emmip (mG RP3, studyarm ~ mean indivhorz, cov.reduce = range)
4714
       emmip(mG_RP3, studyarm ~ mean_indivvertical, cov.reduce = range)
4715
       emmip (mG RP3, studyarm ~ mean collvertical, cov.reduce = range)
4716
4717
      mG RP4 v <- emmeans (mG RP4, ~studyarm|edhi)
4718
      mG RP4 v
4719
      pairs (mG RP4 v)
4720
      mG RP4 e <- emmeans (mG RP4, ~edhi|studyarm)
4721
       mG RP4 e
4722
       pairs (mG_RP4_e)
4723
4724
       emmeans (mG RP5, ~studyarm|edhi)
4725
4726
4727
4728
4729
       # Now running models on imputed data.
4730
       #CHANGELOG ASJ: No missing data for mean riskperception2 6, no model with imputation
       performed, 21-09-20.
4731
4732
4733
```

#### + Measles ####

```
4734
4735
       # Model 1: Check for direct effects of factors without any covariates
4736
       mM RP26 1 <- lm(mean riskperception2 6 ~ studyarm, data=datMeasles)
4737
       Anova (mM RP26 1, type="III")
4738
       summary(mM RP26 1)
4739
4740
       # Model 2: Check for direct effects of factors with adjustment for other covariates
4741 mM RP26 2 <-
4742
         lm (
4743
           mean riskperception2 6 ~
4744
             studyarm +
4745
             mean indivhorz +
4746
             mean indivvertical +
4747
             mean collhorz +
4748
             mean collvertical +
4749
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
4750
             language 1 +
4751
             language 2 +
4752
             Asian group +
4753
             White group +
4754
             disability any +
4755
             genderidentity +
4756
             income +
4757
             edhi +
4758
             age,
4759
           data = datMeasles
4760
         )
4761
      Anova(mM RP26 2, type="III")
4762
      summary(mM RP26 2)
4763
4764
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
4765
       mM RP26 3 <-
4766
         lm(
4767
           mean riskperception2 6 ~
4768
             studyarm * mean indivhorz +
4769
             studyarm * mean_indivvertical +
4770
             studyarm * mean collhorz +
4771
             studyarm * mean_collvertical +
4772
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
4773
             language 1 +
4774
             language 2 +
4775
             Asian group +
4776
             White group +
4777
             disability any +
4778
             genderidentity +
4779
             income +
4780
             edhi +
4781
             age,
4782
           data = datMeasles
4783
         )
4784
      Anova (mM RP26 3, type="III")
4785
       summary(mM RP26 3)
4786
4787
       # CHANGELOG: Model 4 + 5 : To check the interaction between the study arm and education
4788
       # Model 4: Check for interaction studyarm*edhi
4789
       mM RP26 4 <- lm(mean riskperception2 6 ~ studyarm*edhi, data=datMeasles)
4790
       Anova (mM RP26 4, type="III")
4791
       summary(mM RP26 4)
4792
4793
       # Model 5: Check for interaction studyarm*edhi with adjustment for other covariates
4794
       mM RP26 5 <- lm(mean riskperception2 6 ~ studyarm*edhi +
4795
                         mean indivhorz +
4796
                         mean indivvertical +
4797
                         mean collhorz +
4798
                         mean collvertical +
4799
                         bornincanada +
4800
                         language 1 +
4801
                         language 2 +
```

```
4802
                         Asian group +
4803
                         White group +
4804
                         disability any +
4805
                         genderidentity +
4806
                         income +
4807
                         age, data=datMeasles)
4808
      Anova (mM RP26 5, type="III")
4809
      summary(mM RP26 5)
4810
4811
      #### ++ Validating assumptions ####
4812
     # Check to see if the assumptions of the models are respected. If not, we will
4813
      transform the
4814
      # outcome.
4815
4816
      checkassumptions (mM RP26 1)
4817 checkassumptions (mM RP26 2)
4818 checkassumptions (mM RP26 3)
4819 checkassumptions (mM RP26 4)
4820 checkassumptions (mM RP26 5)
4821
4822
     #### ++ Interpretation ####
4823 #CHANGELOG ASJ: adapt relevant functions depending on results of global tests,
      2021-08-11.
4824
      mM RP26 1 arm <- emmeans (mM RP26 1,~studyarm)
      mM RP26 1 arm
4825
4826
      pairs (mM RP26 1 arm)
4827
4828
      emmeans (mM RP26 2,~studyarm)
4829
4830
       emmip (mM RP26 3, studyarm ~ mean indivvertical, cov.reduce = range)
4831
4832
       emmeans (mM RP26 4, ~studyarm|edhi)
4833
4834
       emmeans (mM RP26 5, ~studyarm|edhi)
4835
4836
4837
4838
       # Now running models on imputed data.
4839
       #CHANGELOG ASJ: No missing data for mean riskperception2 6, no model with imputation
       performed, 21-09-20.
4840
4841
4842
4843
      #### + Flu ####
4844
4845
      # Model 1: Check for direct effects of factors without any covariates
4846
      mF RP26 1 <- lm(mean riskperception2 6 ~ studyarm, data=datFlu)
4847
      Anova (mF_RP26_1, type="III")
4848
      summary(mF RP26 1)
4849
4850
      # Model 2: Check for direct effects of factors with adjustment for other covariates
4851
      mF RP26 2 <-
4852
         lm (
4853
           mean riskperception2 6 ~
4854
             studyarm +
4855
             mean indivhorz +
4856
             mean indivvertical +
4857
             mean collhorz +
4858
             mean collvertical +
4859
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
4860
             language 1 +
4861
             language 2 +
4862
             Asian group +
4863
             White group +
4864
            disability any +
4865
             genderidentity +
4866
             income +
4867
             edhi +
```

```
4868
             age,
4869
           data = datFlu
4870
         )
4871
      Anova (mF RP26 2, type="III")
4872
       summary(mF RP26 2)
4873
4874
     # Model 3: Check for moderating effects of individualism & collectivism with adjustment
      for other covariates
4875
     mF RP26 3 <-
4876
        lm (
4877
           mean riskperception2 6 ~
4878
             studyarm * mean indivhorz +
4879
             studyarm * mean indivvertical +
             studyarm * mean collhorz +
4880
             studyarm * mean collvertical +
4881
4882
             bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
4883
             language_1 +
4884
             language 2 +
4885
             Asian group +
4886
            White group +
4887
            disability any +
4888
             genderidentity +
4889
            income +
4890
            edhi +
4891
             age,
4892
           data = datFlu
4893
        )
4894
     Anova(mF_RP26_3,type="III")
4895
      summary(mF RP26 3)
4896
4897
4898
       # CHANGELOG: Model 4 + 5 : To check the interaction between the study arm and education
4899
     # Model 4: Check for interaction studyarm*edhi
4900 mF RP26 4 <- lm(mean riskperception2 6 ~ studyarm*edhi, data=datFlu)
4901
       Anova (mF RP26 4, type="III")
4902
       summary (mF RP26 4)
4903
4904
       # Model 5: Check for interaction studyarm*edhi with adjustment for other covariates
4905
       mF RP26 5 <- lm(mean riskperception2 6 ~ studyarm*edhi +
4906
                         mean indivhorz +
4907
                         mean indivvertical +
4908
                         mean collhorz +
4909
                         mean collvertical +
4910
                         bornincanada +
4911
                         language 1 +
4912
                         language 2 +
4913
                         Asian group +
4914
                         White group +
4915
                         disability any +
4916
                         genderidentity +
4917
                         income +
4918
                         age, data=datFlu)
4919
      Anova (mF RP26 5, type="III")
4920
       summary(mF RP26 5)
4921
4922
4923
       #### ++ Validating assumptions ####
4924
4925
       # Check to see if the assumptions of the models are respected. If not, we will
       transform the
       # outcome.
4926
4927
4928
       checkassumptions (mF RP26 1)
4929 checkassumptions (mF RP26 2)
4930 checkassumptions (mF RP26 3)
4931
      checkassumptions (mF RP26 4)
4932
      checkassumptions (mF RP26 5)
4933
4934
      #### ++ Interpretation ####
```

```
#CHANGELOG ASJ: adapt relevant functions depending on results of global tests,
4935
       2021-08-11.
4936
4937
      mF RP26 1 arm <- emmeans (mF RP26 1,~studyarm)
4938
      mF RP26 1 arm
4939
      pairs (mF_RP26_1_arm)
4940
4941 mF RP26 2 arm <- emmeans(mF RP26 2,~studyarm)
4942 mF RP26 2 arm
4943
      pairs (mF RP26 2 arm)
4944
4945
      emmip (mF RP26 3, studyarm ~ mean indivhorz, cov.reduce = range)
4946
       emmip (mF RP26 3, studyarm ~ mean indivvertical, cov.reduce = range)
4947
4948
       emmeans (mF RP26 4,~studyarm|edhi)
4949
4950
       emmeans (mF RP26 5, ~studyarm|edhi)
4951
4952
4953
4954
4955
      # Now running models on imputed data.
4956
      #CHANGELOG ASJ: No missing data for mean riskperception2 6, no model with imputation
       performed, 21-09-20.
4957
4958
4959
      #CHANGELOG ASJ: Added for secondary outcomes, 21-09-03.
4960
4961 #### +++ ONE WAY ANOVA FOR EMOTIONS ####
4962
      #### + Generic ####
4963
4964 # Model 1: Check for direct effects of factors without any covariates
4965 options(contrasts=c("contr.sum", "contr.poly"))
4966 mG E1 <- lm(mean emotion ~ studyarm, data=datGeneric)
4967
      Anova (mG E1, type="III")
4968
      summary (mG E1)
4969
4970
      # Model 2: Check for direct effects of factors with adjustment for other covariates
4971
      mG E2 <-
4972
         lm(
4973
          mean emotion ~
4974
           studyarm +
4975
            mean indivhorz +
4976
            mean indivvertical +
4977
            mean collhorz +
4978
            mean collvertical +
4979
            bornincanada +
4980
            language 1 +
4981
            language_2 +
4982
            Asian_group +
4983
            White group +
4984
            disability any +
4985
            genderidentity +
4986
            income +
4987
            edhi +
4988
            age,
4989
           data = datGeneric
4990
         )
4991
       Anova (mG E2, type="III")
4992
      summary(mG E2)
4993
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
4994
       for other covariates
4995
      mG E3 <-
4996
        1m (
4997
          mean emotion ~
4998
             studyarm * mean_indivhorz +
4999
             studyarm * mean indivvertical +
5000
             studyarm * mean collhorz +
```

```
5001
             studyarm * mean collvertical +
5002
             bornincanada +
5003
             language 1 +
5004
             language 2 +
5005
             Asian group +
5006
             White_group +
5007
             disability any +
5008
             genderidentity +
5009
             income +
5010
             edhi +
5011
             age,
           data = datGeneric
5012
5013
         )
5014
       Anova (mG E3, type="III")
5015
       summary(mG E3)
5016
5017
       # CHANGELOG: Model 4 + 5 : To check the interaction between the study arm and education
5018
       # Model 4: Check for interaction studyarm*edhi
       mG E4 <- lm(mean emotion ~ studyarm*edhi, data=datGeneric)
5019
5020
       Anova (mG E4, type="III")
5021
       summary (mG E4)
5022
5023
       # Model 5: Check for interaction studyarm*edhi with adjustment for other covariates
5024
       mG E5 <- lm(mean emotion ~ studyarm*edhi +
5025
                     mean indivhorz +
5026
                     mean indivvertical +
5027
                     mean collhorz +
5028
                     mean collvertical +
5029
                     bornincanada +
5030
                     language 1 +
5031
                     language 2 +
5032
                     Asian group +
5033
                     White group +
5034
                     disability any +
5035
                     genderidentity +
5036
                     income +
5037
                     age, data=datGeneric)
5038
       Anova (mG E5, type="III")
5039
       summary(mG E5)
5040
5041
       #### ++ Validating assumptions ####
5042
5043
       # Check to see if the assumptions of the models are respected. If not, we will
       transform the
5044
      # outcome.
5045
5046
      checkassumptions (mG E1)
5047
      checkassumptions (mG E2)
5048
      checkassumptions (mG E3)
5049
      checkassumptions (mG E4)
5050
      checkassumptions (mG E5)
5051
5052
       #### ++ Interpretation ####
5053
5054
      mG E1 arm <- emmeans (mG E1, ~studyarm)
5055
       mG E1 arm
5056
       plot (mG_E1_arm)
5057
5058
       mG E2 arm <- emmeans (mG E2, ~studyarm)
5059
       mG E2 arm
5060
       plot(mG E2 arm)
5061
5062
       emmip(mG_E3, studyarm ~ mean_indivhorz, cov.reduce = range)
5063
       emmip (mG E3, studyarm ~ mean collhorz, cov.reduce = range)
5064
5065
       emmeans (mG E4, ~studyarm|edhi)
5066
5067
       emmeans (mG E5, ~studyarm|edhi)
5068
```

```
5069
5070
5071
5072
       # Now running models on imputed data.
5073
       #CHANGELOG ASJ: No missing data for mean emotion, no model with imputation performed,
       21-09-20.
5074
5075
5076
5077
       #### + Measles ####
5078
5079
      # Model 1: Check for direct effects of factors without any covariates
5080
      mM E 1 <- lm(mean emotion ~ studyarm, data=datMeasles)</pre>
5081
       Anova (mM E 1, type="III")
5082
       summary(mM E 1)
5083
5084
       # Model 2: Check for direct effects of factors with adjustment for other covariates
5085
      mM E 2 <-
5086
       lm (
5087
          mean emotion ~
5088
             studyarm +
5089
             mean indivhorz +
5090
             mean indivvertical +
5091
             mean collhorz +
5092
             mean collvertical +
5093
             bornincanada +
5094
             language 1 +
             language 2 +
5095
5096
             Asian group +
5097
             White group +
5098
             disability any +
5099
             genderidentity +
5100
             income +
5101
             edhi +
5102
             age,
5103
           data = datMeasles
5104
         )
5105
       Anova (mM E 2, type="III")
5106
      summary(mM E 2)
5107
5108
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
5109
      mM E 3 <-
5110
         lm(
5111
           mean emotion ~
             studyarm * mean_indivhorz +
5112
5113
             studyarm * mean indivvertical +
5114
             studyarm * mean collhorz +
5115
             studyarm * mean collvertical +
5116
             bornincanada +
5117
             language 1 +
5118
             language 2 +
5119
             Asian group +
5120
             White group +
5121
             disability any +
5122
             genderidentity +
5123
             income +
5124
             edhi +
5125
             age,
5126
           data = datMeasles
5127
         )
5128
       Anova (mM E 3, type="III")
5129
      summary(mM E 3)
5130
5131
       # CHANGELOG: Model 4 + 5 : To check the interaction between the study arm and education
5132
      # Model 4: Check for interaction studyarm*edhi
5133
      mM_E_4 <- lm(mean_emotion ~ studyarm*edhi, data=datMeasles)</pre>
5134
       Anova (mM E 4, type="III")
5135
       summary (mM E 4)
```

```
5136
5137
       # Model 5: Check for interaction studyarm*edhi with adjustment for other covariates
5138
       mM E 5 <- lm (mean emotion ~ studyarm*edhi +
5139
                      mean indivhorz +
                      mean_indivvertical +
5140
5141
                      mean collhorz +
                      mean collvertical +
5142
5143
                      bornincanada +
5144
                      language 1 +
5145
                      language 2 +
5146
                      Asian group +
5147
                      White group +
5148
                      disability any +
5149
                      genderidentity +
5150
                      income +
                      age, data=datMeasles)
5151
5152
       Anova (mM_E_5, type="III")
5153
      summary(mM E 5)
5154
5155
       #### ++ Validating assumptions ####
5156
5157
       # Check to see if the assumptions of the models are respected. If not, we will
       transform the
5158
      # outcome.
5159
5160
      checkassumptions (mM E 1)
      checkassumptions (mM E 2)
5161
      checkassumptions (mM_E_3)
5162
5163
      checkassumptions (mM E 4)
5164
      checkassumptions (mM E 5)
5165
5166
      #### ++ Interpretation ####
5167 #CHANGELOG ASJ: adapt relevant functions depending on results of global tests,
       2021-08-11.
5168
      mM_E_1_arm <- emmeans(mM_E_1,~studyarm)</pre>
5169
       mM E 1 arm
5170
      pairs (mM E 1 arm)
5171
5172
      mM_E_2_arm <- emmeans(mM E 2,~studyarm)</pre>
5173
      mM E 2 arm
5174
      pairs (mM E 2 arm)
5175
5176
       emmeans (mM E 4,~studyarm|edhi)
5177
5178
       emmeans (mM E 5, ~studyarm|edhi)
5179
5180
5181
5182
       # Now running models on imputed data.
5183
       #CHANGELOG ASJ: No missing data for mean emotion, no model with imputation performed,
       21-09-20.
5184
5185
5186
       #### + Flu ####
5187
5188
       # Model 1: Check for direct effects of factors without any covariates
5189
       mF E 1 <- lm(mean emotion ~ studyarm, data=datFlu)
       Anova (mF E 1, type="III")
5190
5191
       summary(mF E 1)
5192
5193
       # Model 2: Check for direct effects of factors with adjustment for other covariates
5194
      mF E 2 <-
5195
         lm (
5196
           mean emotion ~
5197
             studyarm +
5198
             mean indivhorz +
5199
             mean_indivvertical +
5200
             mean collhorz +
5201
             mean collvertical +
```

```
bornincanada +
5202
5203
             language 1 +
5204
             language 2 +
5205
             Asian group +
5206
             White group +
5207
             disability any +
5208
             genderidentity +
5209
             income +
5210
             edhi +
5211
             age,
5212
           data = datFlu
5213
         )
5214 Anova (mF E 2, type="III")
5215
      summary(mF E 2)
5216
5217
      # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
5218
      mF E 3 <-
       \overline{1}m (
5219
5220
           mean emotion ~
5221
             studyarm * mean indivhorz +
5222
             studyarm * mean indivvertical +
            studyarm * mean collhorz +
5223
5224
             studyarm * mean collvertical +
5225
             bornincanada +
5226
             language 1 +
             language 2 +
5227
5228
             Asian_group +
5229
             White group +
5230
             disability any +
5231
             genderidentity +
5232
             income +
5233
             edhi +
5234
             age,
5235
           data = datFlu
5236
         )
5237
       Anova (mF E 3, type="III")
5238
       summary(mF E 3)
5239
5240
5241
       \# CHANGELOG: Model 4 + 5 : To check the interaction between the study arm and education
5242
      # Model 4: Check for interaction studyarm*edhi
5243 mF E 4 <- lm(mean emotion ~ studyarm*edhi, data=datFlu)
5244
      Anova (mF E 4, type="III")
5245
      summary(mF E 4)
5246
5247
       # Model 5: Check for interaction studyarm*edhi with adjustment for other covariates
5248
      mF E 5 <- lm(mean emotion ~ studyarm*edhi +
5249
                      mean indivhorz +
5250
                      mean_indivvertical +
5251
                      mean collhorz +
5252
                      mean collvertical +
5253
                      bornincanada +
5254
                      language 1 +
5255
                      language 2 +
5256
                      Asian group +
5257
                      White group +
5258
                      disability any +
5259
                      genderidentity +
5260
                      income +
5261
                      age, data=datFlu)
5262
      Anova(mF E 5, type="III")
5263
      summary(mF E 5)
5264
5265
5266
      #### ++ Validating assumptions ####
5267
5268
       # Check to see if the assumptions of the models are respected. If not, we will
       transform the
```

```
5269
       # outcome.
5270
5271
       checkassumptions (mF E 1)
5272
       checkassumptions (mF E 2)
5273
       checkassumptions (mF E 3)
5274
      checkassumptions (mF_E_4)
5275
      checkassumptions (mF E 5)
5276
5277
       #### ++ Interpretation ####
5278
      #CHANGELOG ASJ: adapt relevant functions depending on results of global tests,
       2021-08-11.
5279
5280
       emmeans (mF E 1,~studyarm)
5281
5282
       emmeans (mF E 2, ~studyarm)
5283
5284
      mF E4 s<-emmeans (mF E 4,~studyarm|edhi)
      mF E4 s
5285
      pairs (mF E4 s)
5286
5287
5288
      mF E4 e<-emmeans(mF E 4,~edhi|studyarm)
5289
      pairs (mF E4 e)
5290
5291
       emmeans (mF E 5,~studyarm|edhi)
5292
5293
5294
5295
5296
       # Now running models on imputed data.
       #CHANGELOG ASJ: No missing data for mean emotion, no model with imputation performed,
5297
       21-09-20.
5298
5299
      #### +++ ONE WAY ANOVA FOR KNOWLEDGE ####
5300
5301
       #### + Generic ####
5302
5303
       # Model 1: Check for direct effects of factors without any covariates
5304
       options(contrasts=c("contr.sum", "contr.poly"))
5305
       mG_K1 <- lm(sum_knowledge ~ studyarm, data=datGeneric)</pre>
5306
      Anova (mG K1, type="III")
5307
      summary(mG K1)
5308
5309
      # Model 2: Check for direct effects of factors with adjustment for other covariates
5310
      mG K2 <-
5311
         lm(
5312
          sum knowledge ~
5313
             studyarm +
5314
             mean indivhorz +
5315
             mean_indivvertical +
5316
             mean collhorz +
5317
             mean collvertical +
5318
             bornincanada +
5319
             language 1 +
5320
             language 2 +
5321
             Asian group +
5322
             White group +
5323
             disability any +
5324
             genderidentity +
5325
             income +
5326
             edhi +
5327
             age,
5328
           data = datGeneric
5329
         )
5330
       Anova (mG_ K2, type="III")
5331
       summary(mG K2)
5332
5333
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
5334
       mG K3 <-
```

```
lm(
5335
5336
           sum knowledge ~
5337
             studyarm * mean indivhorz +
5338
             studyarm * mean indivvertical +
5339
             studyarm * mean_collhorz +
5340
             studyarm * mean collvertical +
             bornincanada +
5341
5342
             language 1 +
5343
             language 2 +
5344
             Asian group +
5345
             White group +
5346
             disability any +
5347
             genderidentity +
5348
             income +
5349
             edhi +
5350
             age,
5351
           data = datGeneric
5352
         )
5353
       Anova (mG K3, type="III")
5354
       summary(mG K3)
5355
5356
       # CHANGELOG: Model 4 + 5 : To check the interaction between the study arm and education
5357
       # Model 4: Check for interaction studyarm*edhi
5358
       mG K4 <- lm(sum knowledge ~ studyarm*edhi, data=datGeneric)
5359
       Anova (mG K4, type="III")
5360
       summary(mG K4)
5361
       # Model 5: Check for interaction studyarm*edhi with adjustment for other covariates
5362
5363
       mG K5 <- lm(sum knowledge ~ studyarm*edhi +
5364
                     mean indivhorz +
5365
                      mean indivvertical +
5366
                      mean collhorz +
5367
                     mean collvertical +
5368
                     bornincanada +
5369
                      language 1 +
5370
                      language_2 +
5371
                     Asian group +
5372
                     White_group +
5373
                      disability_any +
5374
                      genderidentity +
5375
                      income +
5376
                      age, data=datGeneric)
5377
       Anova (mG K5, type="III")
5378
       summary(mG K5)
5379
5380
       #### ++ Validating assumptions ####
5381
5382
       # Check to see if the assumptions of the models are respected. If not, we will
       transform the
5383
       # outcome.
5384
5385
      checkassumptions (mG K1)
5386 checkassumptions (mG K2)
5387
       checkassumptions (mG K3)
5388
       checkassumptions (mG K4)
5389
       checkassumptions (mG K5)
5390
5391
       #### ++ Interpretation ####
5392
       mG_K1_arm <- emmeans(mG K1,~studyarm)</pre>
5393
5394
       mG K1 arm
5395
       pairs (mG K1 arm)
5396
5397
       mG K2 arm <- emmeans (mG K2,~studyarm)
5398
       mG K2 arm
5399
       pairs (mG K2 arm)
5400
5401
       emmeans (mG_K4,~studyarm|edhi)
5402
```

```
5403
       emmeans (mG K5, ~studyarm|edhi)
5404
5405
5406
       # Now running models on imputed data.
5407
       #CHANGELOG ASJ: No missing data for sum knowledge, no model with imputation performed,
       21-09-20.
5408
5409
5410
5411
       #### + Measles ####
5412
5413
      # Model 1: Check for direct effects of factors without any covariates
5414
      mM K 1 <- lm(sum knowledge ~ studyarm, data=datMeasles)</pre>
       Anova (mM K 1, type="III")
5415
5416
       summary (mM K 1)
5417
5418
      # Model 2: Check for direct effects of factors with adjustment for other covariates
5419
      mM K 2 <-
5420
      lm (
5421
          sum knowledge ~
5422
            studyarm +
5423
             mean indivhorz +
5424
            mean indivvertical +
5425
             mean collhorz +
5426
             mean collvertical +
5427
             bornincanada +
5428
             language 1 +
             language 2 +
5429
5430
             Asian group +
5431
             White group +
5432
             disability any +
5433
             genderidentity +
5434
             income +
5435
             edhi +
5436
             age,
5437
           data = datMeasles
5438
         )
5439
      Anova (mM K 2, type="III")
5440
      summary(mM K 2)
5441
5442
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
      for other covariates
5443
      mM K 3 <-
5444
        lm (
5445
           sum knowledge ~
5446
             studyarm * mean indivhorz +
             studyarm * mean_indivvertical +
5447
5448
             studyarm * mean collhorz +
5449
             studyarm * mean collvertical +
5450
             bornincanada +
5451
             language 1 +
5452
             language 2 +
5453
             Asian group +
5454
             White group +
5455
             disability any +
5456
             genderidentity +
5457
             income +
5458
             edhi +
5459
             age,
5460
           data = datMeasles
5461
         )
5462
      Anova(mM K 3, type="III")
5463
      summary(mM K 3)
5464
5465
       # CHANGELOG: Model 4 + 5 : To check the interaction between the study arm and education
5466
      # Model 4: Check for interaction studyarm*edhi
5467
      mM_K_4 <- lm(sum_knowledge ~ studyarm*edhi, data=datMeasles)</pre>
5468
       Anova (mM K 4, type="III")
5469
       summary (mM K 4)
```

```
5470
5471
       # Model 5: Check for interaction studyarm*edhi with adjustment for other covariates
5472
       mM K 5 <- lm(sum knowledge ~ studyarm*edhi +
5473
                      mean indivhorz +
                      mean_indivvertical +
5474
5475
                      mean collhorz +
5476
                      mean collvertical +
5477
                      bornincanada +
5478
                      language 1 +
5479
                      language 2 +
5480
                      Asian group +
5481
                      White group +
5482
                      disability any +
5483
                      genderidentity +
5484
                      income +
5485
                      age, data=datMeasles)
5486
      Anova(mM_K_5,type="III")
5487
      summary(mM K 5)
5488
5489
       #### ++ Validating assumptions ####
5490
5491
       # Check to see if the assumptions of the models are respected. If not, we will
       transform the
5492
      # outcome.
5493
5494
      checkassumptions (mM K 1)
5495
      checkassumptions (mM K 2)
5496
      checkassumptions (mM_K_3)
5497
      checkassumptions (mM K 4)
5498
      checkassumptions (mM K 5)
5499
5500
      #### ++ Interpretation ####
5501 #CHANGELOG ASJ: adapt relevant functions depending on results of global tests,
       2021-08-11.
5502
      mM K 1 arm <- emmeans (mM K 1, ~studyarm)
5503
       mM K 1 arm
5504
      pairs (mM K 1 arm)
5505
      mM_K_2_arm <- emmeans(mM K 2,~studyarm)</pre>
5506
5507
      mM K 2 arm
5508
      pairs(mM K 2 arm)
5509
5510
       emmip (mM K 3, studyarm ~ mean indivvertical, cov.reduce = range)
5511
5512
       emmeans (mM K 4,~studyarm|edhi)
5513
5514
       emmeans (mM K 5, ~studyarm|edhi)
5515
5516
5517
5518
       # Now running models on imputed data.
5519
       #CHANGELOG ASJ: No missing data for sum knowledge, no model with imputation performed,
       21-09-20.
5520
5521
5522
5523
       #### + Flu ####
5524
5525
5526
       # Model 1: Check for direct effects of factors without any covariates
5527
       mF K 1 <- lm(sum knowledge ~ studyarm, data=datFlu)
5528
       Anova (mF K 1, type="III")
5529
       summary(mF K 1)
5530
5531
       # Model 2: Check for direct effects of factors with adjustment for other covariates
5532
      mF K 2 <-
5533
         lm(
5534
           sum knowledge ~
5535
             studyarm +
```
```
5536
             mean indivhorz +
5537
             mean indivvertical +
5538
             mean collhorz +
5539
             mean collvertical +
5540
             bornincanada +
5541
             language 1 +
5542
             language 2 +
5543
             Asian group +
             White group +
5544
5545
             disability any +
5546
             genderidentity +
5547
             income +
5548
             edhi +
5549
             age,
5550
           data = datFlu
5551
         )
5552
      Anova(mF_K_2,type="III")
5553
      summary(mF K 2)
5554
5555
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
5556
      mF K 3 <-
5557
         lm(
5558
           sum knowledge ~
             studyarm * mean indivhorz +
5559
             studyarm * mean_indivvertical +
5560
5561
             studyarm * mean collhorz +
             studyarm * mean collvertical +
5562
5563
             bornincanada +
5564
             language 1 +
5565
             language 2 +
5566
             Asian group +
5567
             White group +
5568
             disability any +
5569
             genderidentity +
5570
             income +
5571
             edhi +
5572
             age,
5573
           data = datFlu
5574
         )
5575
       Anova (mF K 3, type="III")
5576
       summary(mF K 3)
5577
5578
5579
      # CHANGELOG: Model 4 + 5 : To check the interaction between the study arm and education
5580
      # Model 4: Check for interaction studyarm*edhi
5581
      mF K 4 <- lm(sum knowledge ~ studyarm*edhi, data=datFlu)
5582
       Anova (mF K 4, type="III")
5583
       summary(mF_K_4)
5584
5585
       # Model 5: Check for interaction studyarm*edhi with adjustment for other covariates
5586
      mF K 5 <- lm(sum knowledge ~ studyarm*edhi +
5587
                      mean indivhorz +
5588
                      mean indivvertical +
5589
                      mean collhorz +
5590
                      mean collvertical +
5591
                      bornincanada +
5592
                      language 1 +
5593
                      language 2 +
5594
                      Asian_group +
5595
                      White_group +
5596
                      disability any +
5597
                      genderidentity +
5598
                      income +
5599
                      age, data=datFlu)
5600
       Anova (mF K 5, type="III")
5601
       summary(mF_K_5)
5602
5603
```

```
#### ++ Validating assumptions ####
5604
5605
5606
       # Check to see if the assumptions of the models are respected. If not, we will
       transform the
5607
       # outcome.
5608
      checkassumptions (mF K 1)
5609
5610
     checkassumptions (mF K 2)
5611
      checkassumptions (mF K 3)
5612
       checkassumptions (mF K 4)
5613
       checkassumptions (mF K 5)
5614
5615
       #### ++ Interpretation ####
5616
       #CHANGELOG ASJ: adapt relevant functions depending on results of global tests,
       2021-08-11.
5617
5618
       mF K 1 arm <- emmeans (mF K 1,~studyarm)
5619
       mF K 1 arm
5620
       pairs (mF K 1 arm)
5621
5622
       mF K 2 arm <- emmeans (mF K 2,~studyarm)
5623
       mF K 2 arm
5624
       pairs (mF K 2 arm)
5625
5626
       emmip (mF K 3, studyarm ~ mean indivvertical, cov.reduce = range)
5627
5628
       emmeans (mF K 4,~studyarm|edhi)
5629
5630
      mF K 5 arm <- emmeans (mF K 5,~studyarm|edhi)
5631
      mF K 5 arm
5632
      pairs (mF K 5 arm)
5633
       pairs (emmeans (mF K 5, ~edhi|studyarm))
5634
5635
5636
5637
       # Now running models on imputed data.
       #CHANGELOG ASJ: No missing data for sum knowledge, no model with imputation performed,
5638
       21-09-20.
5639
5640
5641
5642
5643
5644
5645
       #CHANGELOG ASJ: Add logistic regression models for dichotomous outcomes, 2021-08-11.
5646
5647
       #### +++ Logistic regression for RP1 ####
5648
5649
       #Create relevel before model to avoid problems with pairs function.
       datGeneric$RP1_dicho <- relevel(datGeneric$RP1 dicho,ref = "Low")</pre>
5650
5651
       datMeasles$RP1 dicho <- relevel(datMeasles$RP1 dicho, ref = "Low")
5652
       datFlu$RP1 dicho <- relevel(datFlu$RP1 dicho, ref = "Low")</pre>
5653
5654
       #### ++ Generic ####
5655
5656
       #### + Model 1: Check for direct effects of factors without any covariates ####
5657
5658
       options(contrasts=c("contr.sum", "contr.poly"))
5659
       rlogG RP1 1 <- glm(RP1 dicho ~ studyarm, data = datGeneric, family=binomial("logit"))</pre>
5660
       Anova(rlogG_RP1_1, type="III")
5661
       summary(rlogG RP1 1)
5662
5663
       mgRP1 <- emmeans(rlogG RP1 1,~studyarm,type = "response") #proportions
5664
5665
       confint (pairs (mgRP1, reverse = TRUE)) #Odds ratios
5666
       pairs (mgRP1, reverse = TRUE, type = "response")
5667
5668
       # Model 2: Check for direct effects of factors with adjustment for other covariates
5669
       rlogG RP1 2 <-
```

```
5670
         glm (RP1 dicho ~ studyarm +
5671
              mean indivhorz +
5672
              mean indivvertical +
5673
              mean collhorz +
5674
              mean collvertical +
5675
              bornincanada +
5676
              language 1 +
5677
              language 2 +
5678
              Asian group +
5679
              White group +
5680
              disability any +
5681
               genderidentity +
5682
               income +
5683
               edhi +
5684
               age,
5685
             data = datGeneric, family=binomial("logit")
5686
         )
5687
       Anova(rlogG RP1 2, type = "III")
5688
      summary(rlogG RP1 2)
5689
5690
      mgRP1 2 <- emmeans(rlogG RP1 2,~studyarm,type = "response")
5691
       mgRP1 2
5692
       confint(pairs(mgRP1 2, reverse = TRUE))
       pairs (mgRP1_2, reverse = TRUE, type = "response")
5693
5694
5695
5696
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
5697
      rlogG_RP1_3 <-
5698
        glm(RP1 dicho
5699
               studyarm * mean indivhorz +
5700
               studyarm * mean indivvertical +
              studyarm * mean collhorz +
5701
5702
              studyarm * mean collvertical +
5703
               bornincanada +
5704
               language 1 +
5705
               language 2 +
5706
               Asian group +
5707
               White_group +
5708
              disability any +
5709
              genderidentity +
5710
              income +
5711
               edhi +
5712
               age,
5713
             data = datGeneric, family=binomial("logit")
5714
         )
       Anova(rlogG_RP1 3, type = "III")
5715
5716
       summary(rlogG RP1 3)
5717
5718
       #No interaction with moderator to interpret
5719
5720
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
5721
5722
       rlogG RP1 4 <- glm(RP1 dicho ~ studyarm * edhi, data =
       datGeneric, family=binomial("logit"))
5723
       Anova(rlogG_RP1_4, type="III")
5724
       summary(rlogG RP1 4)
5725
5726
       mgRP1 4 s <- emmeans(rlogG RP1 4,~studyarm|edhi,type = "response")
5727
       mgRP1 4 s
5728
       confint (pairs (mgRP1_4_s, reverse = TRUE))
5729
5730
       mgRP1 4 e <- emmeans(rlogG RP1 4, ~ edhi|studyarm, type = "response")
5731
       confint(pairs(mgRP1 4 e, reverse = TRUE))
5732
5733
5734
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
5735
5736
       rlogG RP1 5 <-
```

```
5737
         glm (RP1 dicho
                       ~ studyarm*edhi +
5738
              mean indivhorz +
5739
              mean indivvertical +
5740
              mean collhorz +
5741
              mean collvertical +
5742
              bornincanada +
5743
              language 1 +
5744
              language 2 +
5745
              Asian group +
5746
              White group +
5747
              disability any +
5748
               genderidentity +
5749
               income +
5750
               age,
5751
             data = datGeneric, family=binomial("logit")
5752
         )
5753
       Anova(rlogG RP1 5, type = "III")
5754
       summary(rlogG RP1 5)
5755
5756
       mgRP1 5 s <- emmeans(rlogG RP1 5,~studyarm|edhi,type = "response")
5757
       mgRP1 5 s
5758
       confint(pairs(mgRP1 5 s, reverse = TRUE))
5759
5760
       mgRP1 5 e <- emmeans(rlogG RP1 5, ~ edhi|studyarm, type = "response")
5761
       confint(pairs(mgRP1 5 e, reverse = TRUE))
5762
5763
       # Now running models on imputed data.
5764
5765
      imprlogG RP1 1 <-
5766
       with(data = datGenericImputed,
5767
              exp = glm(relevel(RP1 dicho,ref="Low") ~ studyarm,family = binomial("logit")))
5768
      combineimprlogG RP1 1 <- pool(imprlogG RP1 1)</pre>
5769
       summary(combineimprlogG RP1 1)
5770
5771
5772
       #### ++ Measles ####
5773
5774
       #### + Model 1: Check for direct effects of factors without any covariates ####
5775
5776
       options(contrasts=c("contr.sum", "contr.poly"))
5777
       rlogM RP1 1 <- glm(RP1 dicho ~ studyarm, data = datMeasles, family=binomial("logit"))</pre>
5778
       Anova(rlogM RP1 1, type="III")
5779
       summary(rlogM RP1 1)
5780
5781
      mmRP1 <- emmeans(rlogM RP1 1,~studyarm,type = "response") #proportions
5782
       mmRP1
5783
       confint(pairs(mmRP1, reverse = TRUE)) #Odds ratios
5784
       pairs (mmRP1, reverse = TRUE, type = "response")
5785
5786
       # Model 2: Check for direct effects of factors with adjustment for other covariates
5787
      rlogM RP1 2 <-
5788
         glm(RP1 dicho ~ studyarm +
5789
              mean indivhorz +
5790
               mean indivvertical +
5791
              mean collhorz +
5792
              mean collvertical +
5793
               bornincanada +
5794
               language 1 +
5795
               language 2 +
5796
               Asian_group +
5797
              White_group +
5798
              disability any +
5799
              genderidentity +
5800
              income +
5801
              edhi +
5802
5803
             data = datMeasles, family=binomial("logit")
5804
5805
       Anova(rlogM RP1 2, type = "III")
```

```
5806
       summary(rlogM RP1 2)
5807
5808
      mmRP1 2 <- emmeans(rlogM RP1 2,~studyarm,type = "response")
5809
      mmRP1 2
5810
      confint(pairs(mmRP1 2, reverse = TRUE))
5811
      pairs (mmRP1 2, reverse = TRUE, type = "response")
5812
5813
5814
      # Model 3: Check for moderating effects of individualism & collectivism with adjustment
      for other covariates
5815
     rlogM RP1 3 <-
5816
         glm(RP1 dicho ~
5817
               studyarm * mean indivhorz +
5818
               studyarm * mean indivvertical +
5819
               studyarm * mean collhorz +
5820
               studyarm * mean collvertical +
5821
               bornincanada +
5822
               language 1 +
5823
              language 2 +
5824
              Asian group +
5825
              White group +
5826
              disability any +
5827
              genderidentity +
5828
              income +
5829
               edhi +
5830
               age,
5831
             data = datMeasles, family=binomial("logit")
5832
         )
5833
     Anova(rlogM RP1 3, type = "III")
5834
      summary(rlogM RP1 3)
5835
5836
       #No interaction with moderator to interpret
5837
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
5838
5839
5840
       rlogM RP1 4 <- glm(RP1 dicho ~ studyarm * edhi, data =</pre>
       datMeasles, family=binomial("logit"))
5841
      Anova(rlogM RP1 4, type="III")
5842
      summary(rlogM RP1 4)
5843
5844
     mmRP1 4 s <- emmeans(rlogM RP1 4,~studyarm|edhi,type = "response")
5845
     mmRP1 4 s
5846
      confint(pairs(mmRP1 4 s, reverse = TRUE))
5847
5848
      mmRP1 4 e <- emmeans(rlogM RP1 4, ~ edhi|studyarm, type = "response")
5849
      confint(pairs(mmRP1 4 e, reverse = TRUE))
5850
5851
5852
      # Model 5: Check for interaction viz*edhi with adjustment for other covariates
5853
5854
     rlogM RP1 5 <-
5855
       glm(RP1 dicho
                        ~ studyarm*edhi +
5856
              mean indivhorz +
5857
               mean indivvertical +
5858
              mean collhorz +
5859
              mean collvertical +
5860
               bornincanada +
5861
               language 1 +
5862
               language 2 +
5863
               Asian_group +
5864
               White_group +
5865
              disability any +
5866
              genderidentity +
5867
              income +
5868
               age,
5869
             data = datMeasles, family=binomial("logit")
5870
         )
5871
       Anova(rlogM_RP1 5, type = "III")
5872
      summary(rlogM RP1 5)
```

```
5873
5874
       mmRP1 5 s <- emmeans(rlogM RP1 5,~studyarm|edhi,type = "response")
5875
       mmRP1 5 s
5876
       confint (pairs (mmRP1 5 s, reverse = TRUE))
5877
      mmRP1_5_e <- emmeans(rlogM_RP1_5, ~ edhi|studyarm, type = "response")
5878
5879
      confint(pairs(mmRP1 5 e, reverse = TRUE))
5880
5881
       # Now running models on imputed data.
5882
5883
      imprlogM RP1 1 <-
5884
         with(data = datMeaslesImputed,
5885
              exp = glm(relevel(RP1 dicho,ref="Low") ~ studyarm,family = binomial("logit")))
       combineimprlogM RP1 1 <- pool(imprlogM_RP1_1)</pre>
5886
5887
       summary(combineimprlogM RP1 1)
5888
5889
5890
       #### ++ Flu ####
5891
5892
       #### + Model 1: Check for direct effects of factors without any covariates ####
5893
5894
      options(contrasts=c("contr.sum", "contr.poly"))
5895
      rlogF RP1 1 <- glm(RP1 dicho ~ studyarm, data = datFlu, family=binomial("logit"))</pre>
5896
       Anova(rlogF RP1 1, type="III")
5897
       summary(rlogF RP1 1)
5898
5899
      mfRP1 1 <- emmeans(rlogF RP1 1,~studyarm,type = "response") #proportions
5900
     mfRP1_1
      confint(pairs(mfRP1 1, reverse = TRUE)) #Odds ratios
5901
5902
      pairs (mfRP1 1, reverse = TRUE, type = "response")
5903
5904
      # Model 2: Check for direct effects of factors with adjustment for other covariates
5905
      rlogF RP1 2 <-
         glm (RP1 dicho ~ studyarm +
5906
5907
               mean indivhorz +
5908
               mean indivvertical +
5909
               mean collhorz +
5910
               mean collvertical +
5911
               bornincanada +
5912
               language 1 +
5913
               language 2 +
5914
              Asian group +
5915
              White group +
5916
              disability any +
5917
               genderidentity +
5918
               income +
5919
               edhi +
5920
               age,
5921
             data = datFlu, family=binomial("logit")
5922
         )
5923
      Anova(rlogF RP1 2, type = "III")
5924
      summary(rlogF RP1 2)
5925
5926
      mfRP1 2 <- emmeans(rlogF RP1 2,~studyarm,type = "response")
5927
      mfRP1 2
5928
       confint(pairs(mfRP1_2, reverse = TRUE))
5929
       pairs (mfRP1 2, reverse = TRUE, type = "response")
5930
5931
5932
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
       rlogF_RP1_3 <-
5933
5934
         glm(RP1 dicho ~
5935
               studyarm * mean indivhorz +
5936
               studyarm * mean indivvertical +
5937
              studyarm * mean collhorz +
5938
               studyarm * mean collvertical +
5939
               bornincanada +
5940
               language 1 +
```

```
5941
              language 2 +
5942
              Asian group +
5943
              White group +
5944
              disability any +
5945
               genderidentity +
5946
               income +
5947
               edhi +
5948
               age,
5949
             data = datFlu, family=binomial("logit")
5950
         )
       Anova(rlogF RP1 3, type = "III")
5951
5952
       summary(rlogF RP1 3)
5953
5954
       emmip(rlogF RP1 3, studyarm ~ mean collhorz, cov.reduce = range, type = "response")
5955
       emmip(rlogF RP1 3, studyarm ~ mean collvertical, cov.reduce = range, type = "response")
5956
5957
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
5958
5959
5960
     rlogF RP1 4 <- glm(RP1 dicho ~ studyarm * edhi, data =</pre>
       datMeasles, family=binomial("logit"))
5961
       Anova (rlogF RP1 4, type="III")
5962
       summary(rlogF RP1 4)
5963
5964
       mfRP1 4 s <- emmeans(rlogF RP1 4,~studyarm|edhi,type = "response")
      mfRP1 4 s
5965
5966
      confint(pairs(mfRP1 4 s, reverse = TRUE))
5967
5968
      mfRP1 4 e <- emmeans(rlogF RP1 4, ~ edhi|studyarm, type = "response")
5969
      confint(pairs(mfRP1 4 e, reverse = TRUE))
5970
5971
5972
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
5973
5974
       rlogF RP1 5 <-
5975
       glm(RP1 dicho
                        ~ studyarm*edhi +
5976
               mean indivhorz +
5977
               mean indivvertical +
5978
              mean collhorz +
5979
              mean collvertical +
5980
              bornincanada +
5981
              language 1 +
5982
              language 2 +
5983
              Asian group +
5984
              White group +
5985
              disability any +
5986
               genderidentity +
5987
               income +
5988
               age,
5989
             data = datFlu, family=binomial("logit")
5990
         )
5991
      Anova(rlogF RP1 5, type = "III")
5992
      summary(rlogF RP1 5)
5993
5994
      mfRP1 5 s <- emmeans(rlogF RP1 5,~studyarm|edhi,type = "response")
5995
      mfRP1 5 s
5996
       confint(pairs(mfRP1 5 s, reverse = TRUE))
5997
5998
       mfRP1 5 e <- emmeans(rlogF RP1 5, ~ edhi|studyarm, type = "response")
5999
       confint (pairs (mfRP1_5_e, reverse = TRUE))
6000
6001
       # Now running models on imputed data.
6002
6003
       imprlogF RP1 1 <-
6004
         with(data = datFluImputed,
6005
              exp = glm(relevel(RP1 dicho,ref="Low") ~ studyarm,family = binomial("logit")))
6006
       combineimprlogF RP1 1 <- pool(imprlogF RP1 1)</pre>
6007
       summary(combineimprlogF RP1 1)
6008
```

```
6009
6010
       #### +++ Logistic regression for VaxIntention ####
6011
6012
       #Create relevel before model to avoid problems with pairs function.
6013
       datGeneric$vaxintent <- relevel(datGeneric$vaxintent,ref = "Low")</pre>
6014
       datMeasles$vaxintent <- relevel(datMeasles$vaxintent,ref = "Low")</pre>
6015
       datFlu$vaxintent <- relevel(datFlu$vaxintent, ref = "Low")</pre>
6016
6017
       #### ++ Generic ####
6018
6019
       #### + Model 1: Check for direct effects of factors without any covariates ####
6020
6021
       options(contrasts=c("contr.sum", "contr.poly"))
6022
       rlogG vi 1 <- glm(vaxintent ~ studyarm, data = datGeneric,family=binomial("logit"))</pre>
6023
       Anova(rlogG vi 1, type="III")
6024
       summary(rlogG vi 1)
6025
6026
      mgvi 1 <- emmeans(rlogG vi 1,~studyarm, type = "response") #proportions
6027
       mgvi 1
       confint(pairs(mgvi 1, reverse = TRUE)) #Odds ratios
6028
6029
6030
       # Model 2: Check for direct effects of factors with adjustment for other covariates
6031
      rlogG vi 2 <-
6032
         glm(vaxintent ~ studyarm +
6033
               mean indivhorz +
6034
               mean indivvertical +
               mean collhorz +
6035
6036
               mean collvertical +
6037
               bornincanada +
6038
               language 1 +
6039
               language 2 +
6040
               Asian group +
6041
               White group +
6042
               disability any +
6043
               genderidentity +
6044
               income +
6045
               edhi +
6046
               age,
6047
             data = datGeneric, family=binomial("logit")
6048
         )
6049
       Anova(rlogG vi 2, type = "III")
6050
       summary(rlogG vi 2)
6051
6052
       mgvi 2 <- emmeans(rlogG vi 2,~studyarm,type = "response")</pre>
6053
       mqvi 2
6054
       confint(pairs(mgvi 2, reverse = TRUE))
6055
6056
6057
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
6058
      rlogG vi 3 <-
6059
         glm (vaxintent
6060
               studyarm * mean indivhorz +
6061
               studyarm * mean indivvertical +
               studyarm * mean collhorz +
6062
6063
               studyarm * mean collvertical +
6064
               bornincanada +
6065
               language 1 +
6066
               language 2 +
6067
               Asian_group +
6068
               White_group +
6069
               disability any +
6070
               genderidentity +
6071
               income +
6072
               edhi +
6073
6074
             data = datGeneric, family=binomial("logit")
6075
6076
       Anova(rlogG vi 3, type = "III")
```

```
6077
       summary(rlogG vi 3)
6078
6079
       #No interaction with moderator to interpret
6080
6081
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
6082
       rlogG_vi_4 <- glm(vaxintent ~ studyarm * edhi, data =</pre>
6083
       datGeneric, family=binomial("logit"))
6084
       Anova(rlogG vi 4, type="III")
6085
       summary(rlogG vi 4)
6086
6087
      mgvi 4 s <- emmeans(rlogG vi 4,~studyarm|edhi,type = "response")
6088
       mqvi 4 s
6089
       confint(pairs(mgvi 4 s,reverse = TRUE))
6090
6091
       mgvi 4 e <- emmeans(rlogG vi 4, ~ edhi|studyarm, type = "response")
6092
       confint(pairs(mgvi 4 e, reverse = TRUE))
6093
6094
6095
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
6096
6097
      rlogG vi 5 <-
6098
         glm (vaxintent
                         ~ studyarm*edhi +
6099
               mean indivhorz +
               \label{eq:mean_indivvertical} \ \ \textbf{+}
6100
6101
               mean collhorz +
6102
               mean collvertical +
6103
               bornincanada +
6104
               language 1 +
6105
               language 2 +
               Asian group +
6106
6107
               White group +
6108
               disability any +
6109
               genderidentity +
6110
               income +
6111
               age,
             data = datGeneric, family=binomial("logit")
6112
6113
         )
6114
       Anova(rlogG_vi_5, type = "III")
6115
       summary(rlogG vi 5)
6116
6117
       mgvi 5 s <- emmeans(rlogG vi 5,~studyarm|edhi,type = "response")
6118
6119
       confint(pairs(mgvi 5 s,reverse = TRUE))
6120
6121
       mgvi 5 e <- emmeans(rlogG vi 5, ~ edhi|studyarm, type = "response")
6122
       confint (pairs (mgvi 5 e, reverse = TRUE))
6123
6124
       # Now running models on imputed data.
6125
6126
      imprlogG vi 1 <-
6127
        with (data = datGenericImputed,
              exp = glm(relevel(vaxintent,ref="Low") ~ studyarm,family = binomial("logit")))
6128
6129
       combineimprlogG vi 1 <- pool(imprlogG vi 1)</pre>
6130
       summary(combineimprlogG vi 1)
6131
6132
       #CHANGELOG ASJ: add test to check if global test result changes or not, 21-09-20.
6133
       imprlogG vi vide <-</pre>
6134
        with(data = datGenericImputed,
6135
              exp = glm(relevel(vaxintent,ref="Low") ~ 1,family = binomial("logit"))) #model
              with intercept only
6136
       combineimprlogG vi vide <- pool(imprlogG vi vide)</pre>
6137
       summary(combineimprlogG vi vide)
6138
       test sig<-D2(imprlogG vi 1,imprlogG vi vide) #compare model with studyarm vs model with
       intercept only
6139
       summary(test sig)
6140
6141
```

6142

```
6144
       #### ++ Measles ####
6145
6146
       #### + Model 1: Check for direct effects of factors without any covariates ####
6147
6148
      options(contrasts=c("contr.sum", "contr.poly"))
6149
      rlogM vi 1 <- glm(vaxintent ~ studyarm, data = datMeasles, family=binomial("logit"))</pre>
6150
      Anova(rlogM vi 1, type="III")
6151
      summary(rlogM vi 1)
6152
6153
      mmvi <- emmeans(rlogM vi 1,~studyarm, type = "response") #proportions
6154
6155
      confint(pairs(mmvi, reverse = TRUE)) #Odds ratios
6156
       pairs (mmvi, reverse = TRUE, type = "response")
6157
6158
       # Model 2: Check for direct effects of factors with adjustment for other covariates
6159
      rlogM vi 2 <-
6160
         glm(vaxintent ~ studyarm +
6161
               mean indivhorz +
6162
               mean indivvertical +
6163
               mean collhorz +
6164
               mean collvertical +
6165
               bornincanada +
6166
               language 1 +
6167
               language 2 +
6168
               Asian group +
6169
               White group +
6170
               disability any +
6171
               genderidentity +
6172
               income +
6173
               edhi +
6174
6175
             data = datMeasles, family=binomial("logit")
6176
         )
       Anova(rlogM_vi 2, type = "III")
6177
6178
       summary(rlogM vi 2)
6179
6180
       mmvi 2 <- emmeans (rlogM vi 2, ~studyarm, type = "response")
6181
6182
       confint(pairs(mmvi 2, reverse = TRUE))
6183
6184
6185
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
6186
      rlogM vi 3 <-
6187
         glm(vaxintent ~
6188
               studyarm * mean indivhorz +
6189
               studyarm * mean indivvertical +
6190
               studyarm * mean collhorz +
               studyarm * mean collvertical +
6191
6192
               bornincanada +
6193
               language 1 +
6194
               language 2 +
6195
               Asian group +
6196
               White group +
6197
               disability any +
6198
               genderidentity +
6199
               income +
6200
               edhi +
6201
6202
             data = datMeasles, family=binomial("logit")
6203
         )
6204
       Anova(rlogM vi 3, type = "III")
6205
       summary(rlogM vi 3)
6206
6207
       #No interaction with moderator to interpret
6208
6209
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
6210
```

6143

```
6211
       rlogM vi 4 <- glm(vaxintent ~ studyarm * edhi, data =</pre>
       datMeasles, family=binomial("logit"))
6212
       Anova(rlogM vi 4, type="III")
6213
       summary(rlogM vi 4)
6214
6215
      mmvi 4 s <- emmeans(rlogM vi 4,~studyarm|edhi,type = "response")
6216
      mmvi 4 s
6217
      confint (pairs (mmvi 4 s, reverse = TRUE))
6218
6219
      mmvi 4 e <- emmeans(rlogM vi 4, ~ edhi|studyarm, type = "response")
6220
      confint(pairs(mmvi 4 e, reverse = TRUE))
6221
6222
6223
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
6224
6225
      rlogM vi 5 <-
6226
         glm(vaxintent ~ studyarm*edhi +
6227
              mean indivhorz +
6228
               mean indivvertical +
6229
              mean collhorz +
6230
              mean collvertical +
6231
              bornincanada +
6232
              language 1 +
6233
              language 2 +
6234
               Asian group +
6235
               White group +
6236
              disability any +
6237
               genderidentity +
6238
              income +
6239
               age,
6240
             data = datMeasles, family=binomial("logit")
6241
6242
      Anova(rlogM vi 5, type = "III")
6243
      summary(rlogM vi 5)
6244
      mmvi 5 s <- emmeans(rlogM vi 5,~studyarm|edhi,type = "response")</pre>
6245
      mmvi 5 s
6246
6247
      confint(pairs(mmvi 5 s,reverse = TRUE))
6248
6249
      mmvi 5 e <- emmeans(rlogM vi 5, ~ edhi|studyarm, type = "response")
6250
      confint (pairs (mmvi 5 e, reverse = TRUE))
6251
6252
       # Now running models on imputed data.
6253
      imprlogM vi 1 <-
6254
         with(data = datMeaslesImputed,
6255
              exp = glm(relevel(vaxintent,ref="Low") ~ studyarm,family = binomial("logit")))
6256
       combineimprlogM vi 1 <- pool(imprlogM vi 1)</pre>
6257
       summary(combineimprlogM vi 1)
6258
6259
6260
       #### ++ Flu ####
6261
6262
      #### + Model 1: Check for direct effects of factors without any covariates ####
6263
6264
      options(contrasts=c("contr.sum", "contr.poly"))
6265
      rlogF vi 1 <- glm(vaxintent ~ studyarm, data = datFlu, family=binomial("logit"))</pre>
6266
      Anova(rlogF vi 1, type="III")
6267
       summary(rlogF vi 1)
6268
6269
      mfvi 1 <- emmeans(rlogF vi 1,~studyarm,type = "response") #proportions
      mfvi_1
6270
6271
      confint(pairs(mfvi 1, reverse = TRUE)) #Odds ratios
6272
6273
6274
       # Model 2: Check for direct effects of factors with adjustment for other covariates
6275
      rlogF vi 2 <-
6276
         glm(vaxintent ~ studyarm +
6277
               mean indivhorz +
6278
               mean indivvertical +
```

```
6279
              mean collhorz +
6280
              mean collvertical +
6281
              bornincanada +
6282
               language 1 +
6283
               language 2 +
6284
              Asian group +
6285
              White group +
6286
              disability any +
6287
               genderidentity +
6288
               income +
6289
               edhi +
6290
               age,
             data = datFlu, family=binomial("logit")
6291
6292
         )
6293
       Anova(rlogF vi 2, type = "III")
6294
       summary(rlogF vi 2)
6295
6296
      mfvi 2 <- emmeans(rlogF vi 2,~studyarm,type = "response")</pre>
6297
      mfvi 2
6298
       confint(pairs(mfvi 2, reverse = TRUE))
6299
6300
6301
      # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
      rlogF vi 3 <-
6302
6303
        glm (vaxintent ~
6304
               studyarm * mean indivhorz +
6305
               studyarm * mean_indivvertical +
6306
               studyarm * mean collhorz +
6307
              studyarm * mean collvertical +
6308
              bornincanada +
6309
              language 1 +
6310
              language 2 +
6311
              Asian group +
6312
              White group +
6313
               disability any +
6314
               genderidentity +
6315
               income +
6316
               edhi +
6317
               age,
6318
             data = datFlu, family=binomial("logit")
6319
         )
6320
       Anova(rlogF vi 3, type = "III")
6321
       summary(rlogF vi 3)
6322
6323
       emmip(rlogF vi 3, studyarm ~ mean indivvertical, cov.reduce = range, type = "response")
6324
6325
6326
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
6327
6328
      rlogF vi 4 <- glm(vaxintent ~ studyarm * edhi, data = datFlu, family=binomial("logit"))</pre>
6329
      Anova(rlogF vi 4, type="III")
6330
      summary(rlogF vi 4)
6331
6332
      mfvi 4 s <- emmeans(rlogF vi 4,~studyarm|edhi,type = "response")
6333
      mfvi 4 s
6334
       confint(pairs(mfvi 4 s,reverse = TRUE))
6335
6336
       mfvi 4 e <- emmeans(rlogF vi 4, ~ edhi|studyarm, type = "response")
6337
       confint(pairs(mfvi 4 e, reverse = TRUE))
6338
6339
6340
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
6341
6342
      rlogF vi 5 <-
6343
         glm (vaxintent
                        ~ studyarm*edhi +
6344
               mean indivhorz +
6345
               mean indivvertical +
6346
               mean collhorz +
```

```
6347
               mean collvertical +
6348
              bornincanada +
6349
               language 1 +
               language 2 +
6350
6351
               Asian group +
6352
               White_group +
               disability_any +
6353
6354
               genderidentity +
6355
               income +
6356
6357
             data = datFlu, family=binomial("logit")
6358
         )
6359
      Anova(rlogF vi 5, type = "III")
6360
       summary(rlogF vi 5)
6361
6362
      mfvi 5 s <- emmeans(rlogF vi 5,~studyarm|edhi,type = "response")
6363
      mfvi_5_s
6364
      confint(pairs(mfvi 5 s, reverse = TRUE))
6365
6366
      mfvi 5 e <- emmeans(rlogF vi 5, ~ edhi|studyarm, type = "response")
6367
      confint(pairs(mfvi 5 e, reverse = TRUE))
6368
6369
       # Now running models on imputed data.
6370
      imprlogF vi 1 <-
6371
         with (data = datFluImputed,
              exp = glm(relevel(vaxintent,ref="Low") ~ studyarm,family = binomial("logit")))
6372
6373
      combineimprlogF vi 1 <- pool(imprlogF vi 1)</pre>
6374
      summary(combineimprlogF vi 1)
6375
6376
       #### +++ Logistic regression for C19VaxIntention ####
6377
6378
      #Create relevel before model to avoid problems with pairs function.
6379
     datGeneric$c19vaxintent <- relevel(datGeneric$c19vaxintent,ref = "Low")</pre>
6380
      datMeasles$c19vaxintent <- relevel(datMeasles$c19vaxintent,ref = "Low")</pre>
6381
       datFlu$c19vaxintent <- relevel(datFlu$c19vaxintent,ref = "Low")</pre>
6382
       #### ++ Generic ####
6383
6384
6385
       #### + Model 1: Check for direct effects of factors without any covariates ####
6386
6387
       options(contrasts=c("contr.sum", "contr.poly"))
6388
       rlogG c19vi 1 <- glm(c19vaxintent ~ studyarm, data =</pre>
       datGeneric, family=binomial("logit"))
6389
       Anova(rlogG c19vi 1, type="III")
6390
      summary(rlogG c19vi 1)
6391
6392
      mgc19vi 1 <- emmeans(rlogG c19vi 1,~studyarm,type = "response") #proportions
6393
      mgc19vi 1
6394
      confint(pairs(mqc19vi 1, reverse = TRUE)) #Odds ratios
6395
6396
     # Model 2: Check for direct effects of factors with adjustment for other covariates
6397
     rlogG c19vi 2 <-
6398
        glm(c19vaxintent ~ studyarm +
6399
               mean indivhorz +
6400
               mean indivvertical +
6401
               mean collhorz +
6402
               mean collvertical +
6403
               bornincanada +
6404
               language 1 +
6405
               language 2 +
6406
               Asian_group +
6407
               White group +
6408
              disability any +
6409
              genderidentity +
6410
              income +
6411
              edhi +
6412
               age,
6413
             data = datGeneric, family=binomial("logit")
6414
         )
```

```
6415
       Anova(rlogG c19vi 2, type = "III")
6416
       summary(rlogG c19vi 2)
6417
6418
      mgc19vi 2 <- emmeans(rlogG c19vi 2,~studyarm,type = "response")
6419
      mgc19vi 2
6420
      confint(pairs(mgc19vi 2, reverse = TRUE))
6421
      pairs (mgc19vi 2, reverse = TRUE, type = "response")
6422
6423
     # Model 3: Check for moderating effects of individualism & collectivism with adjustment
      for other covariates
6424
      rlogG c19vi 3 <-
6425
         glm(c19vaxintent ~
6426
               studyarm * mean indivhorz +
6427
               studyarm * mean indivvertical +
6428
               studyarm * mean collhorz +
6429
               studyarm * mean collvertical +
6430
               bornincanada +
6431
               language 1 +
6432
               language 2 +
6433
               Asian group +
6434
              White group +
6435
              disability any +
6436
               genderidentity +
6437
               income +
6438
               edhi +
6439
               age,
6440
             data = datGeneric, family=binomial("logit")
6441
         )
6442
      Anova(rlogG c19vi 3, type = "III")
6443
      summary(rlogG c19vi 3)
6444
6445
       #No interaction with moderator to interpret
6446
6447
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
6448
6449
       rlogG c19vi 4 <- glm(c19vaxintent ~ studyarm * edhi, data =</pre>
       datGeneric, family=binomial("logit"))
6450
       Anova(rlogG c19vi 4, type="III")
6451
      summary(rlogG_c19vi_4)
6452
6453
      mgc19vi 4 s <- emmeans(rlogG c19vi 4,~studyarm|edhi,type = "response")
6454
      mgc19vi 4 s
6455
      confint(pairs(mgc19vi 4 s, reverse = TRUE))
6456
6457
       mgc19vi 4 e <- emmeans(rlogG c19vi 4, ~ edhi|studyarm, type = "response")
6458
       confint(pairs(mgc19vi 4 e,reverse = TRUE))
6459
6460
6461
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
6462
6463
      rlogG c19vi 5 <-
6464
       glm(c19vaxintent
                            ~ studyarm*edhi +
6465
               mean indivhorz +
6466
               mean indivvertical +
6467
               mean collhorz +
6468
               mean collvertical +
6469
               bornincanada +
6470
               language 1 +
6471
               language 2 +
6472
               Asian_group +
6473
               White_group +
6474
               disability any +
6475
               genderidentity +
6476
               income +
6477
               age,
6478
             data = datGeneric, family=binomial("logit")
6479
         )
6480
       Anova(rlogG c19vi 5, type = "III")
6481
       summary(rlogG c19vi 5)
```

```
6482
6483
      mgc19vi 5 s <- emmeans(rlogG c19vi 5,~studyarm|edhi,type = "response")
6484
       mgc19vi 5 s
6485
       confint(pairs(mgc19vi 5 s, reverse = TRUE))
6486
      mgc19vi_5_e <- emmeans(rlogG_c19vi_5, ~ edhi|studyarm, type = "response")</pre>
6487
6488
      confint(pairs(mgc19vi 5 e, reverse = TRUE))
6489
6490
       #### ++ Measles ####
6491
6492
       #### + Model 1: Check for direct effects of factors without any covariates ####
6493
       options(contrasts=c("contr.sum", "contr.poly"))
6494
       rlogM c19vi 1 <- glm(c19vaxintent ~ studyarm, data =</pre>
6495
       datMeasles, family=binomial("logit"))
6496
       Anova(rlogM c19vi 1, type="III")
6497
       summary(rlogM c19vi 1)
6498
6499
      mmc19vi 1 <- emmeans(rlogM c19vi 1,~studyarm,type = "response") #proportions
6500
      mmc19vi 1
6501
      confint(pairs(mmc19vi 1, reverse = TRUE)) #Odds ratios
6502
6503
       # Model 2: Check for direct effects of factors with adjustment for other covariates
6504
      rlogM c19vi 2 <-
6505
         glm(c19vaxintent ~ studyarm +
6506
               mean indivhorz +
               mean indivvertical +
6507
6508
               mean collhorz +
6509
              mean collvertical +
6510
              bornincanada +
6511
              language 1 +
6512
              language 2 +
6513
              Asian group +
6514
              White group +
6515
               disability any +
6516
               genderidentity +
6517
               income +
6518
               edhi +
6519
               age,
6520
             data = datMeasles, family=binomial("logit")
6521
         )
6522
       Anova(rlogM c19vi 2, type = "III")
6523
      summary(rlogM c19vi 2)
6524
6525
      mmc19vi 2 <- emmeans(rlogM c19vi 2,~studyarm,type = "response")
6526
      mmc19vi 2
6527
       confint(pairs(mmc19vi 2, reverse = TRUE))
6528
6529
6530
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
6531
      rlogM c19vi 3 <-
6532
        glm(c19vaxintent
6533
               studyarm * mean indivhorz +
6534
               studyarm * mean indivvertical +
6535
               studyarm * mean collhorz +
6536
               studyarm * mean collvertical +
6537
               bornincanada +
6538
               language 1 +
6539
               language_2 +
6540
               Asian_group +
6541
               White group +
6542
              disability any +
6543
              genderidentity +
6544
              income +
6545
              edhi +
6546
               age,
6547
             data = datMeasles, family=binomial("logit")
6548
         )
```

```
6549
       Anova(rlogM c19vi 3, type = "III")
6550
       summary(rlogM c19vi 3)
6551
6552
       #No interaction with moderator to interpret
6553
6554
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
6555
      rlogM c19vi 4 <- glm(c19vaxintent ~ studyarm * edhi, data =
6556
       datMeasles, family=binomial("logit"))
6557
      Anova(rlogM c19vi 4, type="III")
6558
      summary(rlogM c19vi 4)
6559
6560
      mmc19vi 4 s <- emmeans(rlogM c19vi 4,~studyarm|edhi,type = "response")
6561
       mmc19vi 4 s
6562
       confint(pairs(mmc19vi 4 s, reverse = TRUE))
6563
      mmc19vi_4_e <- emmeans(rlogM_c19vi_4, ~ edhi|studyarm, type = "response")</pre>
6564
6565
       confint(pairs(mmc19vi 4 e,reverse = TRUE))
6566
6567
6568
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
6569
6570
      rlogM c19vi 5 <-
6571
         glm(c19vaxintent ~ studyarm*edhi +
6572
               mean indivhorz +
               mean indivvertical +
6573
6574
              mean collhorz +
6575
              mean collvertical +
6576
              bornincanada +
6577
              language 1 +
6578
              language 2 +
6579
              Asian group +
6580
              White group +
6581
              disability any +
6582
               genderidentity +
6583
               income +
6584
               age,
6585
             data = datMeasles, family=binomial("logit")
6586
         )
6587
       Anova(rlogM c19vi 5, type = "III")
6588
      summary(rlogM c19vi 5)
6589
6590
      mmc19vi 5 s <- emmeans(rlogM c19vi 5,~studyarm|edhi,type = "response")
6591
      mmc19vi 5 s
6592
      confint(pairs(mmc19vi 5 s,reverse = TRUE))
6593
6594
      mmc19vi 5 e <- emmeans(rlogM c19vi 5, ~ edhi|studyarm, type = "response")
6595
       confint(pairs(mmc19vi 5 e, reverse = TRUE))
6596
6597
6598
6599
       #### ++ Flu ####
6600
6601
       #### + Model 1: Check for direct effects of factors without any covariates ####
6602
6603
      options(contrasts=c("contr.sum", "contr.poly"))
6604
       rlogF c19vi 1 <- glm(c19vaxintent ~ studyarm, data = datFlu,family=binomial("logit"))</pre>
6605
       Anova (rlogF c19vi 1, type="III")
6606
       summary(rlogF c19vi 1)
6607
6608
      mfc19vi 1 <- emmeans(rlogF c19vi 1,~studyarm,type = "response") #proportions
6609
      mfc19vi 1
6610
      confint(pairs(mfc19vi 1, reverse = TRUE)) #Odds ratios
6611
6612
6613
       # Model 2: Check for direct effects of factors with adjustment for other covariates
6614
      rlogF c19vi 2 <-
6615
         glm(c19vaxintent ~ studyarm +
6616
               mean indivhorz +
```

```
6617
              mean indivvertical +
6618
              mean collhorz +
6619
              mean collvertical +
6620
              bornincanada +
6621
               language 1 +
              language_2 +
6622
6623
              Asian group +
6624
              White_group +
6625
              disability any +
6626
               genderidentity +
6627
               income +
6628
               edhi +
6629
               age,
6630
             data = datFlu, family=binomial("logit")
6631
         )
6632
      Anova(rlogF c19vi 2, type = "III")
6633
      summary(rlogF c19vi 2)
6634
6635
     mfc19vi 2 <- emmeans(rlogF c19vi 2,~studyarm,type = "response")
6636 mfc19vi 2
6637
      confint(pairs(mfc19vi 2, reverse = TRUE))
6638
6639
6640
      # Model 3: Check for moderating effects of individualism & collectivism with adjustment
      for other covariates
6641
      rlogF c19vi 3 <-
6642
        glm(c19vaxintent ~
6643
               studyarm * mean_indivhorz +
6644
               studyarm * mean indivvertical +
6645
              studyarm * mean collhorz +
6646
              studyarm * mean collvertical +
6647
              bornincanada +
6648
               language 1 +
               language 2 +
6649
6650
               Asian group +
6651
               White group +
6652
               disability any +
6653
               genderidentity +
6654
               income +
6655
               edhi +
6656
               age,
6657
             data = datFlu, family=binomial("logit")
6658
6659
       Anova(rlogF c19vi 3, type = "III")
6660
       summary(rlogF c19vi 3)
6661
6662
       #No interaction with moderator to interpret
6663
6664
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
6665
6666
     rlogF c19vi 4 <- glm(c19vaxintent ~ studyarm * edhi, data =</pre>
       datFlu, family=binomial("logit"))
6667
      Anova(rlogF c19vi 4, type="III")
6668
      summary(rlogF c19vi 4)
6669
6670
      mfc19vi 4 s <- emmeans(rlogF c19vi 4,~studyarm|edhi,type = "response")
6671
      mfc19vi 4 s
6672
      confint(pairs(mfc19vi 4 s, reverse = TRUE))
6673
6674
      mfc19vi_4_e <- emmeans(rlogF_c19vi_4, ~ edhi|studyarm, type = "response")</pre>
6675
      confint (pairs (mfc19vi_4_e, reverse = TRUE))
6676
6677
6678
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
6679
6680
      rlogF c19vi 5 <-
6681
         glm(c19vaxintent
                            ~ studyarm*edhi +
6682
               mean indivhorz +
               mean indivvertical +
6683
```

```
6684
              mean collhorz +
6685
              mean collvertical +
6686
              bornincanada +
6687
               language 1 +
6688
               language 2 +
6689
               Asian group +
6690
               White group +
6691
               disability any +
6692
               genderidentity +
6693
               income +
6694
               age.
6695
             data = datFlu, family=binomial("logit")
6696
         )
6697
       Anova(rlogF c19vi 5, type = "III")
6698
       summary(rlogF c19vi 5)
6699
6700
      mfc19vi 5 s <- emmeans(rlogF c19vi 5,~studyarm|edhi,type = "response")
6701
      mfc19vi 5 s
6702
      confint(pairs(mfc19vi 5 s, reverse = TRUE))
6703
6704
      mfc19vi 5 e <- emmeans(rlogF c19vi 5, ~ edhi|studyarm, type = "response")
6705
       confint(pairs(mfc19vi 5 e, reverse = TRUE))
6706
6707
6708
6709
6710
6711
6712
6713
       #### +++ Logistic regression for Trust Info ####
6714
6715
      #Create relevel before model to avoid problems with pairs function.
6716
      datGeneric$Htrustinfo <- relevel(datGeneric$Htrustinfo,ref = "No")</pre>
6717
       datMeasles$Htrustinfo <- relevel(datMeasles$Htrustinfo,ref = "No")
       datFlu$Htrustinfo <- relevel(datFlu$Htrustinfo,ref = "No")</pre>
6718
6719
6720
       #### ++ Generic ####
6721
6722
       #### + Model 1: Check for direct effects of factors without any covariates ####
6723
6724
       options(contrasts=c("contr.sum", "contr.poly"))
6725
       rlogG_ti_1 <- glm(Htrustinfo ~ studyarm, data = datGeneric, family=binomial("logit"))</pre>
6726
       Anova (rlogG ti 1, type="III")
6727
       summary(rlogG ti 1)
6728
6729
      mgti 1 <- emmeans(rlogG ti 1,~studyarm,type = "response") #proportions
6730
      mgti 1
6731
       confint(pairs(mgti 1, reverse = TRUE)) #Odds ratios
6732
      pairs (mgti 1, reverse = TRUE, type="response")
6733
6734
      # Model 2: Check for direct effects of factors with adjustment for other covariates
6735
     rlogG ti 2 <-
6736
        glm(Htrustinfo ~ studyarm +
6737
               mean indivhorz +
6738
               mean indivvertical +
6739
               mean collhorz +
6740
               mean collvertical +
6741
               bornincanada +
6742
               language 1 +
6743
               language 2 +
6744
               Asian_group +
6745
               White group +
6746
              disability any +
6747
              genderidentity +
6748
              income +
6749
              edhi +
6750
               age,
6751
             data = datGeneric, family=binomial("logit")
6752
         )
```

```
6753
       Anova(rlogG ti 2, type = "III")
6754
       summary(rlogG ti 2)
6755
6756
       mgti 2 <- emmeans(rlogG ti 2,~studyarm,type = "response")
6757
6758
       confint(pairs(mgti 2, reverse = TRUE))
6759
      pairs (mgti 2, reverse = TRUE, type="response")
6760
6761
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
6762
       rlogG ti 3 <-
6763
         glm (Htrustinfo ~
6764
               studyarm * mean indivhorz +
6765
               studyarm * mean indivvertical +
               studyarm * mean collhorz +
6766
6767
               studyarm * mean collvertical +
6768
               bornincanada +
6769
               language 1 +
6770
               language 2 +
6771
               Asian group +
6772
               White group +
6773
               disability any +
6774
               genderidentity +
6775
               income +
6776
               edhi +
6777
               age,
6778
             data = datGeneric, family=binomial("logit")
6779
         )
6780
       Anova(rlogG ti 3, type = "III")
6781
       summary(rlogG_ti_3)
6782
6783
       #No interaction with moderator to interpret
6784
6785
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
6786
6787
       rlogG ti 4 <- glm(Htrustinfo ~ studyarm * edhi, data =</pre>
       datGeneric, family=binomial("logit"))
6788
       Anova(rlogG ti 4, type="III")
6789
       summary(rlogG ti 4)
6790
6791
       mgti 4 s <- emmeans(rlogG ti 4,~studyarm|edhi,type = "response")
6792
       mgti 4 s
6793
       confint(pairs(mgti 4 s,reverse = TRUE))
6794
6795
       mgti_4_e <- emmeans(rlogG_ti_4, ~ edhi|studyarm, type = "response")</pre>
       confint(pairs(mgti_4_e,reverse = TRUE))
6796
6797
6798
6799
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
6800
6801
      rlogG ti 5 <-
6802
         glm (Htrustinfo
                         ~ studyarm*edhi +
6803
               mean indivhorz +
6804
               mean indivvertical +
6805
               mean collhorz +
6806
               mean collvertical +
6807
               bornincanada +
6808
               language 1 +
6809
               language 2 +
6810
               Asian_group +
6811
               White_group +
6812
               disability any +
6813
               genderidentity +
6814
               income +
6815
               age,
6816
             data = datGeneric, family=binomial("logit")
6817
         )
6818
       Anova(rlogG_ti_5, type = "III")
6819
       summary(rlogG ti 5)
```

```
6820
6821
      mgti 5 s <- emmeans(rlogG ti 5,~studyarm|edhi,type = "response")
6822
      mgti 5 s
6823
      confint(pairs(mgti 5 s, reverse = TRUE))
6824
6825
      mgti 5 e <- emmeans(rlogG ti 5, ~ edhi|studyarm, type = "response")
6826
      confint(pairs(mgti 5 e, reverse = TRUE))
6827
6828
      # Now running models on imputed data.
6829
     imprlogG ti 1 <-
6830
         with (data = datGenericImputed,
              exp = glm(relevel(Htrustinfo,ref="No") ~ studyarm,family = binomial("logit")))
6831
       combineimprlogG ti 1 <- pool(imprlogG_ti_1)</pre>
6832
6833
       summary(combineimprlogG ti 1)
6834
6835
6836
       #### ++ Measles ####
6837
6838
       #### + Model 1: Check for direct effects of factors without any covariates ####
6839
6840
      options(contrasts=c("contr.sum", "contr.poly"))
6841
      rlogM ti 1 <- glm(Htrustinfo ~ studyarm, data = datMeasles, family=binomial("logit"))
6842
      Anova(rlogM ti 1, type="III")
6843
      summary(rlogM ti 1)
6844
6845
      mmti 1 <- emmeans(rlogM ti 1,~studyarm,type = "response") #proportions
      mmti 1
6846
6847
      confint(pairs(mmti 1, reverse = TRUE)) #Odds ratios
6848
      pairs (mmti 1, reverse = TRUE, type = "response")
6849
6850
      # Model 2: Check for direct effects of factors with adjustment for other covariates
6851
      rlogM ti 2 <-
6852
         glm (Htrustinfo ~ studyarm +
6853
               mean indivhorz +
6854
               mean indivvertical +
6855
               mean collhorz +
6856
               mean collvertical +
6857
               bornincanada +
6858
               language_1 +
6859
               language 2 +
6860
              Asian group +
6861
              White group +
6862
              disability any +
6863
               genderidentity +
6864
               income +
6865
               edhi +
6866
               age,
6867
             data = datMeasles, family=binomial("logit")
6868
         )
6869
      Anova(rlogM_ti_2, type = "III")
6870
      summary(rlogM ti 2)
6871
6872
      mmti 2 <- emmeans(rlogM ti 2,~studyarm,type = "response")</pre>
6873
6874
      confint(pairs(mmti 2, reverse = TRUE))
6875
       pairs (mmti 2, reverse = TRUE, type = "response")
6876
6877
      # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
6878
       rlogM_ti_3 <-</pre>
6879
         glm(Htrustinfo ~
6880
               studyarm * mean indivhorz +
6881
               studyarm * mean indivvertical +
6882
              studyarm * mean collhorz +
6883
              studyarm * mean collvertical +
6884
              bornincanada +
6885
               language 1 +
               language 2 +
6886
6887
               Asian group +
```

```
6888
               White group +
6889
               disability any +
6890
               genderidentity +
6891
               income +
6892
               edhi +
6893
               age,
6894
             data = datMeasles, family=binomial("logit")
6895
         )
6896
      Anova(rlogM ti 3, type = "III")
6897
       summary(rlogM ti 3)
6898
       #No interaction with moderator to interpret
6899
6900
6901
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
6902
6903
       rlogM ti 4 <- glm(Htrustinfo ~ studyarm * edhi, data =</pre>
       datMeasles, family=binomial("logit"))
6904
       Anova(rlogM ti 4, type="III")
6905
      summary(rlogM ti 4)
6906
6907
      mmti 4 s <- emmeans(rlogM ti 4,~studyarm|edhi,type = "response")
6908
      mmti 4 s
6909
       confint(pairs(mmti 4 s, reverse = TRUE))
6910
6911
       mmti 4 e <- emmeans(rlogM ti 4, ~ edhi|studyarm, type = "response")
6912
       confint(pairs(mmti 4 e, reverse = TRUE))
6913
6914
       \# Model 5: Check for interaction viz*edhi with adjustment for other covariates
6915
6916
6917
      rlogM ti 5 <-
6918
         glm (Htrustinfo
                         ~ studyarm*edhi +
6919
               mean indivhorz +
6920
               mean indivvertical +
6921
               mean collhorz +
6922
               mean collvertical +
6923
               bornincanada +
6924
               language 1 +
6925
               language_2 +
6926
               Asian group +
6927
               White group +
6928
               disability any +
6929
               genderidentity +
6930
               income +
6931
               age,
             data = datMeasles,family=binomial("logit")
6932
6933
6934
      Anova(rlogM ti 5, type = "III")
6935
      summary(rlogM ti 5)
6936
6937
      mmti 5 s <- emmeans(rlogM ti 5,~studyarm|edhi,type = "response")
6938
      mmti 5 s
6939
      confint(pairs(mmti 5 s, reverse = TRUE))
6940
6941
      mmti 5 e <- emmeans(rlogM ti 5, ~ edhi|studyarm, type = "response")
6942
      confint(pairs(mmti 5 e, reverse = TRUE))
6943
6944
       # Now running models on imputed data.
6945
       #CHANGELOG ASJ: No missing data for htrustinfo in measles, no model with imputation
       performed, 21-09-20.
6946
6947
6948
6949
       #### ++ Flu ####
6950
6951
       #### + Model 1: Check for direct effects of factors without any covariates ####
6952
6953
       options(contrasts=c("contr.sum", "contr.poly"))
6954
       rlogF ti 1 <- glm(Htrustinfo ~ studyarm, data = datFlu,family=binomial("logit"))</pre>
```

```
6955
       Anova(rlogF ti 1, type="III")
6956
       summary(rlogF ti 1)
6957
6958
       mfti 1 <- emmeans (rlogF ti 1,~studyarm, type = "response") #proportions
6959
6960
      confint(pairs(mfti 1, reverse = TRUE)) #Odds ratios
6961
      pairs (mfti 1, reverse = TRUE, type="response")
6962
6963
     # Model 2: Check for direct effects of factors with adjustment for other covariates
6964 rlogF ti 2 <-
6965
         glm(Htrustinfo ~ studyarm +
6966
               mean indivhorz +
               mean indivvertical +
6967
6968
               mean collhorz +
6969
               mean collvertical +
6970
               bornincanada +
6971
               language_1 +
6972
               language 2 +
6973
               Asian group +
6974
               White group +
6975
               disability any +
6976
               genderidentity +
6977
               income +
6978
               edhi +
6979
               age,
             data = datFlu, family=binomial("logit")
6980
6981
         )
6982
      Anova(rlogF_ti_2, type = "III")
6983
      summary(rlogF ti 2)
6984
6985
      mfti 2 <- emmeans(rlogF ti 2,~studyarm,type = "response")</pre>
6986
      mfti 2
6987
      confint(pairs(mfti 2, reverse = TRUE))
6988
       pairs (mfti 2, reverse = TRUE, type="response")
6989
6990
6991
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
6992
       rlogF_ti_3 <-</pre>
6993
         glm(Htrustinfo ~
6994
               studyarm * mean indivhorz +
6995
               studyarm * mean indivvertical +
6996
               studyarm * mean collhorz +
6997
               studyarm * mean collvertical +
6998
               bornincanada +
6999
               language 1 +
7000
               language 2 +
7001
               Asian group +
7002
               White_group +
7003
               disability any +
7004
               genderidentity +
7005
               income +
7006
               edhi +
7007
7008
             data = datFlu, family=binomial("logit")
7009
         )
7010
       Anova(rlogF_ti_3, type = "III")
7011
       summary(rlogF ti 3)
7012
7013
       #No interaction with moderators to interpret
7014
7015
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
7016
7017
       rlogF ti 4 <- glm(Htrustinfo ~ studyarm * edhi, data = datFlu, family=binomial("logit"))</pre>
7018
       Anova(rlogF ti 4, type="III")
7019
       summary(rlogF ti 4)
7020
7021
       mfti_4_s <- emmeans(rlogF_ti_4,~studyarm|edhi,type = "response")</pre>
7022
       mfti 4 s
```

```
7023
       confint(pairs(mfti 4 s,reverse = TRUE))
7024
7025
       mfti 4 e <- emmeans(rlogF ti 4, ~ edhi|studyarm, type = "response")
7026
       confint(pairs(mfti 4 e, reverse = TRUE))
7027
7028
7029
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
7030
7031
     rlogF ti 5 <-
7032
         glm (Htrustinfo
                         ~ studyarm*edhi +
7033
               mean indivhorz +
7034
               mean indivvertical +
7035
              mean collhorz +
7036
               mean collvertical +
7037
               bornincanada +
7038
               language 1 +
7039
               language_2 +
7040
               Asian group +
7041
               White group +
7042
               disability any +
7043
               genderidentity +
7044
               income +
7045
               age,
             data = datFlu, family=binomial("logit")
7046
7047
         )
7048
       Anova(rlogF ti 5, type = "III")
7049
       summary(rlogF ti 5)
7050
7051
      mfti 5 s <- emmeans(rlogF ti 5,~studyarm|edhi,type = "response")</pre>
7052
      mfti 5 s
7053
      confint(pairs(mfti 5 s, reverse = TRUE))
7054
7055
      mfti 5 e <- emmeans(rlogF ti 5, ~ edhi|studyarm, type = "response")
7056
      confint(pairs(mfti 5 e, reverse = TRUE))
7057
7058
       # Now running models on imputed data.
7059
       #CHANGELOG ASJ: No missing data for htrustinfo in flu, no model with imputation
       performed, 21-09-20.
7060
7061
7062
7063
       #### +++ Logistic regression for C5 Confidence ####
7064
7065
       #Create relevel before model to avoid problems with pairs function.
7066
       datGeneric$mean C5 conf2 <- relevel(as.factor(datGeneric$mean C5 conf2), ref = "0")
7067
       datMeasles$mean C5 conf2 <- relevel(as.factor(datMeasles$mean C5 conf2),ref = "0")</pre>
       datFlu$mean C5 conf2 <- relevel(as.factor(datFlu$mean C5 conf2), ref = "0")
7068
7069
7070
       #### ++ Generic ####
7071
7072
       #### + Model 1: Check for direct effects of factors without any covariates ####
7073
       options(contrasts=c("contr.sum", "contr.poly"))
7074
7075
       rlogG C5conf 1 <- glm(mean C5 conf2 ~ studyarm, data =</pre>
       datGeneric, family=binomial("logit"))
7076
       Anova(rlogG C5conf 1, type="III")
7077
       summary(rlogG C5conf 1)
7078
7079
       mgC5conf <- emmeans(rlogG C5conf 1,~studyarm,type = "response") #proportions
7080
7081
      confint(pairs(mgC5conf,reverse = TRUE)) #Odds ratios
7082
7083
       # Model 2: Check for direct effects of factors with adjustment for other covariates
7084
      rlogG C5conf 2 <-
7085
         glm (mean C5 conf2 ~ studyarm +
7086
               mean indivhorz +
7087
               mean_indivvertical +
7088
               mean collhorz +
7089
               mean collvertical +
```

```
bornincanada +
7090
7091
               language 1 +
7092
               language 2 +
7093
               Asian group +
7094
               White group +
7095
              disability any +
7096
               genderidentity +
7097
              income +
               edhi +
7098
7099
               age,
7100
             data = datGeneric, family=binomial("logit")
7101
         )
7102
       Anova(rlogG C5conf 2, type = "III")
7103
       summary(rlogG C5conf 2)
7104
7105
      mgC5conf 2 <- emmeans(rlogG C5conf 2,~studyarm,type = "response")</pre>
7106
       mgC5conf 2
7107
       confint(pairs(mgC5conf 2, reverse = TRUE))
7108
7109
7110
     # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
7111
      rlogG C5conf 3 <-
7112
         glm(mean C5 conf2 ~
7113
               studyarm * mean indivhorz +
7114
               studyarm * mean indivvertical +
7115
               studyarm * mean collhorz +
               studyarm * mean_collvertical +
7116
7117
              bornincanada +
7118
              language 1 +
7119
              language 2 +
7120
              Asian group +
7121
              White group +
7122
              disability any +
7123
               genderidentity +
7124
               income +
7125
               edhi +
7126
               age,
7127
             data = datGeneric, family=binomial("logit")
7128
         )
7129
       Anova(rlogG C5conf 3, type = "III")
7130
       summary(rlogG C5conf 3)
7131
7132
       #No interaction with moderator to interpret
7133
7134
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
7135
7136
       rlogG C5conf 4 <- glm(mean C5 conf2 ~ studyarm * edhi, data =</pre>
       datGeneric, family=binomial("logit"))
7137
       Anova(rlogG_C5conf_4,type="III")
7138
       summary(rlogG C5conf 4)
7139
7140
      mgC5conf 4 s <- emmeans(rlogG C5conf 4,~studyarm|edhi,type = "response")
7141
      mgC5conf 4 s
7142
       confint(pairs(mgC5conf 4 s,reverse = TRUE))
7143
7144
       mgC5conf 4 e <- emmeans(rlogG C5conf 4, ~ edhi|studyarm, type = "response")
7145
       confint(pairs(mgC5conf 4 e,reverse = TRUE))
7146
7147
7148
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
7149
7150
       rlogG C5conf 5 <-
7151
         glm (mean C5 conf2
                             ~ studyarm*edhi +
7152
               mean indivhorz +
7153
               mean indivvertical +
7154
               mean collhorz +
7155
               mean collvertical +
7156
               bornincanada +
```

```
7157
               language 1 +
7158
               language 2 +
7159
               Asian group +
7160
               White group +
7161
               disability any +
7162
               genderidentity +
7163
               income +
7164
               age,
7165
             data = datGeneric, family=binomial("logit")
7166
         )
7167
       Anova(rlogG C5conf 5, type = "III")
7168
       summary(rlogG C5conf 5)
7169
7170
       mgC5conf 5 s <- emmeans(rlogG C5conf 5,~studyarm|edhi,type = "response")
7171
       mgC5conf 5 s
7172
       confint(pairs(mgC5conf 5 s,reverse = TRUE))
7173
7174
       mgC5conf 5 e <- emmeans(rlogG C5conf 5, ~ edhi|studyarm, type = "response")
       confint(pairs(mgC5conf 5 e,reverse = TRUE))
7175
7176
7177
       # Now running models on imputed data.
7178
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
7179
7180
7181
7182
       #### ++ Measles ####
7183
7184
       #### + Model 1: Check for direct effects of factors without any covariates ####
7185
      options(contrasts=c("contr.sum", "contr.poly"))
7186
7187
      rlogM C5conf 1 <- glm(mean C5 conf2 ~ studyarm, data =</pre>
       datMeasles, family=binomial("logit"))
7188
       Anova(rlogM C5conf 1, type="III")
7189
       summary(rlogM C5conf 1)
7190
7191
       mmC5conf <- emmeans(rlogM C5conf 1,~studyarm,type = "response") #proportions
7192
       mmC5conf
7193
       confint(pairs(mmC5conf,reverse = TRUE)) #Odds ratios
7194
7195
       # Model 2: Check for direct effects of factors with adjustment for other covariates
7196
       rlogM C5conf 2 <-
7197
         glm(mean C5 conf2 ~ studyarm +
7198
               mean indivhorz +
7199
               mean indivvertical +
7200
               mean collhorz +
7201
               mean collvertical +
7202
               bornincanada +
7203
               language 1 +
7204
               language_2 +
7205
               Asian group +
7206
              White group +
7207
              disability any +
7208
               genderidentity +
7209
               income +
7210
               edhi +
7211
7212
             data = datMeasles, family=binomial("logit")
7213
7214
       Anova(rlogM C5conf 2, type = "III")
7215
       summary(rlogM C5conf 2)
7216
7217
       mmC5conf 2 <- emmeans(rlogM C5conf 2,~studyarm,type = "response")
7218
       mmC5conf 2
7219
       confint(pairs(mmC5conf 2, reverse = TRUE))
7220
7221
7222
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
7223
       rlogM_C5conf_3 <-</pre>
```

```
7224
         glm (mean C5 conf2 ~
7225
              studyarm * mean indivhorz +
               studyarm * mean indivvertical +
7226
7227
               studyarm * mean collhorz +
7228
               studyarm * mean collvertical +
7229
              bornincanada +
7230
               language 1 +
7231
               language 2 +
7232
               Asian group +
7233
               White group +
7234
               disability any +
7235
               genderidentity +
7236
               income +
7237
               edhi +
7238
               age,
7239
             data = datMeasles, family=binomial("logit")
7240
         )
7241
       Anova(rlogM C5conf 3, type = "III")
7242
       summary(rlogM C5conf 3)
7243
7244
       #No interaction with moderator to interpret
7245
7246
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
7247
7248
       rlogM C5conf 4 <- glm(mean C5 conf2 ~ studyarm * edhi, data =</pre>
       datMeasles, family=binomial("logit"))
7249
       Anova(rlogM C5conf 4, type="III")
7250
       summary(rlogM C5conf 4)
7251
7252
      mmC5conf 4 s <- emmeans(rlogM C5conf 4,~studyarm|edhi,type = "response")
7253
      mmC5conf 4 s
7254
      confint(pairs(mmC5conf 4 s,reverse = TRUE))
7255
7256
      mmC5conf 4 e <- emmeans(rlogM C5conf 4, ~ edhi|studyarm, type = "response")
7257
       confint(pairs(mmC5conf 4 e, reverse = TRUE))
7258
7259
7260
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
7261
7262
       rlogM C5conf 5 <-
7263
         glm (mean C5 conf2
                             ~ studyarm*edhi +
7264
               mean indivhorz +
7265
               mean indivvertical +
7266
               mean collhorz +
7267
               mean collvertical +
7268
               bornincanada +
7269
               language 1 +
7270
               language 2 +
7271
               Asian group +
7272
               White_group +
7273
               disability any +
7274
               genderidentity +
7275
               income +
7276
7277
             data = datMeasles, family=binomial("logit")
7278
         )
7279
       Anova(rlogM C5conf 5, type = "III")
7280
       summary(rlogM_C5conf 5)
7281
7282
       mmC5conf 5 s <- emmeans(rlogM C5conf 5,~studyarm|edhi,type = "response")
7283
       mmC5conf_5_s
7284
       confint (pairs (mmC5conf 5 s, reverse = TRUE))
7285
7286
       mmC5conf 5 e <- emmeans(rlogM C5conf 5, ~ edhi|studyarm, type = "response")
7287
       confint(pairs(mmC5conf 5 e, reverse = TRUE))
7288
7289
       # Now running models on imputed data.
7290
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
7291
```

```
7292
7293
       #### ++ Flu ####
7294
7295
       #### + Model 1: Check for direct effects of factors without any covariates ####
7296
7297
       options(contrasts=c("contr.sum", "contr.poly"))
7298
       rlogF C5conf 1 <- glm(mean C5 conf2 ~ studyarm, data = datFlu,family=binomial("logit"))</pre>
7299
       Anova(rlogF C5conf 1, type="III")
7300
       summary(rlogF C5conf 1)
7301
7302
      mfC5conf 1 <- emmeans(rlogF C5conf 1,~studyarm,type = "response") #proportions
7303
      mfC5conf 1
7304
       confint(pairs(mfC5conf 1, reverse = TRUE)) #Odds ratios
7305
7306
       # Model 2: Check for direct effects of factors with adjustment for other covariates
       rlogF C5conf 2 <-
7307
7308
         glm(mean C5 conf2 ~ studyarm +
7309
               mean indivhorz +
7310
               mean indivvertical +
7311
               mean collhorz +
7312
               mean collvertical +
7313
               bornincanada +
7314
               language 1 +
7315
               language 2 +
7316
               Asian group +
7317
               White group +
7318
               disability any +
7319
               genderidentity +
7320
               income +
7321
               edhi +
7322
               age,
7323
             data = datFlu, family=binomial("logit")
7324
         )
7325
       Anova(rlogF C5conf 2, type = "III")
7326
       summary(rlogF C5conf 2)
7327
7328
       mfC5conf 2 <- emmeans(rlogF C5conf 2,~studyarm,type = "response")
7329
       mfC5conf 2
7330
       confint(pairs(mfC5conf 2, reverse = TRUE))
7331
7332
7333
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
7334
       rlogF C5conf 3 <-
7335
         glm (mean C5 conf2 ~
7336
               studyarm * mean indivhorz +
7337
               studyarm * mean indivvertical +
7338
               studyarm * mean collhorz +
7339
               studyarm * mean_collvertical +
7340
               bornincanada +
7341
               language 1 +
7342
               language 2 +
7343
               Asian group +
7344
               White group +
7345
               disability any +
7346
               genderidentity +
7347
               income +
7348
               edhi +
7349
               age,
7350
             data = datFlu, family=binomial("logit")
7351
         )
7352
       Anova(rlogF C5conf 3, type = "III")
7353
       summary(rlogF C5conf 3)
7354
7355
       emmip(rlogF C5conf 3, studyarm ~ mean indivvertical, cov.reduce = range, type =
       "response")
7356
7357
7358
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
```

```
7359
7360
       rlogF C5conf 4 <- glm(mean C5 conf2 ~ studyarm * edhi, data =</pre>
       datFlu, family=binomial("logit"))
7361
       Anova(rlogF_C5conf 4,type="III")
7362
       summary(rlogF C5conf 4)
7363
7364
      mfC5conf 4 s <- emmeans(rlogF C5conf 4,~studyarm|edhi,type = "response")
7365
      mfC5conf 4 s
7366
      confint(pairs(mfC5conf 4 s,reverse = TRUE))
7367
7368
       mfC5conf 4 e <- emmeans(rlogF C5conf 4, ~ edhi|studyarm, type = "response")
7369
       confint(pairs(mfC5conf 4 e, reverse = TRUE))
7370
7371
7372
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
7373
7374
       rlogF C5conf 5 <-
7375
         glm (mean C5 conf2
                            ~ studyarm*edhi +
7376
               mean indivhorz +
7377
               mean indivvertical +
7378
              mean collhorz +
7379
              mean collvertical +
7380
              bornincanada +
7381
               language 1 +
7382
               language 2 +
7383
               Asian group +
7384
               White group +
7385
              disability any +
7386
               genderidentity +
7387
               income +
7388
               age,
7389
             data = datFlu, family=binomial("logit")
7390
         )
7391
       Anova(rlogF C5conf 5, type = "III")
7392
       summary(rlogF C5conf 5)
7393
7394
       mfC5conf 5 s <- emmeans(rlogF C5conf 5,~studyarm|edhi,type = "response")
7395
       mfC5conf 5 s
7396
       confint(pairs(mfC5conf 5 s,reverse = TRUE))
7397
7398
       mfC5conf 5 e <- emmeans(rlogF C5conf 5, ~ edhi|studyarm, type = "response")
7399
       confint (pairs (mfC5conf 5 e, reverse = TRUE))
7400
7401
       # Now running models on imputed data.
7402
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
7403
7404
       #### +++ Logistic regression for C5 Complacency ####
7405
7406
       #Create relevel before model to avoid problems with pairs function.
       datGeneric$mean_C5_comp2 <- relevel(as.factor(datGeneric$mean C5 comp2),ref = "0")</pre>
7407
7408
       datMeasles$mean C5 comp2 <- relevel(as.factor(datMeasles$mean C5 comp2),ref = "0")
7409
       datFlu$mean C5 comp2 <- relevel(as.factor(datFlu$mean C5 comp2), ref = "0")
7410
7411
       #### ++ Generic ####
7412
7413
       #### + Model 1: Check for direct effects of factors without any covariates ####
7414
       options(contrasts=c("contr.sum", "contr.poly"))
7415
7416
       rlogG C5comp 1 <- glm(mean C5 comp2 ~ studyarm, data =</pre>
       datGeneric, family=binomial("logit"))
7417
       Anova(rlogG_C5comp_1, type="III")
7418
       summary(rlogG C5comp 1)
7419
7420
      mgC5comp 1 <- emmeans(rlogG C5comp 1,~studyarm,type = "response") #proportions
7421
      mgC5comp 1
7422
       confint(pairs(mgC5comp 1, reverse = TRUE)) #Odds ratios
7423
       pairs (mgC5comp_1, reverse = TRUE)
7424
7425
       # Model 2: Check for direct effects of factors with adjustment for other covariates
```

```
7426
      rlogG C5comp 2 <-
7427
         glm(mean C5 comp2 ~ studyarm +
7428
               mean indivhorz +
7429
               mean indivvertical +
7430
               mean collhorz +
7431
               mean_collvertical +
7432
               bornincanada +
7433
               language 1 +
7434
               language 2 +
7435
               Asian group +
7436
               White group +
7437
               disability any +
7438
               genderidentity +
7439
               income +
7440
               edhi +
7441
               age,
7442
             data = datGeneric, family=binomial("logit")
7443
         )
7444
       Anova(rlogG C5comp 2, type = "III")
7445
       summary(rlogG C5comp 2)
7446
7447
       mgC5comp 2 <- emmeans(rlogG C5comp 2,~studyarm,type = "response")
7448
       mqC5comp 2
7449
       confint(pairs(mgC5comp 2, reverse = TRUE))
7450
       pairs (mgC5comp 2, reverse = TRUE)
7451
7452
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
7453
      rlogG C5comp 3 <-
7454
         glm (mean C5 comp2
7455
               studyarm * mean indivhorz +
7456
               studyarm * mean indivvertical +
7457
               studyarm * mean collhorz +
               studyarm * mean collvertical +
7458
7459
               bornincanada +
7460
               language 1 +
7461
               language 2 +
7462
               Asian group +
7463
               White_group +
7464
               disability any +
7465
               genderidentity +
7466
               income +
7467
               edhi +
7468
               age,
7469
             data = datGeneric, family=binomial("logit")
7470
         )
7471
       Anova(rlogG C5comp 3, type = "III")
7472
       summary(rlogG C5comp 3)
7473
7474
       #No interaction with moderator to interpret
7475
7476
       #### + Model 4: Check for interaction viz*edhi without any covariates
7477
7478
       rlogG C5comp 4 <- glm (mean C5 comp2 ~ studyarm * edhi, data =</pre>
       datGeneric, family=binomial("logit"))
7479
       Anova(rlogG C5comp 4, type="III")
7480
       summary(rlogG C5comp 4)
7481
7482
       mgC5comp 4 s <- emmeans(rlogG C5comp 4,~studyarm|edhi,type = "response")
7483
       mgC5comp_4_s
7484
       confint(pairs(mgC5comp_4_s,reverse = TRUE))
7485
       pairs (mgC5comp 4 s,reverse = TRUE)
7486
7487
       mgC5comp 4 e <- emmeans(rlogG C5comp 4, ~ edhi|studyarm, type = "response")
7488
       confint(pairs(mgC5comp 4 e,reverse = TRUE))
7489
       pairs (mgC5comp 4 e, reverse = TRUE)
7490
7491
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
7492
```

```
7493
       rlogG C5comp 5 <-
7494
         glm (mean C5 comp2 ~ studyarm*edhi +
7495
               mean indivhorz +
7496
               mean indivvertical +
7497
               mean collhorz +
7498
               mean_collvertical +
               bornincanada +
7499
7500
               language 1 +
7501
               language 2 +
7502
               Asian group +
7503
               White group +
7504
               disability any +
7505
               genderidentity +
7506
               income +
7507
               age,
7508
             data = datGeneric, family=binomial("logit")
7509
         )
7510
       Anova(rlogG C5comp 5, type = "III")
7511
       summary(rlogG C5comp 5)
7512
7513
       mgC5comp 5 s <- emmeans(rlogG C5comp 5,~studyarm|edhi,type = "response")
7514
       mqC5comp 5 s
7515
       confint(pairs(mgC5comp 5 s,reverse = TRUE))
7516
7517
       mgC5comp 5 e <- emmeans(rlogG C5comp 5, ~ edhi|studyarm, type = "response")
7518
       confint(pairs(mgC5comp 5 e,reverse = TRUE))
7519
7520
       # Now running models on imputed data.
7521
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
7522
7523
7524
       #### ++ Measles ####
7525
7526
       #### + Model 1: Check for direct effects of factors without any covariates ####
7527
7528
       options(contrasts=c("contr.sum", "contr.poly"))
7529
       rlogM C5comp 1 <- glm(mean C5 comp2 ~ studyarm, data =</pre>
       datMeasles, family=binomial("logit"))
7530
       Anova(rlogM C5comp 1, type="III")
7531
       summary(rlogM C5comp 1)
7532
7533
       mmC5comp 1 <- emmeans(rlogM C5comp 1,~studyarm,type = "response") #proportions
7534
7535
       confint(pairs(mmC5comp 1, reverse = TRUE)) #Odds ratios
7536
7537
       # Model 2: Check for direct effects of factors with adjustment for other covariates
7538
       rlogM C5comp 2 <-
7539
         glm(mean C5 comp2 ~ studyarm +
               mean_indivhorz +
7540
7541
               mean indivvertical +
               mean collhorz +
7542
7543
               mean collvertical +
7544
               bornincanada +
7545
               language 1 +
7546
               language 2 +
7547
               Asian_group +
7548
               White group +
7549
               disability any +
7550
               genderidentity +
7551
               income +
7552
               edhi +
7553
               age,
7554
             data = datMeasles, family=binomial("logit")
7555
7556
       Anova(rlogM C5comp 2, type = "III")
7557
       summary(rlogM C5comp 2)
7558
7559
       mmC5comp 2 <- emmeans(rlogM C5comp 2,~studyarm,type = "response")
7560
       mmC5comp 2
```

```
7561
       confint(pairs(mmC5comp 2, reverse = TRUE))
7562
7563
7564
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
7565
      rlogM_C5comp_3 <-
7566
         glm (mean C5 comp2 ~
7567
               studyarm * mean indivhorz +
7568
               studyarm * mean indivvertical +
7569
               studyarm * mean collhorz +
               studyarm * mean collvertical +
7570
7571
               bornincanada +
7572
               language 1 +
7573
               language 2 +
7574
               Asian group +
7575
               White group +
7576
               disability_any +
7577
               genderidentity +
7578
               income +
7579
               edhi +
7580
               age,
7581
             data = datMeasles, family=binomial("logit")
7582
         )
       Anova(rlogM_C5comp_3, type = "III")
7583
7584
       summary(rlogM C5comp 3)
7585
7586
       #No interaction with moderator to interpret
7587
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
7588
7589
7590
       rlogM C5comp 4 <- glm(mean C5 comp2 ~ studyarm * edhi, data =</pre>
       datMeasles, family=binomial("logit"))
7591
       Anova(rlogM C5comp 4, type="III")
7592
       summary(rlogM C5comp 4)
7593
7594
       mmC5comp 4 s <- emmeans(rlogM C5comp 4,~studyarm|edhi,type = "response")
7595
       mmC5comp 4 s
7596
       confint(pairs(mmC5comp 4 s,reverse = TRUE))
7597
7598
       mmC5comp 4 e <- emmeans(rlogM C5comp 4, ~ edhi|studyarm, type = "response")
7599
       confint(pairs(mmC5comp 4 e, reverse = TRUE))
7600
7601
7602
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
7603
7604
      rlogM C5comp 5 <-
7605
         glm (mean C5 comp2 ~ studyarm*edhi +
7606
               mean indivhorz +
7607
               mean_indivvertical +
7608
              mean collhorz +
              mean collvertical +
7609
7610
              bornincanada +
7611
              language 1 +
7612
              language 2 +
7613
              Asian group +
7614
               White_group +
7615
               disability any +
7616
               genderidentity +
7617
               income +
7618
               age,
7619
             data = datMeasles, family=binomial("logit")
7620
7621
       Anova(rlogM C5comp 5, type = "III")
7622
       summary(rlogM C5comp 5)
7623
7624
       mmC5comp 5 s <- emmeans(rlogM C5comp 5,~studyarm|edhi,type = "response")
7625
       mmC5comp 5 s
7626
       confint(pairs(mmC5comp_5_s,reverse = TRUE))
7627
```

```
7628
       mmC5comp 5 e <- emmeans(rlogM C5comp 5, ~ edhi|studyarm, type = "response")
7629
       confint(pairs(mmC5comp 5 e, reverse = TRUE))
7630
7631
       # Now running models on imputed data.
7632
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
7633
7634
7635
       #### ++ Flu ####
7636
7637
       #### + Model 1: Check for direct effects of factors without any covariates ####
7638
7639
       options(contrasts=c("contr.sum", "contr.poly"))
7640
       rlogF C5comp 1 <- glm(mean C5 comp2 ~ studyarm, data = datFlu,family=binomial("logit"))</pre>
7641
       Anova(rlogF C5comp 1,type="III")
7642
       summary(rlogF C5comp 1)
7643
7644
      mfC5comp 1 <- emmeans(rlogF C5comp 1,~studyarm,type = "response") #proportions
7645
      mfC5comp 1
7646
      confint(pairs(mfC5comp 1, reverse = TRUE)) #Odds ratios
7647
      pairs (mfC5comp 1, reverse = TRUE)
7648
7649
       # Model 2: Check for direct effects of factors with adjustment for other covariates
7650
      rlogF C5comp 2 <-
7651
         glm(mean C5 comp2 ~ studyarm +
7652
               mean indivhorz +
7653
               mean indivvertical +
7654
              mean collhorz +
7655
              mean_collvertical +
7656
              bornincanada +
7657
              language 1 +
7658
              language 2 +
7659
              Asian group +
7660
              White group +
7661
              disability any +
7662
               genderidentity +
7663
               income +
7664
               edhi +
7665
               age,
7666
             data = datFlu, family=binomial("logit")
7667
         )
7668
       Anova(rlogF C5comp 2, type = "III")
7669
       summary(rlogF C5comp 2)
7670
7671
       mfC5comp 2 <- emmeans(rlogF C5comp 2,~studyarm,type = "response")</pre>
7672
       mfC5comp 2
7673
       confint (pairs (mfC5comp 2, reverse = TRUE))
7674
      pairs (mfC5comp 2, reverse = TRUE)
7675
7676
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
7677
      rlogF C5comp 3 <-
7678
        glm (mean C5 comp2 ~
7679
               studyarm * mean indivhorz +
7680
               studyarm * mean indivvertical +
7681
               studyarm * mean collhorz +
7682
               studyarm * mean collvertical +
7683
               bornincanada +
7684
               language 1 +
7685
               language 2 +
7686
               Asian_group +
7687
              White_group +
7688
              disability any +
7689
              genderidentity +
7690
              income +
7691
               edhi +
7692
7693
             data = datFlu, family=binomial("logit")
7694
7695
       Anova(rlogF C5comp 3, type = "III")
```

```
7696
       summary(rlogF C5comp 3)
7697
7698
       emmip(rlogF C5comp 3, studyarm ~ mean collhorz, cov.reduce = range, type = "response")
7699
7700
7701
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
7702
7703
       rlogF C5comp 4 <- glm (mean C5 comp2 ~ studyarm * edhi, data =</pre>
       datFlu, family=binomial("logit"))
7704
       Anova(rlogF C5comp 4, type="III")
7705
       summary(rlogF C5comp 4)
7706
7707
      mfC5comp 4 s <- emmeans(rlogF C5comp 4,~studyarm|edhi,type = "response")
7708
       mfC5comp 4 s
7709
       confint(pairs(mfC5comp 4 s,reverse = TRUE))
7710
7711
       mfC5comp_4_e <- emmeans(rlogF_C5comp_4, ~ edhi|studyarm, type = "response")</pre>
7712
       confint(pairs(mfC5comp 4 e,reverse = TRUE))
7713
7714
7715
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
7716
7717
      rlogF C5comp 5 <-
7718
         glm (mean C5 comp2 ~ studyarm*edhi +
7719
               mean indivhorz +
7720
               mean indivvertical +
7721
               mean collhorz +
7722
              mean collvertical +
7723
              bornincanada +
7724
              language 1 +
7725
              language 2 +
7726
              Asian group +
7727
              White group +
7728
              disability any +
7729
               genderidentity +
7730
               income +
7731
7732
             data = datFlu, family=binomial("logit")
7733
         )
7734
       Anova(rlogF C5comp 5, type = "III")
7735
       summary(rlogF C5comp 5)
7736
7737
      mfC5comp 5 s <- emmeans(rlogF C5comp 5,~studyarm|edhi,type = "response")
7738
      mfC5comp 5 s
7739
       confint (pairs (mfC5comp 5 s, reverse = TRUE))
7740
7741
       mfC5comp 5 e <- emmeans(rlogF C5comp 5, ~ edhi|studyarm, type = "response")
7742
       confint(pairs(mfC5comp 5 e,reverse = TRUE))
7743
7744
       # Now running models on imputed data.
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
7745
7746
7747
7748
       #### +++ Logistic regression for C5 Constraints ####
7749
7750
       #Create relevel before model to avoid problems with pairs function.
7751
       datGeneric$mean C5 cons2 <- relevel(as.factor(datGeneric$mean C5 cons2),ref = "0")
7752
       datMeasles$mean C5 cons2 <- relevel(as.factor(datMeasles$mean C5 cons2),ref = "0")
7753
       datFlu$mean C5 cons2 <- relevel(as.factor(datFlu$mean C5 cons2), ref = "0")
7754
7755
       #### ++ Generic ####
7756
7757
       #### + Model 1: Check for direct effects of factors without any covariates ####
7758
7759
       options(contrasts=c("contr.sum", "contr.poly"))
7760
       rlogG C5cons 1 <- glm(mean C5 cons2 ~ studyarm, data =</pre>
       datGeneric, family=binomial("logit"))
7761
       Anova(rlogG C5cons 1,type="III")
7762
       summary(rlogG C5cons 1)
```

```
7763
7764
       mgC5cons 1 <- emmeans(rlogG C5cons 1,~studyarm,type = "response") #proportions
7765
       mgC5cons 1
7766
       confint(pairs(mgC5cons 1, reverse = TRUE)) #Odds ratios
7767
       pairs (mgC5cons 1, reverse = TRUE)
7768
7769
      # Model 2: Check for direct effects of factors with adjustment for other covariates
7770
      rlogG C5cons 2 <-
7771
         glm(mean C5 cons2 ~ studyarm +
7772
               mean indivhorz +
7773
               mean indivvertical +
7774
               mean collhorz +
7775
               mean collvertical +
7776
               bornincanada +
7777
               language 1 +
7778
               language 2 +
7779
               Asian_group +
7780
               White group +
7781
               disability any +
7782
               genderidentity +
7783
               income +
7784
               edhi +
7785
               age,
7786
             data = datGeneric, family=binomial("logit") )
7787
       Anova(rlogG C5cons 2, type = "III")
7788
       summary(rlogG C5cons 2)
7789
7790
      mgC5cons 2 <- emmeans(rlogG C5cons 2,~studyarm,type = "response")
7791
      mgC5cons 2
7792
      confint (pairs (mgC5cons 2, reverse = TRUE))
7793
      pairs (mgC5cons 2, reverse = TRUE)
7794
7795
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
7796
       rlogG C5cons 3 <-
7797
         glm (mean C5 cons2 ~
7798
               studyarm * mean indivhorz +
7799
               studyarm * mean indivvertical +
7800
               studyarm * mean_collhorz +
7801
               studyarm * mean_collvertical +
7802
               bornincanada +
7803
               language 1 +
7804
               language 2 +
7805
               Asian group +
7806
               White group +
7807
               disability any +
7808
               genderidentity +
7809
               income +
7810
               edhi +
7811
               age,
7812
             data = datGeneric, family=binomial("logit")
7813
         )
7814
       Anova(rlogG C5cons 3, type = "III")
7815
       summary(rlogG C5cons 3)
7816
7817
       emmip(rlogG C5cons 3, studyarm ~ mean indivvertical, cov.reduce = range, type =
       "response")
7818
7819
7820
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
7821
7822
       rlogG C5cons 4 <- glm(mean C5 cons2 ~ studyarm * edhi, data =</pre>
       datGeneric, family=binomial("logit"))
7823
       Anova(rlogG C5cons 4, type="III")
7824
       summary(rlogG C5cons 4)
7825
7826
       mgC5cons_4_s <- emmeans(rlogG_C5cons_4,~studyarm|edhi,type = "response")</pre>
7827
       mgC5cons 4 s
7828
       confint(pairs(mgC5cons 4 s,reverse = TRUE))
```

```
7829
7830
       mgC5cons 4 e <- emmeans(rlogG C5cons 4, ~ edhi|studyarm, type = "response")
7831
       confint(pairs(mgC5cons 4 e,reverse = TRUE))
7832
7833
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
7834
7835
      rlogG C5cons 5 <-
7836
                             ~ studyarm*edhi +
         glm (mean C5 cons2
7837
              mean indivhorz +
7838
               mean indivvertical +
7839
              mean collhorz +
7840
              mean collvertical +
7841
              bornincanada +
7842
               language 1 +
               language 2 +
7843
7844
               Asian group +
7845
               White_group +
7846
               disability any +
7847
               genderidentity +
7848
               income +
7849
               age,
7850
             data = datGeneric, family=binomial("logit")
7851
         )
      Anova(rlogG_C5cons 5, type = "III")
7852
7853
       summary(rlogG C5cons 5)
7854
7855
      mgC5cons 5 s <- emmeans(rlogG C5cons 5,~studyarm|edhi,type = "response")
7856
      mgC5cons_5_s
7857
      confint(pairs(mgC5cons 5 s,reverse = TRUE))
7858
7859
      mgC5cons 5 e <- emmeans(rlogG C5cons 5, ~ edhi|studyarm, type = "response")
7860
      confint(pairs(mgC5cons 5 e, reverse = TRUE))
7861
      # Now running models on imputed data.
7862
7863
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
7864
7865
7866
       #### ++ Measles ####
7867
7868
       #### + Model 1: Check for direct effects of factors without any covariates ####
7869
7870
       options(contrasts=c("contr.sum", "contr.poly"))
7871
       rlogM C5cons 1 <- glm(mean C5 cons2 ~ studyarm, data =
       datMeasles,family=binomial("logit"))
7872
       Anova(rlogM C5cons 1,type="III")
7873
       summary(rlogM C5cons 1)
7874
7875
       mmC5cons 1 <- emmeans(rlogM C5cons 1,~studyarm,type = "response") #proportions
7876
       mmC5cons 1
7877
      confint(pairs(mmC5cons 1, reverse = TRUE)) #Odds ratios
7878
7879
       # Model 2: Check for direct effects of factors with adjustment for other covariates
7880
      rlogM C5cons 2 <-
7881
         glm (mean C5 cons2 ~ studyarm +
7882
               mean indivhorz +
7883
               mean indivvertical +
7884
               mean collhorz +
7885
               mean collvertical +
7886
               bornincanada +
7887
               language_1 +
               language_2 +
7888
7889
              Asian group +
7890
              White_group +
7891
              disability any +
7892
              genderidentity +
7893
              income +
7894
              edhi +
7895
               age,
7896
            data = datMeasles, family=binomial("logit")
```

```
7897
7898
       Anova(rlogM C5cons 2, type = "III")
7899
       summary(rlogM C5cons 2)
7900
7901
       mmC5cons 2 <- emmeans(rlogM C5cons 2,~studyarm,type = "response")
7902
      mmC5cons 2
7903
      confint(pairs(mmC5cons 2, reverse = TRUE))
7904
7905
7906
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
7907
       rlogM C5cons 3 <-
7908
         glm (mean C5 cons2 ~
7909
               studyarm * mean indivhorz +
               studyarm * mean indivvertical +
7910
7911
               studyarm * mean_collhorz +
7912
               studyarm * mean_collvertical +
7913
               bornincanada +
7914
               language 1 +
7915
              language 2 +
7916
              Asian group +
7917
              White group +
7918
              disability any +
7919
               genderidentity +
7920
               income +
7921
               edhi +
7922
               age,
7923
             data = datMeasles, family=binomial("logit")
7924
         )
7925
      Anova(rlogM_C5cons_3, type = "III")
7926
      summary(rlogM C5cons 3)
7927
7928
       emmip(rlogM C5cons 3, studyarm ~ mean indivvertical, cov.reduce = range, type =
       "response")
7929
7930
7931
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
7932
7933
       rlogM_C5cons_4 <- glm(mean_C5_cons2 ~ studyarm * edhi, data =</pre>
       datMeasles, family=binomial("logit"))
7934
       Anova(rlogM C5cons 4, type="III")
7935
       summary(rlogM C5cons 4)
7936
7937
       mmC5cons 4 s <- emmeans(rlogM C5cons 4,~studyarm|edhi,type = "response")
7938
       mmC5cons 4 s
7939
       confint (pairs (mmC5cons 4 s, reverse = TRUE))
7940
7941
       mmC5cons 4 e <- emmeans(rlogM C5cons 4, ~ edhi|studyarm, type = "response")
7942
       confint(pairs(mmC5cons 4 e,reverse = TRUE))
7943
7944
7945
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
7946
7947
      rlogM C5cons 5 <-
7948
         glm (mean C5 cons2
                             ~ studyarm*edhi +
7949
               mean indivhorz +
7950
               mean indivvertical +
7951
               mean collhorz +
7952
               mean collvertical +
7953
               bornincanada +
7954
               language_1 +
7955
              language 2 +
7956
              Asian group +
7957
              White group +
7958
              disability any +
7959
              genderidentity +
7960
              income +
7961
               age,
7962
             data = datMeasles, family=binomial("logit")
```
```
7963
7964
       Anova(rlogM C5cons 5, type = "III")
7965
       summary(rlogM C5cons 5)
7966
7967
       mmC5cons 5 s <- emmeans(rlogM C5cons 5,~studyarm|edhi,type = "response")
7968
      mmC5cons_5_s
7969
      confint(pairs(mmC5cons 5 s,reverse = TRUE))
7970
7971
      mmC5cons 5 e <- emmeans(rlogM C5cons 5, ~ edhi|studyarm, type = "response")
7972
      confint(pairs(mmC5cons 5 e, reverse = TRUE))
7973
7974
       # Now running models on imputed data.
7975
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
7976
7977
7978
       #### ++ Flu ####
7979
7980
       #### + Model 1: Check for direct effects of factors without any covariates ####
7981
7982
       options(contrasts=c("contr.sum", "contr.poly"))
7983
       rlogF C5cons 1 <- glm (mean C5 cons2 ~ studyarm, data = datFlu, family=binomial("logit"))
7984
       Anova(rlogF C5cons 1, type="III")
7985
       summary(rlogF C5cons 1)
7986
7987
       mfC5cons 1 <- emmeans(rlogF C5cons 1,~studyarm,type = "response") #proportions
7988
       mfC5cons 1
7989
       confint(pairs(mfC5cons 1, reverse = TRUE)) #Odds ratios
7990
7991
       # Model 2: Check for direct effects of factors with adjustment for other covariates
7992
      rlogF C5cons 2 <-
7993
         glm (mean C5 cons2 ~ studyarm +
7994
               mean indivhorz +
7995
               mean indivvertical +
7996
               mean collhorz +
7997
               mean collvertical +
7998
               bornincanada +
7999
               language 1 +
8000
               language 2 +
8001
               Asian_group +
8002
               White group +
8003
               disability any +
8004
               genderidentity +
8005
               income +
8006
               edhi +
8007
               age,
8008
             data = datFlu, family=binomial("logit")
8009
8010
       Anova(rlogF C5cons 2, type = "III")
8011
       summary(rlogF_C5cons_2)
8012
8013
      mfC5cons 2 <- emmeans(rlogF C5cons 2,~studyarm,type = "response")
8014
      mfC5cons 2
8015
      confint(pairs(mfC5cons 2, reverse = TRUE))
8016
      pairs (mfC5cons 2, reverse = TRUE)
8017
8018
      # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
       rlogF C5cons_3 <-</pre>
8019
8020
         glm (mean C5 cons2 ~
8021
               studyarm * mean_indivhorz +
8022
               studyarm * mean_indivvertical +
8023
               studyarm * mean collhorz +
8024
               studyarm * mean collvertical +
8025
               bornincanada +
8026
               language 1 +
8027
              language 2 +
8028
              Asian_group +
8029
               White group +
8030
               disability any +
```

```
8031
               genderidentity +
8032
               income +
8033
               edhi +
8034
               age.
8035
             data = datFlu, family=binomial("logit")
8036
         )
8037
      Anova(rlogF C5cons 3, type = "III")
8038
       summary(rlogF C5cons 3)
8039
8040
       emmip(rlogF C5cons 3, studyarm ~ mean collhorz, cov.reduce = range, type = "response")
8041
8042
8043
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
8044
       rlogF C5cons 4 <- glm(mean C5 cons2 ~ studyarm * edhi, data =</pre>
8045
       datFlu, family=binomial("logit"))
       Anova(rlogF_C5cons_4,type="III")
8046
8047
       summary(rlogF C5cons 4)
8048
8049
      mfC5cons 4 s <- emmeans(rlogF C5cons 4,~studyarm|edhi,type = "response")
8050
      mfC5cons 4 s
8051
      confint(pairs(mfC5cons 4 s,reverse = TRUE))
8052
8053
      mfC5cons 4 e <- emmeans(rlogF C5cons 4, ~ edhi|studyarm, type = "response")
       confint (pairs (mfC5cons 4 e, reverse = TRUE))
8054
8055
8056
8057
      # Model 5: Check for interaction viz*edhi with adjustment for other covariates
8058
8059
      rlogF C5cons 5 <-
8060
         glm (mean C5 cons2
                             ~ studyarm*edhi +
8061
               mean indivhorz +
8062
               mean indivvertical +
8063
               mean collhorz +
               mean collvertical +
8064
8065
               bornincanada +
8066
               language 1 +
8067
               language 2 +
8068
               Asian group +
8069
               White group +
8070
               disability any +
8071
               genderidentity +
8072
               income +
8073
               age,
8074
             data = datFlu, family=binomial("logit")
8075
         )
8076
       Anova(rlogF C5cons 5, type = "III")
8077
       summary(rlogF C5cons 5)
8078
8079
      mfC5cons 5 s <- emmeans(rlogF C5cons 5,~studyarm|edhi,type = "response")
8080
      mfC5cons 5 s
8081
      confint(pairs(mfC5cons 5 s, reverse = TRUE))
8082
8083
      mfC5cons 5 e <- emmeans(rlogF C5cons 5, ~ edhi|studyarm, type = "response")
8084
       confint(pairs(mfC5cons 5 e, reverse = TRUE))
8085
8086
8087
       # Now running models on imputed data.
8808
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
8089
8090
       #### +++ Logistic regression for C5 Calculation ####
8091
8092
       #Create relevel before model to avoid problems with pairs function.
       datGeneric$mean_C5_calc2 <- relevel(as.factor(datGeneric$mean C5 calc2),ref = "0")</pre>
8093
8094
       datMeasles$mean C5 calc2 <- relevel(as.factor(datMeasles$mean C5 calc2),ref = "0")
8095
       datFlu$mean C5 calc2 <- relevel(as.factor(datFlu$mean C5 calc2),ref = "0")
8096
8097
       #### ++ Generic ####
8098
```

```
#### + Model 1: Check for direct effects of factors without any covariates ####
8099
8100
8101
       options(contrasts=c("contr.sum", "contr.poly"))
8102
       rlogG C5calc 1 <- glm(mean C5 calc2 ~ studyarm, data =</pre>
       datGeneric, family=binomial("logit"))
       Anova(rlogG_C5calc_1,type="III")
8103
8104
      summary(rlogG C5calc 1)
8105
8106
      mgC5calc 1 <- emmeans(rlogG C5calc 1,~studyarm,type = "response") #proportions
8107
8108
       confint(pairs(mgC5calc 1, reverse = TRUE)) #Odds ratios
8109
8110
      # Model 2: Check for direct effects of factors with adjustment for other covariates
8111
       rlogG C5calc 2 <-
8112
         glm(mean C5 calc2 \sim studyarm +
8113
               mean indivhorz +
8114
               mean_indivvertical +
               mean_collhorz +
8115
8116
               mean collvertical +
8117
               bornincanada +
8118
               language 1 +
8119
               language 2 +
8120
              Asian group +
8121
               White group +
8122
               disability any +
8123
               genderidentity +
8124
               income +
8125
               edhi +
8126
               age,
8127
             data = datGeneric, family=binomial("logit") )
8128
      Anova(rlogG C5calc 2, type = "III")
8129
      summary(rlogG C5calc 2)
8130
8131
      mgC5calc 2 <- emmeans(rlogG C5calc 2,~studyarm,type = "response")
8132
       mgC5calc 2
       confint (pairs (mgC5calc_2, reverse = TRUE))
8133
8134
8135
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
8136
       rlogG C5calc 3 <-
8137
         glm (mean C5 calc2 ~
8138
               studyarm * mean indivhorz +
8139
               studyarm * mean indivvertical +
8140
               studyarm * mean collhorz +
8141
               studyarm * mean collvertical +
8142
               bornincanada +
8143
               language 1 +
8144
               language 2 +
8145
               Asian group +
8146
               White_group +
8147
               disability any +
8148
               genderidentity +
8149
               income +
8150
               edhi +
8151
               age,
8152
             data = datGeneric, family=binomial("logit")
8153
         )
       Anova(rlogG C5calc 3, type = "III")
8154
8155
       summary(rlogG C5calc 3)
8156
8157
       #No interaction to interpret
8158
8159
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
8160
8161
       rlogG C5calc 4 <- glm(mean C5 calc2 ~ studyarm * edhi, data =</pre>
       datGeneric, family=binomial("logit"))
8162
       Anova(rlogG C5calc 4,type="III")
8163
       summary(rlogG C5calc 4)
8164
```

```
8165
      mgC5calc 4 s <- emmeans(rlogG C5calc 4,~studyarm|edhi,type = "response")
8166
      mgC5calc 4 s
8167
       confint(pairs(mgC5calc 4 s,reverse = TRUE))
8168
8169
      mgC5calc 4 e <- emmeans(rlogG C5calc 4, ~ edhi|studyarm, type = "response")
8170
      confint(pairs(mgC5calc 4 e, reverse = TRUE))
8171
8172
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
8173
8174
      rlogG C5calc 5 <-
         glm (mean C5 calc2
8175
                           ~ studyarm*edhi +
8176
               mean indivhorz +
8177
               mean indivvertical +
8178
               mean collhorz +
8179
               mean collvertical +
8180
               bornincanada +
8181
               language_1 +
              language 2 +
8182
8183
              Asian group +
8184
              White group +
8185
              disability any +
8186
               genderidentity +
8187
              income +
8188
               age,
             data = datGeneric, family=binomial("logit")
8189
8190
8191
      Anova(rlogG C5calc 5, type = "III")
8192
      summary(rlogG C5calc 5)
8193
8194
     mgC5calc 5 s <- emmeans(rlogG C5calc 5,~studyarm|edhi,type = "response")
8195
      mgC5calc 5 s
8196
      confint(pairs(mgC5calc 5 s,reverse = TRUE))
8197
8198
      mgC5calc 5 e <- emmeans(rlogG C5calc 5, ~ edhi|studyarm, type = "response")
8199
      confint(pairs(mgC5calc 5 e,reverse = TRUE))
8200
8201
       # Now running models on imputed data.
8202
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
8203
8204
8205
       #### ++ Measles ####
8206
8207
       #### + Model 1: Check for direct effects of factors without any covariates ####
8208
8209
       options(contrasts=c("contr.sum", "contr.poly"))
8210
       rlogM C5calc 1 <- glm(mean C5 calc2 ~ studyarm, data =</pre>
       datMeasles, family=binomial("logit"))
8211
       Anova(rlogM C5calc 1, type="III")
8212
      summary(rlogM C5calc 1)
8213
8214 mmC5calc 1 <- emmeans(rlogM C5calc 1,~studyarm,type = "response") #proportions
8215 mmC5calc 1
8216
      confint(pairs(mmC5calc 1, reverse = TRUE)) #Odds ratios
8217
      pairs (mmC5calc 1, reverse = TRUE)
8218
8219
      # Model 2: Check for direct effects of factors with adjustment for other covariates
8220
       rlogM C5calc 2 <-
8221
         glm(mean C5 calc2 \sim studyarm +
8222
               mean indivhorz +
8223
               mean_indivvertical +
              mean_collhorz +
8224
8225
              mean collvertical +
8226
              bornincanada +
8227
              language 1 +
8228
              language 2 +
8229
              Asian group +
              White_group +
8230
8231
               disability any +
8232
               genderidentity +
```

```
8233
               income +
8234
               edhi +
8235
               age,
8236
             data = datMeasles, family=binomial("logit")
8237
         )
8238
      Anova(rlogM C5calc 2, type = "III")
8239
      summary(rlogM C5calc 2)
8240
8241 mmC5calc 2 <- emmeans(rlogM C5calc 2,~studyarm,type = "response")
8242 mmC5calc 2
8243
      confint(pairs(mmC5calc 2, reverse = TRUE))
8244
8245
8246
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
8247
       rlogM_C5calc_3 <-
         glm (mean C5 calc2 ~
8248
8249
               studyarm * mean indivhorz +
8250
               studyarm * mean indivvertical +
8251
              studyarm * mean collhorz +
8252
              studyarm * mean collvertical +
8253
              bornincanada +
8254
              language 1 +
8255
              language 2 +
8256
              Asian group +
8257
              White group +
8258
              disability any +
8259
              genderidentity +
8260
              income +
8261
              edhi +
8262
               age,
8263
             data = datMeasles, family=binomial("logit")
8264
         )
       Anova(rlogM C5calc 3, type = "III")
8265
8266
       summary(rlogM C5calc 3)
8267
8268
       #No interaction to interpret
8269
8270
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
8271
8272
       rlogM C5calc 4 <- glm(mean C5 calc2 ~ studyarm * edhi, data =</pre>
       datMeasles, family=binomial("logit"))
8273
       Anova(rlogM C5calc 4, type="III")
8274
       summary(rlogM C5calc 4)
8275
8276
       mmC5calc 4 s <- emmeans(rlogM C5calc 4,~studyarm|edhi,type = "response")
8277
       mmC5calc 4 s
8278
       confint(pairs(mmC5calc 4 s,reverse = TRUE))
8279
8280
      mmC5calc 4 e <- emmeans(rlogM C5calc 4, ~ edhi|studyarm, type = "response")
8281
       confint (pairs (mmC5calc 4 e, reverse = TRUE))
8282
8283
8284
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
8285
8286
       rlogM C5calc 5 <-
8287
         glm (mean C5 calc2
                             ~ studyarm*edhi +
8288
               mean indivhorz +
8289
               mean indivvertical +
8290
               mean_collhorz +
               mean_collvertical +
8291
8292
               bornincanada +
8293
               language 1 +
8294
              language 2 +
8295
              Asian group +
8296
              White group +
8297
              disability_any +
8298
               genderidentity +
8299
               income +
```

```
8300
               age,
8301
             data = datMeasles, family=binomial("logit")
8302
         )
8303
       Anova(rlogM C5calc 5, type = "III")
8304
       summary(rlogM C5calc 5)
8305
8306
      mmC5calc 5 s <- emmeans(rlogM C5calc 5,~studyarm|edhi,type = "response")
8307
      mmC5calc 5 s
8308
      confint(pairs(mmC5calc 5 s,reverse = TRUE))
8309
8310
      mmC5calc 5 e <- emmeans(rlogM C5calc 5, ~ edhi|studyarm, type = "response")
8311
       confint(pairs(mmC5calc 5 e,reverse = TRUE))
8312
8313
       # Now running models on imputed data.
8314
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
8315
8316
8317
       #### ++ Flu ####
8318
       #### + Model 1: Check for direct effects of factors without any covariates ####
8319
8320
8321
       options(contrasts=c("contr.sum", "contr.poly"))
8322
       rlogF C5calc 1 <- glm(mean C5 calc2 ~ studyarm, data = datFlu, family=binomial("logit"))</pre>
8323
       Anova(rlogF C5calc 1, type="III")
8324
       summary(rlogF C5calc 1)
8325
8326
      mfC5calc 1 <- emmeans(rlogF C5calc 1,~studyarm,type = "response") #proportions
      mfC5calc 1
8327
8328
      confint(pairs(mfC5calc 1, reverse = TRUE)) #Odds ratios
8329
8330
       # Model 2: Check for direct effects of factors with adjustment for other covariates
8331
      rlogF C5calc 2 <-
         glm(mean C5 calc2 ~ studyarm +
8332
8333
               mean indivhorz +
8334
               mean indivvertical +
8335
               mean collhorz +
8336
               mean collvertical +
8337
               bornincanada +
8338
               language_1 +
8339
               language 2 +
8340
              Asian group +
8341
              White group +
8342
              disability any +
8343
               genderidentity +
8344
               income +
8345
               edhi +
8346
               age,
8347
             data = datFlu, family=binomial("logit")
8348
         )
8349
      Anova(rlogF_C5calc_2, type = "III")
8350
      summary(rlogF C5calc 2)
8351
8352
      mfC5calc 2 <- emmeans(rlogF C5calc 2,~studyarm,type = "response")
8353
8354
       confint(pairs(mfC5calc 2, reverse = TRUE))
8355
8356
      # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
8357
       rlogF C5calc 3 <-
8358
         glm (mean_C5_calc2 ~
8359
               studyarm * mean_indivhorz +
8360
               studyarm * mean indivvertical +
8361
               studyarm * mean collhorz +
8362
               studyarm * mean collvertical +
8363
              bornincanada +
8364
               language 1 +
8365
               language_2 +
8366
               Asian group +
8367
               White group +
```

```
8368
               disability any +
8369
               genderidentity +
8370
               income +
8371
               edhi +
8372
               age,
8373
             data = datFlu, family=binomial("logit")
8374
         )
8375
      Anova(rlogF C5calc 3, type = "III")
8376
      summary(rlogF C5calc 3)
8377
8378
       #No interaction to interpret
8379
8380
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
8381
8382
      rlogF C5calc 4 <- glm(mean C5 calc2 ~ studyarm * edhi, data =</pre>
       datFlu, family=binomial("logit"))
8383
       Anova(rlogF_C5calc_4,type="III")
8384
      summary(rlogF C5calc 4)
8385
8386
      mfC5calc 4 s <- emmeans(rlogF C5calc 4,~studyarm|edhi,type = "response")
8387
      mfC5calc 4 s
8388
      confint (pairs (mfC5calc 4 s, reverse = TRUE))
8389
8390
      mfC5calc 4 e <- emmeans(rlogF C5calc 4, ~ edhi|studyarm, type = "response")
8391
       confint(pairs(mfC5calc 4 e,reverse = TRUE))
8392
8393
      # Model 5: Check for interaction viz*edhi with adjustment for other covariates
8394
8395
8396
     rlogF C5calc 5 <-
8397
         glm (mean C5 calc2
                             ~ studyarm*edhi +
8398
               mean indivhorz +
8399
               mean indivvertical +
              mean collhorz +
8400
8401
              mean collvertical +
8402
               bornincanada +
8403
               language 1 +
8404
               language 2 +
8405
               Asian_group +
8406
              White group +
8407
              disability any +
8408
              genderidentity +
8409
              income +
8410
               age,
8411
             data = datFlu, family=binomial("logit")
8412
         )
8413
      Anova(rlogF C5calc 5, type = "III")
8414
      summary(rlogF C5calc 5)
8415
8416
      mfC5calc 5 s <- emmeans(rlogF C5calc 5,~studyarm|edhi,type = "response")
8417
      mfC5calc 5 s
8418
      confint(pairs(mfC5calc 5 s, reverse = TRUE))
8419
8420
      mfC5calc 5 e <- emmeans(rlogF C5calc 5, ~ edhi|studyarm, type = "response")
8421
      confint(pairs(mfC5calc 5 e, reverse = TRUE))
8422
8423
      # Now running models on imputed data.
8424
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
8425
8426
8427
8428
       #### +++ Logistic regression for C5 Collective Response ####
8429
8430
       #Create relevel before model to avoid problems with pairs function.
8431
       datGeneric$mean C5 coll2 <- relevel(as.factor(datGeneric$mean C5 coll2),ref = "0")
8432
       datMeasles$mean C5 coll2 <- relevel(as.factor(datMeasles$mean C5 coll2),ref = "0")
8433
      datFlu$mean C5 coll2 <- relevel(as.factor(datFlu$mean C5 coll2),ref = "0")
8434
8435
       #### ++ Generic ####
```

```
8436
8437
       #### + Model 1: Check for direct effects of factors without any covariates ####
8438
       options(contrasts=c("contr.sum", "contr.poly"))
8439
8440
       rlogG C5coll 1 <- glm(mean C5 coll2 ~ studyarm, data =</pre>
       datGeneric, family=binomial("logit"))
8441
       Anova(rlogG C5coll 1,type="III")
8442
      summary(rlogG C5coll 1)
8443
8444
      mgC5coll 1 <- emmeans(rlogG C5coll 1,~studyarm,type = "response") #proportions
8445
      mgC5coll 1
8446
      confint(pairs(mgC5coll 1, reverse = TRUE)) #Odds ratios
       pairs (mgC5coll 1, reverse = TRUE)
8447
8448
8449
8450
       # Model 2: Check for direct effects of factors with adjustment for other covariates
8451
       rlogG C5coll 2 <-
8452
         glm(mean C5 coll2 ~ studyarm +
8453
               mean indivhorz +
8454
               mean indivvertical +
8455
               mean collhorz +
8456
               mean collvertical +
8457
               bornincanada +
8458
               language 1 +
8459
               language 2 +
8460
               Asian group +
               White_group +
8461
8462
               disability any +
8463
               genderidentity +
8464
               income +
8465
               edhi +
8466
               age,
8467
             data = datGeneric, family=binomial("logit") )
8468
      Anova(rlogG C5coll 2, type = "III")
8469
      summary(rlogG C5coll 2)
8470
8471
      mgC5coll 2 <- emmeans(rlogG C5coll 2,~studyarm,type = "response")
8472
      mqC5coll 2
8473
      confint(pairs(mgC5coll_2, reverse = TRUE))
8474
      pairs (mgC5coll 2, reverse = TRUE)
8475
8476
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
8477
       rlogG C5coll 3 <-
8478
         glm (mean C5 coll2 ~
8479
               studyarm * mean indivhorz +
8480
               studyarm * mean indivvertical +
               studyarm * mean collhorz +
8481
8482
               studyarm * mean_collvertical +
8483
               bornincanada +
8484
               language 1 +
8485
               language 2 +
8486
               Asian group +
8487
               White group +
8488
               disability any +
8489
               genderidentity +
8490
               income +
8491
               edhi +
8492
               age,
8493
             data = datGeneric, family=binomial("logit")
8494
         )
8495
       Anova(rlogG C5coll 3, type = "III")
8496
       summary(rlogG C5coll 3)
8497
8498
       emmip(rlogG C5coll 3, studyarm ~ mean indivvertical, cov.reduce = range, type =
       "response")
8499
       emmip(rlogG_C5coll_3, studyarm ~ mean_collhorz, cov.reduce = range, type = "response")
8500
8501
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
```

```
8502
8503
       rlogG C5coll 4 <- glm(mean C5 coll2 ~ studyarm * edhi, data =</pre>
       datGeneric, family=binomial("logit"))
8504
       Anova(rlogG C5coll 4, type="III")
8505
       summary(rlogG C5coll 4)
8506
8507
      mgC5coll 4 s <- emmeans(rlogG C5coll 4,~studyarm|edhi,type = "response")
8508
      mgC5coll 4 s
8509
       confint(pairs(mgC5coll 4 s,reverse = TRUE))
8510
       pairs (mgC5coll 4 s, reverse = TRUE)
8511
8512
      mgC5coll 4 e <- emmeans(rlogG C5coll 4, ~ edhi|studyarm, type = "response")
8513
       confint(pairs(mgC5coll 4 e, reverse = TRUE))
8514
       pairs (mgC5coll 4 e, reverse = TRUE)
8515
8516
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
8517
8518
       rlogG C5coll 5 <-
8519
                             ~ studyarm*edhi +
         glm (mean C5 coll2
8520
               mean indivhorz +
8521
               mean indivvertical +
8522
               mean collhorz +
8523
               mean collvertical +
8524
               bornincanada +
8525
               language 1 +
               language 2 +
8526
8527
               Asian group +
8528
               White_group +
8529
               disability any +
8530
               genderidentity +
8531
               income +
8532
               age,
8533
             data = datGeneric, family=binomial("logit")
8534
         )
8535
       Anova(rlogG C5coll 5, type = "III")
8536
       summary(rlogG C5coll 5)
8537
8538
       mgC5coll 5 s <- emmeans(rlogG C5coll 5,~studyarm|edhi,type = "response")
8539
       mgC5coll_5_s
8540
       confint(pairs(mgC5coll 5 s,reverse = TRUE))
8541
8542
       mgC5coll 5 e <- emmeans(rlogG C5coll 5, ~ edhi|studyarm, type = "response")
8543
       confint(pairs(mgC5coll 5 e,reverse = TRUE))
8544
8545
       # Now running models on imputed data.
8546
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
8547
8548
8549
       #### ++ Measles ####
8550
8551
       #### + Model 1: Check for direct effects of factors without any covariates ####
8552
8553
       options(contrasts=c("contr.sum", "contr.poly"))
8554
       rlogM C5coll 1 <- glm(mean C5 coll2 ~ studyarm, data =</pre>
       datMeasles, family=binomial("logit"))
8555
       Anova(rlogM C5coll 1, type="III")
8556
       summary(rlogM C5coll 1)
8557
8558
       mmC5coll 1 <- emmeans(rlogM C5coll 1,~studyarm,type = "response") #proportions
8559
       mmC5coll 1
8560
       confint(pairs(mmC5coll 1, reverse = TRUE)) #Odds ratios
8561
8562
       # Model 2: Check for direct effects of factors with adjustment for other covariates
8563
       rlogM C5coll 2 <-
8564
         glm (mean C5 coll2 ~ studyarm +
8565
               mean indivhorz +
8566
               mean indivvertical +
8567
               mean collhorz +
8568
               mean collvertical +
```

```
8569
              bornincanada +
8570
               language 1 +
8571
              language 2 +
8572
              Asian group +
8573
              White group +
8574
              disability any +
8575
              genderidentity +
8576
              income +
8577
               edhi +
8578
               age,
8579
             data = datMeasles, family=binomial("logit")
8580
        )
8581
      Anova(rlogM C5coll 2, type = "III")
8582
       summary(rlogM C5coll 2)
8583
8584
      mmC5coll 2 <- emmeans(rlogM C5coll 2,~studyarm,type = "response")
8585
      mmC5coll 2
8586
      confint(pairs(mmC5coll 2,reverse = TRUE))
8587
8588
8589
     # Model 3: Check for moderating effects of individualism & collectivism with adjustment
      for other covariates
8590
     rlogM C5coll 3 <-
8591
         glm(mean C5 coll2 ~
8592
               studyarm * mean indivhorz +
               studyarm * mean indivvertical +
8593
8594
               studyarm * mean collhorz +
              studyarm * mean_collvertical +
8595
8596
              bornincanada +
8597
              language 1 +
8598
              language 2 +
8599
              Asian group +
8600
              White group +
8601
              disability any +
8602
              genderidentity +
8603
               income +
8604
               edhi +
8605
               age,
8606
             data = datMeasles, family=binomial("logit")
8607
         )
8608
       Anova(rlogM C5coll 3, type = "III")
8609
      summary(rlogM C5coll 3)
8610
8611
       #No interaction to interpret
8612
8613
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
8614
8615
       rlogM C5coll 4 <- glm(mean C5 coll2 ~ studyarm * edhi, data =
       datMeasles, family=binomial("logit"))
8616
      Anova(rlogM_C5coll_4, type="III")
8617
      summary(rlogM C5coll 4)
8618
8619
      mmC5coll 4 s <- emmeans(rlogM C5coll 4,~studyarm|edhi,type = "response")
8620
      mmC5coll 4 s
8621
      confint(pairs(mmC5coll 4 s,reverse = TRUE))
8622
8623
      mmC5coll 4 e <- emmeans(rlogM C5coll 4, ~ edhi|studyarm, type = "response")
8624
       confint(pairs(mmC5coll 4 e, reverse = TRUE))
8625
8626
8627
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
8628
8629
      rlogM C5coll 5 <-
8630
         glm (mean C5 coll2
                           ~ studyarm*edhi +
8631
              mean indivhorz +
8632
              mean indivvertical +
8633
              mean collhorz +
8634
               mean collvertical +
8635
               bornincanada +
```

```
8636
               language 1 +
8637
               language 2 +
8638
               Asian group +
8639
               White group +
8640
               disability any +
8641
               genderidentity +
8642
               income +
8643
               age,
8644
             data = datMeasles, family=binomial("logit")
8645
         )
8646
      Anova(rlogM C5coll 5, type = "III")
8647
       summary(rlogM C5coll 5)
8648
8649
      mmC5coll 5 s <- emmeans(rlogM C5coll 5,~studyarm|edhi,type = "response")
       mmC5coll 5 s
8650
8651
      confint(pairs(mmC5coll 5 s, reverse = TRUE))
8652
8653
      mmC5coll 5 e <- emmeans(rlogM C5coll 5, ~ edhi|studyarm, type = "response")
8654
      confint(pairs(mmC5coll 5 e, reverse = TRUE))
8655
8656
       # Now running models on imputed data.
8657
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
8658
8659
8660
       #### ++ Flu ####
8661
8662
       #### + Model 1: Check for direct effects of factors without any covariates ####
8663
8664
      options(contrasts=c("contr.sum", "contr.poly"))
8665
      rlogF C5coll 1 <- glm(mean C5 coll2 ~ studyarm, data = datFlu, family=binomial("logit"))
8666
      Anova(rlogF C5coll 1, type="III")
8667
       summary(rlogF C5coll 1)
8668
8669
      mfC5coll 1 <- emmeans(rlogF C5coll 1,~studyarm,type = "response") #proportions
8670
      mfC5coll 1
8671
       confint(pairs(mfC5coll 1, reverse = TRUE)) #Odds ratios
8672
8673
       # Model 2: Check for direct effects of factors with adjustment for other covariates
8674
       rlogF_C5coll_2 <-</pre>
8675
         glm(mean C5 coll2 ~ studyarm +
8676
               mean indivhorz +
8677
               mean indivvertical +
8678
               mean collhorz +
8679
               mean collvertical +
8680
              bornincanada +
               language 1 +
8681
8682
               language 2 +
8683
               Asian group +
8684
               White_group +
8685
               disability any +
8686
               genderidentity +
8687
               income +
8688
               edhi +
8689
8690
             data = datFlu, family=binomial("logit")
8691
         )
8692
       Anova(rlogF C5coll 2, type = "III")
8693
       summary(rlogF_C5coll 2)
8694
8695
      mfC5coll 2 <- emmeans(rlogF C5coll 2,~studyarm,type = "response")</pre>
       mfC5coll 2
8696
8697
       confint (pairs (mfC5coll 2, reverse = TRUE))
8698
8699
       # Model 3: Check for moderating effects of individualism & collectivism with adjustment
       for other covariates
8700
      rlogF C5coll 3 <-
8701
         glm (mean C5 coll2 ~
8702
               studyarm * mean indivhorz +
8703
               studyarm * mean indivvertical +
```

```
8704
               studyarm * mean collhorz +
8705
              studyarm * mean collvertical +
8706
              bornincanada +
8707
               language 1 +
8708
               language 2 +
8709
               Asian_group +
8710
               White group +
8711
              disability any +
8712
               genderidentity +
8713
               income +
8714
               edhi +
8715
               age,
8716
             data = datFlu, family=binomial("logit")
8717
         )
8718
       Anova(rlogF C5coll 3, type = "III")
       summary(rlogF_C5coll 3)
8719
8720
8721
       emmip(rlogF C5coll 3, studyarm ~ mean collhorz, cov.reduce = range, type = "response")
8722
8723
8724
       #### + Model 4: Check for interaction viz*edhi without any covariates ####
8725
8726
       rlogF C5coll 4 <- glm(mean C5 coll2 ~ studyarm * edhi, data =</pre>
       datFlu, family=binomial("logit"))
8727
       Anova(rlogF C5coll 4, type="III")
8728
       summary(rlogF C5coll 4)
8729
8730
      mfC5coll 4 s <- emmeans(rlogF C5coll 4,~studyarm|edhi,type = "response")
8731
      mfC5coll 4 s
8732
      confint(pairs(mfC5coll 4 s, reverse = TRUE))
8733
8734
      mfC5coll 4 e <- emmeans(rlogF C5coll 4, ~ edhi|studyarm, type = "response")
8735
      confint(pairs(mfC5coll 4 e,reverse = TRUE))
8736
8737
8738
       # Model 5: Check for interaction viz*edhi with adjustment for other covariates
8739
8740
       rlogF C5coll 5 <-
8741
         glm (mean C5 coll2
                             ~ studyarm*edhi +
8742
               mean indivhorz +
8743
              mean indivvertical +
8744
              mean collhorz +
8745
              mean collvertical +
8746
              bornincanada +
8747
               language 1 +
8748
               language 2 +
8749
               Asian group +
8750
               White group +
8751
               disability any +
8752
               genderidentity +
               income +
8753
8754
               age,
8755
             data = datFlu, family=binomial("logit")
8756
         )
8757
       Anova(rlogF C5coll 5, type = "III")
8758
       summary(rlogF C5coll 5)
8759
8760
      mfC5coll 5 s <- emmeans(rlogF C5coll 5,~studyarm|edhi,type = "response")
8761
       mfC5coll 5 s
8762
      confint (pairs (mfC5coll_5_s, reverse = TRUE))
8763
8764
      mfC5coll_5_e <- emmeans(rlogF_C5coll_5, ~ edhi|studyarm, type = "response")</pre>
       confint(pairs(mfC5coll 5 e,reverse = TRUE))
8765
8766
8767
       # Now running models on imputed data.
8768
       #CHANGELOG ASJ: No missing data for c5conf, no model with imputation performed, 21-09-20.
8769
8770
```

8771

#### COMPLETES VS INCOMPLETES ####

```
8772
8773
       # Here we test for differences between people who finished the survey (completes) and
       those who
       # started but did not finish (incompletes) to explore potential issues or limitations
8774
       introduced by
8775
       # imputing missing data. To do this, we run Chi-squared tests on categorical variables
       and Wilcoxon
      # tests on continuous variables, comparing people who did and did not complete the
8776
      survey. We ran
8777
      # the sociodemographic panel of questions first to maximally enable this comparison but
8778
      # able to compare with people who never clicked on the survey or who started to read
       and didn't
8779
       # answer anything.
8780
8781
       #CHANGELOG ASJ: Compare people analysed who finished with quality answer VS (did not
       finished or finished with poor quality), 2021-08-06.
8782
       table (datConsent$used) #CHANGELOG ASJ: changed finished to used, and everywhere below
       2021-08-06
8783
       prop.table(table(datConsent$used))*100
8784
8785
       #CHANGELOG ASJ: Apply the same changes to the variables as in the dataset dat, 2021-09-01
8786
       datConsent$yearofbirth <- as.numeric(datConsent$yearofbirth)</pre>
8787
       datConsent$yearofbirth[datConsent$yearofbirth==888] <- NA
8788
       datConsent$age <- 2021 - datConsent$yearofbirth</pre>
8789
8790
      cols.num <-
8791
8792
       C (
           "bornincanada",
8793
8794
           "language 1",
           "language 2",
8795
           "language 3",
8796
           "language 888",
8797
8798
           "ethnicity 1",
           "ethnicity 2",
8799
           "ethnicity 3",
8800
8801
           "ethnicity 4",
           "ethnicity_5",
8802
8803
           "ethnicity 6",
           "ethnicity_7",
8804
           "ethnicity 8",
8805
8806
          "ethnicity 9",
8807
          "ethnicity 10",
          "ethnicity 11",
8808
8809
          "ethnicity 12",
8810
          "ethnicity 13",
          "ethnicity 14",
8811
          "ethnicity_15",
8812
          "ethnicity_16",
8813
8814
          "ethnicity_17",
           "ethnicity 888",
8815
8816
           "disability",
8817
           "techdisability",
8818
           "sexatbirth",
8819
           "genderidentity",
8820
           "supportedbyincome",
           "educationlevel",
8821
8822
           "studyarm",
           "viz",
8823
8824
           "disease",
           "immune",
8825
           "c19vax"
8826
8827
8828
       datConsent[cols.num] <- lapply(datConsent[cols.num],as.numeric)</pre>
8829
8830
       datConsent$language_1[is.na(datConsent$language_1)] <- 0</pre>
8831
       datConsent$language 2[is.na(datConsent$language 2)] <- 0</pre>
8832
       datConsent$language 3[is.na(datConsent$language 3)] <- 0</pre>
```

```
8833
8834
           datConsent$language 1[datConsent$language 888==1&datConsent$language 1==0&datConsent$language 1
           uage 2==0&datConsent$language 3==0] <- NA
8835
           datConsent$language 2[datConsent$language 888==1&datConsent$language 1==0&datConsent$language 1
           uage 2==0&datConsent$language 3==0] <- NA</pre>
           \label{language} \verb| datConsent| anguage 888 == 1 & datConsent| anguage 1 == 0 & datConsent| anguage 1
8836
           uage_2==0&datConsent$language 3==0] <- NA</pre>
8837
           datConsent$ethnicity 1[is.na(datConsent$ethnicity 1)] <- 0</pre>
8838
8839
           datConsent$ethnicity 2[is.na(datConsent$ethnicity 2)] <- 0</pre>
8840
           datConsent$ethnicity 3[is.na(datConsent$ethnicity 3)] <- 0</pre>
8841
           datConsent$ethnicity 4[is.na(datConsent$ethnicity 4)] <- 0</pre>
           datConsent$ethnicity 5[is.na(datConsent$ethnicity 5)] <- 0</pre>
8842
           datConsent$ethnicity_6[is.na(datConsent$ethnicity_6)] <- 0</pre>
8843
           datConsent$ethnicity_7[is.na(datConsent$ethnicity_7)] <- 0</pre>
8844
8845
           datConsent$ethnicity_8[is.na(datConsent$ethnicity_8)] <- 0</pre>
           datConsent$ethnicity_9[is.na(datConsent$ethnicity_9)] <- 0</pre>
8846
           datConsent$ethnicity_10[is.na(datConsent$ethnicity 10)] <- 0</pre>
8847
8848
           datConsent$ethnicity 11[is.na(datConsent$ethnicity 11)] <- 0</pre>
8849
           datConsent$ethnicity 12[is.na(datConsent$ethnicity 12)] <- 0</pre>
8850
           datConsent$ethnicity 13[is.na(datConsent$ethnicity 13)] <- 0</pre>
8851
           datConsent$ethnicity 14[is.na(datConsent$ethnicity 14)] <- 0</pre>
8852
           datConsent$ethnicity 15[is.na(datConsent$ethnicity 15)] <- 0</pre>
8853
           datConsent$ethnicity 16[is.na(datConsent$ethnicity 16)] <- 0</pre>
8854
           datConsent$ethnicity 17[is.na(datConsent$ethnicity 17)] <- 0</pre>
8855
8856
8857
          datConsent ethnicity <-
8858
              subset (
8859
                 datConsent,
8860
                 select = c(
8861
                     ethnicity 1,
8862
                     ethnicity 2,
                     ethnicity 3,
8863
8864
                     ethnicity 4,
8865
                     ethnicity
8866
                     ethnicity 6,
8867
                     ethnicity 7,
8868
                     ethnicity 8,
8869
                     ethnicity 9,
8870
                     ethnicity 10,
8871
                     ethnicity 11,
8872
                     ethnicity 12,
8873
                     ethnicity 13,
8874
                     ethnicity 14,
8875
                     ethnicity 15,
8876
                     ethnicity 16,
8877
                     ethnicity 17
8878
8879
8880
8881
           datConsent$sum ethnicity <-rowSums(datConsent ethnicity,na.rm=T)</pre>
8882
8883
           datConsent$ethnicity 1[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
8884
           datConsent$ethnicity 2[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
           datConsent$ethnicity_3[datConsent$ethnicity_888==1&datConsent$sum_ethnicity==0] <- NA
8885
8886
           datConsent$ethnicity 4[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
8887
           datConsent$ethnicity 5[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
8888
           datConsent$ethnicity 6[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
8889
           datConsent$ethnicity_7[datConsent$ethnicity_888==1&datConsent$sum_ethnicity==0] <- NA
8890
           datConsent$ethnicity_8[datConsent$ethnicity_888==1&datConsent$sum_ethnicity==0] <- NA
8891
           datConsent$ethnicity 9[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
8892
           datConsent$ethnicity 10[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
8893
           datConsent$ethnicity 11[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
           datConsent$ethnicity_12[datConsent$ethnicity 888==1&datConsent$sum_ethnicity==0] <- NA
8894
8895
           datConsent$ethnicity 13[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
           datConsent$ethnicity_14[datConsent$ethnicity_888==1&datConsent$sum_ethnicity==0] <- NA
8896
8897
           datConsent$ethnicity 15[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
           datConsent$ethnicity 16[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
8898
```

```
datConsent$ethnicity 17[datConsent$ethnicity 888==1&datConsent$sum ethnicity==0] <- NA
8900
8901
      datConsent$Asian group <-
8902
        ifelse(
8903
           datConsent$ethnicity 1 == 1 |
8904
             datConsent$ethnicity_2 == 1 |
8905
             datConsent$ethnicity_3 == 1 |
8906
             datConsent$ethnicity 4 == 1,
8907
8908
           0
8909
         )
8910
8911
8912
      datConsent$White group <-
8913
        ifelse(
8914
           datConsent$ethnicity 6 == 1 |
             datConsent$ethnicity 7 == 1,
8915
8916
8917
8918
         )
8919
8920
       datConsent$edhi <- ifelse(datConsent$educationlevel == 4 |</pre>
                                   datConsent$educationlevel == 5|
8921
8922
                                   datConsent$educationlevel == 6|
8923
                                   datConsent$educationlevel == 7, TRUE,
                                 ifelse(datConsent$educationlevel == 8 |
8924
                                 datConsent$educationlevel == 888, NA, FALSE))
8925
8926
8927
       datConsent$bornincanada[datConsent$bornincanada==888] <- NA
8928
      datConsent$disability[datConsent$disability==888] <- NA
8929
      datConsent$techdisability[datConsent$techdisability==888] <- NA
8930 datConsent$sexatbirth[datConsent$sexatbirth==888] <- NA
      datConsent$genderidentity[datConsent$genderidentity==888] <- NA
8931
8932
      datConsent$income[datConsent$income==888] <- NA</pre>
8933
       datConsent$income[datConsent$income==5] <- NA</pre>
8934
       datConsent$supportedbyincome[datConsent$supportedbyincome==888] <- NA
8935
       datConsent$educationlevel==888] <- NA
8936
      datConsent$educationlevel[datConsent$educationlevel==8] <- NA
8937
8938
       datConsent$agecat[datConsent$agecat==888 | datConsent$agecat==1] <- NA</pre>
8939
8940
8941
      datConsent$bornincanada <-
8942
         factor(datConsent$bornincanada,
8943
                levels = c(1, 0),
8944
                labels = c("Yes", "No"))
8945
      datConsent$language 1 <-
8946
8947
         factor(datConsent$language 1,
8948
                levels = c(1, 0),
8949
                labels = c("Yes", "No"))
8950
8951
      datConsent$language 2 <-
8952
         factor(datConsent$language 2,
8953
                levels = c(1, 0),
                labels = c("Yes", "No"))
8954
8955
8956
       datConsent$Asian group <-
         factor(datConsent$Asian group,
8957
                levels = c(1, 0),
8958
                labels = c("Yes", "No"))
8959
8960
8961
8962
      datConsent$White group <-
8963
         factor(datConsent$White group,
8964
                levels = c(1, 0),
8965
                labels = c("Yes", "No"))
```

8899

8966

```
8967
8968
      datConsent$disability <-
8969
         factor(
8970
           datConsent$disability,
8971
           levels = c(0, 1),
8972
           labels = c("No disability", "yes, at least one")
8973
         )
8974
8975
      datConsent$techdisability <-
8976
         factor (datConsent$techdisability,
                levels = c(0, 1),
8977
                labels = c("No", "Yes"))
8978
8979
8980
       datConsent$sexatbirth <-</pre>
8981
       factor(datConsent$sexatbirth,
                levels = c(1, 2),
8982
8983
                labels = c("Female", "Male"))
8984
8985
      datConsent$genderidentity <- factor(</pre>
8986
       datConsent$genderidentity,
8987
         levels = c(1, 2, 3, 4),
8988
         labels = c(
8989
           "Female",
           "Male",
8990
8991
          "Indigenous or other cultural gender minority identity",
           "Something else"
8992
8993
8994
      )
8995
8996 datConsent$income <-
8997
       factor(
8998
           datConsent$income,
8999
           levels = c(1, 2, 3, 4),
           labels = c("24 999 or less", "25 000 to 49 999",
9000
                       "50 000 to 99 999", "100 000 or more")
9001
9002
         )
9003
9004
      datConsent$educationlevel <- factor(</pre>
9005
         datConsent$educationlevel,
9006
         levels = c(1, 2, 3, 4, 5, 6, 7),
9007
         labels = c(
9008
           "Some Elementary School",
9009
           "High School Diploma",
9010
           "Apprenticeship or trade certificate or diploma",
9011
           "College or polytechnical school certificate or diploma",
9012
           "University degree bachelor level or below",
9013
           "University graduate degree Master level",
9014
           "University graduate degree Doctorate level"
9015
9016
      )
9017
9018
      datConsent$agecat<-
9019
       factor(
9020
           datConsent$agecat,
9021
           levels = c(2, 3, 4),
9022
           labels = c("18-34 \text{ years}", "35-49 \text{ years}", "50 \text{ years and more}")
9023
         )
9024
9025
       datConsent$UserLanguage <- as.factor(datConsent$UserLanguage)</pre>
9026
9027
      datConsent$studyarm <-
9028
         factor (
9029
           datConsent$studyarm,
9030
           levels = c(0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 11, 12, 13),
9031
           labels = c(
9032
             "controlgeneric",
            "controlmeasles",
9033
             "controlpertussis",
9034
             "controlflu",
9035
```

```
"herdimmgeneric",
9036
9037
             "herdimmmeasles",
9038
             "herdimmpertussis",
9039
             "herdimmflu",
9040
             "robertkochgeneric",
9041
             "sbsnewsgeneric",
9042
             "quardianmeasles",
9043
             "theotheredmundmeasles",
9044
             "publichealthagencycanadaflu"
9045
9046
         )
9047
9048
      datConsent$viz <- factor (
9049
         datConsent$viz,
9050
         levels = c(0, 1, 2, 3, 5, 6, 7),
9051
         labels = c(
9052
          "no visualization",
           "herdimm",
9053
           "robertkoch",
9054
9055
           "sbsnews",
          "guardian",
9056
9057
           "theotheredmund",
9058
           "publichealthagencycanada"
9059
        )
9060
      )
9061
      datConsent$disease <-
9062
9063
       factor (
9064
          datConsent$disease,
9065
           levels = c(0, 1, 2, 3),
9066
           labels = c("Generic", "Measles", "Pertussis", "Flu")
9067
         )
9068
9069
9070
       datConsent$genderidentity[datConsent$genderidentity == "Something else" |
                                    datConsent$genderidentity == "Indigenous or other cultural
9071
                                    gender minority identity"] <- NA
9072
       datConsent$genderidentity <- droplevels(datConsent$genderidentity)</pre>
9073
9074
9075
       datConsent$disability any <-ifelse(datConsent$disability =="yes,at least one" |</pre>
       datConsent$techdisability == "Yes", 1, 0)
9076
       datConsent$disability any <-</pre>
9077
         factor (
9078
           datConsent$disability any,
9079
           levels = c(1, 0),
9080
           labels = c("Yes", "No")
9081
9082
9083
      datConsent$agecat <- as.numeric(datConsent$agecat)</pre>
9084
9085
     datConsent$used <-
9086
       factor(
9087
           datConsent$used,
9088
           levels = c(1, 0),
           labels = c("Yes", "No")
9089
9090
         )
9091
9092
       # For each categorical demographic to do along with the next step of chi square
9093
       #CHANGELOG ASJ: Add table for other demographic variables 21-08-31
9094
       t1<-data.frame(datConsent$used,datConsent$studyarm)</pre>
9095
       table(t1)
9096
      prop.table(table(t1), 1) * 100
9097
9098
       t1<-data.frame(datConsent$used,datConsent$viz)
9099
      table(t1)
9100
      prop.table(table(t1), 1) * 100
9101
9102
       t1<-data.frame(datConsent$used,datConsent$disease)
```

```
9103
       table (t1)
9104
       prop.table(table(t1), 1) * 100
9105
9106
       t1<-data.frame (datConsent$used, datConsent$bornincanada)
9107
       table(t1)
9108
      prop.table(table(t1), 1) * 100
9109
9110
      t1<-data.frame(datConsent$used,datConsent$language 1)
9111
      table(t1)
9112
      prop.table(table(t1), 1) * 100
9113
9114
      t1<-data.frame(datConsent$used,datConsent$language 2)
9115
      table(t1)
9116
       prop.table(table(t1), 1) * 100
9117
9118
       t1<-data.frame(datConsent$used,datConsent$White group)
9119
       table(t1)
9120
      prop.table(table(t1), 1) * 100
9121
9122
       t1<-data.frame(datConsent$used,datConsent$Asian group)
9123
      table(t1)
9124
      prop.table(table(t1), 1) * 100
9125
9126
       t1<-data.frame(datConsent$used, datConsent$disability)</pre>
9127
       table(t1)
9128
      prop.table(table(t1), 1) * 100
9129
9130
      t1<-data.frame(datConsent$used,datConsent$techdisability)
9131
      table(t1)
9132
      prop.table(table(t1), 1) * 100
9133
9134
      t1<-data.frame(datConsent$used,datConsent$disability any)
9135
      table(t1)
9136
       prop.table(table(t1), 1) * 100
9137
9138
       t1<-data.frame(datConsent$used, datConsent$sexatbirth)</pre>
9139
       table (t1)
9140
       prop.table(table(t1), 1) * 100
9141
9142
       t1<-data.frame(datConsent$used,datConsent$genderidentity)
9143
       table(t1)
9144
      prop.table(table(t1), 1) * 100
9145
9146
       t1<-data.frame(datConsent$used, datConsent$income)</pre>
9147
       table(t1)
9148
       prop.table(table(t1), 1) * 100
9149
9150
       t1<-data.frame(datConsent$used,datConsent$educationlevel)
9151
       table(t1)
9152
      prop.table(table(t1), 1) * 100
9153
9154
      t1<-data.frame(datConsent$used, datConsent$edhi)</pre>
9155
      table(t1)
9156
       prop.table(table(t1), 1) * 100
9157
9158
       #Comparison for continuous demographics
9159
       describeBy (datConsent$age, datConsent$used)
9160
       wilcox.test(datConsent$age~datConsent$used)
9161
9162
       #CHANGELOG ASJ: Only keep variables analysed with >5% and dichotomous versions 2021-08-06
9163
       chisq.test(datConsent$used,datConsent$studyarm, correct=FALSE)
9164
       chisq.test(datConsent$used,datConsent$viz, correct=FALSE)
9165
       chisq.test(datConsent$used, datConsent$disease, correct=FALSE)
9166
       chisq.test(datConsent$used,datConsent$bornincanada, correct=FALSE)
9167
       chisq.test(datConsent$used, datConsent$language 1, correct=FALSE)
       chisq.test(datConsent$used,datConsent$language 2, correct=FALSE)
9168
9169
       chisq.test(datConsent$used,datConsent$Asian_group, correct=FALSE)
9170
       chisq.test(datConsent$used,datConsent$White group, correct=FALSE)
9171
       chisq.test(datConsent$used,datConsent$disability, correct=FALSE)
```

```
chisq.test(datConsent$used, datConsent$techdisability, correct=FALSE)
9172
9173
       chisq.test(datConsent$used,datConsent$disability any, correct=FALSE)
9174
       chisq.test(datConsent$used, datConsent$sexatbirth, correct=FALSE)
9175
       chisq.test(datConsent$used, datConsent$genderidentity, correct=FALSE)
9176
       chisq.test(datConsent$used,datConsent$income, correct=FALSE)
9177
       chisq.test(datConsent$used, datConsent$educationlevel, correct=FALSE)
9178
       chisq.test(datConsent$used,datConsent$edhi, correct=FALSE)
9179
9180
9181
       #### RESEARCH QUESTION 4: Effects of male vs female voice ####
9182
       # Recall: Research question 4 (add-on, may be reported separately from Hina Hakim's
9183
       thesis): Are the
9184
       # effects of the herdimm intervention different when the narration uses a female or
       male voice?
9185
       # Force this variable to be read as a factor and define the labels (this could be up in
9186
       the data
9187
       # cleaning section but we are keeping it separate in case we don't include this in
       Hina's thesis.)
9188
9189
       dat$voice <- factor(dat$voice, levels = c(1,2), labels = c("Male", "Female"))
9190
9191
       # Create 2 new variables combining voice and study arm to facilitate analyses
9192
9193
       dat$viz voice <- as.factor(paste(dat$viz,dat$voice,sep=" "))</pre>
9194
       dat$studyarm voice <- as.factor(paste(dat$studyarm,dat$voice,sep=" "))</pre>
9195
9196
       # Effect of male versus female voice in herdimm narration
9197
9198
      datHerdimm <-
9199
        subset (
9200
           dat,
9201
           dat$studyarm == "herdimmgeneric" |
9202
             dat$studyarm == "herdimmmeasles" |
             dat$studyarm == "herdimmpertussis" |
9203
             dat$studyarm == "herdimmflu"
9204
9205
         )
9206
9207
       # Analysis for risk perception, adjusted for covariates and moderators, with
       interaction of gender
9208
      # of respondents
9209
       options (contrasts=c("contr.sum", "contr.poly")) # CHANGELOG: Added to calculate
       properly the type III sum of squares with 1m 2021-07-27
9210
      mHV RP <- lm(
9211
         mean riskperception2 6 ~
9212
           studyarm * voice * genderidentity +
9213
           mean indivhorz +
9214
           mean_indivvertical +
9215
           mean collhorz +
9216
           mean collvertical +
9217
           bornincanada + #CHANGELOG ASJ: covariate list shortened 2021-08-04
9218
           language 1 +
9219
           language 2 +
9220
           Asian group +
9221
           White group +
9222
           disability any +
9223
           income +
9224
           edhi +
9225
           age,
9226
         data = datHerdimm
9227
9228
       Anova (mHV RP, type="III")
9229
       summary(mHV RP)
9230
9231
9232
       # The same analysis will be done for the other outcomes, and the model will be
       validated as for the
9233
       # main analyses. If there is an effect of voice in the above model, the 2-way ANOVA
```

```
9234
     # (viz*disease) and one-way anova model (studyarm) per disease will be done again. In
      these new
       # models, Herdimm technique will be divided according to the voice gender. The factors
9235
      for the
9236
      # two-way anova will be viz voice and disease. The factor for the one-way anova will be
      # studyarm_voice.
9237
9238
9239
      #CHANGELOG ASJ: Add this model for other continuous outcomes, 2021-08-05.
9240
9241 mHV_emot <- lm(
9242
       mean emotion ~
9243
          studyarm * voice * genderidentity +
9244
          mean indivhorz +
          mean indivvertical +
9245
          mean_collhorz +
9246
9247
          mean_collvertical +
9248
          bornincanada +
9249
          language 1 +
9250
          language 2 +
9251
         Asian group +
9252
          White group +
9253
          disability any +
9254
          income +
9255
          edhi +
9256
          age,
9257
       data = datHerdimm
9258
     )
9259
     Anova (mHV emot, type="III")
9260
9261 mHV know <- lm(
9262
      sum knowledge ~
9263
          studyarm * voice * genderidentity +
9264
          mean indivhorz +
9265
          mean indivvertical +
9266
          mean collhorz +
9267
          mean collvertical +
9268
          bornincanada +
9269
          language_1 +
9270
          language 2 +
9271
          Asian group +
9272
          White group +
9273
          disability any +
9274
          income +
9275
          edhi +
9276
          age,
9277
         data = datHerdimm
9278
9279
     Anova(mHV know, type="III")
9280
9281 #Logistic regressions
9282 rlHV_RP1 <- glm(
9283
       relevel(RP1 dicho, ref="Low") ~
9284
          studyarm * voice * genderidentity +
9285
          mean indivhorz +
9286
          mean indivvertical +
9287
          mean collhorz +
9288
          mean collvertical +
9289
          bornincanada +
9290
          language_1 +
9291
          language 2 +
9292
          Asian group +
9293
          White group +
9294
          disability any +
9295
          income +
9296
          edhi +
9297
          age,
9298
         data = datHerdimm, family=binomial("logit")
9299
```

```
9300
      Anova(rlHV RP1, type="III")
9301
9302
      rlHV c19vi <- glm(
9303
       relevel(c19vaxintent, ref="Low") ~
9304
          studyarm * voice * genderidentity +
9305
          mean indivhorz +
9306
          mean indivvertical +
9307
          mean collhorz +
9308
          mean collvertical +
9309
          bornincanada +
9310
          language 1 +
9311
          language 2 +
9312
          Asian group +
9313
          White group +
9314
          disability any +
9315
          income +
9316
          edhi +
9317
          age,
9318
         data = datHerdimm, family=binomial("logit")
9319
9320
      Anova(rlHV c19vi,type="III")
9321
9322
9323
     rlHV vi <- glm(
9324
       relevel(vaxintent, ref="Low") ~
9325
          studyarm * voice * genderidentity +
          mean indivhorz +
9326
9327
          mean_indivvertical +
          mean collhorz +
9328
9329
          mean collvertical +
9330
          bornincanada +
9331
          language 1 +
9332
          language 2 +
9333
          Asian group +
9334
          White group +
9335
          disability_any +
9336
          income +
9337
          edhi +
9338
           age,
9339
         data = datHerdimm, family=binomial("logit")
9340
9341
      Anova(rlHV vi,type="III")
9342
9343 rlHV Hti <- qlm(
9344
       relevel(Htrustinfo, ref="No") ~
9345
          studyarm * voice * genderidentity +
9346
          mean indivhorz +
9347
          mean indivvertical +
          mean collhorz +
9348
9349
          mean collvertical +
9350
          bornincanada +
9351
          language 1 +
9352
          language 2 +
9353
          Asian group +
9354
          White group +
9355
          disability any +
9356
          income +
9357
          edhi +
9358
           age,
9359
         data = datHerdimm, family=binomial("logit")
9360
       )
9361
      Anova(rlHV Hti,type="III")
9362
9363 #CHANGELOG ASJ: Add same analysis for C5 subscales, 21-09-20.
9364 rlHV C5conf <- glm(
9365
         relevel(as.factor(mean C5 conf2), ref="0") ~
9366
          studyarm * voice * genderidentity +
9367
          mean indivhorz +
9368
          mean indivvertical +
```

```
9369
          mean collhorz +
9370
          mean collvertical +
9371
          bornincanada +
9372
           language 1 +
9373
          language 2 +
9374
          Asian group +
9375
          White group +
9376
          disability_any +
9377
          income +
9378
          edhi +
9379
          age,
         data = datHerdimm, family=binomial("logit")
9380
9381
9382
      Anova(rlHV C5conf, type="III")
9383
      rlHV C5cons <- glm(
9384
      relevel(as.factor(mean C5 cons2), ref="0") ~
9385
9386
          studyarm * voice * genderidentity +
9387
          mean indivhorz +
9388
          mean indivvertical +
9389
          mean collhorz +
9390
          mean collvertical +
9391
          bornincanada +
          language 1 +
9392
9393
          language 2 +
9394
          Asian group +
          White_group +
9395
9396
          disability any +
9397
          income +
9398
          edhi +
9399
          age,
9400
         data = datHerdimm, family=binomial("logit")
9401
9402
      Anova(rlHV C5cons, type="III")
9403
9404
     rlHV C5comp <- glm(
9405
       relevel(as.factor(mean C5 comp2), ref="0") ~
9406
          studyarm * voice * genderidentity +
9407
          mean_indivhorz +
9408
          mean indivvertical +
9409
          mean collhorz +
9410
          mean collvertical +
9411
          bornincanada +
9412
          language 1 +
9413
          language 2 +
9414
          Asian group +
9415
          White group +
9416
          disability any +
9417
          income +
9418
          edhi +
9419
          age,
9420
       data = datHerdimm, family=binomial("logit")
9421
9422
      Anova(rlHV C5comp, type="III")
9423
9424
9425
      rlHV C5calc <- glm(
9426
        relevel(as.factor(mean C5 calc2), ref="0") ~
9427
           studyarm * voice * genderidentity +
9428
          mean_indivhorz +
9429
          mean_indivvertical +
9430
          mean collhorz +
9431
          mean collvertical +
9432
          bornincanada +
9433
          language 1 +
9434
          language 2 +
9435
          Asian_group +
          White group +
9436
9437
          disability any +
```

```
9438
         income +
9439
         edhi +
9440
          age,
9441
       data = datHerdimm, family=binomial("logit")
9442
     Anova(rlHV_C5calc,type="III")
9443
9444
9445
9446 rlHV_C5coll <- glm(
9447 relevel(as.factor(mean C5 coll2), ref="0") ~
       studyarm * voice * genderidentity +
mean_indivhorz +
9448
9449
         mean indivvertical +
9450
         mean_collhorz +
9451
          mean collvertical +
9452
9453
          bornincanada +
9454
          language_1 +
9455
         language 2 +
9456
         Asian group +
9457
         White group +
         disability_any +
9458
9459
         income +
9460
         edhi +
9461
          age,
9462
       data = datHerdimm, family=binomial("logit")
9463
     Anova(rlHV_C5coll,type="III")
9464
9465
9466
9467
      #### END ####
9468
9469
```